Official Title: A Phase 3, Randomized, Double-blind, Multicenter, Placebo-controlled,

Parallel-group Trial Evaluating the Efficacy, Safety, and Tolerability of Centanafadine Sustained-release Tablets in Adults With Attention-

deficit/Hyperactivity Disorder

NCT Number: NCT03605836

**Document Date:** SAP Final Version : 26 May 2020

# **Table of Contents**

| Table of Contents |
|---|
| Statistical Analysis Plan; Final: 26 May 2020 |
| STAT-1.1 Adjusted Mean Change from Baseline in AISRS Line Items at Day 42 - MMRM (Efficacy Sample) |
| STAT-1.2 Adjusted Mean Change from Baseline in ASRS Line Items at Day 42 - MMRM (Efficacy Sample) |
| STAT-3.1 MMRM Output for Test on Treatment by Sex Interaction at Day 42 (Efficacy Sample) |
| STAT-3.2 MMRM Output for Test on Treatment by Race Interaction at Day 42 (Efficacy Sample) |
| STAT-4.1.1 Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=KENWARDROGER (Efficacy Sample) |
| STAT-4.1.2 Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=SATTERTHWAITE (Efficacy Sample)131 |
| STAT-4.2 Proc GLM Output for Change from Baseline to Day 42 in AISRS Total Score, LOCF (Efficacy Sample) |
| STAT-4.3 Proc GLM Output for Change from Baseline to Day 42 in AISRS Total Score, OC (Efficacy Sample) |
| STAT-4.4 Proc GLM Output for Treatment by Center Interaction at Day 42 in AISRS Total Score, LOCF (Efficacy Sample) |
| STAT-4.5.1 Summary of Mean Change at Day 42 from Baseline in AISRS Total Score By Center - LOCF (Efficacy Sample) |
| STAT-4.5.2 Differences in Unadjusted Mean Changes of AISRS Total Score at Day 42 Among Treatment Groups By Center - LOCF (Efficacy Sample) |
| STAT-4.6 Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, LOCF (Efficacy Sample) |
| STAT-4.7 Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, OC (Efficacy Sample) |
| STAT-4.8 Non-Parametric Stratified by Center Analysis of Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, LOCF (Efficacy Sample) |
| STAT-4.9 Residual at Day 42 from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample) |
| STAT-4.10 Proc Mixed Output Using Heterogeneous Variance Structure for Treatment Groups (Efficacy Sample)230 |

| (Efficacy Sample)25 | 56 |
|---|---|
| STAT-5.2 Proc GLM Output for Change from Baseline to Day 42 in CGI-S Scale, LOCF (Efficacy Sample) | 70 |
| STAT-5.3 Proc GLM Output for Change from Baseline to Day 42 in CGI-S Scale, OC (Efficacy Sample) | 76 |
| STAT-6.1.1 Shapiro-Wilk Test for Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample) 28 | 82 |
| STAT-6.1.2 Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample) | 83 |

# Otsuka Pharmaceutical Development & Commercialization, Inc.

**Investigational Medicinal Product** 

Centanafadine (EB-1020)

A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled Evaluation the Efficacy, Safety and Tolerability of Centanafadine Sustained-release in Adults with Attention-deficit/Hyperactivity Disorder

Protocol No. 405-201-00014 IND No. 119,361

# **Statistical Analysis Plan**

**Version: Final** 

Date: May 26, 2020

CONFIDENTIAL – PROPRIETARY INFORMATION

Confidential

May not be used, divulged, published or otherwise disclosed
without the consent of Otsuka Pharmaceutical Development & Commercialization, Inc.

# **Table of Contents**

| I ab | ie of Contents | <u>4</u> |
|---|---|---|
| 1 | Introduction | 5 |
| 2 | Study Objectives | |
| 3 | Study Design | |
| 4 | Sample Size and Power Justification | <mark>7</mark> |
| 5 | Data Sets for Analysis and Missing Data | |
| 5.1 | Data Sets for Analysis | |
| 5.2 | Handling of Missing Data | 8 |
| 6 | Study Conduct | 9 |
| 6.1 | Subject Disposition, Completion Rate and Reasons for Discontinuation | 9 |
| 6.2 | Treatment Compliance | 9 |
| 6.3 | Protocol Deviation | 10 |
| 7 | Baseline Characteristics | 10 |
| 7.1 | Baseline Definition | 10 |
| 7.2 | Demographic Characteristics | 10 |
| 7.3 | Medical and Psychiatric History | 10 |
| 7.4 | Neuropsychiatric Diagnosis | 11 |
| 7.5 | Baseline Psychiatric Evaluation | 11 |
| 8 | Efficacy Analysis | 11 |
| 8.1 | Primary Efficacy Endpoint | 11 |
| 8.1.1 | Primary Efficacy Analysis | 11 |
| 8.1.2 | Technical Computation Details for Primary Efficacy Analysis | 13 |
| 8.1.3 | Sensitivity Analyses | 14 |
| 8.1.3 | .1 Sensitivity Analyses for Missing at Random (MAR) Assumption | 14 |
| 8.1.3 | .2 Per Protocol Analyses | 15 |
| 8.1.3 | Other Sensitivity Analyses | 15 |
| 8.1.3 | 3 3 | |
| 8.1.4 | Subgroup Analyses | |
| 8.2 | Key Secondary Efficacy Endpoint | |
| 8.3 | Other Efficacy Endpoints | 18 |

| C | A | P | 4 | Ŋ٠ | ۲. | _ 🤈 | n | ١1 | l _( | በ | n | ۱ | ١ | ١1 | 14 | L |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| J. | $\overline{}$ | | - | v. | , - | -/. | u | ч | - | 11 | u | ,, | ш | ч | - | ۰ |

| 8.4 Exploratory Efficacy Endpoints | | |
|---|---|---|
| 8.5 | Exploratory Analysis | 19 |
| 9 | Safety Analysis | 20 |
| 9.1 | Adverse Events | 20 |
| 9.1.1 | Adverse Events in the Double-Blind Treatment Period | 21 |
| 9.1.2 | Adverse Events in the Single-blind Placebo Run-in Period | 21 |
| 9.2 | Clinical Laboratory Tests | 21 |
| 9.2.1 | Clinical Laboratory Tests in Double-Blind Treatment Period | 22 |
| 9.2.2 | Drug Induced Liver Injury (DILI) | 22 |
| 9.2.3 | Clinical Laboratory Tests in the Single-blind Placebo Run-in Period | 22 |
| 9.3 | Vital Signs | 22 |
| 9.3.1 | Vital Signs in the Double-Blind Treatment Period | 22 |
| 9.3.2 | Vital Signs in the Single-blind Placebo Run-in Period | 23 |
| 9.4 | Electrocardiogram (ECG) Data | 23 |
| 9.4.1 | ECG Data in the Double-Blind Treatment Period | 23 |
| 9.4.2 | ECG Data in the Single-blind Placebo Run-in Period | 24 |
| 9.5 | Physical Examinations | 24 |
| 9.5.1 | Body Weight, Waist Circumference and Body Mass Index (BMI) | 24 |
| 9.6 | Suicidality Data | 24 |
| 9.7 | SMWQ | 25 |
| 9.8 | Medication Handling Irregularities (MHIs) and Events Subject to Addition Monitoring (ESAMs) | |
| 9.9 | Concomitant Medications | 25 |
| 9.10 | Extent of Exposure | 26 |
| 10 | Conventions | 26 |
| 10.1 | Study Visit Windows | 26 |
| 10.2 | Pooling of small centers | 27 |
| 10.3 | Scales: Rules for Scoring and Handling of Missing Data | 27 |
| 10.3.1 | Adult ADHD Investigator Symptom Rating Scale (AISRS) | 27 |
| 10.3.2 | Clinical Global Impression Severity of Illness Scale – Modified for Attention-Deficit Hyperactivity Disorder | 28 |
| 10.3.3 | Clinical Global Impression Change from Baseline | 28 |
| 10.3.4 | Attention-Deficit Hyperactivity Disorder Impact Module – Adult (AIM- | A) 28 |

| SAP 405 | 5-201-00014 | |
|-------------|-----------------------------------------------------|----|
| 10.3.5 | | 29 |
| 10.3.6 | Study Medication Withdrawal Questionnaire (SMWQ) | 29 |
| 10.3.7 | Columbia-Suicide Severity Rating Scale (C-SSRS) | 29 |
| <b>11</b> ] | References | 31 |
| <b>12</b> ] | Potential Clinical Relevance Criteria from Protocol | 32 |
| <b>13</b> | Proposed List of Summary Tables | 35 |

## 1 Introduction

This statistical analysis plan (SAP) documents the statistical methodology and data analysis algorithms and conventions to be applied for statistical analysis and reporting of efficacy and safety data of study 405-201-00014. All amendments to the protocol are taken into consideration in developing this SAP.

# 2 Study Objectives

Primary: To confirm the efficacy of centanafadine SR tablets administered BID (200 mg or 400 mg TDDs) compared to placebo in the treatment of adults with ADHD

Secondary: To confirm the safety and tolerability of centanafadine SR tablets administered BID (200 mg or 400 mg TDDs) compared to placebo in the treatment of adults with ADHD

# 3 Study Design

This trial is a phase 3, randomized, double-blind, multicenter, placebo-controlled, parallel-group trial to confirm the efficacy, safety, and tolerability of centanafadine SR (200 mg TDD or 400 mg TDD) compared to placebo for the treatment of adults with ADHD. The trial population will include male and female subjects 18 to 55 years of age (inclusive) with a current diagnosis of ADHD as confirmed by the Adult ADHD Clinical Diagnostic Scale (ACDS) Version 1.2 at screening.

The trial will have 4 periods: (1) screening and washout; (2) 1 week single-blind placebo runin; (3) 6-week double blind treatment; and (4) 7-day follow-up period (follow-up telephone calls at 1, 3, and 5 days after the last dose of IMP, and in-clinic visits 2 and 7 days after the last dose of IMP) for subjects who complete the trial, and decide to enroll in Trial 405-201-00015. For subjects who terminate early, decide to not enroll in Trial 405-201-00015, or who are not eligible to enroll in Trial 405-201-00015, they will be required to participate in the 7-day follow-up period as well as participate in an additional follow-up telephone call 10 days after the last dose of IMP. Subjects randomized to receive a TDD of 200 mg centanafadine SR will start at their target dose at the start of the double-blind treatment period. Subjects randomized to receive a TDD of 400 mg centanafadine SR will start the double-blind treatment period at the TDD of 200 mg centanafadine SR for 7 days, before they are escalated to their target TDD of 400 mg for a total of approximately 42 days of treatment. Subjects will be required to visit the site up to 12 times over the trial. See Figure 3-1 for a schematic of the trial design.

Subjects who complete both the 6-week double-blind treatment period and the 7-day safety follow-up period (follow-up telephone calls at 1, 3, and 5 days after the last dose of IMP, and in-clinic visits 2 and 7 days after the last dose of IMP), and refrain from using prohibited

medications after the IMP is stopped may be eligible to enroll into Trial 405-201-00015, which is a 12-month, observational, open-label trial to evaluate the long-term safety and tolerability of subjects with ADHD who previously participated in Trials 405-201-00013 or 405-201-00014. Subjects who terminate early, decide to not enroll in Trial 405-201-00015, or who are not eligible to enroll in Trial 405-201-00015, will be required to participate in the 7-day follow-up period as well as participate in an additional follow-up telephone call 10 days after the last dose of IMP. For subjects who early terminate or decline participation in the open-label trial, they will be instructed to refrain from utilizing prohibited concomitant medications, including ADHD treatments, until after the follow-up telephone call 10 days after the last dose of IMP.



Figure 3-1 Trial Design Schematic

ASRS = Adult ADHD Self Report Scale; CTN SR = centanafadine sustained release; ET = early termination; P = placebo administration; R = randomization.

During the trial, administration of the investigational medicinal product (IMP) will be double-blinded. In other words, neither the investigator nor the subject will have knowledge of the treatment assignment (e.g., centanafadine SR 200 mg, 400 mg, or placebo). Treatment assignments will be based on a computer-generated randomization code provided by the Otsuka Pharmaceutical Development & Commercialization, Inc (OPDC) Biometrics Department. Sponsor personnel, including those involved in monitoring, data management, and data analysis, will not have access to the treatment code during the trial. The bioanalytical

<sup>&</sup>lt;sup>a</sup>All subjects will be required to participate in the 7-day follow-up period (follow-up telephone calls at 1, 3, and 5 days after the last dose of IMP, and in-clinic follow-up visits at 2 and 7 days after the last dose of IMP). Subjects who terminate early, decide to not enroll in Trial 405-201-00015, or who are not eligible to enroll in Trial 405-201-00015, will be required to participate in an additional follow-up telephone call 10 days after the last dose of IMP.

laboratory will also be sent the randomization code. The randomization will be stratified by trial site and designed to allocate subjects in a 1:1:1 ratio to centanafadine SR 200 mg/day or 400 mg/day or placebo.

# 4 Sample Size and Power Justification

The primary efficacy endpoint is the change from baseline at Day 42 in Adult ADHD Investigator Symptom Rating Scale (AISRS) total score. The trial will compare the placebo arm to the centanafadine dose arms, randomized at a ratio of 1:1:1, with an overall alpha of 0.05 for the primary endpoint.

Based on the results from Phase 2 centanafadine trials, it is reasonable to expect a treatment effect of 5 points with a standard deviation (SD) of 12.5 in the mean change from baseline to Day 42 on AISRS total score. The planned sample size of 405 evaluable subjects (135 in each treatment arm) will yield at least 90% power to detect the treatment effects at a 2-tailed significance level of 0.05.

A sufficient number of subjects will be enrolled and randomized to achieve approximately 405 evaluable subjects in the Double-blind Treatment Phase (i.e., subjects with an AISRS total score at baseline and at least 1 subsequent AISRS total score in the Double-blind Treatment Phase). After allowance of 10% non-evaluable subjects in the Double-blind Treatment Phase, the total number of subjects to be randomized is 450 (150 in each treatment arm). In order to ensure 405 evaluable subjects, the number of non-evaluable subjects will be monitored in a blinded manner on an ongoing basis During the trial. The power and sample size were obtained using the PASS 14 (2015) statistical computing software.

# 5 Data Sets for Analysis and Missing Data

## 5.1 Data Sets for Analysis

The following analysis samples are defined for this trial:

**Enrolled Sample**: comprises all subjects who signed an informed consent form (ICF) for the trial and enrolled into the single-blind placebo run-in period.

**Randomized Sample**: comprises all subjects who were randomized in the double-blind treatment period. Subjects are considered randomized when they are assigned a treatment group by eSource at the end of single-blind placebo run-in period. A subject receiving IMP outside of the eSource will not be considered randomized, but safety will be reported.

**Safety Sample**: comprises those randomized subjects in the double-blind treatment period who received at least one dose of double-blind IMP as indicated on the dosing record. Subjects will only be excluded from this population if there is documented evidence (i.e., drug

dispensed = drug returned or no IMP dispensed) that the subject did not take IMP. If a subject is dispensed IMP and is lost to follow up, he/she will be considered exposed.

**Efficacy Sample**: the Full Analysis Set (FAS) comprises all subjects in the Safety Sample who have a baseline value and at least one valid post-randomization efficacy evaluation for AISRS total score in the double-blind treatment period.

**Per Protocol (PP) Sample:** comprises those subjects in the Efficacy Sample who complete at least the first 2 weeks of double-blind medication ((last day of IMP - first day of IMP + 1)  $\geq$  14 days) and have at least one post baseline AISRS measurement on or after Day 14 visit during the double-blind treatment period without major protocol violations deemed to compromise the assessment of efficacy. These major protocol violations will be any of the followings:

- 1. Subjects who were not at least 80% or were more than 120% compliant with double-blind IMP or missed 7 or more consecutive days of dosing immediately prior to the Day 42/ET AISRS measurement date during the double-blind treatment period based on subject-reported (eCRF) compliance data
- 2. Subjects who reported concomitant medication use that will impact the primary efficacy endpoint
- 3. Subjects who had major protocol deviation as represented on the protocol deviation eCRF page that will impact the primary efficacy endpoint
- 4. Subjects who took the wrong study treatment

The core dataset for all efficacy analyses is the FAS, which is created based on the intent-to-treat (ITT) principle. However, as will be described below, in order to handle missing data and restrictions imposed by different types of analyses (e.g., change from baseline analysis), other datasets derived from the FAS dataset will be used for the efficacy analyses.

## 5.2 Handling of Missing Data

The mixed-effect model repeated measure (MMRM) assumes data are missing at random (MAR), which is a reasonable assumption in longitudinal clinical trials in MDD<sup>1</sup>. However, the possibility of "missing not at random" (MNAR) data can never be ruled out. As sensitivity analyses, selection model<sup>2</sup>, pattern-mixture model<sup>3,4,5,6</sup>, and/or shared parameter model<sup>7</sup> will be used to explore data missing mechanisms of MNAR and investigate the response profile of dropout patients by last dropout reason under MNAR mechanism for the following 3 scenarios: 1) Dropout reasons due to either AE or LOE as MNAR, 2) Dropout reasons due to either AE or LOE or subject withdrew consent as MNAR, 3) All dropouts as MNAR using

both 1) Delta adjustment imputation method which is to departure from MAR assumption by progressively increasing the delta until conclusion from the primary analysis is overturned, and 2) Placebo based imputation methods in which missing data for both placebo and drug group are imputed based on the imputation model derived from placebo data. If drug improved outcomes prior to dropout, this benefit is carried into subsequent imputed values, but will diminish over time in accordance with the correlation structure. Details are provided in Section 8.1.3 Sensitivity Analysis. The observed-cases (OC) data set will consist of actual observations recorded at each visit during the double-blind treatment period and no missing data will be imputed. MMRM, Wu-Bailey, and pattern-mixture model will be performed on the OC dataset.

The last-observation-carried-forward (LOCF) data set will include data recorded at a scheduled double-blind treatment period visit or, if no observation is recorded at that visit, data carried forward from the previous scheduled double-blind treatment period visit. Baseline data (e.g., the last visit of the single-blind placebo run-in period) will not be carried forward to impute missing values for the LOCF data set. The analysis of covariance (ANCOVA) analysis will be performed for the change from baseline to the end of the double-blind treatment period (Day 42, LOCF) in AISRS total score as sensitivity analysis. The ANCOVA\_LOCF model includes treatment and study center as main effects, and baseline value as a covariate.

ANCOVA analysis with OC data will also be conducted on change from baseline for AISRS total score, as well as all continuous change from baseline efficacy endpoints.

For Clinical Global Impression (CGI) Change from Baseline and categorical response/remission variables, OC analyses will be performed in addition to LOCF analyses. Study center will not be included in the models for OC analyses.

# **6** Study Conduct

# 6.1 Subject Disposition, Completion Rate and Reasons for Discontinuation

Subject disposition will be summarized for the Randomized Sample by treatment group, and by center.

Subject completion rate and reasons for discontinuation will be summarized for the Randomized Sample by treatment group for the double-blind treatment period.

# 6.2 Treatment Compliance

For each subject, compliance in taking IMP is calculated by dividing the number of tablets taken by the total number of tablets the patients were scheduled to take during the double-blind

treatment period. Compliance is calculated on double-blind IMP for the double-blind treatment period. For lost-to-follow up patients, the last IMP end date record will be used as the treatment end date.

Summary of Treatment compliance will be provided based on both eCRF data and AiCure captured data, respectively.

#### 6.3 Protocol Deviation

Protocol deviations are summarized by center and type of deviation for randomized subjects by treatment group. Listing of protocol deviation will list the treatment phases during which the deviations occurred. In addition, protocol deviations affected by the COVID-19 will be summarized. Listing of subjects with protocol deviations affected by the COVID-19 will also be provided.

## 7 Baseline Characteristics

#### 7.1 Baseline Definition

Baseline for the single-blind placebo run-in period refers to last available measurement prior to the start of administration of placebo in the single-blind placebo run-in period.

For analyses of the double-blind treatment period data, the baseline is defined as the last available measurement prior to the first dose of double-blind Investigational Medicinal Product (IMP) in the double-blind treatment period.

# 7.2 Demographic Characteristics

For the Randomized Sample, demographic characteristics will be summarized by treatment group. Age, race, ethnicity, height, weight, waist circumference, and body mass index (BMI) will be tabulated by gender and overall using the baseline assessments for the single-blind placebo run-in period.

Mean, range and standard deviation will be used to describe continuous variables such as age. Frequency distributions will be tabulated for categorical variables such as race.

# 7.3 Medical and Psychiatric History

A summary of medical and psychiatric history will be presented for the Randomized Sample by treatment group and overall.

A summary of the Adult ADHD Clinical Diagnostic Scale (ACDS) at screening will also be presented for the Randomized Sample (by treatment group and overall). The number and

percentage of patients with each response to items A23-A41 from Section A (Childhood ADHD Symptoms Summary), B22-B39 from Section B (Adult ADHD Symptoms Summary), and C1-C5 will be presented.

## 7.4 Neuropsychiatric Diagnosis

A summary of MINI International Neuropsychiatric Interview (M.I.N.I.) will be presented for the Randomized Sample by treatment group and overall. Summarized will be the number and percentage of patients who meet each diagnosis criteria, and number and percentage of patients with each primary diagnosis.

## 7.5 Baseline Psychiatric Evaluation

For the Randomized Sample, baseline for the single-blind placebo run-in period and baseline for the double-blind treatment period psychiatric scale evaluation will be summarized by treatment group and overall. The mean, median, range and standard deviation will be used to summarize the assessments of: AISRS total score, ASRS and CGI - Severity of Illness Score (CGI-S).

# 8 Efficacy Analysis

All efficacy analyses pertaining to the double-blind treatment period will be performed on the Efficacy Sample, and patients will be included in the treatment group as randomized.

For analysis of the double-blind treatment period data, the baseline for the double-blind treatment period defined in Section 7.1 will be used. Statistical comparisons are based on 2-sided, 0.05 significance levels.

# 8.1 Primary Efficacy Endpoint

The primary efficacy endpoint is the change from the baseline of the double-blind treatment period to Day 42 in AISRS total score.

# 8.1.1 Primary Efficacy Analysis

The objective of the primary efficacy analysis is to compare the efficacy between centanafadine (SR 200 mg TDD or SR 400 mg TDD) and placebo.

The primary estimand defining the treatment effect of interest in the trial uses the hypothetical strategy specified in the draft ICH E9 (R1) Addendum. The objective of the primary analysis is to evaluate the efficacy of centanafadine SR 400mg TDD in adult subjects with ADHD

versus placebo. The estimand, or target of estimation, following the hypothetical strategy is the pharmacological effect seen, had no withdrawals occurred. This hypothetical estimand is justifiable in this case, since the focus is on the pharmacological effect of the drug additional to non-specific effects. Subjects who withdraw from a symptomatic IMP treatment either could have lost their treatment effect, had the subjects not taken any other symptomatic medication after withdrawal, or could have their treatment effect been masked, had the subjects taken other symptomatic medication after withdrawal. This means that any observations taken after subjects stop IMP will most likely not contribute relevant information about the pharmacological effect of the drug. Due to this strategy, the last collected efficacy assessment after premature trial discontinuation will be done only once at the ET Visit. Every effort will be made to complete all of the ET evaluations prior to administering any additional medications for the treatment of ADHD or other prohibited medications. In the case of terminal or lost to follow-up events, no ET evaluations would be expected, and only scheduled assessments performed before such an event has occurred.

The primary estimand for this trial is defined by the following components:

- Target Population: Efficacy Sample
- Endpoint: Change from baseline to Day 42 in the AISRS total score
- Intercurrent Events: Premature treatment discontinuation
- Measure of Intervention Effect: Difference in endpoint means between centanafadine (SR 200 mg TDD or SR 400 mg TDD) and placebo.

In this hypothetical strategy, the event of withdrawing IMP is considered missing at random (MAR), and the primary endpoint of the trial could be considered as a combination of the responses of on-treatment completers at Day 42 and the imputation of the endpoint to Day 42 following the trend in each treatment group using the MMRM method for subjects who withdraw IMP during the trial. All data collected during the trial treatment period will be used for statistical analysis. For the primary efficacy analysis, the treatment effect will be estimated using the MMRM method described below. Under the MAR assumption, MMRM provides an unbiased estimate of treatment effect for the treatment period. Analyses with missing values imputed by multiple imputation under MNAR and other methods will be performed as sensitivity analyses. The primary analysis will be performed on Efficacy Sample which includes all randomized subjects who took at least 1 dose of IMP in the double-blind treatment period and who have both a baseline for the double-blind treatment period. The primary efficacy analysis will be performed by fitting a MMRM analysis with an unstructured (UN) variance covariance structure in which the change from baseline for the double-blind

treatment period in AISRS total score at the scheduled double-blind treatment period visits will be the dependent variable based on the OC data set. The model will include fixed class effect terms for treatment, study center, visit day, and an interaction term of treatment by visit day. The model will also include the interaction term of baseline values for the double-blind treatment period of AISRS Total score by visit day as covariates. The primary comparison between centanafadine (400 mg TDD group or 200 mg TDD group) and placebo at Day 42 in the double-blind treatment period will be estimated as the difference between Least Squares (LS) means utilizing the computing software SAS procedure PROC MIXED.

In case there is a convergence problem with MMRM model with the unstructured (UN) variance covariance matrix, the following structures other than unstructured will be used in order of 1) heterogeneous toeplitz (TOEPH), 2) heterogeneous autoregressive of order 1 (ARH1), and 3) heterogeneous compound symmetry (CSH) and the first (co)variance structure converging to the best fit will be used as the primary analysis. If a structured covariance has to be used, the empirical "sandwich" estimator of the standard error of the fixed effects parameters will be used in order to deal with possible model misspecification of the covariance matrix.

Small centers will be defined as centers that do not have at least one evaluable subject (evaluable with regard to the primary efficacy variable) in each treatment arm in the double-blind treatment period. All small centers will be pooled to form "pseudo centers" for the purpose of analysis according to the following algorithm. Small centers will be ordered from the largest to the smallest based on the number of evaluable subjects (i.e., subjects who have baseline and at least one post-baseline value for the primary endpoint in the double-blind treatment period). The process will start by pooling the largest of the small centers with the smallest of the small centers until a non-small center is formed. This process will be repeated using the centers left out of the previous pass. In case of ties in center size, the center with the smallest center code will be selected. If any centers are left out at the end of this process, they will be pooled with the smallest pseudo centers, or if no pseudo centers exist, they will be pooled with the smallest non-small center.

# 8.1.2 Technical Computation Details for Primary Efficacy Analysis

The SAS code for the PROC MIXED procedure to carry out the above MMRM analysis with an unstructured variance covariance structure is illustrated as follows:

```
proc mixed;
  class treatment center visit subjid;
  model change=treatment center visit treatment*visit baseline*visit / s cl
ddfm=kenwardroger;
  repeated visit /type=un subject=subjid r rcorr;
```

lsmeans treatment\*visit / pdiff cl alpha=0.05 slice=visit; run;

where baseline is the last AISRS Total score prior to the first dose of double-blind IMP in the double-blind treatment period.

## 8.1.3 Sensitivity Analyses

## 8.1.3.1 Sensitivity Analyses for Missing at Random (MAR) Assumption

Traditionally the dropout mechanisms are divided into three types (Little, 1995): (1) Missing Completely at Random (MCAR), in which the probability of dropout doesn't depend on the observed data and the missing data; (2) Missing at Random (MAR), in which the probability of dropout depends on the observed data, and (3) Missing Not at Random (MNAR), where the probability of dropout depends on the missing data and possibly the observed data.

Most of MNAR methods (Diggle P, Kenward MG, 1994) have treated all observations with dropout as if they fall within the same dropout type. In practice, we would find that different dropout reasons may be related to the outcomes in different ways, for example, detailed dropout reasons for this study are: adverse events (AE), lack of efficacy (LOE), lost to follow-up, protocol deviation, sponsor discontinued study, subject met (protocol specified) withdrawal criteria, subject was withdrawn from participation by the investigator, and subject withdrew consent to participate. Dropout due to an AE and LOE may lead to MNAR dropout. Subject withdrew consent may also lead to MNAR dropout. However, it is debatable whether a dropout caused by subjects withdrew consent is MAR or MNAR. Except AE, LOE, and subject withdrew consent, all the other dropout reasons may be assumed as either MCAR or MAR dropout. Missing data due to COVID-19 will also be assumed as MAR.

As sensitivity analyses for missing at random (MAR) assumption, analyses for missing not at random (MNAR) will be carried out. Pattern Mixture Models (PMM) based on Multiple Imputation (MI) with mixed missing data mechanisms will be used to investigate the response profile of dropout patients by last dropout reason under MNAR mechanism for the following three scenarios:

- 1) Dropout reasons due to either AE or LOE as MNAR
- 2) Dropout reasons due to either AE or LOE or subject withdrew consent as MNAR
- 3) All dropouts as MNAR

### **Delta Adjustment Imputation Methods**

This MNAR sensitivity analysis is to departure from MAR assumption by progressively increasing the delta until conclusion from the primary analysis is overturned. The delta is 0%, 10%, 20%, 30%, ..., 100% of the expected treatment difference of 5 points and/or the observed

treatment difference between centanafadine and Placebo from the primary analysis of MMRM model until conclusion of the primary analysis is overturned. When delta=0 it is MAR. When delta > 0 it is MNAR.

- 1) Using Monte Carlo Markov Chain (MCMC) methodology from PROC MI to impute the intermittent missing data to a monotone missing pattern;
- 2) Using a standard MAR-based multiple imputation approach from PROC MI to impute the monotone missingness data
- 3) For patients in the treated group and with a dropout reason of AE or LOE or subject withdrew consent, a delta will be added for all the values after the dropout time.
- 4) Using MMRM model in the primary analysis to analyze the completed data using PROC MIXED on the multiple imputed data
- 5) Obtaining the overall results using PROC MIANALYZE.

## **Placebo Based Imputation Methods**

Similar to "Standard" multiple imputations, except parameters for imputation model obtained from only the placebo (control) group. Missing data for both placebo and drug group are imputed based on the imputation model derived from placebo data. If drug improved outcomes prior to dropout, this benefit is carried into subsequent imputed values, but will diminish over time in accordance with the correlation structure.

In addition, model based MNAR methods such as the shared parameter model (Wu and Baily, 1989) and random coefficient pattern mixture model (Hedeker D, Gibbons RD, 1997) will be also performed.

#### **LOCF and OC Analyses**

Change from baseline of the double-blind treatment period for the AISRS total score will be evaluated using ANCOVA with baseline of the double-blind treatment period value as covariate and treatment and, in LOCF analyses, study center as main effects. For the OC analyses, study center will not be included in the model.

# 8.1.3.2 Per Protocol Analyses

Per Protocol analysis will be performed using the Per Protocol Sample.

# 8.1.3.3 Other Sensitivity Analyses

The following analyses will be performed to evaluate of the sensitivity of the results due to the impact of COVID-19.

1. A MMRM analysis (the same model for the primary efficacy analysis) based on the pre-COVID Efficacy Sample using all OC data set during the double-blind treatment

- period. The pre-COVID Efficacy Sample comprises those subjects in the Efficacy Sample who completed or discontinued from the study before March 13, 2020, the National Emergency Announcement on COVID-19<sup>11</sup>.
- 2. A MMRM analysis (the same model for the primary efficacy analysis) based on the Efficacy Sample using pre-COVID data set. The pre-COVID data set consists of actual observations recorded at each visit during the double-blind treatment period before March 13, 2020, the National Emergency Announcement on COVID-19<sup>11</sup>.
- 3. A MMRM analysis (the same model for the primary efficacy analysis) based on the non-COVID Efficacy Sample using all OC data set during the double-blind treatment period. The non-COVID Efficacy Sample comprises those subjects in the Efficacy Sample who had no COVID-19 related PDs.
- 4. A MMRM analysis (the same model for the primary efficacy analysis) based on the Efficacy Sample using non-COVID data set. The non-COVID data set consists of actual observations recorded at each visit during the non-COVID treatment period which represents the time period where subjects did not have any COVID-19 related PDs during the double-blind treatment period. For each subject, the non-COVID treatment period starts from randomization and ends on the Day 42/ET date or the date before the first COVID-19 related PD (if present), whichever occurs earlier.
- 5. A MMRM analysis (the same model for the primary efficacy analysis) based on the Efficacy Sample excluding the assessments performed remotely.

# 8.1.3.4 Sensitivity Analyses for Violation of Normality Assumption

The primary endpoint MMRM analysis is a maximum likelihood method that relies on normality assumption. Residual analyses will be carried out to examine model assumption.

In the case of gross violations of the normality assumptions, nonparametric van Elteren test<sup>8</sup> (van Elteren, 1960) will be performed to compare treatment effect at Week 14 on both LOCF dataset and Multiple Imputation (MI) data. The van Elteren test is a generalized CMH procedure useful for stratified continuous data in non-normal setting. It belongs to a general family of Mantel-Haenszel mean score tests. The test is performed via SAS procedure PROC FREQ, by including CMH2 and SCORES=MODRIDIT options in the TABLE statement. The stratification factor is trial center.

In addition, other methods that are robust to distributional assumption will also be performed to provide different views on the primary efficacy result, these include generalized estimating equations (GEE), weighted GEE (WGEE), and MI-robust regression<sup>9</sup>.

For MI-van Elteren test and MI-robust regression, imputation datasets will be generated with SAS MI procedure, each dataset will be analyzed, then an overall estimate is derived with SAS MIANALYZE procedure.

## 8.1.4 Subgroup Analyses

Subgroup analyses of change from baseline of the double-blind treatment period in AISRS total score to every scheduled visit in the double-blind treatment period will be performed by the following factors:

- Sex (Based on the biological status)
- Race (White and All Other Races)

All subgroup analyses will be conducted using the same MMRM analysis as for the primary efficacy analysis except that the fixed class effect term for trial center will not be included in the model.

Interaction effects of treatment-by-subgroup will be assessed at Day 42 for the subgroups identified in the previous paragraph. MMRM analyses will be performed by adding addition of terms for subgroup-by-day and treatment-by-subgroup-by-day. These treatment-by-subgroup interaction analyses will be presented in statistical documentation.

# 8.2 Key Secondary Efficacy Endpoint

The key secondary efficacy endpoint is the change from baseline of the double-blind treatment period to Day 42 using the CGI-S. This key secondary efficacy endpoint will be analyzed by fitting the same MMRM model described in the primary analysis.

To control the overall experiment-wise type I error at 0.05 level, A fixed sequence testing approach will be applied. The statistical test will be performed in the following order:

- 1) Change from baseline to Day 42 in the double-blind treatment period in AISRS total score between centanafadine 400 mg TDD and placebo;
- 2) Change from baseline to Day 42 in the double-blind treatment period in AISRS total score between centanafadine 200 mg TDD and placebo;
- 3) Change from baseline to Day 42 in CGI-S score between centanafadine 400 mg TDD and placebo;
- 4) Change from baseline to Day 42 in CGI-S score between centanafadine 200 mg TDD and placebo.

The testing procedure will stop at the first comparison where the p-value is  $\geq 0.05$ . None of the subsequent comparisons will be performed.

## 8.3 Other Efficacy Endpoints

Other efficacy analyses are listed below. All other efficacy variables will be evaluated at a nominal 0.05 level (2-sided) without adjusting for multiplicity.

- 1) Change from baseline in AISRS total score for every scheduled visit during the doubleblind treatment period other than the Day 42 visit;
- 2) Change from baseline for the Inattentive subscale and Hyperactive-Impulsive subscale of the AISRS for scheduled visits during the double-blind treatment period, separately at every visit
- 3) Change from baseline in CGI-S for every scheduled visit during the double-blind treatment period other than the Day 42 visit
- 4) CGI Change from Baseline will be collected at each scheduled visit
- 5) Percentage of responders at each post-baseline visit during the double-blind treatment period, where a responder is defined as a subject with a CGI Change from Baseline score of 1 or 2 OR a ≥ 30% improvement in ADHD symptoms compared with baseline as measured by the AISRS total score
- 6) Response rate at each post-baseline visit during the double-blind treatment period, where response is defined as
  - a) a CGI Change from Baseline score of 1 or 2 OR a  $\geq$  20% improvement in ADHD symptoms compared with baseline as measured by the AISRS total score.
  - b) a CGI Change from Baseline score of 1 or 2 OR a  $\geq$  40% improvement in ADHD symptoms compared with baseline as measured by the AISRS total score.
- 7) Remission rate for every scheduled visit during the double-blind treatment period, where remission is defined as AISRS total score  $\leq 18$ .

Variable (1) through variable (3) will be evaluated using the same MMRM model described in the primary analysis. Variable (4) will be evaluated by the Cochran Mantel Haenszel (CMH) Row Mean Score Differ Test controlling, in LOCF analysis, for trial center. Variable (5) through variable (7) will be evaluated by the CMH General Association Test controlling, in LOCF analysis, for study center. An OC analysis will also be conducted for variables (4) through (7) but will not control for trial center. Separate summary and statistical test for response rate based only on the AISRS improvement and only on the CGI Change from Baseline score will be presented for (5) and (6).

### 8.4 Exploratory Efficacy Endpoints

The exploratory efficacy endpoints are listed below. The exploratory efficacy endpoints, when applicable, will be evaluated at a nominal 0.05 level (2-sided) without adjusting for multiplicity.

- 1) Change from baseline for Question 1 (Global Quality of Life) and Questions 9Aa 9Ai and 9Ba 9Bi (Impact of Symptoms) of AIM-A at scheduled visits during the double-blind treatment period, separately at every visit
- 2) Proportion of subjects in each response for the following questions of AIM-A at scheduled visits during the double-blind treatment period, separately at every visit
  - a. Questions 2-4 (Global Quality of Life)
  - b. Questions 5a-5j (Living with ADHD)
  - c. Questions 6a-6k (General Well-Being)
  - d. Questions 7a-7j (Work, Home and School Performance and Daily Functioning)
  - e. Questions 8a-8h (Relationships and Communication)
  - f. Economic impact (5 items)
  - g. Questions 17-23 (Demographics/Medication Status)
- 3) Change from baseline in the total score of (18 item) ADHD Symptoms score of the ASRS and subscale scores for ASRS at scheduled visits during the double-blind treatment period, separately at every visit

Variables (1) and (3) will be evaluated using the same MMRM model described in the primary analysis. Variable (2) will be summarized by descriptive statistics and no statistical comparisons between centanafadine and placebo will be performed.

## 8.5 Exploratory Analysis

Exploratory efficacy analyses will be presented in Statistical Documentation.

Treatment-by-center interaction will be assessed at Day 42 by including the treatment-by-center-by-visit interaction in the model. Results for study centers will be displayed from largest center to smallest center.

Line Item score will be performed for AISRS and ASRS on Change from baseline of the double-blind treatment period to Day 42 using the MMRM model for AISRS and ASRS, where Cohen's D Effect Size<sup>10</sup> is the difference between the two means divided by their standard deviation [as defined by Cohen's D and reviewed on pages 4-6 from the Sage book "Effect Size for ANOVA Designs" (Vol 129) by Cortina and Nouri]. For MMRM (using SAS PROC MIXED), or ANCOVA (Using SAS PROC GLM), LSMean difference of treatment effects for the between centanafadine and placebo groups, and the standard error of the difference (Stderr) will be obtained with an Estimate statement. Let n<sub>1</sub> and n<sub>2</sub> denote the

respective sample sizes of the two groups to compare, Effect Size =  $d = (LSMean_1 - Effect)$ 

LSMean<sub>2</sub>) / 
$$\sigma$$
, where  $\sigma = \frac{\text{Stderr}}{\sqrt{\frac{1}{n_1} + \frac{1}{n_2}}}$ .

# 9 Safety Analysis

Standard safety variables to be analyzed include AEs, clinical laboratory tests, vital signs, electrocardiograms (ECGs), body weight, waist circumference, and BMI. In addition, data from the following safety scales will be evaluated: C-SSRS and Study Medication Withdrawal Questionnaire (SMWQ).

Analyses of the double-blind treatment period safety data will be performed on the Safety Sample unless indicated otherwise.

The Safety Sample will also be analyzed for the single-blind placebo lead-in period safety data, as applicable, by treatment groups the subjects eventually being assigned in the double-blind treatment period.

#### 9.1 Adverse Events

All adverse events (AEs) will be coded by system organ class (SOC) and Medical Dictionary for Regulatory Activities (MedDRA) Preferred Term (PT). The incidence of the following events will be summarized:

- a) Treatment-emergent AEs (TEAEs)
- b) TEAEs by severity
- c) TEAEs potentially causally related to the IMP
- d) TEAEs with an outcome of death
- e) Serious TEAEs
- f) TEAEs leading to discontinuation of the IMP
- g) Treatment-emergent Adverse Events of Special Interest (AESI)
- h) Abuse-related TEAEs and TEAEs involving MHIs (Medication handling irregularities)

AEs will be classified by Primary SOC and PT according to the MedDRA. AEs that are gender-specific, e.g., ovarian cancer, will have their incidence rates evaluated for the specific gender.

Incidence of TEAEs will be summarized by double-blind treatment group for the double-blind treatment period. Incidence of TEAEs by SOC and MedDRA PT will be summarized for sex and race.

## Adverse Events of Special Interest

Newly acquired skin eruptions that are non-traumatic will be considered AESIs. These may include but are not limited to eruptions such as skin rashes, skin irritations, skin reactions, or acneiform lesions. This does not include localized contact irritation at ECG lead sites due to application or removal of lead adhesive.

Refer to the separate rash workup plan for complete details, including reporting forms, and extra measures that must be performed to characterize any skin AESI of a newly acquired skin eruption that is non-traumatic. The trial site will have a local designated dermatologist available for immediate consultation during the trial for these AESIs.

#### 9.1.1 Adverse Events in the Double-Blind Treatment Period

TEAEs in the double-blind treatment period are defined as AEs with an onset date on or after the start of double-blind treatment. In more detail, TEAEs are all adverse events which started after start of double-blind IMP; or if the event was continuous from end of the single-blind placebo run-in period and was worsening, serious, study drug related, or resulted in death, discontinuation, interruption or reduction of study therapy. Adverse Events occurring up to 30 days after the last day of double-blind dosing will be included in the summary tables. The incidence of AEs in the double-blind treatment period will be tabulated by treatment group and overall using the Safety Sample. Incidence of TEAE during the double-blind treatment period of at least 5% in either centanafadine group and also greater than placebo by SOC and MedDRA PT will be provided.

Unless otherwise specified, in general, analysis of safety data will be performed on observed case and for last visit.

### 9.1.2 Adverse Events in the Single-blind Placebo Run-in Period

Adverse Events in the single-blind placebo run-in period will be summarized for patients in the Safety Sample. AEs occurring up to 30 days after the last day of IMP in this period, but prior to the start of the double-blind treatment period, will be included in these summary tables. The incidence of adverse events in the single-blind placebo run-in period will be tabulated by the double-blind treatment patients receive in the double-blind treatment period.

#### 9.2 Clinical Laboratory Tests

Summary statistics for routine clinical laboratory measurements will be provided. For The double-blind treatment period laboratory tests, change from baseline for the double-blind

treatment period will be summarized by treatment group. Potentially clinically relevant results in laboratory tests will also be summarized.

## 9.2.1 Clinical Laboratory Tests in Double-Blind Treatment Period

Potentially clinically relevant laboratory measurement test results in the double-blind treatment period will be identified for the Safety Sample and will be summarized by treatment group and listed. Criteria for identifying laboratory values of potential clinical relevance are provided in Appendix 2.

## 9.2.2 Drug Induced Liver Injury (DILI)

Total bilirubin level should be checked for any subject with increased ALT or AST levels ≥ three times the upper normal limits (ULN) or baseline.

| Reporting a | ll DILI as S <i>i</i> | E to the FDA | based on Hy's Law: |
|-------------|-----------------------|--------------|--------------------|
|-------------|-----------------------|--------------|--------------------|

- $\square$  AST or ALT  $\geq$  3 x ULN or baseline and
- $\Box$  T\_Bili  $\geq 2 \times ULN$  or baseline

A separate incidence table will be provided for DILI cases, and the corresponding listing will be provided for Safety Sample during the double-blind treatment period and the single-blind placebo run-in period.

# 9.2.3 Clinical Laboratory Tests in the Single-blind Placebo Run-in Period

Potentially clinically relevant laboratory measurement test results in the Single-blind Placebo Run-in Period will be summarized for the Safety Sample by treatment group and overall as well as listed by subject and by laboratory test.

# 9.3 Vital Signs

Summary statistics for vital signs will be provided. For the double-blind treatment period vital signs, change from baseline for the double-blind treatment period will be summarized for the Safety Sample by treatment group. Potentially clinically relevant results in vital signs will also be summarized. Similar summaries will be provided for the Safety Sample during the Single-blind Placebo Run-in Period.

## 9.3.1 Vital Signs in the Double-Blind Treatment Period

Potentially clinically relevant vital signs measurements identified in the double-blind treatment period for the Safety Sample will be summarized by treatment group. Criteria for

identifying vital signs of potential clinical relevance are provided in Appendix 1. All potentially clinically relevant events or changes will be listed and included in summary tables.

## 9.3.2 Vital Signs in the Single-blind Placebo Run-in Period

Potentially clinically relevant vital signs measurements identified in the Single-blind Placebo Run-in Period for the Safety Sample will be summarized by treatment group.

## 9.4 Electrocardiogram (ECG) Data

Summary statistics and incidence of potentially clinically relevant changes will be provided for ECG parameters.

For the analysis of QT and QTc, data from three consecutive complexes (representing three consecutive heart beats) will be measured to determine average values. The following QT corrections will be used for reporting purposes in the clinical study report:

- 1) QTcB is the length of the QT interval corrected for heart rate by the Bazett formula: QTcB=QT/(RR)<sup>0.5</sup> and
- 2) QTcF is the length of the QT interval corrected for heart rate by the Fridericia formula:  $QTcF=QT/(RR)^{0.33}$
- 3) QTcN is the length of the QT interval corrected for heart rate by the FDA Neuropharm Division formula: QTcN=QT/(RR)<sup>0.37</sup>

#### 9.4.1 ECG Data in the Double-Blind Treatment Period

Potentially clinically relevant changes in the 12-lead ECG identified in the double-blind treatment period for the Safety Sample will be listed and summarized by treatment group. Criteria for identifying ECG measurements of potential clinical relevance are provided in Appendix 3.

Categorical changes in ECG parameters during the double-blind treatment period will be summarized based on the following criteria:

| Categorical Change Criteria in QT/QTc Parameters | | |
|---|---|---|
| Classification Category Criteria | | |
| QT | New Onset (> 450 Msec) | New onset (>450 msec) in QT means a subject who attains a value > 450 msec during treatment period but not at baseline. |
| QTc * | New Onset (> 450 Msec) | New onset (> 450 msec) in QTc means a subject who attains a value > 450 msec during treatment period but not at baseline. |

| Categorical Change Criteria in QT/QTc Parameters | | |
|---|---|---|
| Classification Category | | Criteria |
| | New Onset (> 450 Msec) | New onset (> 450 msec) and |
| | And > 10% Increase > 10% increase in QTc means a subject who | |
| | | a value > 450 msec and > 10% increase during |
| | | treatment period but not at baseline |
| | New Onset (> 500 Msec) New onset (> 500 msec) in QTc means a | |
| | | who attains a value > 500 msec during treatment |
| | | period but not at baseline. |
| | Increase 30 - 60 Msec Increase from baseline value $> 30$ and $\le 6$ | |
| | QTc | |
| | Increase > 60 Msec | Increase from baseline value > 60 msec in QTc |

<sup>\*</sup> QTc categorical change criteria apply to QTcB, QTcF and QTcN.

## 9.4.2 ECG Data in the Single-blind Placebo Run-in Period

Potentially clinically relevant changes in the 12-lead ECG identified in the Single-blind Placebo Run-in Period for the Safety Sample will be listed and summarized by treatment group.

## 9.5 Physical Examinations

By-patient listings will be provided for physical examination.

# 9.5.1 Body Weight, Waist Circumference and Body Mass Index (BMI)

Analyses of body weight, waist circumference and BMI will be performed for the Safety Sample. The mean change from baseline of the double-blind treatment period to Day 42 (OC) and last visit in the double-blind treatment period in body weight will be tabulated and analyzed using ANCOVA. The ANCOVA models for both the OC and last visit analyses will include the baseline of the double-blind treatment period body weight and the treatment group.

Percentages of patients showing significant weight gain (≥ 7 % increase in weight), as well as percentages of patients showing significant weight loss (≥ 7 % decrease in weight) baseline of the double-blind treatment period to Day 42 (OC and LOCF) will be analyzed using Cochran-Mantel-Haenszel (CMH) General Association Test.

Body mass index is defined as weight in kilograms divided by the square of height in meters.

# 9.6 Suicidality Data

Suicidality will be monitored during the study using the C-SSRS and will be summarized as number and percentage of subjects reporting any suicidal behavior, ideation, behavior by type (4 types), ideation by type (5 types) and treatment emergent suicidal behavior and ideation.

Summary will be provided for the single-blind placebo run-in period and the double-blind treatment period for the Safety Sample.

Suicidality is defined as report of at least one occurrence of any type of suicidal ideation or at least one occurrence of any type of suicidal behavior during assessment period (count each person only once).

Treatment emergent suicidal behavior and ideation is summarized by four types: Emergence of suicidal ideation, Emergence of serious suicidal ideation, Worsening of suicidal ideation, Emergence of suicidal behavior.

Emergence of suicidal behavior/ideation is defined as report of any type of suicidal behavior/ideation during treatment when there was no baseline suicidal behavior/ideation.

Emergence of serious suicidal ideation is defined as observation of suicidal ideation severity rating of 4 or 5 during treatment when there was no baseline suicidal ideation.

Worsening of suicidal ideation is defined as a suicidal ideation severity rating that is more severe than it was at baseline.

For the double-blind treatment period analyses, the last available measurement prior to the first dose of double-blind IMP is being used as "Baseline".

#### 9.7 **SMWQ**

Medication withdrawal symptoms assessed by SMWQ total scores at the scheduled visits during the double-blind treatment period and follow-up period will be summarized for the Safety Sample by treatment group and overall. The number of patients, mean, median, range and standard deviation will be presented.

# 9.8 Medication Handling Irregularities (MHIs) and Events Subject to Additional Monitoring (ESAMs)

MHIs and ESAMs will be summarized for the Safety Sample by treatment group and overall. By-patient listings will be provided.

## 9.9 Concomitant Medications

Number and proportion of patients taking concomitant medications prior to the single-blind placebo run-in period, during the single-blind placebo run-in period, during the double-blind treatment period, and after study therapy are tabulated by drug classification using the World Health Organization (WHO) drug dictionary. For the double-blind treatment period Randomized Sample, data will be presented by treatment group and overall.

## 9.10 Extent of Exposure

The start date of double-blind IMP - centanafadine or placebo - will be the first day of double-blind dosing. The number and percentage of subjects who receive double-blind IMP, will be presented by week and by treatment group. Each dosing week will be based on the actual week; i.e., Day 1-7 in Week 1, Day 8-14 in Week 2, etc. This summary will be performed on the Safety Sample.

The mean daily dosage will be summarized by week and treatment group using descriptive statistics. The mean daily dosage per subject per week will be determined for each week of the study. This will be calculated by dividing the sum of individual total doses by the number of days in the week interval. The summary will contain for each treatment group the number of patients receiving double-blind IMP, and the mean and range of the mean daily dose for each week.

## 10 Conventions

# 10.1 Study Visit Windows

Study visit windows will be used to map visits using study day intervals. This visit window convention applies to tables and listings for all efficacy and safety scales (AISRS, CGI-S, AIM-A, ASRS and CGI Change from Baseline). This derived study window variable will be named as DAY and will be footnoted. In listings it will be listed along with the eCRF study visit.

Table 10-1 shows classifications for study day intervals in the double-blind treatment period. The variable "target day" is defined using the number of days since the start of double-blind dosing in the double-blind treatment period. The first day of double-blind dosing is defined as "Day 1".

If more than one observation falls within a particular study day interval, then the last observation within that interval is used. Evaluations occurring more than three days after the last double-blind dosing date and evaluations occurring during the follow-up period will not be mapped into study visit windows and will be excluded from the double-blind treatment period analysis.

Table 10-1: Study Day and Visit Windows in the Double-Blind Treatment Period

| | Day | Target Day <sup>a</sup> | Study Day Interval <sup>a</sup> |
|-----|-----|-------------------------|---------------------------------|
| - 1 | | | |

SAP 405-201-00014

| 7 | 7 | 2-10 |
|----|----|---------|
| 14 | 14 | 11-17 |
| 21 | 21 | 18-24 |
| 28 | 28 | 25-31 |
| 35 | 35 | 32-38 |
| 42 | 42 | 39-49 b |

<sup>&</sup>lt;sup>a</sup> Relative to the first day of double-blind IMP in the double-blind treatment period.

## 10.2 Pooling of small centers

Primary efficacy analysis will be performed on the Efficacy Sample which comprises those subjects in the Randomized Sample who have a baseline value for the double-blind treatment period and at least one post-randomization value for AISRS total score in the double-blind treatment period. Small centers will be defined as centers that do not have at least one evaluable subject (evaluable with regard to the primary efficacy variable) in each treatment arm in the double-blind treatment period. All small centers will be pooled to form "pseudo centers" for the purpose of analysis according to the following algorithm. Small centers will be ordered from the largest to the smallest based on the number of evaluable subjects (i.e., subjects who have a baseline value for the double-blind treatment period value and at least one post-randomization value for AISRS total score in the double-blind treatment period). The process will start by pooling the largest of the small centers with the smallest of the small centers until a non-small center is formed. This process will be repeated using the centers left out of the previous pass. In case of ties in center size, the center with the smallest center code will be selected. If any centers are left out at the end of this process, they will be pooled with the smallest pseudo centers, or if no pseudo centers exist, they will be pooled with the smallest non-small center.

## 10.3 Scales: Rules for Scoring and Handling of Missing Data

# 10.3.1 Adult ADHD Investigator Symptom Rating Scale (AISRS)

The AISRS is utilized as the primary efficacy assessment of a subject's level of ADHD symptoms. It is a modified version of the ADHD Rating Scale that reflects the impact and severity of ADHD among adults and will be administered at each scheduled visit in the screening period, the single-blind placebo run-in period, the double-blind treatment period, and at 2 and 7 days after the last dose of IMP in the follow-up period. It is a clinician-administered scale that measures the 18 symptoms of adult ADHD using a Likert scale: 0

b Evaluations occurring more than three days after the last double-blind dosing date and evaluations occurring during the follow-up period will be excluded from the double-blind treatment period analyses.

(none); 1 (mild); 2 (moderate); and 3 (severe) and uses a semi-structured interview methodology with suggested prompts for each item to improve interrater reliability. The scale's 18 items directly correspond to the 18 DSM-5 symptoms of ADHD where 9 inattentive items alternate with 9 hyperactive impulsive items. The maximum total score for the scale is 54 points, with 27 points for each subscale. The total score is the sum of both the Inattentive and Hyperactive Impulsive subscales.

The AISRS inattentive subscale score and hyperactive-impulsive subscale score, as well as the AISRS total score is set to be missing if more than one item of a subscale is missing for inattentive subscale or hyperactive-impulsive subscale, separately. If one item is missing for a given subscale (inattentive or hyperactive-impulsive), then the subscale score is derived as the mean of scores from the 8 non-missing items multiplied by 9. All imputed scores are rounded to the first decimal place. The 9 inattentive items consist of the 9 odd numbered items and the 9 hyperactive impulsive items consist of the 9 even numbered items.

# 10.3.2 Clinical Global Impression Severity of Illness Scale – Modified for Attention-Deficit Hyperactivity Disorder

The CGI-S modified is an observer-rated scale that will be used to measure symptom severity. To perform this assessment, the investigator or rater will respond to the following question: "Considering your total clinical experience with adult ADHD, how mentally ill is the patient at this time?" Response choices include: 1 = normal, not at all ill; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; and 7 = among the most extremely ill patients. CGI-S is assessed at each scheduled visit in the double-blind treatment period.

# 10.3.3 Clinical Global Impression Change from Baseline

The CGI Change from Baseline is an observer-rated scale that will be used to measure the subject's total improvement compared to before trial drug treatment was initiated. The rater or investigator will rate the subject's total improvement relative to baseline. Response choices include: 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, and 7 = very much worse. CGI Change from Baseline is assessed at each scheduled visit in the double-blind treatment period except for the Day -1 visit.

# 10.3.4 Attention-Deficit Hyperactivity Disorder Impact Module – Adult (AIM-A)

The AIM-A is a subject self-report questionnaire which assesses quality of life in adults with ADHD. The questionnaire has 4 global quality of life items, 5 economic impact items, and

5 multi-item scales that assess the following key concepts: Living with ADHD, General Well-Being, Work, Home and School Performance and Daily Functioning. Additionally, Relationships and Communication, and Impact of Symptoms are also included.

## 10.3.5 Adult ADHD Self Report Scale (ASRS)

The ASRS is a self-report questionnaire developed by the WHO. The subject will answer 18 questions about the frequency of recent ADHD symptoms that are consistent with the DSM-IV criteria. The ASRS is assessed at the scheduled visits during the screening period, the single-blind placebo run-in period, and at Days -1, 28 and 42/ET during the double-blind treatment period.

The total score of (18 item) ADHD Symptoms score of the ASRS is set to be missing if more than one item of a subscale is missing for inattentive subscale or hyperactive-impulsive subscale, separately. If one item is missing for a given subscale (inattentive or hyperactive-impulsive), then the subscale score is derived as the mean of scores from the 8 non-missing items multiplied by 9. All imputed scores are rounded to the first decimal place. The 9 inattentive items consist of items 1-4 and 7-11 and the 9 hyperactive impulsive items consist of items 5-6 and 12-18.

## 10.3.6 Study Medication Withdrawal Questionnaire (SMWQ)

The SMWQ is a questionnaire to assess withdrawal symptoms. The SMWQ is a modification of the Amphetamine Withdrawal Questionnaire in which the terms "amphetamines and methamphetamine" are replaced with the term "the study medication." The SMWQ is assessed at Day 35 and Day 42/ET in the double-blind treatment period and at 1, 2, 3, 5, 7, and 10 days after the last dose of IMP in the follow-up period.

# 10.3.7 Columbia-Suicide Severity Rating Scale (C-SSRS)

Suicidality will be monitored during the trial using the C-SSRS. The C-SSRS is a semi-structured interview that captures the occurrence, severity, and frequency of suicide-related thoughts and behaviors during the assessment period. The interview includes definitions and suggested questions to solicit the type of information needed to determine if a suicide-related thought or behavior has occurred. The interview and rating for the C-SSRS must be completed by a licensed clinician who has been successfully trained to rate this scale by the sponsor or a designee and is medically responsible for the subject. Documentation of trial training should be maintained in the investigational site's files.

The C-SSRS has a "Screening/Baseline" version, which will be completed at screening and a "Since Last Visit" version that will be completed at all other visits (including the ET visit, if applicable). There are a maximum of 19 items to be completed: 7 required, 10 potential

additional items if there is a positive response to a required item, and 2 items for suicide/suicide behavior present during the interview. The C-SSRS uses dichotomous scales (i.e., yes or no), Likert scales, and text or narrative to further describe the thoughts or behaviors.

The C-SSRS is assessed at each scheduled visit in the screening period, the single-blind placebo run-in period, the double-blind treatment period, and at 2 and 7 days after the last dose of IMP in the follow-up period.

## 11 References

- Siddiqui O, Hung JHM, O'Neill R. MMRM vs. LOCF: A comprehensive comparison based on simulation study and 25 NDA datasets. J Biopharmaceutical Stats. 2009; 19(2):227-46.
- Diggle P, Kenward MG. Informative drop-out in longitudinal data analysis. Applied Statistics. 1994; 43:49-93.
- Little RJA. Pattern-mixture models for multivariate incomplete data. J Am Stat Assoc. 1993; 88:125-34.
- Little RJA. Modeling the drop-out mechanism in repeated measures studies. J Am Stat Assoc. 1995; 90:1112-21.
- Hedeker D, Gibbons RD. Application of random effects pattern-mixture models for missing data in longitudinal studies. Psychological Methods. 1997; 2:64-78.
- Ali MW, Siddiqui O. Multiple imputation compared with some information dropout procedures in the estimation and comparison of rates of change in longitudinal clinical trials with dropouts. J Biopharmaceutical Stats. 2000;10(2):165-81.
- Wu MC, Bailey KR. Estimation and comparison of changes in the presence of informative right censoring: Conditional linear model. Biometrics. 1989; 45:939-55.
- van Elteren, PH. On the combination of independent two sample tests of Wilcoxon. Bull Int Stat Inst. 1960; 37:351-61.
- Mehrotra D, Li X, Liu J, Lu K. Analysis of Longitudinal Clinical Trials with Missing Data Using Multiple Imputation in Conjunction with Robust Regression. Biometrics 2012; 68:1250-1259.
- Cortina, J. M., & Nouri, H. (2000). Effect size for ANOVA designs. Thousand Oaks, Calif.: Sage Publications.
- https://www.whitehouse.gov/presidential-actions/proclamation-declaring-national-emergency-concerning-novel-coronavirus-disease-covid-19-outbreak/

## 12 Potential Clinical Relevance Criteria from Protocol

# Appendix 1 Criteria for Identifying Vital Signs of Potential Clinical Relevance

| Variable | Criterion Value <sup>a</sup> | Change Relative to Baseline <sup>a</sup> |
|---|---|---|
| Heart Rate <sup>b</sup> | > 100 bpm<br>< 50 bpm | ≥ 10 bpm increase<br>≥ 10 bpm decrease |
| Systolic Blood Pressure <sup>b</sup> | ≥ 140 mmHg<br>< 90 mmHg | ≥ 20 mmHg increase<br>≥ 20 mmHg decrease |
| Diastolic Blood Pressure <sup>b</sup> | $\geq$ 90 mmHg < 60 mmHg | ≥ 10 mmHg increase<br>≥ 10 mmHg decrease |
| Orthostatic Hypotension | ≥ 30 mmHg decrease in systolic blood<br>pressure or a ≥ 20 mmHg<br>in diastolic blood pressure after at least<br>3 minutes of standing compared to the<br>previous supine blood pressure. | Not Applicable (baseline status not considered) |
| Orthostatic Tachycardia | ≥ 25 bpm increase in heart rate from supine to standing | Not Applicable (baseline status not considered) |
| Weight | - | ≥ 7% increase<br>≥ 7% decrease |

<sup>&</sup>lt;sup>a</sup> In order to be identified as potentially clinically relevant, an on-treatment value must meet the "Criterion Value" and also represent a change from the subject's baseline value of at least the magnitude shown in the "Change Relative to Baseline" column.

<sup>&</sup>lt;sup>b</sup> As defined in "Supplementary Suggestions for Preparing an Integrated Summary of Safety Information in an Original NDA Submission and for Organizing Information in Periodic Safety Updates," FDA Division of Neuropharmacological Drug Products draft (2/27/87).

# Appendix 2 Criteria for Identifying Laboratory Values of Potential Clinical Relevance

| Laboratory Tests | Criteria |
|---|---|
| Chemistry | |
| AST (SGOT) | $\geq$ 3 x upper limit of normal (ULN) |
| ALT (SGPT) | $\geq 3 \times ULN$ |
| Alkaline phosphatase | $\geq 3 \times ULN$ |
| BUN | $\geq 30 \text{ mg/dL}$ |
| Creatinine | $\geq 2.0 \text{ mg/dL}$ |
| Uric Acid | |
| Men | $\geq 10.5 \text{ mg/dL}$ |
| Women | $\geq 8.5 \text{ mg/dL}$ |
| Bilirubin (total) | $\geq 2.0 \text{ mg/dL}$ |
| Creatine Phosphokinase (CPK) | > 3 x ULN |
| Hematology | |
| Hematocrit | |
| Men | $\leq$ 37 % and decrease of $\geq$ 3 percentage points from Baseline |
| Women | $\leq$ 32 % and decrease of $\geq$ 3 percentage points from Baseline |
| Hemoglobin | |
| Men | $\leq 11.5 \text{ g/dL}$ |
| Women | $\leq 9.5 \text{ g/dL}$ |
| White blood count | $\leq 2,800/ \text{ mm}^3 \text{ or } \geq 16,000/ \text{ mm}^3$ |
| Eosinophils | ≥ 10% |
| Neutrophils | ≤ 15% |
| Absolute neutrophil count | $\leq 1,500/\mathrm{mm}^3$ |
| Platelet count | $\leq$ 75,000/ mm <sup>3</sup> or $\geq$ 700,000/ mm <sup>3</sup> |
| Urinalysis | |
| Protein | Increase of $\geq 2$ units |
| Glucose | Increase of $\geq 2$ units |
| Additional Criteria | |
| Chloride | $\leq$ 90 mEq/L or $\geq$ 118 mEq/L |
| Potassium | $\leq 2.5 \text{ mEq/L or} \geq 6.5 \text{ mEq/L}$ |
| Sodium | $\leq 126 \text{ mEq/L or} \geq 156 \text{ mEq/L}$ |
| Calcium | $\leq 8.2 \text{ mg/dL or} \geq 12 \text{ mg/dL}$ |
| Glucose | |
| Fasting | $\geq 100 \text{ mg/dL}$ |
| Non-Fasting | $\geq$ 200 mg/dL |
| Total Cholesterol, Fasting | $\geq$ 240 mg/dL |
| LDL Cholesterol, Fasting | $\geq 160 \text{ mg/dL}$ |
| HDL Cholesterol, Fasting | |
| Men | < 40 mg/dL |
| Women | < 50 mg/dL |
| Triglycerides, Fasting | ≥ 150 mg/dL |
## Appendix 3 Relevance

## Criteria for Identifying ECG Measurements of Potential Clinical

| Variable | Criterion Value <sup>a</sup> | Change Relative to Baseline <sup>a</sup> |
|---|---|---|
| Rate | | |
| Tachycardia | ≥ 120 bpm | increase of $\geq 15$ bpm |
| Bradycardia | ≤ 50 bpm | decrease of $\geq 15$ bpm |
| Rhythm | | |
| Sinus tachycardia <sup>b</sup> | ≥ 120 bpm | increase of ≥ 15 bpm |
| Sinus bradycardia <sup>c</sup> | ≤ 50 bpm | decrease of ≥ 15 bpm |
| Supraventricular premature beat | all | not present → present |
| Ventricular premature beat | all | not present → present |
| Supraventricular tachycardia | all | not present → present |
| Ventricular tachycardia | all | not present $\rightarrow$ present |
| Atrial fibrillation | all | not present $\rightarrow$ present |
| Atrial flutter | all | not present $\rightarrow$ present |
| Conduction | | |
| 1° atrioventricular block | $PR \ge 200 \text{ msec}$ | increase of $\geq 50$ msec |
| 2° atrioventricular block | all | not present → present |
| 3° atrioventricular block | all | not present $\rightarrow$ present |
| Left bundle-branch block | all | not present $\rightarrow$ present |
| Right bundle-branch block | all | not present $\rightarrow$ present |
| Pre-excitation syndrome | all | not present $\rightarrow$ present |
| Other intraventricular conduction block <sup>d</sup> | QRS $\geq$ 120 msec | increase of $\geq 20$ msec |
| Infarction | | |
| Acute or subacute | all | not present $\rightarrow$ present |
| Old | all | not present $\rightarrow$ present |
| CENTER A LA LA | | ≥ 12 weeks post study entry |
| ST/T Morphological | | |
| Myocardial Ischemia | all | not present → present |
| Symmetrical T-wave inversion | all | not present $\rightarrow$ present |
| Increase in QTc | QTcF > 450 msec (men) | |
| | QTcF > 470 msec | |
| | (women) | |

<sup>&</sup>lt;sup>a</sup> In order to be identified as potentially clinically relevant, an on-treatment value must meet the "Criterion Value" and also represent a change from the subject's baseline value of at least the magnitude shown in the "Change Relative to Baseline" column.

<sup>&</sup>lt;sup>b</sup> No current diagnosis of supraventricular tachycardia, ventricular tachycardia, atrial fibrillation, atrial flutter, or other rhythm abnormality.

<sup>&</sup>lt;sup>c</sup> No current diagnosis of atrial fibrillation, atrial flutter, or other rhythm abnormality.

<sup>&</sup>lt;sup>d</sup> No current diagnosis of left bundle branch block or right bundle branch block.

## 13 Proposed List of Summary Tables

- CT-1.1 Subject Disposition
- CT-1.2 Subject Disposition by Center
- CT-1.3 Subject Completion Rates by Week During the Double-Blind Treatment Period (Randomized Sample)
- CT-1.4.1 Subject Enrollment by Country (Randomized Sample)
- CT-1.4.2 Subject Enrollment by Country by Age Group (Randomized Sample)
- CT-2 Reasons for Discontinuation in the Double-Blind Treatment Period (Randomized Sample)
- CT-3.1 Demographic Characteristics (Randomized Sample)
- CT-3.2.1 Medical History (Randomized Sample)
- CT-3.2.2 Psychiatric History (Randomized Sample)
- CT-3.2.3 Summary of Adult ADHD Clinical Diagnostic Scale (ACDS) (Randomized Sample)
- CT-3.3 MINI International Neuropsychiatric Interview (M.I.N.I.) (Randomized Sample)
- CT-3.4.1 Baseline Psychiatric Scale Evaluations for the Single-Blind Placebo Run-in Period (Randomized Sample)
- CT-3.4.2 Baseline Psychiatric Scale Evaluations for the Double-Blind Treatment Period (Randomized Sample)
- CT-4.1 Concomitant Medications: Medications Taken Prior to Start of Double-Blind Treatment (Safety Sample)
- CT-4.2 Concomitant Medications: Medications Taken During the Double-Blind Treatment Period (Safety Sample)
- CT-4.3 Concomitant Medications: Medications Taken Post Study Period (Safety Sample)
- CT-5.1 Summary of Efficacy Results at Day 42 in the Double-Blind Treatment Period (Efficacy Sample)
- CT-5.2.1.1 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in Adult ADHD Investigator Symptom Rating Scale (AISRS) Total Score MMRM, UN (Efficacy Sample)
- CT-5.2.1.2 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in Adult ADHD Investigator Symptom Rating Scale (AISRS) Total Score MMRM, UN (Per Protocol Sample)
- CT-5.2.1.3 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in Adult ADHD Investigator Symptom Rating Scale (AISRS) Total Score MMRM, UN (Pre-COVID Efficacy Sample)
- CT-5.2.1.4 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in Adult ADHD Investigator Symptom Rating Scale (AISRS) Total Score MMRM, UN Pre-COVID Data Set (Efficacy Sample)
- CT-5.2.1.5 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in Adult ADHD Investigator Symptom Rating Scale (AISRS) Total Score MMRM, UN (Non-COVID Efficacy Sample)
- CT-5.2.1.6 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in Adult ADHD Investigator Symptom Rating Scale (AISRS) Total Score MMRM, UN Non-COVID Data Set (Efficacy Sample)
- CT-5.2.1.7 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in Adult ADHD Investigator Symptom Rating Scale (AISRS) Total Score MMRM, UN Excluding Remote Assessments (Efficacy Sample)
- CT-5.2.2 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in Adult ADHD Investigator Symptom Rating Scale (AISRS) Total Score MMRM, TOEPH Empirical (Efficacy Sample)
- CT-5.2.3 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in Adult ADHD Investigator Symptom Rating Scale (AISRS) Total Score MMRM, ARH1 Empirical (Efficacy Sample)

- CT-5.2.4 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in Adult ADHD Investigator Symptom Rating Scale (AISRS) Total Score MMRM, CSH Empirical (Efficacy Sample)
- CT-5.2.5 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in Adult ADHD Investigator Symptom Rating Scale (AISRS) Total Score -MMRM, DDFM=SATTERTHWAITE (Efficacy Sample)
- CT-5.2.6.1 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in Adult ADHD Investigator Symptom Rating Scale (AISRS) Total Score LOCF (Efficacy Sample)
- CT-5.2.6.2 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in Adult ADHD Investigator Symptom Rating Scale (AISRS) Total Score OC (Efficacy Sample)
- CT-5.2.7 Summary of Mean Change from Baseline to End of the Single-Blind Run-in Period by Study Day in Adult ADHD Investigator Symptom Rating Scale (AISRS) Total Score OC (Efficacy Sample)
- CT-5.2.8 Summary of Mean Change from Baseline to End of the Follow-up Period by Study Day in Adult ADHD Investigator Symptom Rating Scale (AISRS) Total Score OC (Efficacy Sample)
- CT-5.3.1 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in AISRS Inattentive Subscale MMRM, UN (Efficacy Sample)
- CT-5.3.2 Summary of Mean Change Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in AISRS Inattentive Subscale LOCF (Efficacy Sample)
- CT-5.3.3 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day AISRS Inattentive Subscale OC (Efficacy Sample)
- CT-5.3.4 Summary of Mean Change from Baseline to End of Single-Blind Placebo Run-in Period in AISRS Inattentive Subscale OC (Efficacy Sample)
- CT-5.3.5 Summary of Mean Change from Baseline to End of the Follow-up Period in AISRS Inattentive Subscale OC (Efficacy Sample)
- CT-5.3.6 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in AISRS Hyperactive-Impulsive Subscale MMRM, UN (Efficacy Sample)
- CT-5.3.7 Summary of Mean Change Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in AISRS Hyperactive-Impulsive Subscale LOCF (Efficacy Sample)
- CT-5.3.8 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day AISRS Hyperactive-Impulsive Subscale OC (Efficacy Sample)
- CT-5.3.9 Summary of Mean Change from Baseline to End of Single-Blind Placebo Run-in Period in AISRS Hyperactive-Impulsive Subscale OC (Efficacy Sample)
- CT-5.3.10 Summary of Mean Change from Baseline to End of the Follow-up Period in AISRS Hyperactive-Impulsive Subscale - OC (Efficacy Sample)
- CT-5.4.1 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in Clinical Global Impression Severity of Illness Modified for ADHD (CGI-S) Scale MMRM, UN (Efficacy Sample)
- CT-5.4.2 Summary of Mean Change Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in Clinical Global Impression - Severity of Illness Modified for ADHD (CGI-S) Scale - LOCF (Efficacy Sample)
- CT-5.4.3 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in Clinical Global Impression Severity of Illness Modified for ADHD (CGI-S) Scale OC (Efficacy Sample)
- CT-5.5.1 Summary of Mean Clinical Global Impression Change from Baseline Scale by Study Day in the Double-Blind Treatment Period LOCF (Efficacy Sample)

- CT-5.5.2 Summary of Mean Clinical Global Impression Improvement Change from Baseline Scale by Study Day in the Double-Blind Treatment Period OC (Efficacy Sample)
- CT-5.6.1 Summary of Proportion of Responders to Treatment During the Double-Blind Treatment Period Relative to the End of the Single-Blind Run-in Period LOCF (Efficacy Sample)
- CT-5.6.2 Summary of Proportion of Responders to Treatment During the Double-Blind Treatment Period Relative to the End of the Single-Blind Run-in Period OC (Efficacy Sample)
- CT-5.6.3 Summary of Proportion of Subjects with an Adult ADHD Investigator Symptom Rating Scale (AISRS) Total Score or a CGI Change from Baseline Response During the Double-Blind Treatment Period LOCF (Efficacy Sample)
- CT-5.6.4 Summary of Proportion of Subjects with an Adult ADHD Investigator Symptom Rating Scale (AISRS) Total Score or a CGI Change from Baseline Response During the Double-Blind Treatment Period OC (Efficacy Sample)
- CT-5.6.5 Summary of Proportion of Subjects with an Adult ADHD Investigator Symptom Rating Scale (AISRS) Total Score Remission During the Double-Blind Treatment Period LOCF (Efficacy Sample)
- CT-5.6.6 Summary of Proportion of Subjects with an Adult ADHD Investigator Symptom Rating Scale (AISRS) Total Score Remission During the Double-Blind Treatment Period OC (Efficacy Sample)
- CT-5.7.1 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in Attention-Deficit Hyperactivity Disorder Impact Module Adult (AIM-A) Scale MMRM, UN (Efficacy Sample)
- CT-5.7.2 Summary of Mean Change Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in Attention-Deficit Hyperactivity Disorder Impact Module Adult (AIM-A) Scale LOCF (Efficacy Sample)
- CT-5.7.3 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in Attention-Deficit Hyperactivity Disorder Impact Module Adult (AIM-A) Scale OC (Efficacy Sample)
- CT-5.7.4 Summary of Mean Change from Baseline to End of Single-Blind Placebo Run-in Period in Attention-Deficit Hyperactivity Disorder Impact Module - Adult (AIM-A) Scale - OC (Efficacy Sample)
- CT-5.7.5 Summary of Proportion of Subjects in Each Category During the Single-Blind Run-in Period and Double-Blind Treatment Period by Study Day in Attention-Deficit Hyperactivity Disorder Impact Module Adult (AIM-A) Scale OC (Efficacy Sample)
- CT-5.8.1 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in Adult ADHD Self Report Scale (ASRS) Scale MMRM, UN (Efficacy Sample)
- CT-5.8.2 Summary of Mean Change Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in Adult ADHD Self Report Scale (ASRS) Scale LOCF (Efficacy Sample)
- CT-5.8.3 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in Adult ADHD Self Report Scale (ASRS) Scale OC (Efficacy Sample)
- CT-5.8.4 Summary of Mean Change from Baseline to End of Single-Blind Placebo Run-in Period in Adult ADHD Self Report Scale (ASRS) Scale OC (Efficacy Sample)
- CT-5.9.1 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in ASRS Inattentive Subscale MMRM, UN (Efficacy Sample)
- CT-5.9.2 Summary of Mean Change Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in ASRS Inattentive Subscale LOCF (Efficacy Sample)
- CT-5.9.3 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in ASRS Inattentive Subscale OC (Efficacy Sample)
- CT-5.9.4 Summary of Mean Change from Baseline to End of Single-Blind Placebo Run-in Period in ASRS Inattentive Subscale OC (Efficacy Sample)
- CT-5.9.5 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in ASRS Hyperactive-Impulsive Subscale MMRM, UN (Efficacy Sample)

- CT-5.9.6 Summary of Mean Change Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in ASRS Hyperactive-Impulsive Subscale LOCF (Efficacy Sample)
- CT-5.9.7 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in ASRS Hyperactive-Impulsive Subscale OC (Efficacy Sample)
- CT-5.9.8 Summary of Mean Change from Baseline to End of Single-Blind Placebo Run-in Period in ASRS Hyperactive-Impulsive Subscale OC (Efficacy Sample)
- CT-5.10.1 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in Adult ADHD Investigator Symptom Rating Scale (AISRS) Total Score MI, VAN ELTEREN TEST (Efficacy Sample)
- CT-5.10.2 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in Adult ADHD Investigator Symptom Rating Scale (AISRS) Total Score GEE (Efficacy Sample)
- CT-5.10.3 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in Adult ADHD Investigator Symptom Rating Scale (AISRS) Total Score WGEE (Efficacy Sample)
- CT-5.11.1 Sensitivity Analysis of MNAR using Pattern Mixture Model with Multiple Imputation (Delta Method 1) in AISRS Total Score Assume All Dropouts as MNAR (Efficacy Sample)
- CT-5.11.2 Sensitivity Analysis of MNAR using Pattern Mixture Model with Multiple Imputation (Delta Method 2) in AISRS Total Score Assume All Dropouts as MNAR (Efficacy Sample)
- CT-5.11.3 Sensitivity Analysis of MNAR using Pattern Mixture Model with Multiple Imputation (Delta Method 1) in AISRS Total Score Dropout due to AE or LOE or Withdrew Consent as MNAR (Efficacy Sample)
- CT-5.11.4 Sensitivity Analysis of MNAR using Pattern Mixture Model with Multiple Imputation (Delta Method 2) in AISRS Total Score Dropout due to AE or LOE or Withdrew Consent as MNAR (Efficacy Sample)
- CT-5.11.5 Sensitivity Analysis of MNAR using Pattern Mixture Model with Multiple Imputation (Delta Method 1) in AISRS Total Score Dropouts due to AE or Lack of Efficacy (LOE) as MNAR (Efficacy Sample)
- CT-5.11.6 Sensitivity Analysis of MNAR using Pattern Mixture Model with Multiple Imputation (Delta Method 2) in AISRS Total Score Dropouts due to AE or Lack of Efficacy (LOE) as MNAR (Efficacy Sample)
- CT-5.11.7 Sensitivity Analysis of MNAR using Placebo Based Imputation in AISRS Total Score (Efficacy Sample)
- CT-5.11.8 Sensitivity Analysis of MNAR using Pattern Mixture Model with Multiple Imputation (Delta Method 1) in CGI-S Score Assume All Dropouts as MNAR (Efficacy Sample)
- CT-5.11.9 Sensitivity Analysis of MNAR using Pattern Mixture Model with Multiple Imputation (Delta Method 2) in CGI-S Score Assume All Dropouts as MNAR (Efficacy Sample)
- CT-5.11.10 Sensitivity Analysis of MNAR using Pattern Mixture Model with Multiple Imputation (Delta Method 1) in CGI-S Score Dropout due to AE or LOE or Withdrew Consent as MNAR (Efficacy Sample)
- CT-5.11.11 Sensitivity Analysis of MNAR using Pattern Mixture Model with Multiple Imputation (Delta Method 2) in CGI-S Score Dropout due to AE or LOE or Withdrew Consent as MNAR (Efficacy Sample)
- CT-5.11.12 Sensitivity Analysis of MNAR using Pattern Mixture Model with Multiple Imputation (Delta Method 1) in SDS Mean Score Dropouts due to AE or Lack of Efficacy (LOE) as MNAR (Efficacy Sample)
- CT-5.11.13 Sensitivity Analysis of MNAR using Pattern Mixture Model with Multiple Imputation (Delta Method 2) in CGI-S Score Dropouts due to AE or Lack of Efficacy (LOE) as MNAR (Efficacy Sample)
- CT-5.11.14 Sensitivity Analysis of MNAR using Placebo Based Imputation in CGI-S Score (Efficacy Sample)
- CT-5.11.15 Sensitivity Analysis of MNAR Using Model Based Methods: Shared Parameter Model and Random Coefficient Pattern Mixture Model –OC (Efficacy Sample)
- CT-6.1.1 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in Adult ADHD Investigator Symptom Rating Scale (AISRS)Total Score in the Subgroup of Females MMRM (Efficacy Sample)
- CT-6.1.2 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in Adult ADHD Investigator Symptom Rating Scale (AISRS) Total Score in the Subgroup of Males MMRM (Efficacy Sample)

- CT-6.2.1 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in Adult ADHD Investigator Symptom Rating Scale (AISRS) Total Score in the Subgroup of Whites MMRM (Efficacy Sample)
- CT-6.2.2 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in Adult ADHD Investigator Symptom Rating Scale (AISRS) Total Score in the Subgroup of All Other Races MMRM (Efficacy Sample)
- CT-7.1 Extent of Exposure to Study Medication During the Double-Blind Treatment Period (Safety Sample)
- CT-7.2 Number and Percentage of Subjects Receiving Study Medication and Mean and Range of Average Daily Dose in the Double-Blind Treatment Period (Safety Sample)
- CT-8.1.1 Adverse Events During the Double-Blind Treatment Period (All Causalities) (Safety Sample)
- CT-8.1.2 Adverse Events During the Single-Blind Placebo Run-in Period (All Causalities) (Safety Sample)
- CT-8.2.1.1 Incidence of TEAEs During the Double-Blind Treatment Period by System Organ Class and MedDRA Preferred Term (Safety Sample)
- CT-8.2.1.2 Incidence of TEAEs During the Double-Blind Treatment Period by System Organ Class, MedDRA Preferred Term and Severity (Safety Sample)
- CT-8.2.1.3 Incidence of TEAE During the Double-Blind Treatment Period of at Least 5% in Any Centanafadine Group and Greater Than Placebo by System Organ Class and MedDRA Preferred Term (Safety Sample)
- CT-8.2.1.4 Incidence of TEAEs During the Double-Blind Treatment Period by System Organ Class and MedDRA Preferred Term, by Sex (Safety Sample)
- CT-8.2.1.5 Incidence of TEAEs During the Double-Blind Treatment Period by System Organ Class and MedDRA Preferred Term, by Race (Safety Sample)
- CT-8.2.1.6 Incidence of Non-Serious TEAEs During the Double-Blind Treatment Period of at Least 5% in Any Centanafadine Group and Greater Than Placebo by System Organ Class and MedDRA Preferred Term (Safety Sample)
- CT-8.2.1.7 Incidence of TEAE During the Double-Blind Treatment Period of at Least 2% in Any Centanafadine Group and Greater Than Placebo by System Organ Class and MedDRA Preferred Term (Safety Sample)
- CT-8.2.1.8 Incidence and Occurrence (Number of Events) of Serious TEAEs by System Organ Class and MedDRA Preferred Term (Safety Sample)
- CT-8.2.1.9 Incidence and Occurrence (Number of Events) of Potentially Drug-Related Serious TEAEs by System Organ Class and MedDRA Preferred Term (Safety Sample)
- CT-8.2.1.10 Incidence and Occurrence (Number of Events) of Non-Serious TEAEs by System Organ Class and MedDRA Preferred Term (Safety Sample)
- CT-8.2.2 Incidence of AEs During the Single-Blind Placebo Run-in Period by System Organ Class and MedDRA Preferred Term (Safety Sample)
- CT-8.3.1 Incidence of Potentially Drug-Related TEAEs During the Double-Blind Treatment Period by System Organ Class and MedDRA Preferred Term (Safety Sample)
- CT-8.3.2 Incidence of Potentially Drug-Related TEAEs During the Double-Blind Treatment Period by System Organ Class, MedDRA Preferred Term and Severity (Safety Sample)
- CT-8.4.1.1 Incidence of Deaths Due to TEAEs During the Double-Blind Treatment Period by System Organ Class and MedDRA Preferred Term (Safety Sample)
- CT-8.4.1.2 Incidence of Deaths Due to TEAEs During the Double-Blind Treatment Period by System Organ Class and MedDRA Preferred Term and Severity (Safety Sample)
- CT-8.4.2 Incidence of Deaths Due to AEs During the Single-Blind Placebo Run-in Period by System Organ Class and MedDRA Preferred Term (Safety Sample)
- CT-8.5.1.1 Incidence of Serious TEAEs During the Double-Blind Treatment Period by System Organ Class and MedDRA Preferred Term (Safety Sample)
- CT-8.5.1.2 Incidence of Serious TEAEs During the Double-Blind Treatment Period by System Organ Class, MedDRA Preferred Term and Severity (Safety Sample)

- SAP 405-201-00014
- CT-8.5.2.1 Incidence of Serious AEs During the Single-Blind Placebo Run-in Period by System Organ Class and MedDRA Preferred Term (Safety Sample)
- CT-8.6.1 Incidence of TEAEs Resulting in Discontinuation of Study Medication During the Double-Blind Treatment Period by System Organ Class and MedDRA Preferred Term (Safety Sample)
- CT-8.6.2 Incidence of TEAEs Resulting in Discontinuation of Study Medication During the Double-Blind Treatment Period by System Organ Class, MedDRA Preferred Term and Severity (Safety Sample)
- CT-8.7.1 Incidence of Treatment-Emergent Adverse Events of Special Interests (AESIs) During the Double-Blind Treatment Period by System Organ Class and MedDRA Preferred Term (Safety Sample)
- CT-8.7.2 Incidence of Treatment-Emergent Adverse Events of Special Interests (AESIs) During the Double-Blind Treatment Period by System Organ Class and MedDRA Preferred Term and Severity (Safety Sample)
- CT-8.7.3 Listing of Treatment-Emergent Adverse Events of Special Interests (AESIs) During the Double-Blind Treatment Period (Safety Sample)
- CT-8.8.1 Incidence of Treatment-Emergent Abuse Potential-Related Adverse Events During the Double-Blind Treatment Period by System Organ Class and MedDRA Preferred Term (Safety Sample)
- CT-8.8.2 Incidence of Treatment-Emergent Abuse Potential-Related Adverse Events During the Double-Blind Treatment Period by System Organ Class and MedDRA Preferred Term and Severity (Safety Sample)
- CT-8.8.3 Listing of Treatment-Emergent Abuse Potential-Related Adverse Events During the Double-Blind Treatment Period (Safety Sample)
- CT-9.1.1 Listing of Deaths During the Double-Blind Treatment Period
- CT-9.1.2 Listing of Deaths During the Single-Blind Placebo Run-in Period
- CT-9.2.1 Listing of Serious Adverse Events During the Double-Blind Treatment Period
- CT-9.2.2 Listing of Serious Adverse Events During the Single-Blind Placebo Run-in Period
- CT-9.3 Listing of Discontinuations of Study Medication Due to Adverse Events During the Double-Blind Treatment Period
- CT-9.4 Listing of Adverse Events for Subjects Discontinued from Study Due to Adverse Events During the Double-Blind Treatment Period
- CT-10.1 Criteria for Laboratory Test Values with Potential Clinical Relevance
- CT-10.2.1.1 Listing of Laboratory Test Values with Potential Clinical Relevance During the Double-Blind Treatment Period by Subject (Safety Sample)
- CT-10.2.1.2 Listing of Laboratory Test Values with Potential Clinical Relevance During the Double-Blind Treatment Period by Test (Safety Sample)
- CT-10.2.2 Incidence of Laboratory Test Values with Potential Clinical Relevance During the Double-Blind Treatment Period (Safety Sample)
- CT-10.2.3.1 Mean Change from Baseline of the Double-Blind Treatment Period in Clinical Laboratory Test Results - Serum Chemistry (Safety Sample)
- CT-10.2.3.2 Mean Change from Baseline of the Double-Blind Treatment Period in Clinical Laboratory Test Results Hematology (Safety Sample)
- CT-10.2.3.3 Mean Change from Baseline of the Double-Blind Treatment Period in Clinical Laboratory Test Results Urinalysis (Safety Sample)
- CT-10.3.1.1 Listing of Laboratory Test Values with Potential Clinical Relevance During the Single-Blind Placebo Run-in Period by Subject (Safety Sample)
- CT-10.3.1.2 Listing of Laboratory Test Values with Potential Clinical Relevance During the Single-Blind Placebo Run-in Period by Test (Safety Sample)
- CT-10.3.2 Incidence of Laboratory Test Values with Potential Clinical Relevance During the Single-Blind Placebo Run-in Period (Safety Sample)
- CT-10.3.3.1 Mean Change from Baseline of the Single-Blind Placebo Run-in Period in Clinical Laboratory Test Results During the Single-Blind Placebo Run-in Period Serum Chemistry (Safety Sample)
- CT-10.3.3.2 Mean Change from Baseline of the Single-Blind Placebo Run-in Period in Clinical Laboratory Test Results During the Single-Blind Placebo Run-in Period Hematology (Safety Sample)

- CT-10.3.3.3 Mean Change from Baseline of the Single-Blind Placebo Run-in Period in Clinical Laboratory Test Results During the Single-Blind Placebo Run-in Period Urinalysis (Safety Sample)
- CT-10.4.1 Incidence of Potentially Liver Injury Related Laboratory Test Abnormalities During the Double-Blind Treatment Period (Safety Sample)
- CT-10.4.2 Incidence of Potentially Liver Injury Related Laboratory Test Abnormalities During the Single-Blind Placebo Run-in Period (Safety Sample)
- CT-10.5.1 Listing of Potentially Liver Injury Related Laboratory Test Abnormalities During the Double-Blind Treatment Period (Safety Sample)
- CT-10.5.2 Listing of Potentially Liver Injury Related Laboratory Test Abnormalities During the Single-Blind Placebo Run-in Period (Safety Sample)
- CT-11.1 Criteria for Potentially Clinically Relevant Abnormalities in Vital Signs
- CT-11.2.1 Listing of Potentially Clinically Relevant Abnormalities in Vital Signs During the Double-Blind Treatment Period (Safety Sample)
- CT-11.2.2 Incidence of Potentially Clinically Relevant Abnormalities in Vital Signs During the Double-Blind Treatment Period (Safety Sample)
- CT-11.2.3 Mean Change from Baseline of the Double-Blind Treatment Period in Vital Signs During the Double-Blind Treatment Period (Safety Sample)
- CT-11.3.1 Listing of Potentially Clinically Relevant Abnormalities in Vital Signs During the Single-Blind Placebo Run-in Period (Safety Sample)
- CT-11.3.2 Incidence of Potentially Clinically Relevant Abnormalities in Vital Signs During the Single-Blind Placebo Run-in Period (Safety Sample)
- CT-11.3.3 Mean Change from Baseline of the Single-Blind Placebo Run-in Period in Vital Signs During the Single-Blind Placebo Run-in Period (Safety Sample)
- CT-12.1 Criteria for Potentially Clinically Relevant Abnormalities in ECG Evaluations
- CT-12.2.1 Listing of Potentially Clinically Relevant Abnormalities in ECG Evaluations During the Double-Blind Treatment Period (Safety Sample)
- CT-12.2.2 Incidence of Potentially Clinically Relevant Changes in ECG Evaluations During the Double-Blind Treatment Period (Safety Sample)
- CT-12.2.3 Mean Change from Baseline of the Double-Blind Treatment Period in Electrocardiogram Results During the Double-Blind Treatment Period (Safety Sample)
- CT-12.3.1 Listing of Categorical Changes in QT/QTc During the Double-Blind Treatment Period (Safety Sample)
- CT-12.3.2 Incidence of Categorical Changes in QT/QTc During the Double-Blind Treatment Period (Safety Sample)
- CT-12.4.1 Listing of Potentially Clinically Relevant Abnormalities in ECG Evaluations During the Single-Blind Placebo Run-in Period (Safety Sample)
- CT-12.4.2 Incidence of Potentially Clinically Relevant Changes in ECG Evaluations During the Single-Blind Placebo Run-in Period (Safety Sample)
- CT-12.4.3 Mean Change from Baseline of the Single-Blind Placebo Run-in Period in Electrocardiogram Results During the Single-Blind Placebo Run-in Period (Safety Sample)
- CT-12.5.1 Listing of Categorical Changes in QT/QTc During the Single-Blind Placebo Run-in Period (Safety Sample)
- CT-12.5.2 Incidence of Categorical Changes in QT/QTc During the Single-Blind Placebo Run-in Period (Safety Sample)
- CT-13.1.1 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in Body Weight (kg) (Safety Sample)

- CT-13.1.2 Summary of Proportion of Patients with Potentially Clinically Relevant Weight Gain or Weight Loss During the Double-Blind Treatment Period (Safety Sample)
- CT-13.2 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in Waist Circumference (cm) (Safety Sample)
- CT-13.3 Summary of Mean Change from Baseline of the Double-Blind Treatment Period to the Double-Blind Treatment Period by Study Day in BMI (kg/m2) (Safety Sample)
- CT-14.1.1 Columbia-Suicide Severity Rating Scale(C-SSRS) During the Double-Blind Treatment Period, Suicidality (Safety Sample)
- CT-14.1.2 Columbia-Suicide Severity Rating Scale(C-SSRS) During the Double-Blind Treatment Period, Suicidal Behavior by Type (Safety Sample)
- CT-14.1.3 Columbia-Suicide Severity Rating Scale(C-SSRS) During the Double-Blind Treatment Period, Suicidal Ideation by Type (Safety Sample)
- CT-14.1.4 Columbia-Suicide Severity Rating Scale(C-SSRS) During the Double-Blind Treatment Period, Treatment Emergent Suicidal Behavior and Ideation (Safety Sample)
- CT-14.1.5 Columbia-Suicide Severity Rating Scale (C-SSRS) Listing of Treatment Emergent Suicidal Ideation During the Double-Blind Treatment Period (Safety Sample)
- CT-14.1.6 Columbia-Suicide Severity Rating Scale (C-SSRS) Listing of Treatment Emergent Suicidal Behavior During the Double-Blind Treatment Period (Safety Sample)
- CT-14.1.7 Columbia-Suicide Severity Rating Scale (C-SSRS) Listing of Treatment Emergent Serious Suicidal Ideation During the Double-Blind Treatment Period (Safety Sample)
- CT-14.1.8 Columbia-Suicide Severity Rating Scale (C-SSRS) Listing of Worsening Suicidal Ideation During the Double-Blind Treatment Period (Safety Sample)
- CT-14.2.1 Columbia-Suicide Severity Rating Scale (C-SSRS) During the Single-Blind Placebo Run-in Period, Suicidality (Safety Sample)
- CT-14.2.2 Columbia-Suicide Severity Rating Scale (C-SSRS) During the Single-Blind Placebo Run-in Period, Suicidal Behavior by Type (Safety Sample)
- CT-14.2.3 Columbia-Suicide Severity Rating Scale (C-SSRS) During the Single-Blind Placebo Run-in Period, Suicidal Ideation by Type (Safety Sample)
- CT-14.2.4 Columbia-Suicide Severity Rating Scale (C-SSRS) During the Single-Blind Placebo Run-in Period, Treatment Emergent Suicidal Behavior and Ideation (Safety Sample)
- CT-14.2.5 Columbia-Suicide Severity Rating Scale (C-SSRS) Listing of Treatment Emergent Suicidal Ideation During the Single-Blind Placebo Run-in Period (Safety Sample)
- CT-14.2.6 Columbia-Suicide Severity Rating Scale (C-SSRS) Listing of Treatment Emergent Suicidal Behavior During the Single-Blind Placebo Run-in Period (Safety Sample)
- CT-14.2.7 Columbia-Suicide Severity Rating Scale (C-SSRS) Listing of Treatment Emergent Serious Suicidal Ideation During the Single-Blind Placebo Run-in Period (Safety Sample)
- CT-14.2.8 Columbia-Suicide Severity Rating Scale (C-SSRS) Listing of Worsening Suicidal Ideation During the Single-Blind Placebo Run-in Period (Safety Sample)
- CT-15 Summary of Mean Study Medication Withdrawal Questionnaire (SMWQ) Total Score During the Double-Blind Treatment Period and Follow-up Period by Study Day (Safety Sample)
- CT-16 Summary of Medication Handling Irregularity (Safety Sample)
- CT-17.1 Summary of ESAMs Reported as Abuse Potential AEs During the Double-Blind Treatment Period by System Organ Class and MedDRA Preferred Term (Safety Sample)
- CT-17.2 Summary of Non-Adverse Events Reported as Findings (ESAM) During the Double-Blind Treatment Period (Safety Sample)
- CT-17.3 Summary of ESAMs Reported as Abuse Potential AEs During the Single-Blind Placebo Run-in Period by System Organ Class and MedDRA Preferred Term (Safety Sample)
- CT-17.4 Summary of Non-Adverse Events Reported as Findings (ESAM) During the Single-Blind Placebo Run-in Period (Safety Sample)

This Page has been intentionally left blank.



### This page is a manifestation of an electronically captured signature

### SIGNATURE PAGE

Document Name: 405-201-00014\_Statistical\_Analysis\_Plan

Document Number: 1000047007

**Document Version: 8.0** 

| Signed by | Meaning of Signature | Server Date (dd-MMM- yyyyy hh:min) - UTC timezone |
|---|---|---|
| | Clinical Approval | 26-May-2020<br>18:40:37 |
| | Biostatistics Approval | 26-May-2020<br>19:20:14 |

CENTANAFADINE 1 OF 5
PROTOCOL 405-201-00014

 $\begin{array}{c} {\rm STAT-1.1} \\ {\rm Adjusted~Mean~Change~from~Baseline~in~AISRS~Line~Items~at~Day~42~-~MMRM} \\ {\rm (Efficacy~Sample)} \end{array}$ 

| AISRS<br>Line Items | | IN SR<br>MEAN<br>Base | 200MG<br>LSMean<br>Change <sup>1</sup> | C'<br>N | TN SR<br>MEAN<br>Base | 400MG<br>LSMean<br>Change <sup>1</sup> | N | PLAC<br>MEAN<br>Base | LSMean | TREATMENT<br>COMPARISON | ESTIMATED<br>TREATMENT<br>EFFECT <sup>1</sup> | P-VALUE <sup>1</sup> | COHEN'S D<br>EFFECT<br>SIZE |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| MAKE CARELESS MISTAKES | 140 | 2.15 | -0.75 | 140 | 2.19 | -0.72 | 141 | 2.18 | -0.44 | EB-1020 200mg VS<br>PLACEBO | -0.32 | 0.0059 | -0.33 |
| | | | | | | | | | | EB-1020 400mg VS<br>PLACEBO | -0.29 | 0.0149 | -0.29 |
| FIDGET OR SQUIRM WITH<br>YOUR HANDS OR FEET | 140 | 2.21 | -0.50 | 140 | 2.28 | -0.51 | 141 | 2.18 | -0.50 | EB-1020 200mg VS<br>PLACEBO | -0.00 | 0.9973 | -0.00 |
| | | | | | | | | | | EB-1020 400mg VS<br>PLACEBO | -0.01 | 0.9113 | -0.01 |
| DIFFICULTY KEEPING<br>YOUR ATTENTION | 140 | 2.57 | -0.78 | 140 | 2.54 | -0.73 | 141 | 2.54 | -0.49 | EB-1020 200mg VS<br>PLACEBO | -0.29 | 0.0113 | -0.30 |
| | | | | | | | | | | EB-1020 400mg VS<br>PLACEBO | -0.24 | 0.0450 | -0.24 |
| LEAVE YOUR SEAT | 140 | 1.72 | -0.59 | 140 | 1.78 | -0.65 | 141 | 1.64 | -0.50 | EB-1020 200mg VS<br>PLACEBO | -0.09 | 0.4319 | -0.09 |
| | | | | | | | | | | EB-1020 400mg VS<br>PLACEBO | -0.15 | 0.1936 | -0.16 |
| DIFFICULTY<br>CONCENTRATING ON | 140 | 2.29 | -0.80 | 140 | 2.30 | -0.75 | 141 | 2.29 | -0.50 | EB-1020 200mg VS<br>PLACEBO | -0.30 | 0.0104 | -0.31 |

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, (POOLED) STUDY CENTER, VISIT, TREATMENT BY VISIT AND BASELINE BY VISIT INTERACTIO

CENTANAFADINE 2 OF 5

 ${\tt STAT-1.1} \\ {\tt Adjusted Mean Change from Baseline in AISRS Line Items at Day 42 - MMRM} \\ ({\tt Efficacy Sample})$ 

CTN SR 200MG CTN SR 400MG PLACEBO ESTIMATED COHEN'S AISRS MEAN LSMean MEAN LSMean MEAN LSMean TREATMENT TREATMENT EFFECT SIZE COMPARISON FOR TREATMENT SIZE COMPARISON OF TREATMENT SIZE COMPA COHEN's D EFFECT EB-1020 400mg VS DIFFICULTY -0.25 0.0356 -0.25 CONCENTRATING ON PLACEBO FEEL RESTLESS OR 140 1.93 -0.44 140 2.15 -0.62 141 2.06 -0.41 EB-1020 200mg VS -0.04 0.7284 -0.04 FIDGETY EB-1020 400mg VS -0.22 0.0486 -0.24 PLACEBO TROUBLE WRAPPING UP 140 2.40 -0.67 140 2.44 -0.73 141 2.55 -0.47 EB-1020 200mg VS -0.20 0.0649 -0.22 THE FINAL DETAILS PLACEBO EB-1020 400mg VS -0.26 0.0202 -0.28 PLACEBO -0.09 0.4355 DIFFICULTY UNWINDING 140 1.87 -0.44 140 1.91 -0.41 141 1.80 -0.34 EB-1020 200mg VS -0.09 AND RELAXING PLACEBO -0.06 0.5941 EB-1020 400mg VS -0.06 PLACEBO EB-1020 200mg VS DIFFICULTY GETTING 140 2.36 -0.74 140 2.54 -0.84 141 2.53 -0.62 -0.13 0.2832 -0.13 THINGS IN ORDER PLACEBO EB-1020 400mg VS -0.22 0.0627 -0.22 PLACEBO

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, (POOLED) STUDY CENTER, VISIT, TREATMENT BY VISIT AND BASELINE BY VISIT INTERACTIO

CENTANAFADINE 3 OF 5

 $$\tt STAT-1.1$$  Adjusted Mean Change from Baseline in AISRS Line Items at Day 42 - MMRM (Efficacy Sample)

| AISRS<br>Line Items | | TN SR<br>MEAN<br>Base | 200MG<br>LSMean<br>Change <sup>1</sup> | | TN SR<br>MEAN<br>Base | 400MG<br>LSMean<br>Change¹ | N | PLAC<br>MEAN<br>Base | LSMean | TREATMENT<br>COMPARISON | ESTIMATED<br>TREATMENT<br>EFFECT <sup>1</sup> | P-VALUE <sup>1</sup> | COHEN'S D<br>EFFECT<br>SIZE |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| OVERLY ACTIVE AND COMPELLED TO DO THINGS | 140 | 1.79 | -0.49 | 140 | 1.92 | -0.61 | 141 | 1.75 | -0.46 | EB-1020 200mg VS<br>PLACEBO | -0.02 | 0.8394 | -0.02 |
| | | | | | | | | | | EB-1020 400mg VS<br>PLACEBO | -0.14 | 0.2203 | -0.15 |
| AVOID OR DELAY<br>GETTING STARTED | 140 | 2.51 | -0.67 | 140 | 2.52 | -0.59 | 141 | 2.50 | -0.44 | EB-1020 200mg VS<br>PLACEBO | -0.23 | 0.0473 | -0.24 |
| | | | | | | | | | | EB-1020 400mg VS<br>PLACEBO | -0.15 | 0.2113 | -0.15 |
| TALKING TOO MUCH | 140 | 1.71 | -0.61 | 140 | 1.85 | -0.68 | 141 | 1.71 | -0.47 | EB-1020 200mg VS<br>PLACEBO | -0.14 | 0.1981 | -0.15 |
| | | | | | | | | | | EB-1020 400mg VS<br>PLACEBO | -0.21 | 0.0668 | -0.22 |
| MISPLACE OR HAVE<br>DIFFICULTY FINDING | 140 | 2.20 | -0.77 | 140 | 2.21 | -0.78 | 141 | 2.12 | -0.41 | EB-1020 200mg VS<br>PLACEBO | -0.35 | 0.0022 | -0.37 |
| | | | | | | | | | | EB-1020 400mg VS<br>PLACEBO | -0.37 | 0.0017 | -0.38 |
| FINISHING THE<br>SENTENCES OF THE<br>PEOPLE | 140 | 1.90 | -0.84 | 140 | 1.92 | -0.77 | 141 | 1.80 | -0.42 | EB-1020 200mg VS<br>PLACEBO | -0.42 | 0.0002 | -0.45 |

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, (POOLED) STUDY CENTER, VISIT, TREATMENT BY VISIT AND BASELINE BY VISIT INTERACTIO

CENTANAFADINE

4 OF 5

 ${\tt STAT-1.1} \\ {\tt Adjusted Mean Change from Baseline in AISRS Line Items at Day 42 - MMRM} \\ ({\tt Efficacy Sample})$ 

CTN SR 200MG CTN SR 400MG PLACEBO ESTIMATED COHEN'S AISRS MEAN LSMean MEAN LSMean MEAN LSMean TREATMENT TREATMENT EFFECT SIZE COMPARISON FOR TREATMENT SIZE COMPARISON OF TREATMENT SIZE COMPA COHEN's D EFFECT FINISHING THE EB-1020 400mg VS -0.35 0.0025 -0.36 SENTENCES OF THE PLACEBO PEOPLE BEING DISTRACTED BY 140 2.39 -0.75 140 2.47 -0.60 141 2.53 -0.35 EB-1020 200mg VS -0.41 0.0001 -0.46 ACTIVITY OR NOISE PLACEBO -0.25 EB-1020 400mg VS 0.0191 -0.28 PLACEBO 140 1.87 -0.74 140 1.91 -0.77 141 1.79 -0.48 -0.26 DIFFICULTY WAITING EB-1020 200mg VS 0.0176 -0.28 YOUR TURN PLACEBO EB-1020 400mg VS -0.29 0.0100 -0.31 PLACEBO PROBLEMS REMEMBERING 140 2.01 -0.81 140 2.11 -0.67 141 2.11 -0.44 EB-1020 200mg VS -0.37 0.0026 -0.36 PLACEBO EB-1020 400mg VS -0.23 0.0648 -0.22 PLACEBO INTERRUPT OTHERS WHEN 140 1.71 -0.71 140 1.73 -0.82 141 1.57 -0.43 EB-1020 200mg VS -0.29 0.0068 -0.32 THEY ARE BUSY PLACEBO EB-1020 400mg VS -0.39 0.0004 -0.43 PLACEBO

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, (POOLED) STUDY CENTER, VISIT, TREATMENT BY VISIT AND BASELINE BY VISIT INTERACTIO

CENTANAFADINE 5 OF 5 PROTOCOL 405-201-00014

# $$\tt STAT-1.1$$ Adjusted Mean Change from Baseline in AISRS Line Items at Day 42 - MMRM (Efficacy Sample)

| AISRS<br>Line Items | CTN SR 200MG<br>MEAN LSMean<br>N Base Change <sup>1</sup> | CTN SR 400MG<br>MEAN LSMean<br>N Base Change <sup>1</sup> | PLACEBO<br>MEAN LSMean<br>N Base Change <sup>1</sup> | TREATMENT<br>COMPARISON | ESTIMATED<br>TREATMENT<br>EFFECT <sup>1</sup> P-VALU | COHEN'S D<br>EFFECT<br>E¹ SIZE |
|---|---|---|---|---|---|---|
| AISRS TOTAL SCORE (DERIVED) | 140 37.59 -12.1 | 140 38.76 -12.5 | 141 37.65 -8.07 | EB-1020 200mg VS<br>PLACEBO<br>EB-1020 400mg VS | -4.01 0.002<br>-4.42 0.000 | |

<sup>&</sup>lt;sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, (POOLED) STUDY CENTER, VISIT, TREATMENT BY VISIT AND BASELINE BY VISIT INTERACTIO

CENTANAFADINE 1 OF 5

## $\begin{array}{c} {\rm STAT-1.2} \\ {\rm Adjusted~Mean~Change~from~Baseline~in~ASRS~Line~Items~at~Day~42~-MMRM} \\ {\rm (Efficacy~Sample)} \end{array}$

CTN SR 200MG CTN SR 400MG PLACEBO ESTIMATED COHEN'S
ASRS MEAN LSMean MEAN LSMean MEAN LSMean TREATMENT TREATMENT FOR SIZE
Line Items N Base Change¹ N Base Change¹ N Base Change¹ COMPARISON EFFECT¹ P-VALUE¹ SIZE COHEN's D EFFECT EB-1020 200mg VS ASRS-TROUBLE TO WRAP 124 2.85 -0.67 114 2.73 -0.57 130 2.95 -0.29 -0.38 0.0015 -0.40 DETAILS OF PROJECT PLACEBO -0.29 0.0213 EB-1020 400mg VS -0.30 PLACEBO ASRS-DIFFICULTY 124 2.81 -0.72 114 2.90 -0.62 130 3.00 -0.30 EB-1020 200mg VS -0.42 0.0008 -0.43 GETTING THINGS IN PLACEBO ORDER EB-1020 400mg VS -0.33 0.0100 -0.33 PLACEBO ASRS-PROBLEM 124 2.56 -0.82 114 2.67 -0.70 130 2.72 -0.42 EB-1020 200mg VS -0.40 0.0022 -0.39 REMEMBERING APPTS/OBLIGATNS EB-1020 400mg VS -0.28 0.0330 -0.27 PLACEBO 0.0685 ASRS-AVOID/DELAY 124 3.06 -0.63 114 3.22 -0.72 130 3.19 -0.40 EB-1020 200mg VS -0.22 -0.23 GETTNG STARTD ON PLACEBO THGHTS EB-1020 400mg VS -0.32 0.0128 -0.32 PLACEBO

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, (POOLED) STUDY CENTER, VISIT, TREATMENT BY VISIT AND BASELINE BY VISIT INTERACTIO

CENTANAFADINE 2 OF 5

 $\begin{array}{c} {\rm STAT-1.2} \\ {\rm Adjusted\ Mean\ Change\ from\ Baseline\ in\ ASRS\ Line\ Items\ at\ Day\ 42\ -\ MMRM} \\ {\rm (Efficacy\ Sample)} \end{array}$ 

CTN SR 200MG CTN SR 400MG PLACEBO ESTIMATED COHEN'S
ASRS MEAN LSMean MEAN LSMean MEAN LSMean TREATMENT TREATMENT FOR SIZE
Line Items N Base Change¹ N Base Change¹ N Base Change¹ COMPARISON EFFECT¹ P-VALUE¹ SIZE COHEN's D EFFECT ASRS-FIDGET/SQUIRM 124 3.01 -0.59 114 2.99 -0.56 130 3.00 -0.47 EB-1020 200mg VS -0.12 0.3314 -0.12 WITH HANDS/FEET PLACEBO EB-1020 400mg VS -0.09 0.4849 -0.09 PLACEBO ASRS-FEEL OVERLY 124 2.56 -0.52 114 2.56 -0.56 130 2.55 -0.46 EB-1020 200mg VS -0.07 0.6162 -0.06 ACTIVE TO DO THINGS PLACEBO -0.10 EB-1020 400mg VS 0.4410 -0.10 PLACEBO EB-1020 200mg VS 124 2.69 -0.73 114 2.76 -0.79 130 2.81 -0.40 -0.33 0.0104 ASRS-MAKE CARELESS -0.32 MISTAKES PLACEBO EB-1020 400mg VS -0.39 0.0034 -0.38 PLACEBO 124 3.18 -0.84 114 3.28 -0.75 130 3.38 -0.37 -0.46 0.0004 ASRS-DIFFICULTY EB-1020 200mg VS -0.45 KEEPING ATTENTION PLACEBO EB-1020 400mg VS -0.38 0.0042 -0.37 PLACEBO ASRS-DIFFICULTY 124 2.76 -0.81 114 2.89 -0.79 130 2.96 -0.30 EB-1020 200mg VS -0.50 0.0000 -0.52 KEEPING CONCENTRATION PLACEBO

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, (POOLED) STUDY CENTER, VISIT, TREATMENT BY VISIT AND BASELINE BY VISIT INTERACTIO

CENTANAFADINE 3 OF 5 PROTOCOL 405-201-00014

 $$\tt STAT-1.2$$  Adjusted Mean Change from Baseline in ASRS Line Items at Day 42 - MMRM (Efficacy Sample)

| | C | IN SR | | | | 400MG | | PLAC | | | ESTIMATED | | COHEN's D |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| ASRS Line Items | N | | LSMean<br>Change <sup>1</sup> | | MEAN<br>Base | LSMean<br>Change <sup>1</sup> | N | | LSMean<br>Change <sup>1</sup> | TREATMENT<br>COMPARISON | TREATMENT<br>EFFECT <sup>1</sup> | P-VALUE <sup>1</sup> | EFFECT<br>SIZE |
| ASRS-DIFFICULTY KEEPING CONCENTRATION | | | | | | | | | | EB-1020 400mg VS<br>PLACEBO | -0.49 | 0.0001 | -0.50 |
| ASRS-MISPLACE/DIFFICUL<br>TY FINDING THINGS | 124 | 2.74 | -0.83 | 114 | 3.00 | -0.85 | 130 | 2.90 | -0.40 | EB-1020 200mg VS<br>PLACEBO | -0.42 | 0.0009 | -0.42 |
| | | | | | | | | | | EB-1020 400mg VS<br>PLACEBO | -0.44 | 0.0007 | -0.44 |
| ASRS-DISTRACTED BY<br>ACTIVITY OR NOISE | 124 | 3.10 | -0.73 | 114 | 3.09 | -0.61 | 130 | 3.15 | -0.27 | EB-1020 200mg VS<br>PLACEBO | -0.47 | 0.0001 | -0.48 |
| | | | | | | | | | | EB-1020 400mg VS<br>PLACEBO | -0.35 | 0.0061 | -0.35 |
| ASRS-LEAVE SEAT IN<br>MEETNGS/ORDR SITUATNS | 124 | 1.95 | -0.59 | 114 | 2.10 | -0.76 | 130 | 1.90 | -0.32 | EB-1020 200mg VS<br>PLACEBO | -0.26 | 0.0347 | -0.27 |
| | | | | | | | | | | EB-1020 400mg VS<br>PLACEBO | -0.44 | 0.0008 | -0.44 |
| ASRS-FEELING RESTLESS<br>OR FIDGETY | 124 | 2.92 | -0.65 | 114 | 2.89 | -0.70 | 130 | 2.89 | -0.46 | EB-1020 200mg VS<br>PLACEBO | -0.19 | 0.1224 | -0.19 |
| | | | | | | | | | | EB-1020 400mg VS<br>PLACEBO | -0.24 | 0.0623 | -0.24 |

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, (POOLED) STUDY CENTER, VISIT, TREATMENT BY VISIT AND BASELINE BY VISIT INTERACTIO

CENTANAFADINE

4 OF 5

 $\begin{array}{c} {\rm STAT-1.2} \\ {\rm Adjusted\ Mean\ Change\ from\ Baseline\ in\ ASRS\ Line\ Items\ at\ Day\ 42\ -\ MMRM} \\ {\rm (Efficacy\ Sample)} \end{array}$ 

CTN SR 200MG CTN SR 400MG PLACEBO ESTIMATED COHEN'S
ASRS MEAN LSMean MEAN LSMean MEAN LSMean TREATMENT TREATMENT FOR SIZE
Line Items N Base Change¹ N Base Change¹ N Base Change¹ COMPARISON EFFECT¹ P-VALUE¹ SIZE COHEN's D EFFECT ASRS-DIFF UNWINDING 124 2.56 -0.57 114 2.61 -0.61 130 2.64 -0.42 EB-1020 200mg VS -0.15 0.2810 -0.14 AND RELAXING PLACEBO -0.19 0.1729 EB-1020 400mg VS -0.18 PLACEBO ASRS-FIND YOURSELF 124 2.52 -0.75 114 2.61 -0.70 130 2.58 -0.45 EB-1020 200mg VS -0.31 0.0119 -0.32 TALKING TOO MUCH PLACEBO EB-1020 400mg VS -0.26 0.0408 -0.26 PLACEBO EB-1020 200mg VS ASRS-FINISH SENTENCES 124 2.62 -0.87 114 2.65 -0.86 130 2.68 -0.54 -0.33 0.0103 -0.32 OF PEOPLE PLACEBO EB-1020 400mg VS -0.32 0.0165 -0.31 PLACEBO ASRS-DIFFCULTY 124 2.30 -0.72 114 2.55 -0.74 130 2.42 -0.45 -0.26 0.0433 EB-1020 200mg VS -0.25 WAITING YOUR TURN PLACEBO EB-1020 400mg VS -0.28 0.0355 -0.27 PLACEBO ASRS-INTERRUPT OTHERS 124 2.21 -0.67 114 2.33 -0.83 130 2.47 -0.54 EB-1020 200mg VS -0.13 0.2921 -0.13 WHEN THEY ARE BUSY PLACEBO

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, (POOLED) STUDY CENTER, VISIT, TREATMENT BY VISIT AND BASELINE BY VISIT INTERACTIO


# $\begin{array}{c} {\rm STAT-1.2} \\ {\rm Adjusted~Mean~Change~from~Baseline~in~ASRS~Line~Items~at~Day~42~-MMRM} \\ {\rm (Efficacy~Sample)} \end{array}$

------

| ASRS<br>Line Items | CTN SR 200MG<br>MEAN LSMean<br>N Base Change | CTN SR 400MG<br>MEAN LSMean<br>N Base Change <sup>1</sup> | PLACEBO<br>MEAN LSMean<br>N Base Change <sup>1</sup> | TREATMENT<br>COMPARISON | ESTIMATED<br>TREATMENT<br>EFFECT <sup>1</sup> P | COHEN'S D<br>EFFECT<br>-VALUE¹ SIZE |
|---|---|---|---|---|---|---|
| ASRS-INTERRUPT OTHERS<br>WHEN THEY ARE BUSY | | | | EB-1020 400mg VS<br>PLACEBO | -0.28 | 0.0211 -0.30 |
| ASRS TOTAL SCORE OF<br>18 ITEMS (DERIVED) | 124 48.39 -12.2 | 114 49.83 -12.6 | 130 50.21 -7.28 | EB-1020 200mg VS<br>PLACEBO | | 0.0016 -0.40 |
| | | | | EB-1020 400mg VS<br>PLACEBO | -5.33 | 0.0009 -0.43 |

<sup>1</sup> MIXED MODEL REPEATED MEASURES METHOD WITH MODEL TERMS: TREATMENT, (POOLED) STUDY CENTER, VISIT, TREATMENT BY VISIT AND BASELINE BY VISIT INTERACTIO

CENTANAFADINE 1 OF 28 PROTOCOL 405-201-00014

STAT-3.1 MMRM Output for Test on Treatment by Sex Interaction at Day 42 (Efficacy Sample)

The Mixed Procedure

Model Information

WORK.INDATA Data Set Dependent Variable CHG Dependent Variable Covariance Structure Unstructured Subject Effect SUBJID Estimation Method REML Residual Variance Method Fixed Effects SE Method Kenward-Roger

Degrees of Freedom Method Kenward-Roger

Class Level Information

Class Levels Values 6 7 14 21 28 35 42 AVISITN TRTPN 3 POOLCNTR 39

CENTANAFADINE 2 OF 28 PROTOCOL 405-201-00014

 $$\tt STAT-3.1$$  MMRM Output for Test on Treatment by Sex Interaction at Day 42 (Efficacy Sample)

The Mixed Procedure

Class Level Information

Class Levels Values

SUBJID 421



CENTANAFADINE


 $$\tt STAT-3.1$$  MMRM Output for Test on Treatment by Sex Interaction at Day 42 (Efficacy Sample)

\_\_\_\_\_

The Mixed Procedure



CENTANAFADINE 4 OF 28 PROTOCOL 405-201-00014

 $$\tt STAT-3.1$$  MMRM Output for Test on Treatment by Sex Interaction at Day 42 (Efficacy Sample)

\_\_\_\_\_

The Mixed Procedure



CENTANAFADINE 5 OF 28 PROTOCOL 405-201-00014

 $$\tt STAT-3.1$$  MMRM Output for Test on Treatment by Sex Interaction at Day 42 (Efficacy Sample)

The Mixed Procedure



CENTANAFADINE


 $$\tt STAT-3.1$$  MMRM Output for Test on Treatment by Sex Interaction at Day 42 (Efficacy Sample)

The Mixed Procedure



CENTANAFADINE 7 OF 28 PROTOCOL 405-201-00014

 $$\tt STAT-3.1$$  MMRM Output for Test on Treatment by Sex Interaction at Day 42 (Efficacy Sample)

The Mixed Procedure



FILE: stat2a.lis, RUN: 31AUG2020 08:32; ANALYSIS DATASET CREATED: 16JUN2020 08:14

PROGRAM: /opt/sas/Data/DAP/EB1020/P40520100014/STAT/Program.dev/DOC\_STAT/stat2.sas

OPDC, NEW DRUG APPLICATION, IND # 119,361 CENTANAFADINE STAT-3.1 FINAL

SEX

CENTANAFADINE

STAT-3.1

MMRM Output for Test on Treatment by Sex Interaction at Day 42 (Efficacy Sample)

The Mixed Procedure

Dimensions

Covariance Parameters 21
Columns in X 129
Columns in Z 0
Subjects 421
Max Obs per Subject 6

Number of Observations

Number of Observations Read 2227
Number of Observations Used 2227
Number of Observations Not Used 0

Iteration History

 Iteration
 Evaluations
 -2 Res Log Like
 Criterion

 0
 1
 15728.87827870
 0.00033945

 1
 2
 13520.41397294
 0.00033945

 2
 1
 13518.67561888
 0.00000469

 3
 1
 13518.65293347
 0.00000000

CENTANAFADINE 9 OF 28 PROTOCOL 405-201-00014

 $$\tt STAT-3.1$$  MMRM Output for Test on Treatment by Sex Interaction at Day 42 (Efficacy Sample)

The Mixed Procedure

Convergence criteria met.

Covariance Parameter Estimates

| Cov Parm | Subject | Estimate |
|----------|---------|----------|
| UN(1,1) | SUBJID | 43.3236 |
| UN(2,1) | SUBJID | 38.2897 |
| UN(2,2) | SUBJID | 70.3806 |
| UN(3,1) | SUBJID | 37.4535 |
| UN(3,2) | SUBJID | 60.2826 |
| UN(3,3) | SUBJID | 81.6833 |
| UN(4,1) | SUBJID | 38.9483 |
| UN(4,2) | SUBJID | 59.0458 |
| UN(4,3) | SUBJID | 73.8743 |
| UN(4,4) | SUBJID | 89.8024 |
| UN(5,1) | SUBJID | 38.5482 |
| UN(5,2) | SUBJID | 60.6062 |
| UN(5,3) | SUBJID | 72.6270 |
| UN(5,4) | SUBJID | 82.3083 |
| UN(5,5) | SUBJID | 97.7229 |
| UN(6,1) | SUBJID | 37.9468 |
| UN(6,2) | SUBJID | 60.5956 |
| UN(6,3) | SUBJID | 74.6496 |

CENTANAFADINE 10 OF 28 PROTOCOL 405-201-00014

STAT-3.1

MMRM Output for Test on Treatment by Sex Interaction at Day 42  $$({\tt Efficacy\ Sample})$$ 

The Mixed Procedure

Covariance Parameter Estimates

| Cov Parm | Subject | Estimate |
|----------|---------|----------|
| UN(6,4) | SUBJID | 84.5321 |
| UN(6,5) | SUBJID | 91.9940 |
| UN(6,6) | SUBJID | 109.35 |

### Fit Statistics

| -2 Res Log Likelihood | 13518.7 |
|--------------------------|---------|
| AIC (Smaller is Better) | 13560.7 |
| AICC (Smaller is Better) | 13561.1 |
| RTC (Smaller is Retter) | 13645 5 |

### Null Model Likelihood Ratio Test

| DF | Chi-Square | Pr > ChiSo |
|----|------------|------------|
| 20 | 2210 23 | < 000 |

CENTANAFADINE 11 OF 28 PROTOCOL 405-201-00014

# $$\tt STAT-3.1$$ MMRM Output for Test on Treatment by Sex Interaction at Day 42 (Efficacy Sample)

The Mixed Procedure

#### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|-------------------|-----------|-----------|---------|--------|
| POOLCNTR | 38 | 377 | 2.08 | 0.0003 |
| AVISITN | 5 | 348 | 1.04 | 0.3931 |
| TRTPN | 2 | 375 | 10.16 | <.0001 |
| AVISITN*TRTPN | 10 | 518 | 1.60 | 0.1019 |
| SEX | 1 | 389 | 0.50 | 0.4820 |
| AVISITN*SEX | 5 | 346 | 1.55 | 0.1739 |
| TRTPN*SEX | 2 | 391 | 1.17 | 0.3101 |
| AVISITN*TRTPN*SEX | 10 | 518 | 0.43 | 0.9331 |
| BASE*AVISITN | 6 | 376 | 1.86 | 0.0859 |

Coefficients for 1 vs. 3 BY SEX AT DAY 42

Pooled Analysis Planned
Center Visit Treatment
Effect Number Sex (N) (N) Row1

Intercept POOLCNTR POOLCNTR



CENTANAFADINE 12 OF 28 PROTOCOL 405-201-00014

 $$\tt STAT-3.1$$  MMRM Output for Test on Treatment by Sex Interaction at Day 42 (Efficacy Sample)

The Mixed Procedure

Coefficients for 1 vs. 3 BY SEX AT DAY 42

| Effect | Pooled<br>Center<br>Number | Sex | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|
| POOLCNTR | | | | | |

CENTANAFADINE 13 OF 28 PROTOCOL 405-201-00014

 $$\tt STAT-3.1$$  MMRM Output for Test on Treatment by Sex Interaction at Day 42 (Efficacy Sample)

The Mixed Procedure

Coefficients for 1 vs. 3 BY SEX AT DAY 42

| | Pooled<br>Center | | Analysis<br>Visit | Planned<br>Treatment | |
|---|---|---|---|---|---|
| Effect | Number | Sex | (N) | (N) | Row1 |
| POOLCNTR | | | | | |
| POOLCNTR | | | _ | | |
| AVISITN | | | 7 | | |

CENTANAFADINE 14 OF 28 PROTOCOL 405-201-00014

# $$\tt STAT-3.1$$ MMRM Output for Test on Treatment by Sex Interaction at Day 42 (Efficacy Sample)

### The Mixed Procedure

### Coefficients for 1 vs. 3 BY SEX AT DAY 42

| | Pooled | | Analysis | Planned | |
|---------------|--------|-----|----------|-----------|------|
| | Center | | Visit | Treatment | |
| Effect | Number | Sex | (N) | (N) | Row1 |
| AVISITN | | | 14 | | |
| AVISITN | | | 21 | | |
| AVISITN | | | 28 | | |
| AVISITN | | | 35 | | |
| AVISITN | | | 42 | | |
| TRTPN | | | | 1 | |
| TRTPN | | | | 2 | |
| TRTPN | | | | 3 | |
| AVISITN*TRTPN | | | 7 | 1 | |
| AVISITN*TRTPN | | | 7 | 2 | |
| AVISITN*TRTPN | | | 7 | 3 | |
| AVISITN*TRTPN | | | 14 | 1 | |
| AVISITN*TRTPN | | | 14 | 2 | |
| AVISITN*TRTPN | | | 14 | 3 | |
| AVISITN*TRTPN | | | 21 | 1 | |
| AVISITN*TRTPN | | | 21 | 2 | |
| AVISITN*TRTPN | | | 21 | 3 | |
| AVISITN*TRTPN | | | 28 | 1 | |
| AVISITN*TRTPN | | | 28 | 2 | |

CENTANAFADINE 15 OF 28 PROTOCOL 405-201-00014

# $$\tt STAT-3.1$$ MMRM Output for Test on Treatment by Sex Interaction at Day 42 (Efficacy Sample)

### The Mixed Procedure

Coefficients for 1 vs. 3 BY SEX AT DAY 42

| | Pooled | | Analysis | Planned | |
|---------------|--------|-----|----------|-----------|------|
| | Center | | Visit | Treatment | |
| Effect | Number | Sex | (N) | (N) | Row1 |
| AVISITN*TRTPN | | | 28 | 3 | |
| AVISITN*TRTPN | | | 35 | 1 | |
| AVISITN*TRTPN | | | 35 | 2 | |
| AVISITN*TRTPN | | | 35 | 3 | |
| AVISITN*TRTPN | | | 42 | 1 | |
| AVISITN*TRTPN | | | 42 | 2 | |
| AVISITN*TRTPN | | | 42 | 3 | |
| SEX | | F | | | |
| SEX | | M | | | |
| AVISITN*SEX | | F | 7 | | |
| AVISITN*SEX | | M | 7 | | |
| AVISITN*SEX | | F | 14 | | |
| AVISITN*SEX | | M | 14 | | |
| AVISITN*SEX | | F | 21 | | |
| AVISITN*SEX | | M | 21 | | |
| AVISITN*SEX | | F | 28 | | |
| AVISITN*SEX | | M | 28 | | |
| AVISITN*SEX | | F | 35 | | |
| AVISITN*SEX | | M | 35 | | |
CENTANAFADINE 16 OF 28


# $$\operatorname{STAT-3.1}$$ MMRM Output for Test on Treatment by Sex Interaction at Day 42 (Efficacy Sample)

Parameter Code=AISRSTOT ------

#### The Mixed Procedure

Coefficients for 1 vs. 3 BY SEX AT DAY 42

| | Pooled | | Analysis | Planned | |
|-------------------|--------|-----|----------|-----------|------|
| | Center | | Visit | Treatment | |
| Effect | Number | Sex | (N) | (N) | Row1 |
| AVISITN*SEX | | F | 42 | | |
| AVISITN*SEX | | M | 42 | | |
| TRTPN*SEX | | F | | 1 | 1 |
| TRTPN*SEX | | M | | 1 | -1 |
| TRTPN*SEX | | F | | 2 | |
| TRTPN*SEX | | M | | 2 | |
| TRTPN*SEX | | F | | 3 | -1 |
| TRTPN*SEX | | M | | 3 | 1 |
| AVISITN*TRTPN*SEX | | F | 7 | 1 | |
| AVISITN*TRTPN*SEX | | M | 7 | 1 | |
| AVISITN*TRTPN*SEX | | F | 7 | 2 | |
| AVISITN*TRTPN*SEX | | M | 7 | 2 | |
| AVISITN*TRTPN*SEX | | F | 7 | 3 | |
| AVISITN*TRTPN*SEX | | M | 7 | 3 | |
| AVISITN*TRTPN*SEX | | F | 14 | 1 | |
| AVISITN*TRTPN*SEX | | M | 14 | 1 | |
| AVISITN*TRTPN*SEX | | F | 14 | 2 | |
| AVISITN*TRTPN*SEX | | M | 14 | 2 | |
| AVISITN*TRTPN*SEX | | F | 14 | 3 | |

CENTANAFADINE 17 OF 28 PROTOCOL 405-201-00014

# $$\tt STAT-3.1$$ MMRM Output for Test on Treatment by Sex Interaction at Day 42 (Efficacy Sample)

------

The Mixed Procedure

Coefficients for 1 vs. 3 BY SEX AT DAY 42

| | Pooled | | Analysis | Planned | |
|-------------------|--------|-----|----------|-----------|------|
| | Center | | Visit | Treatment | |
| Effect | Number | Sex | (N) | (N) | Row1 |
| AVISITN*TRTPN*SEX | | M | 14 | 3 | |
| AVISITN*TRTPN*SEX | | F | 21 | 1 | |
| AVISITN*TRTPN*SEX | | M | 21 | 1 | |
| AVISITN*TRTPN*SEX | | F | 21 | 2 | |
| AVISITN*TRTPN*SEX | | M | 21 | 2 | |
| AVISITN*TRTPN*SEX | | F | 21 | 3 | |
| AVISITN*TRTPN*SEX | | M | 21 | 3 | |
| AVISITN*TRTPN*SEX | | F | 28 | 1 | |
| AVISITN*TRTPN*SEX | | M | 28 | 1 | |
| AVISITN*TRTPN*SEX | | F | 28 | 2 | |
| AVISITN*TRTPN*SEX | | M | 28 | 2 | |
| AVISITN*TRTPN*SEX | | F | 28 | 3 | |
| AVISITN*TRTPN*SEX | | M | 28 | 3 | |
| AVISITN*TRTPN*SEX | | F | 35 | 1 | |
| AVISITN*TRTPN*SEX | | M | 35 | 1 | |
| AVISITN*TRTPN*SEX | | F | 35 | 2 | |
| AVISITN*TRTPN*SEX | | M | 35 | 2 | |
| AVISITN*TRTPN*SEX | | F | 35 | 3 | |
| AVISITN*TRTPN*SEX | | M | 35 | 3 | |

CENTANAFADINE 18 OF 28 PROTOCOL 405-201-00014

# $$\tt STAT-3.1$$ MMRM Output for Test on Treatment by Sex Interaction at Day 42 (Efficacy Sample)

-----

#### The Mixed Procedure

Coefficients for 1 vs. 3 BY SEX AT DAY 42

| | Pooled<br>Center | | Analysis<br>Visit | Planned<br>Treatment | |
|---|---|---|---|---|---|
| Effect | Number | Sex | (N) | (N) | Row1 |
| AVISITN*TRTPN*SEX | | F | 42 | 1 | 1 |
| AVISITN*TRTPN*SEX | | M | 42 | 1 | -1 |
| AVISITN*TRTPN*SEX | | F | 42 | 2 | |
| AVISITN*TRTPN*SEX | | M | 42 | 2 | |
| AVISITN*TRTPN*SEX | | F | 42 | 3 | -1 |
| AVISITN*TRTPN*SEX | | M | 42 | 3 | 1 |
| BASE*AVISITN | | | 7 | | |
| BASE*AVISITN | | | 14 | | |
| BASE*AVISITN | | | 21 | | |
| BASE*AVISITN | | | 28 | | |
| BASE*AVISITN | | | 35 | | |
| BASE*AVISITN | | | 42 | | |

CENTANAFADINE 19 OF 28 PROTOCOL 405-201-00014

 $$\tt STAT-3.1$$  MMRM Output for Test on Treatment by Sex Interaction at Day 42 (Efficacy Sample)

The Mixed Procedure

Coefficients for 2 vs. 3 BY SEX AT DAY 42

| | Pooled<br>Center | | Analysis<br>Visit | Planned<br>Treatment | |
|---|---|---|---|---|---|
| Effect | Number | Sex | (N) | (N) | Row1 |
| | | | , | . , | |
| Intercept | | | | | |
| POOLCNTR | | | | | |
| POOLCNTR | | | | | |
| POOLCNTR | | | | | |
| POOLCNTR | | | | | |
| POOLCNTR | | | | | |
| POOLCNTR | | | | | |
| POOLCNTR | | | | | |
| POOLCNTR | | | | | |
| POOLCNTR | | | | | |
| POOLCNTR<br>POOLCNTR | | | | | |
| POOLCNIR | | | | | |
| POOLCNIR | | | | | |
| POOLCNTR | | | | | |
| POOLCNTR | | | | | |
| POOLCNTR | | | | | |
| POOLCNTR | | | | | |
| POOLCNTR | | | | | |

CENTANAFADINE 20 OF 28 PROTOCOL 405-201-00014

 $$\tt STAT-3.1$$  MMRM Output for Test on Treatment by Sex Interaction at Day 42 (Efficacy Sample)

The Mixed Procedure

Coefficients for 2 vs. 3 BY SEX AT DAY 42

| Effect | Pooled<br>Center<br>Number | Sex | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|
| POOLCNTR | | | | | |

CENTANAFADINE 21 OF 28

PROTOCOL 405-201-00014 STAT-3.1 MMRM Output for Test on Treatment by Sex Interaction at Day 42

(Efficacy Sample)

#### The Mixed Procedure

#### Coefficients for 2 vs. 3 BY SEX AT DAY 42

| | Pooled | | Analysis | Planned | |
|---------------|--------|-----|----------|-----------|------|
| | Center | | Visit | Treatment | |
| Effect | Number | Sex | (N) | (N) | Row1 |
| POOLCNTR | | | | | |
| POOLCNTR | | | | | |
| AVISITN | | | 7 | | |
| AVISITN | | | 14 | | |
| AVISITN | | | 21 | | |
| AVISITN | | | 28 | | |
| AVISITN | | | 35 | | |
| AVISITN | | | 42 | | |
| TRTPN | | | | 1 | |
| TRTPN | | | | 2 | |
| TRTPN | | | | 3 | |
| AVISITN*TRTPN | | | 7 | 1 | |
| AVISITN*TRTPN | | | 7 | 2 | |
| AVISITN*TRTPN | | | 7 | 3 | |
| AVISITN*TRTPN | | | 14 | 1 | |
| AVISITN*TRTPN | | | 14 | 2 | |
| AVISITN*TRTPN | | | 14 | 3 | |
| AVISITN*TRTPN | | | 21 | 1 | |
| AVISITN*TRTPN | | | 21 | 2 | |

CENTANAFADINE 22 OF 28 PROTOCOL 405-201-00014

# $$\tt STAT-3.1$$ MMRM Output for Test on Treatment by Sex Interaction at Day 42 (Efficacy Sample)

The Mixed Procedure

Coefficients for 2 vs. 3 BY SEX AT DAY 42

| | Pooled | | Analysis | Planned | |
|---------------|--------|-----|----------|-----------|------|
| | Center | | Visit | Treatment | |
| Effect | Number | Sex | (N) | (N) | Row1 |
| AVISITN*TRTPN | | | 21 | 3 | |
| AVISITN*TRTPN | | | 28 | 1 | |
| AVISITN*TRTPN | | | 28 | 2 | |
| AVISITN*TRTPN | | | 28 | 3 | |
| AVISITN*TRTPN | | | 35 | 1 | |
| AVISITN*TRTPN | | | 35 | 2 | |
| AVISITN*TRTPN | | | 35 | 3 | |
| AVISITN*TRTPN | | | 42 | 1 | |
| AVISITN*TRTPN | | | 42 | 2 | |
| AVISITN*TRTPN | | | 42 | 3 | |
| SEX | | F | | | |
| SEX | | M | | | |
| AVISITN*SEX | | F | 7 | | |
| AVISITN*SEX | | M | 7 | | |
| AVISITN*SEX | | F | 14 | | |
| AVISITN*SEX | | M | 14 | | |
| AVISITN*SEX | | F | 21 | | |
| AVISITN*SEX | | M | 21 | | |
| AVISITN*SEX | | F | 28 | | |

CENTANAFADINE 23 OF 28 PROTOCOL 405-201-00014

# $$\tt STAT-3.1$$ MMRM Output for Test on Treatment by Sex Interaction at Day 42 (Efficacy Sample)

-----

#### The Mixed Procedure

Coefficients for 2 vs. 3 BY SEX AT DAY 42

| Effect | Pooled<br>Center<br>Number | Sex | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|
| AVISITN*SEX | | M | 28 | | |
| AVISITN*SEX | | F | 35 | | |
| AVISITN*SEX | | M | 35 | | |
| AVISITN*SEX | | F | 42 | | |
| AVISITN*SEX | | M | 42 | | |
| TRTPN*SEX | | F | | 1 | |
| TRTPN*SEX | | M | | 1 | |
| TRTPN*SEX | | F | | 2 | 1 |
| TRTPN*SEX | | M | | 2 | -1 |
| TRTPN*SEX | | F | | 3 | -1 |
| TRTPN*SEX | | M | | 3 | 1 |
| AVISITN*TRTPN*SEX | | F | 7 | 1 | |
| AVISITN*TRTPN*SEX | | M | 7 | 1 | |
| AVISITN*TRTPN*SEX | | F | 7 | 2 | |
| AVISITN*TRTPN*SEX | | M | 7 | 2 | |
| AVISITN*TRTPN*SEX | | F | 7 | 3 | |
| AVISITN*TRTPN*SEX | | M | 7 | 3 | |
| AVISITN*TRTPN*SEX | | F | 14 | 1 | |
| AVISITN*TRTPN*SEX | | M | 14 | 1 | |

CENTANAFADINE


 $$\tt STAT-3.1$$  MMRM Output for Test on Treatment by Sex Interaction at Day 42 (Efficacy Sample)

The Mixed Procedure

Coefficients for 2 vs. 3 BY SEX AT DAY 42

| | Pooled | | Analysis | Planned | |
|-------------------|--------|-----|----------|-----------|------|
| | Center | | Visit | Treatment | |
| Effect | Number | Sex | (N) | (N) | Row1 |
| AVISITN*TRTPN*SEX | | F | 14 | 2 | |
| AVISITN*TRTPN*SEX | | M | 14 | 2 | |
| AVISITN*TRTPN*SEX | | F | 14 | 3 | |
| AVISITN*TRTPN*SEX | | M | 14 | 3 | |
| AVISITN*TRTPN*SEX | | F | 21 | 1 | |
| AVISITN*TRTPN*SEX | | M | 21 | 1 | |
| AVISITN*TRTPN*SEX | | F | 21 | 2 | |
| AVISITN*TRTPN*SEX | | M | 21 | 2 | |
| AVISITN*TRTPN*SEX | | F | 21 | 3 | |
| AVISITN*TRTPN*SEX | | M | 21 | 3 | |
| AVISITN*TRTPN*SEX | | F | 28 | 1 | |
| AVISITN*TRTPN*SEX | | M | 28 | 1 | |
| AVISITN*TRTPN*SEX | | F | 28 | 2 | |
| AVISITN*TRTPN*SEX | | M | 28 | 2 | |
| AVISITN*TRTPN*SEX | | F | 28 | 3 | |
| AVISITN*TRTPN*SEX | | M | 28 | 3 | |
| AVISITN*TRTPN*SEX | | F | 35 | 1 | |
| AVISITN*TRTPN*SEX | | M | 35 | 1 | |
| AVISITN*TRTPN*SEX | | F | 35 | 2 | |

CENTANAFADINE 25 OF 28 PROTOCOL 405-201-00014

# $$\tt STAT-3.1$$ MMRM Output for Test on Treatment by Sex Interaction at Day 42 (Efficacy Sample)

-----

#### The Mixed Procedure

Coefficients for 2 vs. 3 BY SEX AT DAY 42

| | Pooled<br>Center | | Analysis<br>Visit | Planned<br>Treatment | |
|---|---|---|---|---|---|
| Effect | Number | Sex | (N) | (N) | Row1 |
| AVISITN*TRTPN*SEX | | М | 35 | 2 | |
| AVISITN*TRTPN*SEX | | F | 35 | 3 | |
| AVISITN*TRTPN*SEX | | M | 35 | 3 | |
| AVISITN*TRTPN*SEX | | F | 42 | 1 | |
| AVISITN*TRTPN*SEX | | M | 42 | 1 | |
| AVISITN*TRTPN*SEX | | F | 42 | 2 | 1 |
| AVISITN*TRTPN*SEX | | M | 42 | 2 | -1 |
| AVISITN*TRTPN*SEX | | F | 42 | 3 | -1 |
| AVISITN*TRTPN*SEX | | M | 42 | 3 | 1 |
| BASE*AVISITN | | | 7 | | |
| BASE*AVISITN | | | 14 | | |
| BASE*AVISITN | | | 21 | | |
| BASE*AVISITN | | | 28 | | |
| BASE*AVISITN | | | 35 | | |
| BASE*AVISITN | | | 42 | | |

CENTANAFADINE 26 OF 28 PROTOCOL 405-201-00014

# $$\operatorname{STAT-3.1}$$ MMRM Output for Test on Treatment by Sex Interaction at Day 42 (Efficacy Sample)

The Mixed Procedure

#### Estimates

Ctandard

| | | Standard | | | |
|--------------------------|----------|----------|-----|---------|---------|
| Label | Estimate | Error | DF | t Value | Pr > t |
| 1 vs. 3 BY SEX AT DAY 42 | 0.2939 | 2.6567 | 383 | 0.11 | 0.9120 |
| 2 vs. 3 BY SEX AT DAY 42 | -2.4115 | 2.6901 | 387 | -0.90 | 0.3706 |

#### Least Squares Means

| | | Analysis<br>Visit | Planned<br>Treatment | | Standard | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Effect | Sex | (N) | (N) | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| AVISITN*TRTPN*SEX | F | 7 | 1 | -5.4027 | 0.8667 | 378 | -6.23 | <.0001 | 0.05 | -7.1068 | -3.6986 |
| AVISITN*TRTPN*SEX | M | 7 | 1 | -6.9479 | 0.8409 | 383 | -8.26 | <.0001 | 0.05 | -8.6013 | -5.2946 |
| AVISITN*TRTPN*SEX | F | 7 | 2 | -7.1868 | 0.8594 | 376 | -8.36 | <.0001 | 0.05 | -8.8767 | -5.4969 |
| AVISITN*TRTPN*SEX | M | 7 | 2 | -5.0335 | 0.8496 | 379 | -5.92 | <.0001 | 0.05 | -6.7041 | -3.3629 |
| AVISITN*TRTPN*SEX | F | 7 | 3 | -3.7852 | 0.8669 | 378 | -4.37 | <.0001 | 0.05 | -5.4897 | -2.0807 |
| AVISITN*TRTPN*SEX | M | 7 | 3 | -4.6461 | 0.8279 | 378 | -5.61 | <.0001 | 0.05 | -6.2739 | -3.0183 |
| AVISITN*TRTPN*SEX | F | 14 | 1 | -7.8481 | 1.0852 | 397 | -7.23 | <.0001 | 0.05 | -9.9815 | -5.7147 |
| AVISITN*TRTPN*SEX | M | 14 | 1 | -10.2218 | 1.0454 | 386 | -9.78 | <.0001 | 0.05 | -12.2771 | -8.1665 |
| AVISITN*TRTPN*SEX | F | 14 | 2 | -9.4956 | 1.1164 | 412 | -8.51 | <.0001 | 0.05 | -11.6901 | -7.3010 |
| AVISITN*TRTPN*SEX | M | 14 | 2 | -8.6092 | 1.0577 | 399 | -8.14 | <.0001 | 0.05 | -10.6885 | -6.5298 |

CENTANAFADINE 27 OF 28 PROTOCOL 405-201-00014

STAT-3.1

MMRM Output for Test on Treatment by Sex Interaction at Day 42

(Efficacy Sample)

\_\_\_\_\_

Parameter Code=AISRSTOT ------

The Mixed Procedure

Least Squares Means

| | | Analysis<br>Visit | Planned<br>Treatment | | Standard | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Effect | Sex | (N) | (N) | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| AVISITN*TRTPN*SEX | F | 14 | 3 | -5.3059 | 1.0908 | 381 | -4.86 | <.0001 | 0.05 | -7.4506 | -3.1612 |
| AVISITN*TRTPN*SEX | M | 14 | 3 | -5.5124 | 1.0340 | 407 | -5.33 | <.0001 | 0.05 | -7.5451 | -3.4797 |
| AVISITN*TRTPN*SEX | F | 21 | 1 | -10.5355 | 1.1670 | 394 | -9.03 | <.0001 | 0.05 | -12.8298 | -8.2411 |
| AVISITN*TRTPN*SEX | M | 21 | 1 | -11.0775 | 1.1325 | 393 | -9.78 | <.0001 | 0.05 | -13.3040 | -8.8510 |
| AVISITN*TRTPN*SEX | F | 21 | 2 | -12.3262 | 1.2227 | 419 | -10.08 | <.0001 | 0.05 | -14.7295 | -9.9229 |
| AVISITN*TRTPN*SEX | M | 21 | 2 | -10.3736 | 1.1476 | 408 | -9.04 | <.0001 | 0.05 | -12.6295 | -8.1176 |
| AVISITN*TRTPN*SEX | F | 21 | 3 | -6.9788 | 1.1675 | 374 | -5.98 | <.0001 | 0.05 | -9.2745 | -4.6830 |
| AVISITN*TRTPN*SEX | М | 21 | 3 | -6.6063 | 1.1096 | 403 | -5.95 | <.0001 | 0.05 | -8.7877 | -4.4249 |
| AVISITN*TRTPN*SEX | F | 28 | 1 | -10.4794 | 1.2327 | 400 | -8.50 | <.0001 | 0.05 | -12.9028 | -8.0561 |
| AVISITN*TRTPN*SEX | М | 28 | 1 | -11.4879 | 1.1864 | 390 | -9.68 | <.0001 | 0.05 | -13.8205 | -9.1553 |
| AVISITN*TRTPN*SEX | F | 28 | 2 | -12.7682 | 1.2871 | 416 | -9.92 | <.0001 | 0.05 | -15.2983 | -10.2381 |
| AVISITN*TRTPN*SEX | M | 28 | 2 | -10.4550 | 1.2036 | 406 | -8.69 | <.0001 | 0.05 | -12.8211 | -8.0890 |
| AVISITN*TRTPN*SEX | F | 28 | 3 | -7.5212 | 1.2256 | 373 | -6.14 | <.0001 | 0.05 | -9.9311 | -5.1113 |
| AVISITN*TRTPN*SEX | M | 28 | 3 | -6.6440 | 1.1591 | 399 | -5.73 | <.0001 | 0.05 | -8.9227 | -4.3652 |
| AVISITN*TRTPN*SEX | F | 35 | 1 | -11.4369 | 1.2920 | 398 | -8.85 | <.0001 | 0.05 | -13.9769 | -8.8969 |
| AVISITN*TRTPN*SEX | М | 35 | 1 | -11.7373 | 1.2478 | 391 | -9.41 | <.0001 | 0.05 | -14.1904 | -9.2842 |
| AVISITN*TRTPN*SEX | F | 35 | 2 | -14.6552 | 1.3521 | 409 | -10.84 | <.0001 | 0.05 | -17.3132 | -11.9971 |
| AVISITN*TRTPN*SEX | M | 35 | 2 | -11.6595 | 1.2727 | 414 | -9.16 | <.0001 | 0.05 | -14.1614 | -9.1577 |
| AVISITN*TRTPN*SEX | F | 35 | 3 | -8.5420 | 1.2828 | 371 | -6.66 | <.0001 | 0.05 | -11.0644 | -6.0196 |

CENTANAFADINE 28 OF 28 PROTOCOL 405-201-00014

# $$\tt STAT-3.1$$ MMRM Output for Test on Treatment by Sex Interaction at Day 42 (Efficacy Sample)

------

Parameter Code=AISRSTOT ------

#### The Mixed Procedure

#### Least Squares Means

| | | Analysis<br>Visit | Planned<br>Treatment | | Standard | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Effect | Sex | (N) | (N) | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| AVISITN*TRTPN*SEX | М | 35 | 3 | -7.1620 | 1.2125 | 396 | -5.91 | <.0001 | 0.05 | -9.5458 | -4.7783 |
| AVISITN*TRTPN*SEX | F | 42 | 1 | -12.3096 | 1.3743 | 401 | -8.96 | <.0001 | 0.05 | -15.0112 | -9.6079 |
| AVISITN*TRTPN*SEX | M | 42 | 1 | -11.8471 | 1.3215 | 389 | -8.96 | <.0001 | 0.05 | -14.4454 | -9.2489 |
| AVISITN*TRTPN*SEX | F | 42 | 2 | -14.1591 | 1.4448 | 408 | -9.80 | <.0001 | 0.05 | -16.9992 | -11.3190 |
| AVISITN*TRTPN*SEX | M | 42 | 2 | -10.9912 | 1.3502 | 412 | -8.14 | <.0001 | 0.05 | -13.6453 | -8.3372 |
| AVISITN*TRTPN*SEX | F | 42 | 3 | -8.4423 | 1.3593 | 370 | -6.21 | <.0001 | 0.05 | -11.1152 | -5.7695 |
| AVISITN*TRTPN*SEX | M | 42 | 3 | -7.6860 | 1.2832 | 394 | -5.99 | <.0001 | 0.05 | -10.2088 | -5.1632 |


STAT-3.2

MMRM Output for Test on Treatment by Race Interaction at Day 42(Efficacy Sample)

The Mixed Procedure

Model Information

WORK.INDATA Data Set Dependent Variable CHG Dependent Variable Covariance Structure Unstructured Subject Effect SUBJID Estimation Method REML Residual Variance Method

Fixed Effects SE Method Kenward-Roger Degrees of Freedom Method Kenward-Roger

Class Level Information

Class Levels Values 6 AVISITN TRTPN 3

POOLCNTR 39

7 14 21 28 35 42

CENTANAFADINE


 $$\tt STAT-3.2$$  MMRM Output for Test on Treatment by Race Interaction at Day 42 (Efficacy Sample)

\_\_\_\_\_

The Mixed Procedure

Class Level Information

Class Levels Values
SUBJID 421



CENTANAFADINE


STAT-3.2

MMRM Output for Test on Treatment by Race Interaction at Day 42

(Efficacy Sample)

The Mixed Procedure



CENTANAFADINE

 $$\tt STAT-3.2$$  MMRM Output for Test on Treatment by Race Interaction at Day 42 (Efficacy Sample)

\_\_\_\_\_\_

The Mixed Procedure




 $$\tt STAT-3.2$$  MMRM Output for Test on Treatment by Race Interaction at Day 42 (Efficacy Sample)

......

The Mixed Procedure



CENTANAFADINE 6 OF 28 PROTOCOL 405-201-00014

 $$\tt STAT-3.2$$  MMRM Output for Test on Treatment by Race Interaction at Day 42 (Efficacy Sample)

\_\_\_\_\_\_

The Mixed Procedure




 $$\tt STAT-3.2$$  MMRM Output for Test on Treatment by Race Interaction at Day 42 (Efficacy Sample)

The Mixed Procedure



FILE: stat2b.lis, RUN: 31AUG2020 08:32; ANALYSIS DATASET CREATED: 16JUN2020 08:14
PROGRAM: /opt/sas/Data/DAP/EB1020/P40520100014/STAT/Program.dev/DOC\_STAT/stat2.sas
OPDC, NEW DRUG APPLICATION, IND # 119,361 CENTANAFADINE STAT-3.2 FINAL

RACEGRP

CENTANAFADINE


STAT-3.2

MMRM Output for Test on Treatment by Race Interaction at Day 42 (Efficacy Sample)

-----

The Mixed Procedure

Dimensions

Covariance Parameters 21
Columns in X 129
Columns in Z 0
Subjects 421
Max Obs per Subject 6

Number of Observations

Number of Observations Read 2227
Number of Observations Used 2227
Number of Observations Not Used 0

Iteration History

 Iteration
 Evaluations
 -2 Res Log Like
 Criterion

 0
 1
 15704.36373766
 0.00024380

 1
 2
 13498.26971465
 0.00024380

 2
 1
 13497.03266047
 0.00000273

 3
 1
 13497.01951942
 0.00000000


STAT-3.2

MMRM Output for Test on Treatment by Race Interaction at Day 42 (Efficacy Sample)

\_\_\_\_\_

The Mixed Procedure

Convergence criteria met.

Covariance Parameter Estimates

| Cov Parm | Subject | Estimate |
|----------|---------|----------|
| UN(1,1) | SUBJID | 43.3078 |
| UN(2,1) | SUBJID | 37.9417 |
| UN(2,2) | SUBJID | 69.5782 |
| UN(3,1) | SUBJID | 36.8986 |
| UN(3,2) | SUBJID | 59.1553 |
| UN(3,3) | SUBJID | 80.0027 |
| UN(4,1) | SUBJID | 38.6686 |
| UN(4,2) | SUBJID | 58.2307 |
| UN(4,3) | SUBJID | 72.5007 |
| UN(4,4) | SUBJID | 88.6310 |
| UN(5,1) | SUBJID | 38.3557 |
| UN(5,2) | SUBJID | 59.4955 |
| UN(5,3) | SUBJID | 71.0718 |
| UN(5,4) | SUBJID | 81.0660 |
| UN(5,5) | SUBJID | 96.3614 |
| UN(6,1) | SUBJID | 37.6519 |
| UN(6,2) | SUBJID | 59.1146 |
| UN(6,3) | SUBJID | 72.6172 |


STAT-3.2

MMRM Output for Test on Treatment by Race Interaction at Day 42  $\,$  (Efficacy Sample)

-----

The Mixed Procedure

Covariance Parameter Estimates

| Cov Parm | Subject | Estimate |
|-----------|---------|----------|
| UN(6,4) | SUBJID | 82.6569 |
| UN(6,5) | SUBJID | 90.2016 |
| IIN (6 6) | SUBJUD | 106 64 |

#### Fit Statistics

| -2 Res Log Likelihood | 13497.0 |
|--------------------------|---------|
| AIC (Smaller is Better) | 13539.0 |
| AICC (Smaller is Better) | 13539.5 |
| BIC (Smaller is Better) | 13623.9 |

### Null Model Likelihood Ratio Test

| DF | Chi-Square | Pr > ChiSc |
|----|------------|------------|
| 20 | 2207 34 | < 0001 |


STAT-3.2

MMRM Output for Test on Treatment by Race Interaction at Day 42  $$({\tt Efficacy}\ {\tt Sample})$$ 

\_\_\_\_\_

The Mixed Procedure

Type 3 Tests of Fixed Effects

| | Num | Den | | |
|----------------------|-----|-----|---------|--------|
| Effect | DF | DF | F Value | Pr > F |
| POOLCNTR | 38 | 377 | 2.15 | 0.0002 |
| AVISITN | 5 | 352 | 1.25 | 0.2856 |
| TRTPN | 2 | 389 | 9.82 | <.0001 |
| AVISITN*TRTPN | 10 | 527 | 2.05 | 0.0272 |
| RACEGRP | 1 | 414 | 8.58 | 0.0036 |
| AVISITN*RACEGRP | 5 | 353 | 2.06 | 0.0695 |
| TRTPN*RACEGRP | 2 | 394 | 0.85 | 0.4284 |
| AVISIT*TRTPN*RACEGRP | 10 | 526 | 1.21 | 0.2828 |
| BASE*AVISITN | 6 | 380 | 2.09 | 0.0534 |

Coefficients for 1 vs. 3 BY RACEGRP AT DAY 42

Pooled Analysis Planned
Center Visit Treatment
Effect Number RACEGRP (N) (N) Row1

Intercept

POOLCNTR POOLCNTR




 $$\tt STAT-3.2$$  MMRM Output for Test on Treatment by Race Interaction at Day 42 (Efficacy Sample)

The Mixed Procedure

Coefficients for 1 vs. 3 BY RACEGRP AT DAY 42

| | Pooled<br>Center | | Analysis<br>Visit | Planned | |
|---|---|---|---|---|---|
| Effect | Number | RACEGRP | (N) | Treatment (N) | Row1 |
| POOLCNTR | | | | | |


 $$\tt STAT-3.2$$  MMRM Output for Test on Treatment by Race Interaction at Day 42 (Efficacy Sample)

The Mixed Procedure

Coefficients for 1 vs. 3 BY RACEGRP AT DAY 42




### STAT-3.2 RM Output for Test on Treatment by Race Interact:

MMRM Output for Test on Treatment by Race Interaction at Day 42  $$({\tt Efficacy\ Sample})$$ 

-----

#### The Mixed Procedure

#### Coefficients for 1 vs. 3 BY RACEGRP AT DAY 42

| | Pooled | | Analysis | Planned | |
|---------------|--------|---------|----------|-----------|------|
| | Center | | Visit | Treatment | |
| Effect | Number | RACEGRP | (N) | (N) | Row1 |
| AVISITN | | | 14 | | |
| AVISITN | | | 21 | | |
| AVISITN | | | 28 | | |
| AVISITN | | | 35 | | |
| AVISITN | | | 42 | | |
| TRTPN | | | | 1 | |
| TRTPN | | | | 2 | |
| TRTPN | | | | 3 | |
| AVISITN*TRTPN | | | 7 | 1 | |
| AVISITN*TRTPN | | | 7 | 2 | |
| AVISITN*TRTPN | | | 7 | 3 | |
| AVISITN*TRTPN | | | 14 | 1 | |
| AVISITN*TRTPN | | | 14 | 2 | |
| AVISITN*TRTPN | | | 14 | 3 | |
| AVISITN*TRTPN | | | 21 | 1 | |
| AVISITN*TRTPN | | | 21 | 2 | |
| AVISITN*TRTPN | | | 21 | 3 | |
| AVISITN*TRTPN | | | 28 | 1 | |
| AVISITN*TRTPN | | | 28 | 2 | |


 $$\operatorname{\mathtt{STAT-3.2}}$$  MMRM Output for Test on Treatment by Race Interaction at Day 42

(Efficacy Sample)

------

The Mixed Procedure

Coefficients for 1 vs. 3 BY RACEGRP AT DAY 42

| | Pooled | | Analysis | Planned | |
|-----------------|--------|-----------------|----------|-----------|------|
| | Center | | Visit | Treatment | |
| Effect | Number | RACEGRP | (N) | (N) | Row1 |
| AVISITN*TRTPN | | | 28 | 3 | |
| AVISITN*TRTPN | | | 35 | 1 | |
| AVISITN*TRTPN | | | 35 | 2 | |
| AVISITN*TRTPN | | | 35 | 3 | |
| AVISITN*TRTPN | | | 42 | 1 | |
| AVISITN*TRTPN | | | 42 | 2 | |
| AVISITN*TRTPN | | | 42 | 3 | |
| RACEGRP | | All Other Races | | | |
| RACEGRP | | White | | | |
| AVISITN*RACEGRP | | All Other Races | 7 | | |
| AVISITN*RACEGRP | | White | 7 | | |
| AVISITN*RACEGRP | | All Other Races | 14 | | |
| AVISITN*RACEGRP | | White | 14 | | |
| AVISITN*RACEGRP | | All Other Races | 21 | | |
| AVISITN*RACEGRP | | White | 21 | | |
| AVISITN*RACEGRP | | All Other Races | 28 | | |
| AVISITN*RACEGRP | | White | 28 | | |
| AVISITN*RACEGRP | | All Other Races | 35 | | |
| AVISITN*RACEGRP | | White | 35 | | |

CENTANAFADINE 16 OF 28 PROTOCOL 405-201-00014

# $$\tt STAT-3.2$$ MMRM Output for Test on Treatment by Race Interaction at Day 42 (Efficacy Sample)

-----

#### The Mixed Procedure

#### Coefficients for 1 vs. 3 BY RACEGRP AT DAY 42

| | Pooled | | Analysis | | |
|---|---|---|---|---|---|
| | Center | | Visit | Treatment | |
| Effect | Number | RACEGRP | (N) | (N) | Row1 |
| AVISITN*RACEGRP | | All Other Races | | | |
| AVISITN*RACEGRP | | White | 42 | | |
| TRTPN*RACEGRP | | All Other Races | | 1 | 1 |
| TRTPN*RACEGRP | | White | | 1 | -1 |
| TRTPN*RACEGRP | | All Other Races | | 2 | |
| TRTPN*RACEGRP | | White | | 2 | |
| TRTPN*RACEGRP | | All Other Races | | 3 | -1 |
| TRTPN*RACEGRP | | White | | 3 | 1 |
| AVISIT*TRTPN*RACEGRP | | All Other Races | 7 | 1 | |
| AVISIT*TRTPN*RACEGRP | | White | 7 | 1 | |
| AVISIT*TRTPN*RACEGRP | | All Other Races | 7 | 2 | |
| AVISIT*TRTPN*RACEGRP | | White | 7 | 2 | |
| AVISIT*TRTPN*RACEGRP | | All Other Races | 7 | 3 | |
| AVISIT*TRTPN*RACEGRP | | White | 7 | 3 | |
| AVISIT*TRTPN*RACEGRP | | All Other Races | 14 | 1 | |
| AVISIT*TRTPN*RACEGRP | | White | 14 | 1 | |
| AVISIT*TRTPN*RACEGRP | | All Other Races | 14 | 2 | |
| AVISIT*TRTPN*RACEGRP | | White | 14 | 2 | |
| AVISIT*TRTPN*RACEGRP | | All Other Races | 14 | 3 | |

CENTANAFADINE 17 OF 28


 $$\tt STAT-3.2$$  MMRM Output for Test on Treatment by Race Interaction at Day 42 (Efficacy Sample)

The Mixed Procedure

Coefficients for 1 vs. 3 BY RACEGRP AT DAY 42

| | Pooled | | Analysis | Planned | |
|----------------|---------|-----------------|----------|-----------|------|
| | Center | | Visit | Treatment | |
| Effect | Number | RACEGRP | (N) | (N) | Row1 |
| AVISIT*TRTPN*R | ACEGRP | White | 14 | 3 | |
| AVISIT*TRTPN*R | ACEGRP | All Other Races | 21 | 1 | |
| AVISIT*TRTPN*R | ACEGRP | White | 21 | 1 | |
| AVISIT*TRTPN*R | ACEGRP | All Other Races | 21 | 2 | |
| AVISIT*TRTPN*R | RACEGRP | White | 21 | 2 | |
| AVISIT*TRTPN*R | RACEGRP | All Other Races | 21 | 3 | |
| AVISIT*TRTPN*R | RACEGRP | White | 21 | 3 | |
| AVISIT*TRTPN*R | ACEGRP | All Other Races | 28 | 1 | |
| AVISIT*TRTPN*R | ACEGRP | White | 28 | 1 | |
| AVISIT*TRTPN*R | RACEGRP | All Other Races | 28 | 2 | |
| AVISIT*TRTPN*R | RACEGRP | White | 28 | 2 | |
| AVISIT*TRTPN*R | RACEGRP | All Other Races | 28 | 3 | |
| AVISIT*TRTPN*R | RACEGRP | White | 28 | 3 | |
| AVISIT*TRTPN*R | RACEGRP | All Other Races | 35 | 1 | |
| AVISIT*TRTPN*R | ACEGRP | White | 35 | 1 | |
| AVISIT*TRTPN*R | ACEGRP | All Other Races | 35 | 2 | |
| AVISIT*TRTPN*R | ACEGRP | White | 35 | 2 | |
| AVISIT*TRTPN*R | ACEGRP | All Other Races | 35 | 3 | |
| AVISIT*TRTPN*R | RACEGRP | White | 35 | 3 | |


 $$\tt STAT-3.2$$  MMRM Output for Test on Treatment by Race Interaction at Day 42 (Efficacy Sample)

Parameter Code=AISRSTOT ------

The Mixed Procedure

Coefficients for 1 vs. 3 BY RACEGRP AT DAY 42

| | Pooled<br>Center | | Analysis<br>Visit | Planned<br>Treatment | |
|---|---|---|---|---|---|
| Effect | Number | RACEGRP | (N) | (N) | Row1 |
| AVISIT*TRTPN*RACEGRP | | All Other Races | 42 | 1 | 1 |
| AVISIT*TRTPN*RACEGRP | | White | 42 | 1 | -1 |
| AVISIT*TRTPN*RACEGRP | | All Other Races | 42 | 2 | |
| AVISIT*TRTPN*RACEGRP | | White | 42 | 2 | |
| AVISIT*TRTPN*RACEGRP | | All Other Races | 42 | 3 | -1 |
| AVISIT*TRTPN*RACEGRP | | White | 42 | 3 | 1 |
| BASE*AVISITN | | | 7 | | |
| BASE*AVISITN | | | 14 | | |
| BASE*AVISITN | | | 21 | | |
| BASE*AVISITN | | | 28 | | |
| BASE*AVISITN | | | 35 | | |
| BASE*AVISITN | | | 42 | | |


STAT-3.2

MMRM Output for Test on Treatment by Race Interaction at Day 42  $$({\tt Efficacy}\ {\tt Sample})$$ 

.------

The Mixed Procedure

Coefficients for 2 vs. 3 BY RACEGRP AT DAY 42

| Effect | Pooled<br>Center<br>Number | RACEGRP | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Row1 |
|---|---|---|---|---|---|
| Intercept | | | | | |
| POOLCNTR | | | | | |


 $$\tt STAT-3.2$$  MMRM Output for Test on Treatment by Race Interaction at Day 42 (Efficacy Sample)

The Mixed Procedure

Coefficients for 2 vs. 3 BY RACEGRP AT DAY 42

| | Pooled | | Analysis<br>Visit | Planned | |
|---|---|---|---|---|---|
| Effect | Center<br>Number | RACEGRP | (N) | Treatment (N) | Row1 |
| Ellect | Number | RACEGRE | (11) | (11) | KOWI |
| POOLCNTR | | | | | |

CENTANAFADINE 21 OF 28 PROTOCOL 405-201-00014

# $$\tt STAT-3.2$$ MMRM Output for Test on Treatment by Race Interaction at Day 42 (Efficacy Sample)

#### The Mixed Procedure

#### Coefficients for 2 vs. 3 BY RACEGRP AT DAY 42

| | Pooled | | Analysis | Planned | |
|---------------|--------|---------|----------|-----------|------|
| | Center | | Visit | Treatment | |
| Effect | Number | RACEGRP | (N) | (N) | Row1 |
| POOLCNTR | | | | | |
| POOLCNTR | | | | | |
| AVISITN | | | 7 | | |
| AVISITN | | | 14 | | |
| AVISITN | | | 21 | | |
| AVISITN | | | 28 | | |
| AVISITN | | | 35 | | |
| AVISITN | | | 42 | | |
| TRTPN | | | | 1 | |
| TRTPN | | | | 2 | |
| TRTPN | | | | 3 | |
| AVISITN*TRTPN | | | 7 | 1 | |
| AVISITN*TRTPN | | | 7 | 2 | |
| AVISITN*TRTPN | | | 7 | 3 | |
| AVISITN*TRTPN | | | 14 | 1 | |
| AVISITN*TRTPN | | | 14 | 2 | |
| AVISITN*TRTPN | | | 14 | 3 | |
| AVISITN*TRTPN | | | 21 | 1 | |
| AVISITN*TRTPN | | | 21 | 2 | |


 $$\tt STAT-3.2$$  MMRM Output for Test on Treatment by Race Interaction at Day 42 (Efficacy Sample)

\_\_\_\_\_

The Mixed Procedure

Coefficients for 2 vs. 3 BY RACEGRP AT DAY 42

| | Pooled | | Analysis | Planned | |
|-----------------|--------|-----------------|----------|-----------|------|
| | Center | | Visit | Treatment | |
| Effect | Number | RACEGRP | (N) | (N) | Row1 |
| | | | 0.1 | 2 | |
| AVISITN*TRTPN | | | 21 | 3 | |
| AVISITN*TRTPN | | | 28 | 1 | |
| AVISITN*TRTPN | | | 28 | 2 | |
| AVISITN*TRTPN | | | 28 | 3 | |
| AVISITN*TRTPN | | | 35 | 1 | |
| AVISITN*TRTPN | | | 35 | 2 | |
| AVISITN*TRTPN | | | 35 | 3 | |
| AVISITN*TRTPN | | | 42 | 1 | |
| AVISITN*TRTPN | | | 42 | 2 | |
| AVISITN*TRTPN | | | 42 | 3 | |
| RACEGRP | | All Other Races | | | |
| RACEGRP | | White | | | |
| AVISITN*RACEGRP | | All Other Races | 7 | | |
| AVISITN*RACEGRP | | White | 7 | | |
| AVISITN*RACEGRP | | All Other Races | 14 | | |
| AVISITN*RACEGRP | | White | 14 | | |
| AVISITN*RACEGRP | | All Other Races | 21 | | |
| AVISITN*RACEGRP | | White | 21 | | |
| AVISITN*RACEGRP | | All Other Races | 28 | | |


# $$\tt STAT-3.2$$ MMRM Output for Test on Treatment by Race Interaction at Day 42 (Efficacy Sample)

\_\_\_\_\_

#### The Mixed Procedure

#### Coefficients for 2 vs. 3 BY RACEGRP AT DAY 42

| | Pooled | | Analysis | Planned | |
|---|---|---|---|---|---|
| | Center | | Visit | Treatment | |
| Effect | Number | RACEGRP | (N) | (N) | Row1 |
| AVISITN*RACEGRP | | White | 28 | | |
| AVISITN*RACEGRP | | All Other Races | 35 | | |
| AVISITN*RACEGRP | | White | 35 | | |
| AVISITN*RACEGRP | | All Other Races | 42 | | |
| AVISITN*RACEGRP | | White | 42 | | |
| TRTPN*RACEGRP | | All Other Races | | 1 | |
| TRTPN*RACEGRP | | White | | 1 | |
| TRTPN*RACEGRP | | All Other Races | | 2 | 1 |
| TRTPN*RACEGRP | | White | | 2 | -1 |
| TRTPN*RACEGRP | | All Other Races | | 3 | -1 |
| TRTPN*RACEGRP | | White | | 3 | 1 |
| AVISIT*TRTPN*RACEGRP | | All Other Races | 7 | 1 | |
| AVISIT*TRTPN*RACEGRP | | White | 7 | 1 | |
| AVISIT*TRTPN*RACEGRP | | All Other Races | 7 | 2 | |
| AVISIT*TRTPN*RACEGRP | | White | 7 | 2 | |
| AVISIT*TRTPN*RACEGRP | | All Other Races | 7 | 3 | |
| AVISIT*TRTPN*RACEGRP | | White | 7 | 3 | |
| AVISIT*TRTPN*RACEGRP | | All Other Races | 14 | 1 | |
| AVISIT*TRTPN*RACEGRP | | White | 14 | 1 | |
CENTANAFADINE


 $$\tt STAT-3.2$$  MMRM Output for Test on Treatment by Race Interaction at Day 42 (Efficacy Sample)

The Mixed Procedure

Coefficients for 2 vs. 3 BY RACEGRP AT DAY 42

| | Pooled | | Analysis | | |
|---|---|---|---|---|---|
| | Center | | Visit | Treatment | |
| Effect | Number | RACEGRP | (N) | (N) | Row1 |
| AVISIT*TRTPN*RACEGRP | | All Other Races | 14 | 2 | |
| AVISIT*TRTPN*RACEGRP | | White | 14 | 2 | |
| AVISIT*TRTPN*RACEGRP | | All Other Races | 14 | 3 | |
| AVISIT*TRTPN*RACEGRP | | White | 14 | 3 | |
| AVISIT*TRTPN*RACEGRP | | All Other Races | 21 | 1 | |
| AVISIT*TRTPN*RACEGRP | | White | 21 | 1 | |
| AVISIT*TRTPN*RACEGRP | | All Other Races | 21 | 2 | |
| AVISIT*TRTPN*RACEGRP | | White | 21 | 2 | |
| AVISIT*TRTPN*RACEGRP | | All Other Races | 21 | 3 | |
| AVISIT*TRTPN*RACEGRP | | White | 21 | 3 | |
| AVISIT*TRTPN*RACEGRP | | All Other Races | 28 | 1 | |
| AVISIT*TRTPN*RACEGRP | | White | | 1 | |
| AVISIT*TRTPN*RACEGRP | | All Other Races | 28 | 2 | |
| AVISIT*TRTPN*RACEGRP | | White | 28 | 2 | |
| AVISIT*TRTPN*RACEGRP | | All Other Races | 28 | 3 | |
| AVISIT*TRTPN*RACEGRP | | White | 28 | 3 | |
| AVISIT*TRTPN*RACEGRP | | All Other Races | 35 | 1 | |
| AVISIT*TRTPN*RACEGRP | | White | 35 | 1 | |
| AVISIT*TRTPN*RACEGRP | | All Other Races | 35 | 2 | |


STAT-3.2

MMRM Output for Test on Treatment by Race Interaction at Day 42  $$({\tt Efficacy\ Sample})$$ 

The Mixed Procedure

Coefficients for 2 vs. 3 BY RACEGRP AT DAY 42

| | Pooled | | Analysis | Planned | |
|---|---|---|---|---|---|
| | Center | | Visit | Treatment | |
| Effect | Number | RACEGRP | (N) | (N) | Row1 |
| AVISIT*TRTPN*RACEGRP | | White | 35 | 2 | |
| AVISIT*TRTPN*RACEGRP | | All Other Races | 35 | 3 | |
| AVISIT*TRTPN*RACEGRP | | White | 35 | 3 | |
| AVISIT*TRTPN*RACEGRP | | All Other Races | 42 | 1 | |
| AVISIT*TRTPN*RACEGRP | | White | 42 | 1 | |
| AVISIT*TRTPN*RACEGRP | | All Other Races | 42 | 2 | 1 |
| AVISIT*TRTPN*RACEGRP | | White | 42 | 2 | -1 |
| AVISIT*TRTPN*RACEGRP | | All Other Races | 42 | 3 | -1 |
| AVISIT*TRTPN*RACEGRP | | White | 42 | 3 | 1 |
| BASE*AVISITN | | | 7 | | |
| BASE*AVISITN | | | 14 | | |
| BASE*AVISITN | | | 21 | | |
| BASE*AVISITN | | | 28 | | |
| BASE*AVISITN | | | 35 | | |
| BASE*AVISITN | | | 42 | | |


# $$\tt STAT-3.2$$ MMRM Output for Test on Treatment by Race Interaction at Day 42 (Efficacy Sample)

#### The Mixed Procedure

#### Estimates

| La | bel | | | | | | | Estimate | Standard<br>Error | DF | t Value | Pr > t |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 1 | vs. | 3 | вч | RACEGRP | AT | DAY | 42 | -1.8375 | 3.1294 | 385 | -0.59 | 0.5574 |
| 2 | vs. | 3 | BY | RACEGRP | AΤ | DAY | 42 | -1.0598 | 3.3731 | 395 | -0.31 | 0.7535 |

#### Least Squares Means

| | | Analysis<br>Visit | Planned<br>Treatment | | Standard | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Effect | RACEGRP | (N) | (N) | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| AVISIT*TRTPN*RACEGRP | All Other Races | 7 | 1 | -7.0994 | 1.2575 | 381 | -5.65 | <.0001 | 0.05 | -9.5720 | -4.6268 |
| AVISIT*TRTPN*RACEGRP | White | 7 | 1 | -5.9784 | 0.6928 | 382 | -8.63 | <.0001 | 0.05 | -7.3405 | -4.6163 |
| AVISIT*TRTPN*RACEGRP | All Other Races | 7 | 2 | -9.0250 | 1.3770 | 376 | -6.55 | <.0001 | 0.05 | -11.7327 | -6.3173 |
| AVISIT*TRTPN*RACEGRP | White | 7 | 2 | -5.4838 | 0.6732 | 378 | -8.15 | <.0001 | 0.05 | -6.8075 | -4.1602 |
| AVISIT*TRTPN*RACEGRP | All Other Races | 7 | 3 | -4.0554 | 1.2955 | 376 | -3.13 | 0.0019 | 0.05 | -6.6028 | -1.5080 |
| AVISIT*TRTPN*RACEGRP | White | 7 | 3 | -4.3810 | 0.6867 | 378 | -6.38 | <.0001 | 0.05 | -5.7311 | -3.0309 |
| AVISIT*TRTPN*RACEGRP | All Other Races | 14 | 1 | -11.5844 | 1.5470 | 394 | -7.49 | <.0001 | 0.05 | -14.6259 | -8.5429 |
| AVISIT*TRTPN*RACEGRP | White | 14 | 1 | -8.3630 | 0.8593 | 397 | -9.73 | <.0001 | 0.05 | -10.0523 | -6.6737 |
| AVISIT*TRTPN*RACEGRP | All Other Races | 14 | 2 | -12.1861 | 1.7791 | 416 | -6.85 | <.0001 | 0.05 | -15.6834 | -8.6889 |
| AVISIT*TRTPN*RACEGRP | White | 14 | 2 | -8.4720 | 0.8445 | 407 | -10.03 | <.0001 | 0.05 | -10.1321 | -6.8120 |


# $$\tt STAT-3.2$$ MMRM Output for Test on Treatment by Race Interaction at Day 42 (Efficacy Sample)

Parameter Code=AISRSTOT ------

# The Mixed Procedure

#### Least Squares Means

| | | Analysis<br>Visit | Planned | | Standard | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Effect | RACEGRP | (N) | Treatment (N) | Estimate | Error | DF | t Value | Pr > t | 7 lmba | Torrow | Ilmnon |
| Filect | RACEGRE | (11) | (11) | ESCIMACE | FILOI | Dr | t value | PI / | Alpha | Lower | Upper |
| AVISIT*TRTPN*RACEGRP | All Other Races | 14 | 3 | -4.3684 | 1.6060 | 390 | -2.72 | 0.0068 | 0.05 | -7.5259 | -1.2109 |
| AVISIT*TRTPN*RACEGRP | White | 14 | 3 | -5.7832 | 0.8529 | 406 | -6.78 | <.0001 | 0.05 | -7.4599 | -4.1064 |
| AVISIT*TRTPN*RACEGRP | All Other Races | 21 | 1 | -13.4900 | 1.6638 | 398 | -8.11 | <.0001 | 0.05 | -16.7608 | -10.2191 |
| AVISIT*TRTPN*RACEGRP | White | 21 | 1 | -10.0518 | 0.9235 | 400 | -10.88 | <.0001 | 0.05 | -11.8674 | -8.2363 |
| AVISIT*TRTPN*RACEGRP | All Other Races | 21 | 2 | -15.6552 | 1.9656 | 433 | -7.96 | <.0001 | 0.05 | -19.5185 | -11.7918 |
| AVISIT*TRTPN*RACEGRP | White | 21 | 2 | -10.4459 | 0.9123 | 409 | -11.45 | <.0001 | 0.05 | -12.2393 | -8.6525 |
| AVISIT*TRTPN*RACEGRP | All Other Races | 21 | 3 | -8.2352 | 1.7156 | 389 | -4.80 | <.0001 | 0.05 | -11.6083 | -4.8622 |
| AVISIT*TRTPN*RACEGRP | White | 21 | 3 | -6.4527 | 0.9087 | 398 | -7.10 | <.0001 | 0.05 | -8.2391 | -4.6662 |
| AVISIT*TRTPN*RACEGRP | All Other Races | 28 | 1 | -13.8665 | 1.7467 | 394 | -7.94 | <.0001 | 0.05 | -17.3004 | -10.4326 |
| AVISIT*TRTPN*RACEGRP | White | 28 | 1 | -10.1758 | 0.9760 | 404 | -10.43 | <.0001 | 0.05 | -12.0944 | -8.2572 |
| AVISIT*TRTPN*RACEGRP | All Other Races | 28 | 2 | -14.8643 | 2.0891 | 437 | -7.12 | <.0001 | 0.05 | -18.9702 | -10.7584 |
| AVISIT*TRTPN*RACEGRP | White | 28 | 2 | -10.8890 | 0.9603 | 407 | -11.34 | <.0001 | 0.05 | -12.7767 | -9.0013 |
| AVISIT*TRTPN*RACEGRP | All Other Races | 28 | 3 | -8.8032 | 1.8058 | 391 | -4.87 | <.0001 | 0.05 | -12.3536 | -5.2529 |
| AVISIT*TRTPN*RACEGRP | White | 28 | 3 | -6.6365 | 0.9533 | 395 | -6.96 | <.0001 | 0.05 | -8.5106 | -4.7624 |
| AVISIT*TRTPN*RACEGRP | All Other Races | 35 | 1 | -14.0585 | 1.8441 | 403 | -7.62 | <.0001 | 0.05 | -17.6837 | -10.4333 |
| AVISIT*TRTPN*RACEGRP | White | 35 | 1 | -10.8714 | 1.0221 | 400 | -10.64 | <.0001 | 0.05 | -12.8808 | -8.8621 |
| AVISIT*TRTPN*RACEGRP | All Other Races | 35 | 2 | -18.2432 | 2.2321 | 447 | -8.17 | <.0001 | 0.05 | -22.6299 | -13.8565 |
| AVISIT*TRTPN*RACEGRP | White | 35 | 2 | -12.0993 | 1.0101 | 407 | -11.98 | <.0001 | 0.05 | -14.0849 | -10.1137 |
| AVISIT*TRTPN*RACEGRP | All Other Races | 35 | 3 | -9.4821 | 1.8927 | 392 | -5.01 | <.0001 | 0.05 | -13.2032 | -5.7609 |


# $$\tt STAT-3.2$$ MMRM Output for Test on Treatment by Race Interaction at Day 42 (Efficacy Sample)

#### The Mixed Procedure

#### Least Squares Means

| | | Analysis<br>Visit | Planned<br>Treatment | | Standard | | | | | _ | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Effect | RACEGRP | (N) | (N) | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| AVISIT*TRTPN*RACEGRP | White | 35 | 3 | -7.4198 | 0.9957 | 392 | -7.45 | <.0001 | 0.05 | -9.3775 | -5.4622 |
| AVISIT*TRTPN*RACEGRP | All Other Races | 42 | 1 | -16.2801 | 1.9359 | 397 | -8.41 | <.0001 | 0.05 | -20.0860 | -12.4743 |
| AVISIT*TRTPN*RACEGRP | White | 42 | 1 | -10.8032 | 1.0812 | 402 | -9.99 | <.0001 | 0.05 | -12.9286 | -8.6777 |
| AVISIT*TRTPN*RACEGRP | All Other Races | 42 | 2 | -16.4160 | 2.3407 | 424 | -7.01 | <.0001 | 0.05 | -21.0168 | -11.8152 |
| AVISIT*TRTPN*RACEGRP | White | 42 | 2 | -11.7167 | 1.0708 | 409 | -10.94 | <.0001 | 0.05 | -13.8216 | -9.6118 |
| AVISIT*TRTPN*RACEGRP | All Other Races | 42 | 3 | -10.9567 | 1.9920 | 390 | -5.50 | <.0001 | 0.05 | -14.8731 | -7.0403 |
| AVISIT*TRTPN*RACEGRP | White | 42 | 3 | -7.3172 | 1.0483 | 390 | -6.98 | <.0001 | 0.05 | -9.3781 | -5.2562 |
| 11/1011 11/11/1 14/02014 | ***** | | 9 | , . 0 = , = | 1.0100 | 000 | 0.00 | | 0.00 | J. 0 / 0 ± | 0.200 |

CENTANAFADINE

STAT-4.1.1

Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=KENWARDROGER (Efficacy Sample)

......

The Mixed Procedure

Model Information

Data Set WORK.INDATA
Dependent Variable CHG
Covariance Structure Unstructured
Subject Effect SUBJID
Estimation Method REML
Residual Variance Method None
Fixed Effects SE Method Kenward-Roger

Fixed Effects SE Method Kenward-Roger
Degrees of Freedom Method Kenward-Roger

Class Level Information

Class Levels Values

AVISITN 6 7 14 21 28 35 42

TRTPN 3 1 2 3

POOLCNTR 39

CENTANAFADINE

2 OF 18

STAT-4.1.1

Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=KENWARDROGER (Efficacy Sample)

The Mixed Procedure

Class Level Information

Class Levels Values

SUBJID 421



CENTANAFADINE 3 OF 18

PROTOCOL 405-201-00014 STAT-4.1.1

Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=KENWARDROGER (Efficacy Sample)

The Mixed Procedure



CENTANAFADINE

4 OF 18

STAT-4.1.1

Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=KENWARDROGER (Efficacy Sample)

......

The Mixed Procedure



CENTANAFADINE 5 OF 18

PROTOCOL 405-201-00014 STAT-4.1.1

Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=KENWARDROGER (Efficacy Sample)

The Mixed Procedure



CENTANAFADINE 6 OF 18 PROTOCOL 405-201-00014

STAT-4.1.1

Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=KENWARDROGER (Efficacy Sample)

The Mixed Procedure



CENTANAFADINE 7 OF 18 PROTOCOL 405-201-00014

STAT-4.1.1

Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=KENWARDROGER (Efficacy Sample)

The Mixed Procedure



| CENTANAFADINE 8 C | OF 18 |
|-------------------|-------|
|-------------------|-------|

PROTOCOL 405-201-00014 STAT-4.1.1

Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=KENWARDROGER (Efficacy Sample)

......

#### The Mixed Procedure

#### Dimensions

| Covariance | Parameters | 21 |
|-------------|------------|-----|
| Columns in | X | 73 |
| Columns in | Z | 0 |
| Subjects | | 421 |
| Max Obs per | Subject | 6 |

## Number of Observations

| Number | of | Observations | Read | 2227 |
|--------|----|--------------|----------|------|
| Number | of | Observations | Used | 2227 |
| Number | of | Observations | Not Used | 0 |

# Iteration History

| Iteration | Evaluations | -2 Res Log Like | Criterion |
|-----------|-------------|-----------------|------------|
| 0 | 1 | 15800.38727426 | |
| 1 | 2 | 13568.79752107 | 0.00031679 |
| 2 | 1 | 13567.17482444 | 0.00000418 |
| 3 | 1 | 13567.15460435 | 0.00000000 |

CENTANAFADINE 9 OF 18 PROTOCOL 405-201-00014

STAT-4.1.1

Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=KENWARDROGER (Efficacy Sample)

\_\_\_\_\_

The Mixed Procedure

Convergence criteria met.

Covariance Parameter Estimates

| Cov Parm | Subject | Estimate |
|----------|---------|----------|
| UN(1,1) | SUBJID | 43.6133 |
| UN(2,1) | SUBJID | 38.4610 |
| UN(2,2) | SUBJID | 70.3656 |
| UN(3,1) | SUBJID | 37.5232 |
| UN(3,2) | SUBJID | 59.9507 |
| UN(3,3) | SUBJID | 81.2761 |
| UN(4,1) | SUBJID | 39.2740 |
| UN(4,2) | SUBJID | 59.0315 |
| UN(4,3) | SUBJID | 73.7748 |
| UN(4,4) | SUBJID | 89.8567 |
| UN(5,1) | SUBJID | 38.9775 |
| UN(5,2) | SUBJID | 60.4118 |
| UN(5,3) | SUBJID | 72.5077 |
| UN(5,4) | SUBJID | 82.3971 |
| UN(5,5) | SUBJID | 97.7856 |
| UN(6,1) | SUBJID | 38.2789 |
| UN(6,2) | SUBJID | 60.0226 |
| UN(6,3) | SUBJID | 74.3151 |

| CENTANAFADINE | 10 OF 18 |
|---------------|----------|
|---------------|----------|


#### STAT-4.1.1

Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=KENWARDROGER (Efficacy Sample)

The Mixed Procedure

#### Covariance Parameter Estimates

| Cov Parm | Subject | Estimate |
|-----------|----------|----------|
| UN(6,4) | SUBJID | 84.3266 |
| UN(6,5) | SUBJID | 91.8307 |
| IIN (6 6) | SIIB.TTD | 108 84 |

## Fit Statistics

| -2 Res Log Likelihood | 13567.2 |
|--------------------------|---------|
| AIC (Smaller is Better) | 13609.2 |
| AICC (Smaller is Better) | 13609.6 |
| BIC (Smaller is Better) | 13694.0 |

# Null Model Likelihood Ratio Test

| DF | Chi-Square | Pr > ChiSq |
|----|------------|------------|
| 20 | 2233.23 | <.0001 |

CENTANAFADINE 11 OF 18 PROTOCOL 405-201-00014

STAT-4.1.1

Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=KENWARDROGER (Efficacy Sample)

\_\_\_\_\_

The Mixed Procedure

Solution for Fixed Effects

| | Pooled | Analysis | Planned | | 01 | | | |
|---|---|---|---|---|---|---|---|---|
| | Center | Visit | Treatment | | Standard | | | |
| Effect | Number | (N) | (N) | Estimate | Error | DF | t Value | Pr > t |
| Intercept | | | | 1.1270 | 4.7691 | 581 | 0.24 | 0.8133 |
| AVISITN | | 7 | | 0.5954 | 2.6832 | 341 | 0.22 | 0.8245 |
| AVISITN | | 14 | | -1.3583 | 2.4093 | 363 | -0.56 | 0.5733 |
| AVISITN | | 21 | | 0.8510 | 2.0449 | 353 | 0.42 | 0.6775 |
| AVISITN | | 28 | | -1.3535 | 1.7676 | 346 | -0.77 | 0.4444 |
| AVISITN | | 35 | | -0.6029 | 1.5610 | 337 | -0.39 | 0.6996 |
| AVISITN | | 42 | | 0 | | | | |
| TRTPN | | | 1 | -4.0055 | 1.2937 | 368 | -3.10 | 0.0021 |
| TRTPN | | | 2 | -4.4192 | 1.3220 | 378 | -3.34 | 0.0009 |
| TRTPN | | | 3 | 0 | | | | |
| AVISITN*TRTPN | | 7 | 1 | 2.0743 | 1.0975 | 335 | 1.89 | 0.0596 |
| AVISITN*TRTPN | | 7 | 2 | 2.6082 | 1.1265 | 339 | 2.32 | 0.0212 |
| AVISITN*TRTPN | | 7 | 3 | 0 | | | | |
| AVISITN*TRTPN | | 14 | 1 | 0.3557 | 0.9813 | 357 | 0.36 | 0.7172 |
| AVISITN*TRTPN | | 14 | 2 | 0.7686 | 1.0094 | 356 | 0.76 | 0.4469 |
| AVISITN*TRTPN | | 14 | 3 | 0 | | | | |
| AVISITN*TRTPN | | 21 | 1 | -0.01500 | 0.8285 | 348 | -0.02 | 0.9856 |
| AVISITN*TRTPN | | 21 | 2 | -0.07966 | 0.8542 | 350 | -0.09 | 0.9258 |
| AVISITN*TRTPN | | 21 | 3 | 0 | | | | |

CENTANAFADINE 12 OF 18 PROTOCOL 405-201-00014

STAT-4.1.1

Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=KENWARDROGER (Efficacy Sample)

\_\_\_\_\_

#### The Mixed Procedure

#### Solution for Fixed Effects

| | Pooled<br>Center | Analysis<br>Visit | Planned<br>Treatment | | Standard | | | |
|---|---|---|---|---|---|---|---|---|
| Effect | Number | (N) | (N) | Estimate | Error | DF | t Value | Pr > t |
| AVISITN*TRTPN | | 28 | 1 | 0.06611 | 0.7137 | 344 | 0.09 | 0.9263 |
| AVISITN*TRTPN | | 28 | 2 | -0.05910 | 0.7352 | 343 | -0.08 | 0.9360 |
| AVISITN*TRTPN | | 28 | 3 | 0 | | | | |
| AVISITN*TRTPN | | 35 | 1 | 0.2307 | 0.6270 | 335 | 0.37 | 0.7131 |
| AVISITN*TRTPN | | 35 | 2 | -0.8321 | 0.6479 | 335 | -1.28 | 0.1999 |
| AVISITN*TRTPN | | 35 | 3 | 0 | | | | |
| AVISITN*TRTPN | | 42 | 1 | 0 | | | | |
| AVISITN*TRTPN | | 42 | 2 | 0 | | | | |
| AVISITN*TRTPN | | 42 | 3 | 0 | | | | |
| POOLCNTR | | | | 1.7152 | 3.7658 | 428 | 0.46 | 0.6490 |
| POOLCNTR | | | | -5.1572 | 5.2435 | 403 | -0.98 | 0.3259 |
| POOLCNTR | | | | 1.6504 | 3.6560 | 432 | 0.45 | 0.6519 |
| POOLCNTR | | | | 0.5885 | 4.4348 | 413 | 0.13 | 0.8945 |
| POOLCNTR | | | | -3.9263 | 4.4129 | 414 | -0.89 | 0.3741 |
| POOLCNTR | | | | 1.2240 | 3.7770 | 428 | 0.32 | 0.7460 |
| POOLCNTR | | | | 0.8833 | 3.7274 | 429 | 0.24 | 0.8128 |
| POOLCNTR | | | | -2.1241 | 4.2789 | 416 | -0.50 | 0.6199 |
| POOLCNTR | | | | 1.9882 | 5.1695 | 403 | 0.38 | 0.7007 |
| POOLCNTR | | | | -3.3736 | 3.8277 | 426 | -0.88 | 0.3786 |

CENTANAFADINE 13 OF 18 PROTOCOL 405-201-00014

STAT-4.1.1

Dooled Applysia Dlanned

Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=KENWARDROGER (Efficacy Sample)

#### The Mixed Procedure

#### Solution for Fixed Effects

| | Pooled<br>Center | Analysis<br>Visit | Planned<br>Treatment | | Standard | | | |
|---|---|---|---|---|---|---|---|---|
| Effect | Number | (N) | (N) | Estimate | Error | DF | t Value | Pr > t |
| POOLCNTR | | | | -2.6399 | 4.1913 | 418 | -0.63 | 0.5291 |
| POOLCNTR | | | | -9.4424 | 5.1658 | 404 | -1.83 | 0.0683 |
| POOLCNTR | | | | -3.1314 | 4.3052 | 416 | -0.73 | 0.4674 |
| POOLCNTR | | | | 3.6852 | 4.0316 | 425 | 0.91 | 0.3612 |
| POOLCNTR | | | | -1.5147 | 4.0615 | 421 | -0.37 | 0.7094 |
| POOLCNTR | | | | -0.7002 | 4.5899 | 411 | -0.15 | 0.8788 |
| POOLCNTR | | | | -3.9140 | 4.1883 | 418 | -0.93 | 0.3506 |
| POOLCNTR | | | | 2.1512 | 4.8016 | 408 | 0.45 | 0.6544 |
| POOLCNTR | | | | -2.5698 | 4.8033 | 408 | -0.54 | 0.5929 |
| POOLCNTR | | | | 0.4082 | 3.9332 | 424 | 0.10 | 0.9174 |
| POOLCNTR | | | | -2.0848 | 4.1288 | 419 | -0.50 | 0.6139 |
| POOLCNTR | | | | 9.2093 | 4.8043 | 408 | 1.92 | 0.0560 |
| POOLCNTR | | | | 3.0940 | 3.9314 | 423 | 0.79 | 0.4317 |
| POOLCNTR | | | | -3.5346 | 3.9635 | 422 | -0.89 | 0.3730 |
| POOLCNTR | | | | -2.2842 | 4.1174 | 419 | -0.55 | 0.5793 |
| POOLCNTR | | | | 6.8249 | 4.3486 | 415 | 1.57 | 0.1173 |
| POOLCNTR | | | | -5.2814 | 4.4034 | 414 | -1.20 | 0.2311 |
| POOLCNTR | | | | -2.7571 | 4.2019 | 417 | -0.66 | 0.5121 |
| POOLCNTR | | | | 2.0058 | 3.6634 | 432 | 0.55 | 0.5843 |

CENTANAFADINE 14 OF 18 PROTOCOL 405-201-00014

STAT-4.1.1

Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=KENWARDROGER (Efficacy Sample)

\_\_\_\_\_

#### The Mixed Procedure

#### Solution for Fixed Effects

| | Pooled<br>Center | Analysis<br>Visit | Planned<br>Treatment | | Standard | | | |
|---|---|---|---|---|---|---|---|---|
| -cc . | | | | | | | | |
| Effect | Number | (N) | (N) | Estimate | Error | DF | t Value | Pr > t |
| POOLCNTR | | | | 3.0549 | 3.6512 | 431 | 0.84 | 0.4032 |
| POOLCNTR | | | | -2.0401 | 4.5650 | 411 | -0.45 | 0.6552 |
| POOLCNTR | | | | 1.7734 | 4.5671 | 411 | 0.39 | 0.6980 |
| POOLCNTR | | | | -4.4210 | 3.9066 | 427 | -1.13 | 0.2584 |
| POOLCNTR | | | | 0.6462 | 4.4087 | 414 | 0.15 | 0.8835 |
| POOLCNTR | | | | -0.5512 | 3.8270 | 427 | -0.14 | 0.8855 |
| POOLCNTR | | | | -1.6096 | 5.1715 | 403 | -0.31 | 0.7558 |
| POOLCNTR | | | | -3.2196 | 4.4113 | 414 | -0.73 | 0.4659 |
| POOLCNTR | | | | -3.8034 | 4.4030 | 413 | -0.86 | 0.3882 |
| POOLCNTR | | | | 0 | | | | |
| BASE*AVISITN | | 7 | | -0.1387 | 0.05917 | 381 | -2.34 | 0.0196 |
| BASE*AVISITN | | 14 | | -0.1179 | 0.07108 | 437 | -1.66 | 0.0979 |
| BASE*AVISITN | | 21 | | -0.2124 | 0.07568 | 436 | -2.81 | 0.0052 |
| BASE*AVISITN | | 28 | | -0.1613 | 0.07907 | 439 | -2.04 | 0.0419 |
| BASE*AVISITN | | 35 | | -0.2010 | 0.08284 | 444 | -2.43 | 0.0156 |
| BASE*AVISITN | | 42 | | -0.2232 | 0.08730 | 443 | -2.56 | 0.0109 |

CENTANAFADINE 15 OF 18 PROTOCOL 405-201-00014

#### STAT-4.1.1

Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=KENWARDROGER (Efficacy Sample)

The Mixed Procedure

Type 3 Tests of Fixed Effects

| | Num | Den | | |
|---------------|-----|-----|---------|--------|
| Effect | DF | DF | F Value | Pr > F |
| AVISITN | 5 | 353 | 1.23 | 0.2932 |
| TRTPN | 2 | 379 | 10.09 | <.0001 |
| AVISITN*TRTPN | 10 | 524 | 1.66 | 0.0881 |
| POOLCNTR | 38 | 380 | 2.12 | 0.0002 |
| BASE*AVISITN | 6 | 382 | 2.15 | 0.0468 |

# Estimates

| Ι | abel | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
|---|---|---|---|---|---|---|---|---|---|
| Ι | AY7 1 vs 3 | -1.9312 | 0.7960 | 381 | -2.43 | 0.0157 | 0.05 | -3.4963 | -0.3661 |
| Ι | AY7 2 vs 3 | -1.8111 | 0.7992 | 379 | -2.27 | 0.0240 | 0.05 | -3.3825 | -0.2396 |
| Ι | AY14 1 vs 3 | -3.6498 | 1.0171 | 373 | -3.59 | 0.0004 | 0.05 | -5.6498 | -1.6497 |
| Ι | AY14 2 vs 3 | -3.6506 | 1.0304 | 381 | -3.54 | 0.0004 | 0.05 | -5.6766 | -1.6246 |
| Ι | AY21 1 vs 3 | -4.0205 | 1.0982 | 369 | -3.66 | 0.0003 | 0.05 | -6.1801 | -1.8609 |
| Ι | AY21 2 vs 3 | -4.4989 | 1.1183 | 380 | -4.02 | <.0001 | 0.05 | -6.6978 | -2.2999 |
| Ι | AY28 1 vs 3 | -3.9394 | 1.1597 | 369 | -3.40 | 0.0008 | 0.05 | -6.2198 | -1.6589 |
| Ι | AY28 2 vs 3 | -4.4783 | 1.1797 | 378 | -3.80 | 0.0002 | 0.05 | -6.7980 | -2.1586 |

CENTANAFADINE 16 OF 18 PROTOCOL 405-201-00014

STAT-4.1.1

Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=KENWARDROGER (Efficacy Sample)

#### The Mixed Procedure

#### Estimates

| | | | Standard | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Label | | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| DAY35 | 1 vs 3 | -3.7747 | 1.2192 | 368 | -3.10 | 0.0021 | 0.05 | -6.1721 | -1.3774 |
| DAY35 | 2 vs 3 | -5.2513 | 1.2437 | 378 | -4.22 | <.0001 | 0.05 | -7.6968 | -2.8058 |
| DAY42 | 1 vs 3 | -4.0055 | 1.2937 | 368 | -3.10 | 0.0021 | 0.05 | -6.5494 | -1.4615 |
| DAY42 | 2 vs 3 | -4.4192 | 1.3220 | 378 | -3.34 | 0.0009 | 0.05 | -7.0186 | -1.8198 |

# Least Squares Means

| Effect | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
|---|---|---|---|---|---|---|---|---|---|---|
| AVISITN*TRTPN | 7 | 1 | -6.2099 | 0.6181 | 385 | -10.05 | <.0001 | 0.05 | -7.4251 | -4.9947 |
| AVISITN*TRTPN | 7 | 2 | -6.0897 | 0.6199 | 381 | -9.82 | <.0001 | 0.05 | -7.3085 | -4.8709 |
| AVISITN*TRTPN | 7 | 3 | -4.2786 | 0.6120 | 381 | -6.99 | <.0001 | 0.05 | -5.4820 | -3.0753 |
| AVISITN*TRTPN | 14 | 1 | -9.0936 | 0.7625 | 402 | -11.93 | <.0001 | 0.05 | -10.5925 | -7.5947 |
| AVISITN*TRTPN | 14 | 2 | -9.0945 | 0.7770 | 415 | -11.70 | <.0001 | 0.05 | -10.6218 | -7.5672 |
| AVISITN*TRTPN | 14 | 3 | -5.4438 | 0.7599 | 405 | -7.16 | <.0001 | 0.05 | -6.9376 | -3.9501 |
| AVISITN*TRTPN | 21 | 1 | -10.8348 | 0.8200 | 407 | -13.21 | <.0001 | 0.05 | -12.4468 | -9.2228 |
| AVISITN*TRTPN | 21 | 2 | -11.3132 | 0.8431 | 423 | -13.42 | <.0001 | 0.05 | -12.9703 | -9.6560 |

SOURCE: MMRMOUT; TABLE: statlaa.lis; RUN: 31AUG2020 08:32; ANALYSIS DATASET CREATED: 16JUN2020 08:14 PROGRAM: /opt/sas/Data/DAP/EB1020/P40520100014/STAT/Program.dev/DOC STAT/statl.sas

OPDC, NEW DRUG APPLICATION, IND # 119,361 CENTANAFADINE STAT-4.1.1 FINAL

CENTANAFADINE 17 OF 18 PROTOCOL 405-201-00014

STAT-4.1.1

Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=KENWARDROGER (Efficacy Sample)

The Mixed Procedure

Least Squares Means

| | Analysis<br>Visit | Planned<br>Treatment | | Standard | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Effect | (N) | (N) | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| AVISITN*TRTPN | 21 | 3 | -6.8143 | 0.8114 | 399 | -8.40 | <.0001 | 0.05 | -8.4095 | -5.2191 |
| AVISITN*TRTPN | 28 | 1 | -11.0222 | 0.8636 | 409 | -12.76 | <.0001 | 0.05 | -12.7198 | -9.3245 |
| AVISITN*TRTPN | 28 | 2 | -11.5611 | 0.8869 | 422 | -13.04 | <.0001 | 0.05 | -13.3044 | -9.8179 |
| AVISITN*TRTPN | 28 | 3 | -7.0828 | 0.8508 | 396 | -8.33 | <.0001 | 0.05 | -8.7554 | -5.4102 |
| AVISITN*TRTPN | 35 | 1 | -11.6110 | 0.9058 | 407 | -12.82 | <.0001 | 0.05 | -13.3916 | -9.8304 |
| AVISITN*TRTPN | 35 | 2 | -13.0876 | 0.9345 | 423 | -14.00 | <.0001 | 0.05 | -14.9245 | -11.2507 |
| AVISITN*TRTPN | 35 | 3 | -7.8362 | 0.8895 | 394 | -8.81 | <.0001 | 0.05 | -9.5850 | -6.0875 |
| AVISITN*TRTPN | 42 | 1 | -12.0791 | 0.9584 | 409 | -12.60 | <.0001 | 0.05 | -13.9632 | -10.1951 |
| AVISITN*TRTPN | 42 | 2 | -12.4928 | 0.9915 | 422 | -12.60 | <.0001 | 0.05 | -14.4418 | -10.5439 |
| AVISITN*TRTPN | 42 | 3 | -8.0736 | 0.9387 | 393 | -8.60 | <.0001 | 0.05 | -9.9192 | -6.2281 |

CENTANAFADINE 18 OF 18 PROTOCOL 405-201-00014

STAT-4.1.1

Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=KENWARDROGER (Efficacy Sample)

The Mixed Procedure

Tests of Effect Slices

| | Analysis | | | | |
|---------------|----------|-----|-----|---------|--------|
| | Visit | Num | Den | | |
| Effect | (N) | DF | DF | F Value | Pr > F |
| AVISITN*TRTPN | 7 | 2 | 380 | 3.70 | 0.0257 |
| AVISITN*TRTPN | 14 | 2 | 378 | 8.52 | 0.0002 |
| AVISITN*TRTPN | 21 | 2 | 377 | 10.00 | <.0001 |
| AVISITN*TRTPN | 28 | 2 | 377 | 8.80 | 0.0002 |
| AVISITN*TRTPN | 35 | 2 | 377 | 9.66 | <.0001 |
| AVISITN*TRTPN | 42 | 2 | 377 | 7.04 | 0.0010 |

CENTANAFADINE

STAT-4.1.2

Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=SATTERTHWAITE (Efficacy Sample)

The Mixed Procedure

Model Information

Data Set

Dependent Variable
CHG
Covariance Structure
Subject Effect
Estimation Method
Residual Variance Method
Fixed Effect SE Method
Degrees of Freedom Method
Satterthwaite

Class Level Information

Class Levels Values

AVISITN 6 7 14 21 28 35 42

TRTPN 3 1 2 3

POOLCNTR 39

CENTANAFADINE 2 OF 14 PROTOCOL 405-201-00014

STAT-4.1.2

Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=SATTERTHWAITE (Efficacy Sample)

.\_\_\_\_\_

------ Parameter Code=AISRSTOT -------

The Mixed Procedure

Class Level Information

Class Levels Values

SUBJID 421



CENTANAFADINE

3 OF 14

STAT-4.1.2

Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=SATTERTHWAITE (Efficacy Sample)

......

The Mixed Procedure




CENTANAFADINE 4 OF 14

STAT-4.1.2

Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=SATTERTHWAITE (Efficacy Sample)

\_\_\_\_\_\_

The Mixed Procedure



CENTANAFADINE 5 OF 14

PROTOCOL 405-201-00014 STAT-4.1.2

Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=SATTERTHWAITE (Efficacy Sample)

......

The Mixed Procedure



CENTANAFADINE 6 OF 14 PROTOCOL 405-201-00014

STAT-4.1.2

Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=SATTERTHWAITE (Efficacy Sample)

The Mixed Procedure



CENTANAFADINE 7 OF 14 PROTOCOL 405-201-00014

STAT-4.1.2

Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=SATTERTHWAITE (Efficacy Sample)

The Mixed Procedure



| CENTANAFADINE 8 OF |
|--------------------|
|--------------------|


STAT-4.1.2

Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=SATTERTHWAITE (Efficacy Sample)

#### The Mixed Procedure

#### Dimensions

| Covariance | Parameters | 21 |
|-------------|------------|-----|
| Columns in | X | 73 |
| Columns in | Z | 0 |
| Subjects | | 421 |
| Max Obs per | Subject | 6 |

## Number of Observations

| Number | of | Observations | Read | 2227 |
|--------|----|--------------|----------|------|
| Number | of | Observations | Used | 2227 |
| Number | of | Observations | Not Used | 0 |

# Iteration History

| Iteration | Evaluations | -2 Res Log Like | Criterion |
|-----------|-------------|-----------------|------------|
| 0 | 1 | 15800.38727426 | |
| 1 | 2 | 13568.79752107 | 0.00031679 |
| 2 | 1 | 13567.17482444 | 0.00000418 |
| 3 | 1 | 13567.15460435 | 0.00000000 |

CENTANAFADINE 9 OF 14 PROTOCOL 405-201-00014

STAT-4.1.2

Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=SATTERTHWAITE (Efficacy Sample)

The Mixed Procedure

Convergence criteria met.

Covariance Parameter Estimates

| Cov Parm | Subject | Estimate |
|----------|---------|----------|
| UN(1,1) | SUBJID | 43.6133 |
| UN(2,1) | SUBJID | 38.4610 |
| UN(2,2) | SUBJID | 70.3656 |
| UN(3,1) | SUBJID | 37.5232 |
| UN(3,2) | SUBJID | 59.9507 |
| UN(3,3) | SUBJID | 81.2761 |
| UN(4,1) | SUBJID | 39.2740 |
| UN(4,2) | SUBJID | 59.0315 |
| UN(4,3) | SUBJID | 73.7748 |
| UN(4,4) | SUBJID | 89.8567 |
| UN(5,1) | SUBJID | 38.9775 |
| UN(5,2) | SUBJID | 60.4118 |
| UN(5,3) | SUBJID | 72.5077 |
| UN(5,4) | SUBJID | 82.3971 |
| UN(5,5) | SUBJID | 97.7856 |
| UN(6,1) | SUBJID | 38.2789 |
| UN(6,2) | SUBJID | 60.0226 |
| UN(6,3) | SUBJID | 74.3151 |

| CENTANAFADINE | 10 OF 14 |
|------------------------|----------|

STAT-4.1.2

Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=SATTERTHWAITE (Efficacy Sample)

The Mixed Procedure

Covariance Parameter Estimates

| Cov Parm | Subject | Estimate |
|-----------|----------|----------|
| UN(6,4) | SUBJID | 84.3266 |
| UN(6,5) | SUBJID | 91.8307 |
| IIN (6 6) | SIIR.TTD | 108 84 |

## Fit Statistics

| -2 Res Log Likelihood | 13567.2 |
|--------------------------|---------|
| AIC (Smaller is Better) | 13609.2 |
| AICC (Smaller is Better) | 13609.6 |
| BIC (Smaller is Better) | 13694.0 |

# Null Model Likelihood Ratio Test

| DF | Chi-Square | Pr > ChiSo |
|----|------------|------------|
| 20 | 2233 23 | < 000 |

CENTANAFADINE 11 OF 14 PROTOCOL 405-201-00014

STAT-4.1.2

Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=SATTERTHWAITE (Efficacy Sample)

The Mixed Procedure

Type 3 Tests of Fixed Effects

| | Num | Den | | |
|---------------|-----|-----|---------|--------|
| Effect | DF | DF | F Value | Pr > F |
| AVISITN | 5 | 357 | 1.25 | 0.2860 |
| TRTPN | 2 | 379 | 10.10 | <.0001 |
| AVISITN*TRTPN | 10 | 356 | 1.68 | 0.0835 |
| POOLCNTR | 38 | 380 | 2.18 | 0.0001 |
| BASE*AVISITN | 6 | 378 | 2.19 | 0.0430 |

#### Estimates

| Label | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
|---|---|---|---|---|---|---|---|---|
| Habel | Boeimace | BITOI | DI | c varac | 11 / (0) | nipna | 50#61 | opper |
| DAY7 1 vs 3 | -1.9312 | 0.7958 | 381 | -2.43 | 0.0157 | 0.05 | -3.4959 | -0.3665 |
| DAY7 2 vs 3 | -1.8111 | 0.7989 | 379 | -2.27 | 0.0240 | 0.05 | -3.3820 | -0.2401 |
| DAY14 1 vs 3 | -3.6498 | 1.0169 | 373 | -3.59 | 0.0004 | 0.05 | -5.6493 | -1.6502 |
| DAY14 2 vs 3 | -3.6506 | 1.0301 | 381 | -3.54 | 0.0004 | 0.05 | -5.6760 | -1.6253 |
| DAY21 1 vs 3 | -4.0205 | 1.0980 | 369 | -3.66 | 0.0003 | 0.05 | -6.1796 | -1.8614 |
| DAY21 2 vs 3 | -4.4989 | 1.1179 | 380 | -4.02 | <.0001 | 0.05 | -6.6970 | -2.3008 |
| DAY28 1 vs 3 | -3.9394 | 1.1594 | 369 | -3.40 | 0.0008 | 0.05 | -6.2192 | -1.6596 |
| DAY28 2 vs 3 | -4.4783 | 1.1792 | 378 | -3.80 | 0.0002 | 0.05 | -6.7970 | -2.1596 |

CENTANAFADINE 12 OF 14 PROTOCOL 405-201-00014

STAT-4.1.2

Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=SATTERTHWAITE (Efficacy Sample)

#### The Mixed Procedure

#### Estimates

| | | | Standard | tandard | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Label | | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| DAY35 | 1 vs 3 | -3.7747 | 1.2186 | 368 | -3.10 | 0.0021 | 0.05 | -6.1711 | -1.3784 |
| DAY35 | 2 vs 3 | -5.2513 | 1.2430 | 378 | -4.22 | <.0001 | 0.05 | -7.6953 | -2.8074 |
| DAY42 | 1 vs 3 | -4.0055 | 1.2930 | 368 | -3.10 | 0.0021 | 0.05 | -6.5480 | -1.4630 |
| DAY42 | 2 vs 3 | -4.4192 | 1.3210 | 378 | -3.35 | 0.0009 | 0.05 | -7.0167 | -1.8217 |

# Least Squares Means

| Effect | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
|---|---|---|---|---|---|---|---|---|---|---|
| AVISITN*TRTPN | 7 | 1 | -6.2099 | 0.6166 | 385 | -10.07 | <.0001 | 0.05 | -7.4223 | -4.9975 |
| AVISITN*TRTPN | 7 | 2 | -6.0897 | 0.6184 | 381 | -9.85 | <.0001 | 0.05 | -7.3056 | -4.8738 |
| AVISITN*TRTPN | 7 | 3 | -4.2786 | 0.6107 | 381 | -7.01 | <.0001 | 0.05 | -5.4793 | -3.0780 |
| AVISITN*TRTPN | 14 | 1 | -9.0936 | 0.7613 | 402 | -11.95 | <.0001 | 0.05 | -10.5902 | -7.5971 |
| AVISITN*TRTPN | 14 | 2 | -9.0945 | 0.7757 | 415 | -11.72 | <.0001 | 0.05 | -10.6193 | -7.5697 |
| AVISITN*TRTPN | 14 | 3 | -5.4438 | 0.7587 | 405 | -7.18 | <.0001 | 0.05 | -6.9353 | -3.9524 |
| AVISITN*TRTPN | 21 | 1 | -10.8348 | 0.8189 | 407 | -13.23 | <.0001 | 0.05 | -12.4445 | -9.2251 |
| AVISITN*TRTPN | 21 | 2 | -11.3132 | 0.8418 | 423 | -13.44 | <.0001 | 0.05 | -12.9677 | -9.6586 |

SOURCE: MMRMOUT; TABLE: statlab.lis; RUN: 31AUG2020 08:32; ANALYSIS DATASET CREATED: 16JUN2020 08:14 PROGRAM: /opt/sas/Data/DAP/EB1020/P40520100014/STAT/Program.dev/DOC STAT/statl.sas

OPDC, NEW DRUG APPLICATION, IND # 119,361 CENTANAFADINE STAT-4.1.2 FINAL

CENTANAFADINE 13 OF 14 PROTOCOL 405-201-00014

STAT-4.1.2

Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=SATTERTHWAITE (Efficacy Sample)

The Mixed Procedure

Least Squares Means

| | Analysis<br>Visit | Planned<br>Treatment | | Standard | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Effect | (N) | (N) | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| AVISITN*TRTPN | 21 | 3 | -6.8143 | 0.8103 | 399 | -8.41 | <.0001 | 0.05 | -8.4073 | -5.2213 |
| AVISITN*TRTPN | 28 | 1 | -11.0222 | 0.8624 | 409 | -12.78 | <.0001 | 0.05 | -12.7175 | -9.3269 |
| AVISITN*TRTPN | 28 | 2 | -11.5611 | 0.8855 | 422 | -13.06 | <.0001 | 0.05 | -13.3017 | -9.8205 |
| AVISITN*TRTPN | 28 | 3 | -7.0828 | 0.8497 | 396 | -8.34 | <.0001 | 0.05 | -8.7533 | -5.4124 |
| AVISITN*TRTPN | 35 | 1 | -11.6110 | 0.9044 | 407 | -12.84 | <.0001 | 0.05 | -13.3890 | -9.8330 |
| AVISITN*TRTPN | 35 | 2 | -13.0876 | 0.9329 | 423 | -14.03 | <.0001 | 0.05 | -14.9214 | -11.2538 |
| AVISITN*TRTPN | 35 | 3 | -7.8362 | 0.8884 | 394 | -8.82 | <.0001 | 0.05 | -9.5828 | -6.0897 |
| AVISITN*TRTPN | 42 | 1 | -12.0791 | 0.9570 | 409 | -12.62 | <.0001 | 0.05 | -13.9603 | -10.1979 |
| AVISITN*TRTPN | 42 | 2 | -12.4928 | 0.9898 | 422 | -12.62 | <.0001 | 0.05 | -14.4384 | -10.5473 |
| AVISITN*TRTPN | 42 | 3 | -8.0736 | 0.9375 | 393 | -8.61 | <.0001 | 0.05 | -9.9168 | -6.2304 |
CENTANAFADINE 14 OF 14 PROTOCOL 405-201-00014

STAT-4.1.2

Proc Mixed Output for Change from Baseline in AISRS Total Score, MMRM (UN), DDFM=SATTERTHWAITE (Efficacy Sample)

The Mixed Procedure

Tests of Effect Slices

| | Analysis | | | | |
|---------------|----------|-----|-----|---------|--------|
| | Visit | Num | Den | | |
| Effect | (N) | DF | DF | F Value | Pr > F |
| AVISITN*TRTPN | 7 | 2 | 380 | 3.70 | 0.0257 |
| AVISITN*TRTPN | 14 | 2 | 378 | 8.52 | 0.0002 |
| AVISITN*TRTPN | 21 | 2 | 377 | 10.01 | <.0001 |
| AVISITN*TRTPN | 28 | 2 | 377 | 8.80 | 0.0002 |
| AVISITN*TRTPN | 35 | 2 | 377 | 9.67 | <.0001 |
| AVISITN*TRTPN | 42 | 2 | 377 | 7.05 | 0.0010 |

CENTANAFADINE 1 OF 6 PROTOCOL 405-201-00014

 $$\tt STAT-4.2$$  Proc GLM Output for Change from Baseline to Day 42 in AISRS Total Score, LOCF (Efficacy Sample)

\_\_\_\_\_

The GLM Procedure

Class Level Information

Class Levels Values
TRTPN 3 1 2 3

POOLCNTR 39

Number of Observations Read 421 Number of Observations Used 421

CENTANAFADINE 2 OF 6


# STAT-4.2 Proc GLM Output for Change from Baseline to Day 42 in AISRS Total Score, LOCF (Efficacy Sample)

The GLM Procedure

Dependent Variable: CHG Change from Baseline

| Source | | DF | Squar | | Mean | Square | F ' | Value | Pr > F |
|---|---|---|---|---|---|---|---|---|---|
| Model | | 41 | 8805.994 | 97 | 214 | .78037 | | 2.07 | 0.0002 |
| Error | | 379 | 39250.456 | 33 | 103 | .56321 | | | |
| Corrected Total | | 420 | 48056.451 | 31 | | | | | |
| | R-Square<br>0.183243 | | f Var<br>.7081 | Root M | | CHG Me | | | |
| Source | | DF | Type III | SS ! | Mean : | Square | F ' | Value | Pr > F |
| TRTPN<br>POOLCNTR | | 2<br>38 | 1454.3280<br>6862.1537 | | | 164026<br>582994 | | 7.02<br>1.74 | 0.0010<br>0.0053 |

280.694601

280.694601 2.71 0.1005

SOURCE: GLMOUT; TABLE: stat1b.lis; RUN: 31AUG2020 08:32; ANALYSIS DATASET CREATED: 16JUN2020 08:14 PROGRAM: /opt/sas/Data/DAP/EB1020/P40520100014/STAT/Program.dev/DOC\_STAT/stat1.sas OPDC, NEW DRUG APPLICATION, IND # 119,361 CENTANAFADINE STAT-4.2 FINAL

BASE

CENTANAFADINE 3 OF 6 PROTOCOL 405-201-00014

STAT-4.2

Proc GLM Output for Change from Baseline to Day 42 in AISRS Total Score, LOCF (Efficacy Sample)

### The GLM Procedure

| Level of | | СНО | } | BAS | SE |
|----------|-----|-------------|------------|------------|------------|
| TRTPN | N | Mean | Std Dev | Mean | Std Dev |
| 1 | 140 | -10.7071429 | 10.8359224 | 37.5857143 | 6.75041775 |
| 2 | 140 | -11.0571429 | 10.7125768 | 38.7642857 | 6.95578090 |
| 3 | 141 | -7.1347518 | 10.1624096 | 37.6453901 | 6.34837972 |

CENTANAFADINE 4 OF 6 PROTOCOL 405-201-00014

### STAT-4.2

Proc GLM Output for Change from Baseline to Day 42 in AISRS Total Score, LOCF (Efficacy Sample)

### The GLM Procedure Least Squares Means

| | | Standard | | LSMEAN |
|-------|-------------|-----------|---------|--------|
| TRTPN | CHG LSMEAN | Error | Pr > t | Number |
| 1 | 11 6011007 | 0.0465643 | . 0001 | 1 |
| 1 | -11.6211087 | 0.9465643 | <.0001 | 1 |
| 2 | -11.7874384 | 0.9518103 | <.0001 | 2 |
| 3 | -7.7408197 | 0.9407099 | <.0001 | 3 |

Least Squares Means for effect TRTPN Pr > |t| for H0: LSMean(i)=LSMean(j)

### Dependent Variable: CHG

| i/j | 1 | 2 | 3 |
|---|---|---|---|
| 1<br>2<br>3 | 0.8926<br>0.0016 | 0.8926 | 0.0016<br>0.0011 |
| TRTPN | CHG LSMEAN | 95% Confidence | ce Limits |
| 1 2 | -11.621109<br>-11.787438 | -13.482284<br>-13.658929 | -9.759933<br>-9.915948 |

CENTANAFADINE 5 OF 6 PROTOCOL 405-201-00014

STAT-4.2

Proc GLM Output for Change from Baseline to Day 42 in AISRS Total Score, LOCF (Efficacy Sample)

The GLM Procedure Least Squares Means

TRTPN CHG LSMEAN 95% Confidence Limits

3 -7.740820 -9.590484 -5.891156

Least Squares Means for Effect TRTPN

Difference
Between 95% Confidence Limits for
LSMean(i)-LSMean(j)

1 2 0.166330 -2.253380 2.586039
1 3 -3.880289 -6.279048 -1.481530
2 3 -4.046619 -6.461174 -1.632064

NOTE: To ensure overall protection level, only probabilities associated with pre-planned comparisons should be used.

CENTANAFADINE 6 OF 6 PROTOCOL 405-201-00014

STAT-4.2

Proc GLM Output for Change from Baseline to Day 42 in AISRS Total Score, LOCF (Efficacy Sample)

The GLM Procedure

Dependent Variable: CHG Change from Baseline

| Parameter | Estimate | Standard<br>Error | t Value | Pr > t |
|-----------|-------------|-------------------|---------|---------|
| 1 vs 3 | -3.88028896 | 1.21997068 | -3.18 | 0.0016 |
| 2 vs 3 | -4.04661870 | 1.22800435 | -3.30 | 0.0011 |

| CENTANAFADINE | 1 OF 6 |
|------------------------|--------|

STAT-4.3

Proc GLM Output for Change from Baseline to Day 42 in AISRS Total Score, OC (Efficacy Sample)

The GLM Procedure

Class Level Information

Class Levels Values
TRTPN 3 1 2 3

Number of Observations Read 421 Number of Observations Used 421

CENTANAFADINE 2 OF 6 PROTOCOL 405-201-00014

STAT-4.3

Proc GLM Output for Change from Baseline to Day 42 in AISRS Total Score, OC

(Efficacy Sample)

The GLM Procedure

Dependent Variable: CHG Change from Baseline

| Source | | DF | Sum<br>Squar | | ean So | quare | FV | /alue | Pr > F |
|---|---|---|---|---|---|---|---|---|---|
| Model | | 3 | 1943.841 | 21 | 647. | 94707 | | 5.86 | 0.0006 |
| Error | | 417 | 46112.610 | 10 | 110. | 58180 | | | |
| Corrected Total | | 420 | 48056.451 | 31 | | | | | |
| | R-Square | | f Var | Root MSI | | CHG Mea | | | |
| | 0.040449 | -109 | .2314 | 10.5157 | 9 | -9.62707 | /8 | | |
| Source | | DF | Type III | SS Me | ean So | quare | F V | /alue | Pr > F |
| TRTPN<br>BASE | | 2<br>1 | 1249.4050<br>618.3653 | | 624.70 | | | 5.65<br>5.59 | 0.0038<br>0.0185 |


STAT-4.3

Proc GLM Output for Change from Baseline to Day 42 in AISRS Total Score, OC (Efficacy Sample)

The GLM Procedure

| Level of | | CHC | G | BAS | SE |
|----------|-----|-------------|------------|------------|------------|
| TRTPN | N | Mean | Std Dev | Mean | Std Dev |
| 1 | 140 | -10.7071429 | 10.8359224 | 37.5857143 | 6.75041775 |
| 2 | 140 | -11.0571429 | 10.7125768 | 38.7642857 | 6.95578090 |
| 3 | 141 | -7.1347518 | 10.1624096 | 37.6453901 | 6.34837972 |


### STAT-4.3

Proc GLM Output for Change from Baseline to Day 42 in AISRS Total Score, OC (Efficacy Sample)

The GLM Procedure Least Squares Means

| | | Standard | LSMEAN | |
|-------|-------------|-----------|---------|--------|
| TRTPN | CHG LSMEAN | Error | Pr > t | Number |
| 1 | -10.7820438 | 0.8893105 | <.0001 | 1 |
| 2 | -10.9177347 | 0.8906994 | <.0001 | 2 |
| 3 | -7.1988014 | 0.8860032 | <.0001 | 3 |

Least Squares Means for effect TRTPN Pr > |t| for H0: LSMean(i)=LSMean(j)

### Dependent Variable: CHG

| i/j | 1 | 2 | 3 |
|---|---|---|---|
| 1<br>2<br>3 | 0.9143<br>0.0045 | 0.9143 | 0.0045<br>0.0033 |
| TRTPN | CHG LSMEAN | 95% Confidence | Limits |
| 1<br>2 | -10.782044<br>-10.917735 | -12.530134<br>-12.668555 | -9.033954<br>-9.166914 |


STAT-4.3

Proc GLM Output for Change from Baseline to Day 42 in AISRS Total Score, OC (Efficacy Sample)

......

The GLM Procedure Least Squares Means

TRTPN CHG LSMEAN 95% Confidence Limits

3 -7.198801 -8.940391 -5.457212

Least Squares Means for Effect TRTPN

Difference
Between 95% Confidence Limits for
i j Means LSMean(i)-LSMean(j)

1 2 0.135691 -2.341328 2.612710
1 3 -3.583242 -6.049479 -1.117006
2 3 -3.718933 -6.190945 -1.246921

NOTE: To ensure overall protection level, only probabilities associated with pre-planned comparisons should be used.


STAT-4.3

Proc GLM Output for Change from Baseline to Day 42 in AISRS Total Score, OC (Efficacy Sample)

The GLM Procedure

Dependent Variable: CHG Change from Baseline

| Parameter | Estimate | Standard<br>Error | t Value | Pr > t |
|-----------|-------------|-------------------|---------|---------|
| 1 vs 3 | -3.58324241 | 1.25465498 | -2.86 | 0.0045 |
| 2 vs 3 | -3.71893327 | 1.25759322 | -2.96 | 0.0033 |

CENTANAFADINE 1 OF 2


STAT-4.4
Proc GLM Output for Treatment by Center Interaction at Day 42 in AISRS Total Score, LOCF

(Efficacy Sample)

\_\_\_\_\_

The GLM Procedure

Class Level Information

Class Levels Values
TRTPN 3 1 2 3

POOLCNTR 39

Number of Observations Read 421 Number of Observations Used 421

CENTANAFADINE 2 OF 2 PROTOCOL 405-201-00014

STAT-4.4

Proc GLM Output for Treatment by Center Interaction at Day 42 in AISRS Total Score, LOCF (Efficacy Sample)

The GLM Procedure

Dependent Variable: CHG Change from Baseline

Sum of

| | DF | Square | s Mean | Square | F Value | Pr > F |
|---|---|---|---|---|---|---|
| | 117 | 17215.3087 | 7 14 | 7.13939 | 1.45 | 0.0067 |
| | 303 | 30841.1425 | 10 | 1.78595 | | |
| | 420 | 48056.4513 | 1 | | | |
| R-Square | Coef | f Var | Root MSE | CHG M | lean | |
| 0.358231 | -104 | .7971 | 10.08890 | -9.627 | 078 | |
| | DF | Type III S | S Mean | Square | F Value | Pr > F |
| | 2 | 475.23497 | 5 237 | .617487 | 2.33 | 0.0986 |
| | 38 | 6881.04792 | 3 181 | .080208 | 1.78 | 0.0046 |
| | 76 | 8409.31379 | 9 110 | .648866 | 1.09 | 0.3087 |
| | • | 303<br>420<br>R-Square Coef<br>0.358231 -104<br>DF<br>2<br>38 | 117 17215.30877 303 30841.14254 420 48056.45133 R-Square Coeff Var II 0.358231 -104.7971 33 DF Type III S8 2 475.234978 38 6881.047923 | 117 17215.30877 14 303 30841.14254 10 420 48056.45131 R-Square Coeff Var Root MSE 0.358231 -104.7971 10.08890 DF Type III SS Mean 2 475.234975 237 38 6881.047923 181 | 117 17215.30877 147.13939 303 30841.14254 101.78595 420 48056.45131 R-Square Coeff Var Root MSE CHG M 0.358231 -104.7971 10.08890 -9.627 DF Type III SS Mean Square 2 475.234975 237.617487 38 6881.047923 181.080208 | 117 17215.30877 147.13939 1.45 303 30841.14254 101.78595 420 48056.45131 R-Square Coeff Var Root MSE CHG Mean 0.358231 -104.7971 10.08890 -9.627078 DF Type III SS Mean Square F Value 2 475.234975 237.617487 2.33 38 6881.047923 181.080208 1.78 |

CENTANAFADINE 1 OF 4 PROTOCOL 405-201-00014

 ${\tt STAT-4.5.1}$  Summary of Mean Change at Day 42 from Baseline in AISRS Total Score By Center - LOCF (Efficacy Sample)

| | CTN SR 200MG | AISRS TOTAL SCORE_<br>CTN SR 400MG | PLACEBO | TREATMENT | |
|---|---|---|---|---|---|
| CENTER | N LS MEAN (SE) | N LS MEAN (SE) | N LS MEAN (SE) | COMPARISON | LS MEAN DIFFERENCE 1 |
| OVERALL | 140 -11.6 (0.95) | 140 -11.8 (0.95) | 141 -7.74 (0.94) | CTN SR 200MG VS. PLACEBO<br>CTN SR 400MG VS. PLACEBO | -3.88 (-6.28, -1.48)<br>-4.05 (-6.46, -1.63) |
| | 8 -5.26 (3.63) | 6 -10.1 (4.15) | 7 -5.83 (3.85) | CTN SR 200MG VS. PLACEBO<br>CTN SR 400MG VS. PLACEBO | 0.57 (-9.71, 10.85)<br>-4.23 (-15.3, 6.82) |
| | 1 -48.7 (10.2) | 1 -8.22 (10.2) | 1 -32.6 (10.2) | CTN SR 200MG VS. PLACEBO<br>CTN SR 400MG VS. PLACEBO | -16.2 (-44.2, 11.92)<br>24.35 (-3.73, 52.44) |
| | 11 -9.62 (3.06) | 13 -9.01 (2.81) | 12 -6.45 (2.91) | CTN SR 200MG VS. PLACEBO<br>CTN SR 400MG VS. PLACEBO | -3.18 (-11.5, 5.13)<br>-2.57 (-10.5, 5.39) |
| | 2 -12.6 (7.24) | 1 -2.74 (10.2) | 3 -7.95 (5.82) | CTN SR 200MG VS. PLACEBO<br>CTN SR 400MG VS. PLACEBO | -4.62 (-22.9, 13.66)<br>5.21 (-17.9, 28.30) |
| | 2 -17.5 (7.14) | 2 -30.1 (7.24) | 2 -2.90 (7.14) | CTN SR 200MG VS. PLACEBO<br>CTN SR 400MG VS. PLACEBO | -14.6 (-34.5, 5.27)<br>-27.2 (-47.2, -7.09) |
| | 7 -13.7 (3.84) | 8 -9.60 (3.58) | , | CTN SR 200MG VS. PLACEBO<br>CTN SR 400MG VS. PLACEBO | -12.0 (-23.0, -0.93)<br>-7.89 (-18.6, 2.84) |
| | 8 -6.71 (3.57) | 8 -11.4 (3.57) | 8 -7.37 (3.60) | CTN SR 400MG VS. PLACEBO | 0.66 (-9.33, 10.65)<br>-4.05 (-14.1, 5.95) |
| | 3 -8.54 (5.84) | 2 -7.61 (7.16) | | CTN SR 200MG VS. PLACEBO CTN SR 400MG VS. PLACEBO | -5.65 (-23.8, 12.48)<br>-4.72 (-24.7, 15.26) |
| | 1 -18.5 (10.1) | 1 6.32 (10.1) | 1 -4.45 (10.1) | CTN SR 400MG VS. PLACEBO | -14.1 (-42.2, 14.12)<br>10.78 (-17.4, 38.94) |
| | 5 -16.8 (4.52) | 6 -9.67 (4.12) | 6 -11.4 (4.12) | CTN SR 400MG VS. PLACEBO | -5.37 (-17.4, 6.67)<br>1.75 (-9.72, 13.21) |
| | 3 -13.7 (5.87) | 3 -11.1 (5.89) | 2 -3.10 (7.14) | CTN SR 200MG VS. PLACEBO<br>CTN SR 400MG VS. PLACEBO | -10.6 (-28.9, 7.57)<br>-7.97 (-26.2, 10.30) |

OVERALL TREATMENT DIFFERENCE IS DERIVED USING ANCOVA MODEL, WITH TREATMENT AND CENTER AS MAIN EFFECT AND BASELINE VALUE AS COVARIATE; BY CENTER DIFFERENCES ARE DERIVED USING ANCOVA MODEL, WITH TREATMENT AND CENTER AS MAIN EFFECT, TREATMENT BY CENTER INTERACTION, AND BASELINE VALUE AS COVARIATE.

NOTE: FOR ANALYSIS PURPOSE, SMALL CENTERS ARE POOLED TOGETHER.

CENTANAFADINE 2 OF 4 PROTOCOL 405-201-00014

STAT-4.5.1 Summary of Mean Change at Day 42 from Baseline in AISRS Total Score By Center - LOCF (Efficacy Sample)

\_\_\_\_AISRS TOTAL SCORE TREATMENT CENTER N LS MEAN (SE) N LS MEAN (SE) N LS MEAN (SE) COMPARISON LS MEAN DIFFERENCE 1 1 -1.84 (10.1) 1 -19.7 (10.1) 1 -18.7 (10.1) CTN SR 200MG VS. PLACEBO 16.84 (-11.2, 44.92) CTN SR 400MG VS. PLACEBO -1.00 (-29.1, 27.08) 2 -25.0 (7.14) 2 -15.6 (7.19) 3 -1.25 (5.84) CTN SR 200MG VS. PLACEBO -23.8 (-41.9, -5.64) CTN SR 400MG VS. PLACEBO -14.4 (-32.5, 3.76) 3 -10.5 (5.85) 4 -8.93 (5.05) 4 -5.67 (5.04) CTN SR 200MG VS. PLACEBO -4.80 (-20.0, 10.39) CTN SR 400MG VS. PLACEBO -3.26 (-17.3, 10.78) 3 -10.4 (5.84) 4 -11.4 (5.04) 3 -6.21 (5.83) CTN SR 200MG VS. PLACEBO -4.19 (-20.4, 12.05) CTN SR 400MG VS. PLACEBO -5.20 (-20.4, 9.96) 28.16 ( 8.31, 48.02) 2 -1.69 (7.15) 1 -17.7 (10.1) 2 -29.9 (7.15) CTN SR 200MG VS. PLACEBO CTN SR 400MG VS. PLACEBO 12.15 (-12.2, 36.47) 3 -16.3 (5.83) 2 -7.29 (7.18) 3 -10.2 (5.83) CTN SR 200MG VS. PLACEBO -6.14 (-22.4, 10.10) CTN SR 400MG VS. PLACEBO 2.89 (-15.4, 21.15) 1 0.55 (10.1) 2 -7.98 (7.14) 1 -9.32 (10.1) CTN SR 200MG VS. PLACEBO 9.87 (-18.2, 37.98) CTN SR 400MG VS. PLACEBO 1.34 (-23.0, 25.65) 1 -10.6 (10.1) 2 -4.48 (7.14) 1 -20.1 (10.1) CTN SR 200MG VS. PLACEBO 9.52 (-18.6, 37.60) CTN SR 400MG VS. PLACEBO 15.65 (-8.68, 39.97) 5 -11.2 (4.54) 5 -10.6 (4.53) 4 1.78 (5.17) CTN SR 200MG VS. PLACEBO -13.0 (-26.4, 0.38) CTN SR 400MG VS. PLACEBO -12.3 (-25.7, 1.06) 3 -14.6 (5.88) 3 -14.9 (5.91) 3 -12.1 (5.87) CTN SR 200MG VS. PLACEBO -2.49 (-18.7, 13.72) CTN SR 400MG VS. PLACEBO -2.76 (-19.0, 13.46) 2 -3.18 (7.14) 1 -13.3 (10.1) 1 6.39 (10.1) CTN SR 200MG VS. PLACEBO -9.56 (-34.0, 14.87) CTN SR 400MG VS. PLACEBO -19.7 (-47.8, 8.40) 4 -14.2 (5.08) 5 -4.19 (4.53) 4 -2.45 (5.05) CTN SR 200MG VS. PLACEBO -11.7 (-25.8, 2.34) CTN SR 400MG VS. PLACEBO -1.73 (-15.1, 11.62)

NOTE: FOR ANALYSIS PURPOSE, SMALL CENTERS ARE POOLED TOGETHER.

<sup>1</sup> OVERALL TREATMENT DIFFERENCE IS DERIVED USING ANCOVA MODEL, WITH TREATMENT AND CENTER AS MAIN EFFECT AND BASELINE VALUE AS COVARIATE; BY CENTER DIFFERENCES ARE DERIVED USING ANCOVA MODEL, WITH TREATMENT AND CENTER AS MAIN EFFECT, TREATMENT BY CENTER INTERACTION, AND BASELINE VALUE AS COVARIATE.

CENTANAFADINE

3 OF 4

 ${\tt STAT-4.5.1}\\ {\tt Summary of Mean Change at Day 42 from Baseline in AISRS Total Score}\\ {\tt By Center - LOCF (Efficacy Sample)}\\$ 

\_\_\_\_AISRS TOTAL SCORE CTN SR 200MG \_\_\_CTN SR 400MG\_\_\_ TREATMENT CENTER N LS MEAN (SE) N LS MEAN (SE) N LS MEAN (SE) COMPARISON LS MEAN DIFFERENCE 1 3 -10.2 (5.90) 5 -14.2 (4.52) 4 -17.8 (5.05) CTN SR 200MG VS. PLACEBO 7.58 (-7.74, 22.91) CTN SR 400MG VS. PLACEBO 3.54 (-9.81, 16.88) 3 -10.8 (5.85) 3 -14.5 (5.83) 3 -2.23 (5.83) CTN SR 200MG VS. PLACEBO -8.58 (-24.8, 7.67) CTN SR 400MG VS. PLACEBO -12.2 (-28.4, 3.98) 4.42 (-15.4, 24.27) 2 2.03 (7.20) 3 3.22 (5.95) 2 -2.39 (7.21) CTN SR 200MG VS. PLACEBO CTN SR 400MG VS. PLACEBO 5.60 (-12.5, 23.73) 6.23 (-13.6, 26.10) 2 -13.9 (7.14) 2 -19.0 (7.19) 2 -20.2 (7.13) CTN SR 200MG VS. PLACEBO 1.21 (-18.7, 21.13) CTN SR 400MG VS. PLACEBO 2 -13.0 (7.19) 3 -7.01 (5.89) 3 -11.3 (5.88) CTN SR 200MG VS. PLACEBO -1.66 (-19.8, 16.46) CTN SR 400MG VS. PLACEBO 4.28 (-11.9, 20.49) 12 -9.45 (2.91) 10 -14.6 (3.19) 11 -0.87 (3.05) CTN SR 200MG VS. PLACEBO -8.58 (-16.9, -0.29) CTN SR 400MG VS. PLACEBO -13.7 (-22.4, -5.01) 12 -5.08 (2.91) 11 -7.96 (3.04) 12 -5.60 (2.91) CTN SR 200MG VS. PLACEBO 0.52 (-7.59, 8.62) CTN SR 400MG VS. PLACEBO -2.37 (-10.7, 5.93) 2 -10.7 (7.15) 1 -0.39 (10.1) 2 -10.1 (7.14) CTN SR 200MG VS. PLACEBO -0.66 (-20.5, 19.19) CTN SR 400MG VS. PLACEBO 9.68 (-14.8, 34.15) 2 -0.69 (7.15) CTN SR 200MG VS. PLACEBO -16.3 (-36.3, 3.80) 2 -17.0 (7.19) 1 -0.29 (10.1) 0.40 (-24.1, 24.86) CTN SR 400MG VS. PLACEBO 5 -15.9 (4.52) 5 -26.3 (4.59) 5 -12.3 (4.55) CTN SR 200MG VS. PLACEBO -3.55 (-16.1, 9.03) CTN SR 400MG VS. PLACEBO -14.0 (-26.5, -1.41) 2 0.08 (7.13) 3 -8.71 (5.83) 1 -13.6 (10.1) CTN SR 200MG VS. PLACEBO 13.69 (-10.7, 38.10) 4.90 (-18.1, 27.88) CTN SR 400MG VS. PLACEBO 6 -16.2 (4.12) 5 -13.8 (4.52) 6 -5.68 (4.13) CTN SR 200MG VS. PLACEBO -10.5 (-22.0, 0.93) CTN SR 400MG VS. PLACEBO -8.17 (-20.2, 3.90)

NOTE: FOR ANALYSIS PURPOSE, SMALL CENTERS ARE POOLED TOGETHER.

<sup>1</sup> OVERALL TREATMENT DIFFERENCE IS DERIVED USING ANCOVA MODEL, WITH TREATMENT AND CENTER AS MAIN EFFECT AND BASELINE VALUE AS COVARIATE; BY CENTER DIFFERENCES ARE DERIVED USING ANCOVA MODEL, WITH TREATMENT AND CENTER AS MAIN EFFECT, TREATMENT BY CENTER INTERACTION, AND BASELINE VALUE AS COVARIATE.

CENTANAFADINE 4 OF 4 PROTOCOL 405-201-00014

 ${\tt STAT-4.5.1}\\ {\tt Summary of Mean Change at Day 42 from Baseline in AISRS Total Score}\\ {\tt By Center - LOCF (Efficacy Sample)}\\$ 

AISRS TOTAL SCORE

CTN SR 200MG
CTN SR 400MG
PLACEBO
TREATMENT

CENTER

N LS MEAN (SE)
N LS MEAN (SE)
N LS MEAN (SE)
COMPARISON
LS MEAN DIFFERENCE

1 -6.32 (10.1)
1 -15.6 (10.1)
1 -1.48 (10.1)
CTN SR 200MG VS. PLACEBO
-4.84 (-32.9, 23.24)
CTN SR 400MG VS. PLACEBO
-14.1 (-42.2, 13.98)
3 -7.77 (5.83)
1 -27.8 (10.1)
2 -14.0 (7.14)
CTN SR 200MG VS. PLACEBO
-14.1 (-42.2, 13.98)
CTN SR 400MG VS. PLACEBO
-13.8 (-38.1, 10.50)
1 -25.6 (10.1)
2 -13.8 (7.14)
3 -16.8 (5.84)
CTN SR 200MG VS. PLACEBO
-8.86 (-31.8, 14.09)

1 3.16 (10.1) 2 -9.65 (7.15) CTN SR 200MG VS. PLACEBO

CTN SR 400MG VS. PLACEBO

CTN SR 400MG VS. PLACEBO

2.93 (-15.2, 21.06)

-8.84 (-33.2, 15.48)

12.81 (-11.5, 37.14)

NOTE: FOR ANALYSIS PURPOSE, SMALL CENTERS ARE POOLED TOGETHER.

FILE: centera.lis, RUN: 31AUG2020 08:32; ANALYSIS DATASET CREATED: 16JUN2020 08:14
PROGRAM: /opt/sas/Data/DAP/EB1020/P40520100014/STAT/Program.dev/DOC\_STAT/center.sas
OPDC, NEW DRUG APPLICATION, IND # 119,361 CENTANAFADINE STAT-4.5.1 FINAL

1 -18.5 (10.1)

OVERALL TREATMENT DIFFERENCE IS DERIVED USING ANCOVA MODEL, WITH TREATMENT AND CENTER AS MAIN EFFECT AND BASELINE VALUE AS COVARIATE; BY CENTER DIFFERENCES ARE DERIVED USING ANCOVA MODEL, WITH TREATMENT AND CENTER AS MAIN EFFECT, TREATMENT BY CENTER INTERACTION, AND BASELINE VALUE AS COVARIATE.

CENTANAFADINE 1 OF 2 PROTOCOL 405-201-00014

 ${\tt STAT-4.5.2}$  Differences in Unadjusted Mean Changes of AISRS Total Score at Day 42 Among Treatment Groups By Center - LOCF (Efficacy Sample)

CTN SR 200MG VS. CTN SR 400MG VS. \_CTN SR 200M CTN SR 400MG \_\_PLACEBO\_\_\_ PLACEBO COUNTRY N MEAN¹ N MEAN¹ N MEAN¹ DIFF² CENTER USA 2 -18.00 2 -32.00 2 -2.50 -15.50

USA 2 -3.50 1 -12.00 1 8.00 -11.50

USA 2 -25.50 2 -17.00 3 -2.00 -33.50

USA 5 -16.20 5 -27.60 5 -13.20 -3.00

USA 12 -9.33 10 -14.70 11 -0.64 -8.70

USA 3 -7.67 1 -28.00 2 -14.50 6.83

USA 1 -6.00 1 -14.00 1 -1.00 -5.00

USA 3 -10.00 3 -14.67 3 -2.33 -7.67

USA 5 -12.00 5 -11.20 4 0.00 -12.00

USA 6 -16.00 5 -14.20 6 -5.17 -10.83

USA 7 -14.43 8 -10.00 6 -2.17 -10.83

USA 7 -14.43 8 -10.00 6 -2.17 -12.26

USA 3 -8.00 2 -8.50 2 -2.00 -6.00

USA 3 -11.00 4 -11.50 3 -6.00 -5.00

USA 8 -6.88 8 -11.63 8 -6.63 -0.25

USA 8 -4.25 6 -9.33 7 -5.00

USA 3 -11.33 4 -9.25 4 -5.75 -5.58

USA 1 -10.09 13 -9.46 12 -6.50 -3.59

USA 3 -13.33 3 -13.33 3 -11.00 -2.33

USA 1 -2.00 1 -20.00 1 -19.00 17.00 -29.50 -20.00 -15.00 -14.40 -14.06 -13.50 -13.00 -12.33 -11.20 -9.03 -7.83 -6.50 -6.17 -5.50 -5.00 -4.33 -3.50 -2.96 -2.55 -2.33 -2.15 -1.00

<sup>&</sup>lt;sup>1</sup> MEAN CHANGE FROM BASELINE AT DAY 42 (LOCF).

 $<sup>^{\</sup>rm 2}$  DIFFERENCE IN MEAN CHANGES AT DAY 42 BETWEEN TWO TREATMENT GROUPS. NOTE: FOR ANALYSIS PURPOSE, SMALL CENTERS ARE POOLED TOGETHER.


STAT-4.5.2

Prences in Unadjusted Mean Changes of AISRS Total Score at Day 42

Differences in Unadjusted Mean Changes of AISRS Total Score at Day 42 Among Treatment Groups By Center - LOCF (Efficacy Sample)

| | | _CTN | SR 200M | CTN | SR 400MG | PI | LACEBO | CTN SR 200MG VS.<br>PLACEBO | CTN SR 400MG VS.<br>PLACEBO |
|---|---|---|---|---|---|---|---|---|---|
| NTER | COUNTRY | N | MEAN 1 | N | MEAN¹ | N | MEAN 1 | DIFF <sup>2</sup> | DIFF <sup>2</sup> |
| | USA | 1 | 2.00 | 2 | -7.50 | 1 | -9.00 | 11.00 | 1.50 |
| | USA | 5 | -16.40 | 6 | -9.83 | 6 | -11.50 | -4.90 | 1.67 |
| | USA | 2 | -14.50 | 2 | -17.50 | 2 | -20.00 | 5.50 | 2.50 |
| | USA | 2 | -15.50 | 1 | 1.00 | 2 | -1.50 | -14.00 | 2.50 |
| | USA | 1 | -24.00 | 2 | -13.50 | 3 | -16.00 | -8.00 | 2.50 |
| | USA | 2 | -14.50 | 1 | -5.00 | 3 | -8.00 | -6.50 | 3.00 |
| | USA | 2 | 0.00 | 3 | -8.33 | 1 | -12.00 | 12.00 | 3.67 |
| | USA | 3 | -8.67 | 5 | -13.80 | 4 | -18.00 | 9.33 | 4.20 |
| | USA | 2 | -11.50 | 3 | -5.67 | 3 | -10.00 | -1.50 | 4.33 |
| | USA | 3 | -16.00 | 2 | -6.00 | 3 | -10.67 | -5.33 | 4.67 |
| | USA | 2 | 0.50 | 3 | 1.33 | 2 | -4.00 | 4.50 | 5.33 |
| | USA | 2 | -10.00 | 1 | -2.00 | 2 | -9.50 | -0.50 | 7.50 |
| | USA | 1 | -19.00 | 1 | 6.00 | 1 | -3.00 | -16.00 | 9.00 |
| | USA | 2 | -2.50 | 1 | -19.00 | 2 | -30.50 | 28.00 | 11.50 |
| | USA | 1 | -18.00 | 1 | 3.00 | 2 | -9.00 | -9.00 | 12.00 |
| | USA | 1 | -9.00 | 2 | -4.00 | 1 | -19.00 | 10.00 | 15.00 |
| | USA | 1 | -51.00 | 1 | -10.00 | 1 | -35.00 | -16.00 | 25.00 |

<sup>&</sup>lt;sup>1</sup> MEAN CHANGE FROM BASELINE AT DAY 42 (LOCF).

 $<sup>^{\</sup>rm 2}$  DIFFERENCE IN MEAN CHANGES AT DAY 42 BETWEEN TWO TREATMENT GROUPS. NOTE: FOR ANALYSIS PURPOSE, SMALL CENTERS ARE POOLED TOGETHER.

CENTANAFADINE 1 OF 24 PROTOCOL 405-201-00014

STAT-4.6

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, LOCF (Efficacy Sample)

The TTEST Procedure

| | Va | riable: CHG | (Change | from Baseline | e) | | |
|---|---|---|---|---|---|---|---|
| TRTI | PN N | Mean | Std Dev | Std Err | Minimum | Maximum | |
| 1<br>3<br>Difi | 137<br>139<br>f (1-2) | -5.3431<br>-3.5612<br>-1.7819 | 7.5542<br>6.6693<br>7.1223 | 0.6454<br>0.5657<br>0.8574 | -27.0000<br>-31.0000 | 12.0000<br>10.0000 | |
| TRTPN | Method | Mean | 95% CL | Mean | Std Dev | 95% CL S | td Dev |
| 1<br>3<br>Diff (1-2)<br>Diff (1-2) | Pooled<br>Satterthwaite | -5.3431<br>-3.5612<br>-1.7819<br>-1.7819 | -6.6194<br>-4.6797<br>-3.4699<br>-3.4716 | -2.4426<br>-0.0939 | 7.5542<br>6.6693<br>7.1223 | 6.7532<br>5.9667<br>6.5726 | 8.5724<br>7.5609<br>7.7730 |
| | Method | Variances | D. | F t Value | Pr > t | | |
| | Pooled<br>Satterthwaite | Equal<br>Unequal | 27<br>268.8 | | 0.0386<br>0.0388 | | |

CENTANAFADINE 2 OF 24


STAT-4.6

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, LOCF (Efficacy Sample)

------ Analysis Visit (N)=7 ------

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > FFolded F 136 138 1.28 0.1458

CENTANAFADINE 3 OF 24


### STAT-4.6

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, LOCF (Efficacy Sample)

### The TTEST Procedure

#### Variable: CHG (Change from Baseline) TRTPN Mean Std Dev Std Err Minimum Maximum 140 -8.1429 9.6018 0.8115 -48.0000 10.0000 141 -4.6879 7.7994 0.6568 -38.0000 8.0000 Diff (1-2) -3.4549 8.7440 1.0432 95% CL Mean TRTPN Method Mean Std Dev 95% CL Std Dev 1 -8.1429 -9.7473 -6.5384 9.6018 8.5936 10.8803 -5.9865 -3.3894 7.7994 -4.6879 6.9830 8.8336 Diff (1-2) Pooled -3.4549 -5.5085 -1.4013 8.7440 8.0747 9.5351 Diff (1-2) Satterthwaite -3.4549 -5.5105 -1.3994 Method Variances t Value Pr > |t| 279 -3.31 0.0010 Pooled Equal 267 -3.31 0.0011 Satterthwaite Unequal

CENTANAFADINE 4 OF 24


STAT-4.6

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, LOCF (Efficacy Sample)

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > FFolded F 139 140 1.52 0.0146

CENTANAFADINE 5 OF 24


### STAT-4.6

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, LOCF (Efficacy Sample)

The TTEST Procedure Variable: CHG (Change from Baseline)

| T | TRTPN | N | Mean | Std Dev | Std Err | Minimum | Maximum |
|---|---|---|---|---|---|---|---|
| 1<br>3<br>1 | L<br>3<br>Diff (1-2) | 140<br>141 | -9.5857<br>-5.8582<br>-3.7276 | 10.1450<br>8.7436<br>9.4678 | 0.8574<br>0.7363<br>1.1296 | -45.0000<br>-40.0000 | 10.0000 |
| TRTPN | Method | | Mean | 95% CL | Mean | Std Dev | 95% CL Std Dev |
| 1<br>3<br>Diff (1-2<br>Diff (1-2 | • | hwaite | -9.5857<br>-5.8582<br>-3.7276<br>-3.7276 | -7.3140 | -7.8905<br>-4.4024<br>-1.5039<br>-1.5025 | 10.1450<br>8.7436<br>9.4678 | 9.0797 11.4957<br>7.8284 9.9031<br>8.7431 10.3244 |

| Method | Variances | DF | t Value | Pr > t |
|---------------|-----------|--------|---------|---------|
| Pooled | Equal | 279 | -3.30 | 0.0011 |
| Satterthwaite | Unequal | 272.48 | -3.30 | 0.0011 |

CENTANAFADINE 6 OF 24


STAT-4.6

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, LOCF (Efficacy Sample)

------ Analysis Visit (N)=21 -----

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > FFolded F 139 140 1.35 0.0801

CENTANAFADINE 7 OF 24 PROTOCOL 405-201-00014

STAT-4.6

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, LOCF (Efficacy Sample)

------ Analysis Visit (N)=28 ------

The TTEST Procedure

| | Va | riable: CHG | (Change | from Baseline | <b>)</b> | |
|---|---|---|---|---|---|---|
| TRTP | N N | Mean S | Std Dev | Std Err | Minimum | Maximum |
| 1 | 140 | -9.8000 | 10.4587 | 0.8839 | -44.0000 | 13.0000 |
| 3 | 141 | -6.2553 | 8.9836 | 0.7566 | -37.0000 | 13.0000 |
| Diff | (1-2) | -3.5447 | 9.7465 | 1.1629 | | |
| TRTPN | Method | Mean | 95% CL | Mean | Std Dev | 95% CL Std Dev |
| 1 | | -9.8000 - | -11.5477 | -8.0523 | 10.4587 | 9.3605 11.8512 |
| 3 | | -6.2553 | -7.7511 | -4.7596 | 8.9836 | 8.0433 10.1749 |
| Diff (1-2) | Pooled | -3.5447 | -5.8338 | -1.2556 | 9.7465 | 9.0005 10.6283 |
| Diff (1-2) | Satterthwaite | -3.5447 | -5.8353 | -1.2541 | | |
| | Method | Variances | DI | f t Value | Pr > t | |
| | Pooled | Equal | 275 | 9 -3.05 | 0.0025 | |
| | Satterthwaite | Unequal | 272.23 | 1 -3.05 | 0.0025 | |

CENTANAFADINE 8 OF 24


STAT-4.6

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, LOCF (Efficacy Sample)

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > FFolded F 139 140 1.36 0.0735

CENTANAFADINE 9 OF 24


### STAT-4.6

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, LOCF (Efficacy Sample)

......

------ Analysis Visit (N)=35 ------

### The TTEST Procedure

## Variable: CHG (Change from Baseline)

| TRTPN | I N | Mean | Std Dev | Std Err | Minimum | Maximum |
|---|---|---|---|---|---|---|
| 1<br>3<br>Diff | 140<br>141<br>(1-2) | -6.9716 | 10.6376<br>9.5086<br>10.0869 | 0.8990<br>0.8008<br>1.2035 | -51.0000<br>-37.0000 | 11.0000<br>12.0000 |
| TRTPN | Method | Mean | 95% CL | Mean | Std Dev | 95% CL Std Dev |
| 1<br>3<br>Diff (1-2)<br>Diff (1-2) | Pooled<br>Satterthwaite | -10.2929<br>-6.9716<br>-3.3212<br>-3.3212 | -12.0704<br>-8.5548<br>-5.6903<br>-5.6914 | -8.5153<br>-5.3885<br>-0.9522<br>-0.9511 | 10.6376<br>9.5086<br>10.0869 | 9.5206 12.0539<br>8.5133 10.7695<br>9.3149 10.9995 |
| | Method | Variances | DI | F t Value | Pr > t | |
| | Pooled<br>Satterthwaite | Equal<br>Unequal | 275<br>275.12 | | 0.0062<br>0.0062 | |

CENTANAFADINE 10 OF 24


STAT-4.6

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, LOCF (Efficacy Sample)

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F Folded F 139 140 1.25 0.1862

CENTANAFADINE 11 OF 24


1

### STAT-4.6

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, LOCF (Efficacy Sample)

------ Analysis Visit (N)=42 ------

# The TTEST Procedure Variable: CHG (Change from Baseline)

#### TRTPN Mean Std Dev Std Err Minimum Maximum 140 -10.7071 10.8359 0.9158 -51.0000 11.0000 141 -7.1348 10.1624 0.8558 -39.0000 12.0000 Diff (1-2) -3.5724 10.5034 1.2532 95% CL Mean TRTPN Method Mean Std Dev 95% CL Std Dev -10.7071 -12.5178 -8.8964 10.8359 9.6981 12.2787 -7.1348 -8.8268 -5.4427 9.0987 11.5100 10.1624 Diff (1-2) Pooled -3.5724 -6.0392 -1.1055

10.5034

9.6995 11.4537

| Method | Variances | DF | t Value | Pr > t |
|---------------|-----------|--------|---------|---------|
| Pooled | Equal | 279 | -2.85 | 0.0047 |
| Satterthwaite | Unequal | 277.59 | -2.85 | 0.0047 |

SOURCE: TTESTLOCF; TABLE: stat1h.lis; RUN: 31AUG2020 08:32; ANALYSIS DATASET CREATED: 16JUN2020 08:14 PROGRAM: /opt/sas/Data/DAP/EB1020/P40520100014/STAT/Program.dev/DOC STAT/stat1.sas OPDC, NEW DRUG APPLICATION, IND # 119,361 CENTANAFADINE STAT-4.6

Diff (1-2) Satterthwaite -3.5724 -6.0399 -1.1049

CENTANAFADINE 12 OF 24


STAT-4.6

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, LOCF (Efficacy Sample)

.....

------ Analysis Visit (N)=42 -----

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F Folded F 139 140 1.14 0.4493

CENTANAFADINE 13 OF 24


STAT-4.6

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, LOCF (Efficacy Sample)

------ Analysis Visit (N)=7 ------

The TTEST Procedure

| | Va | riable: CHG | (Change | from Baseline | ∍) | | |
|---|---|---|---|---|---|---|---|
| TRTPI | N N | Mean | Std Dev | Std Err | Minimum | Maximum | |
| 2 | 139 | -5.4460 | 6.6389 | 0.5631 | -24.0000 | 9.0000 | |
| 3 | 139 | -3.5612 | 6.6693 | 0.5657 | -31.0000 | 10.0000 | |
| Diff | (1-2) | -1.8849 | 6.6541 | 0.7982 | | | |
| TRTPN | Method | Mean | 95% CL | Mean | Std Dev | 95% CL St | d Dev |
| 2 | | -5.4460 | -6.5595 | -4.3326 | 6.6389 | 5.9395 | 7.5264 |
| 3 | | -3.5612 | -4.6797 | -2.4426 | 6.6693 | 5.9667 | 7.5609 |
| Diff (1-2) | Pooled | -1.8849 | -3.4562 | -0.3136 | 6.6541 | 6.1423 | 7.2597 |
| Diff (1-2) | Satterthwaite | -1.8849 | -3.4562 | -0.3136 | | | |
| | Method | Variances | D! | F t Value | Pr > t | | |
| | Pooled | Equal | 27 | | | | |
| | Satterthwaite | Unequal | 275.9 | 9 -2.36 | 0.0189 | | |

CENTANAFADINE 14 OF 24


STAT-4.6

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, LOCF (Efficacy Sample)

------ Analysis Visit (N)=7 ------

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F Folded F 138 138 1.01 0.9572

CENTANAFADINE 15 OF 24


STAT-4.6

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, LOCF (Efficacy Sample)

The TTEST Procedure

| | V | ariable: CHG | (Change | from Baseline | e) | | |
|---|---|---|---|---|---|---|---|
| TRTE | PN N | Mean S | Std Dev | Std Err | Minimum | Maximum | |
| 2<br>3<br>Diff | 140<br>141 | -8.1143<br>-4.6879<br>-3.4263 | 8.1850<br>7.7994<br>7.9938 | 0.6918<br>0.6568<br>0.9537 | -35.0000<br>-38.0000 | 12.0000<br>8.0000 | |
| TRTPN | Method | Mean | 95% CL | Mean | Std Dev | 95% CL Std | l Dev |
| 2<br>3<br>Diff (1-2)<br>Diff (1-2) | Pooled<br>Satterthwaite | -8.1143<br>-4.6879<br>-3.4263<br>-3.4263 | -9.4820<br>-5.9865<br>-5.3038<br>-5.3041 | -6.7466<br>-3.3894<br>-1.5489<br>-1.5485 | 8.1850<br>7.7994<br>7.9938 | 6.9830 8 | 0.2748<br>0.8336<br>0.7171 |
| | Method | Variances | DI | F t Value | Pr > t | | |
| | Pooled<br>Satterthwait | Equal<br>e Unequal | 279<br>278 1 | | 0.0004 | | |
CENTANAFADINE 16 OF 24


STAT-4.6

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, LOCF (Efficacy Sample)

\_\_\_\_\_

------ Analysis Visit (N)=14 ------

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > FFolded F 139 140 1.10 0.5693

CENTANAFADINE 17 OF 24


## STAT-4.6

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, LOCF (Efficacy Sample)

......

### The TTEST Procedure

## Variable: CHG (Change from Baseline)

| TRTPI | ı N | Mean | Std Dev | Std Err | Minimum | Maximum |
|---|---|---|---|---|---|---|
| 2<br>3<br>Diff | 140<br>141<br>(1-2) | -10.1071<br>-5.8582<br>-4.2490 | 9.2088<br>8.7436<br>8.9784 | 0.7783<br>0.7363<br>1.0712 | -34.0000<br>-40.0000 | 17.0000<br>11.0000 |
| TRTPN | Method | Mean | 95% CL | Mean | Std Dev | 95% CL Std Dev |
| 2<br>3<br>Diff (1-2)<br>Diff (1-2) | Pooled<br>Satterthwaite | -10.1071<br>-5.8582<br>-4.2490<br>-4.2490 | -11.6459<br>-7.3140<br>-6.3577<br>-6.3581 | -8.5683<br>-4.4024<br>-2.1403<br>-2.1399 | 9.2088<br>8.7436<br>8.9784 | 8.2418 10.4349<br>7.8284 9.9031<br>8.2912 9.7907 |
| | Method | Variances | s Di | F t Value | Pr > t | |
| | Pooled<br>Satterthwaite | Equal<br>Unequal | 278.03 | | <.0001<br><.0001 | |

CENTANAFADINE 18 OF 24


STAT-4.6

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, LOCF (Efficacy Sample)

------ Analysis Visit (N)=21 ------

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F Folded F 139 140 1.11 0.5411

CENTANAFADINE 19 OF 24


STAT-4.6

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, LOCF (Efficacy Sample)

------ Analysis Visit (N)=28 ------

The TTEST Procedure

Variable: CHG (Change from Baseline)

| | TRTPN | | N | Mean | Std Dev | Std Err | Minimum | Maximum |
|---|---|---|---|---|---|---|---|---|
| | 2<br>3<br>Diff | (1-2) | 140<br>141 | -10.2714<br>-6.2553<br>-4.0161 | 9.6387<br>8.9836<br>9.3157 | 0.8146<br>0.7566<br>1.1115 | -42.0000<br>-37.0000 | 7.0000<br>13.0000 |
| TRTPN | | Method | | Mean | 95% CL | Mean | Std Dev | 95% CL Std Dev |
| 2<br>3<br>Diff (1-<br>Diff (1- | | Pooled<br>Satterth | waite | -10.2714<br>-6.2553<br>-4.0161<br>-4.0161 | -11.8821<br>-7.7511<br>-6.2040<br>-6.2046 | -8.6608<br>-4.7596<br>-1.8282<br>-1.8276 | 9.6387<br>8.9836<br>9.3157 | 8.6266 10.9220<br>8.0433 10.1749<br>8.6028 10.1586 |
| | | Metho | d | Variances | DI | f t Value | Pr > t | |
| | | Poole<br>Satte | d<br>rthwaite | Equal<br>Unequal | 279<br>277.3 | | 0.0004 | |

CENTANAFADINE 20 OF 24


STAT-4.6

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, LOCF (Efficacy Sample)

------ Analysis Visit (N)=28 ------

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F Folded F 139 140 1.15 0.4067

CENTANAFADINE 21 OF 24


2

## STAT-4.6

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, LOCF (Efficacy Sample)

------ Analysis Visit (N)=35 ------

# The TTEST Procedure Variable: CHG (Change from Baseline)

#### TRTPN Mean Std Dev Std Err Minimum Maximum 140 -11.4000 10.1689 0.8594 -40.0000 10.0000 141 -6.9716 9.5086 0.8008 -37.0000 12.0000 Diff (1-2) -4.4284 9.8431 1.1744 95% CL Mean TRTPN Method Mean Std Dev 95% CL Std Dev -11.4000 -13.0992 -9.7008 10.1689 9.1011 11.5229 -6.9716 -8.5548 -5.3885 9.5086 8.5133 10.7695

9.8431 9.0898 10.7337

| Method | Variances | DF | t Value | Pr > t |
|---------------|-----------|--------|---------|---------|
| Pooled | Equal | 279 | -3.77 | 0.0002 |
| Satterthwaite | Unequal | 277.47 | -3.77 | 0.0002 |

SOURCE: TTESTLOCF; TABLE: stat1h.lis; RUN: 31AUG2020 08:32; ANALYSIS DATASET CREATED: 16JUN2020 08:14 PROGRAM: /opt/sas/Data/DAP/EB1020/P40520100014/STAT/Program.dev/DOC STAT/stat1.sas OPDC, NEW DRUG APPLICATION, IND # 119,361 CENTANAFADINE STAT-4.6

Diff (1-2) Pooled -4.4284 -6.7402 -2.1166

Diff (1-2) Satterthwaite -4.4284 -6.7408 -2.1160

CENTANAFADINE 22 OF 24


STAT-4.6

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, LOCF (Efficacy Sample)

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F
Folded F 139 140 1.14 0.4286

CENTANAFADINE 23 OF 24 PROTOCOL 405-201-00014

STAT-4.6

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, LOCF (Efficacy Sample)

The TTEST Procedure

| | | Va | riable: CHG | (Change | from Baselin | e) | |
|---|---|---|---|---|---|---|---|
| TI | RTPN | N | Mean | Std Dev | Std Err | Minimum | Maximum |
| 2<br>3<br>D: | iff (1-2) | 140<br>141 | -7.1348 | 10.7126<br>10.1624<br>10.4401 | 0.9054<br>0.8558<br>1.2456 | -41.0000<br>-39.0000 | 11.0000<br>12.0000 |
| TRTPN | Method | | Mean | 95% CL | Mean | Std Dev | 95% CL Std Dev |
| 2<br>3<br>Diff (1-2)<br>Diff (1-2) | | hwaite | -7.1348 | -12.8472<br>-8.8268<br>-6.3744<br>-6.3749 | -5.4427<br>-1.4704 | 10.7126<br>10.1624<br>10.4401 | 9.5877 12.1389<br>9.0987 11.5100<br>9.6411 11.3847 |
| | Meth | od | Variances | D1 | F t Value | Pr > t | |
| | Pool | ed<br>erthwaite | Equal<br>Unequal | 279<br>278.01 | | | |

CENTANAFADINE 24 OF 24


STAT-4.6

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, LOCF (Efficacy Sample)

------ Analysis Visit (N)=42 ------

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F Folded F 139 140 1.11 0.5341

CENTANAFADINE 1 OF 24


## STAT-4.7

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, OC (Efficacy Sample)

------ Analysis Visit (N)=7 ------

## The TTEST Procedure

| | Va | riable: CHG | (Change | from Baseline | <b>)</b> | |
|---|---|---|---|---|---|---|
| TRTPN | N N | Mean | Std Dev | Std Err | Minimum | Maximum |
| 1 | 137 | -5.3431 | 7.5542 | 0.6454 | -27.0000 | 12.0000 |
| 3 | 139 | -3.5612 | 6.6693 | 0.5657 | -31.0000 | 10.0000 |
| Diff | (1-2) | -1.7819 | 7.1223 | 0.8574 | | |
| TRTPN | Method | Mean | 95% CL | Mean | Std Dev | 95% CL Std Dev |
| 1 | | -5.3431 | -6.6194 | -4.0668 | 7.5542 | 6.7532 8.5724 |
| 3 | | -3.5612 | -4.6797 | -2.4426 | 6.6693 | 5.9667 7.5609 |
| Diff (1-2) | Pooled | -1.7819 | -3.4699 | -0.0939 | 7.1223 | 6.5726 7.7730 |
| Diff (1-2) | Satterthwaite | -1.7819 | -3.4716 | -0.0922 | | |
| | Method | Variances | Di | F t Value | Pr > t | |
| | Pooled | Equal | 27 | 4 -2.08 | 0.0386 | |
| | Satterthwaite | Unequal | 268.8 | 5 -2.08 | 0.0388 | |

CENTANAFADINE 2 OF 24 PROTOCOL 405-201-00014

STAT-4.7

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, OC (Efficacy Sample)

------ Analysis Visit (N)=7 ------

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > FFolded F 136 138 1.28 0.1458

CENTANAFADINE 3 OF 24

PROTOCOL 405-201-00014 STAT-4.7

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, OC (Efficacy Sample)

The TTEST Procedure

| | | | Va | riable: CHG | (Change | from Baseline | ∋) | |
|---|---|---|---|---|---|---|---|---|
| | TRTPN | ī | N | Mean | Std Dev | Std Err | Minimum | Maximum |
| | 1 3 | | 132<br>132 | -8.5606<br>-4.8561 | 9.7042<br>7.9070 | 0.8446<br>0.6882 | -48.0000<br>-38.0000 | 10.0000 |
| | Diff | (1-2) | 132 | -3.7045 | 8.8514 | 1.0895 | -30.0000 | 8.0000 |
| TRTPN | | Method | | Mean | 95% CL | Mean | Std Dev | 95% CL Std Dev |
| 1 3 | | | | -8.5606<br>-4.8561 | -10.2315<br>-6.2175 | -6.8897<br>-3.4946 | 9.7042<br>7.9070 | 8.6579 11.0404<br>7.0545 8.9958 |
| Diff (1 | | Pooled | | -3.7045 | -5.8499 | | 8.8514 | 8.1540 9.6801 |
| Diff (1 | -2) | Satterth | walte | -3.7045 | -5.8503 | -1.5588 | | |
| | | Metho | d | Variances | DI | F t Value | Pr > t | |
| | | Poole<br>Satte | d<br>rthwaite | Equal<br>Unequal | 262<br>251.73 | | | |

CENTANAFADINE 4 OF 24


STAT-4.7

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, OC (Efficacy Sample)

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > FFolded F 131 131 1.51 0.0197

CENTANAFADINE 5 OF 24


STAT-4.7

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, OC (Efficacy Sample)

------ Analysis Visit (N)=21 ------

The TTEST Procedure

| | | | Variable: | CHG (Change | from Baselin | e) | |
|---|---|---|---|---|---|---|---|
| | TRTPN | N | Mean | Std Dev | Std Err | Minimum | Maximum |
| | 1 | 127 | | | 0.9273 | -45.0000 | 10.0000 |
| | 3<br>Diff ( | 132 | -5.9924<br>-3.9761 | | 0.7740<br>1.2041 | -40.0000 | 11.0000 |
| TRTPN | | Method | Mea | n 95% C | L Mean | Std Dev | 95% CL Std Dev |
| 1 | | | -9.968 | 5 -11.8036 | -8.1334 | 10.4501 | 9.3038 11.9212 |
| 3 | | | -5.992 | 4 -7.5236 | -4.4613 | 8.8925 | 7.9337 10.1169 |
| Diff (1- | -2) | Pooled | -3.976 | 1 -6.3473 | -1.6049 | 9.6875 | 8.9175 10.6042 |
| Diff (1- | -2) | Satterthwait | e -3.976 | 1 -6.3551 | -1.5971 | | |
| | | Method | Vari | ances | DF t Value | Pr > t | |
| | | Pooled<br>Satterthw | Equa<br>aite Uneq | | 57 -3.30<br>28 -3.29 | | |

SOURCE: TTESTOC; TABLE: stat1i.lis; RUN: 31AUG2020 08:32; ANALYSIS DATASET CREATED: 16JUN2020 08:14 PROGRAM: /opt/sas/Data/DAP/EB1020/P40520100014/STAT/Program.dev/DOC STAT/stat1.sas OPDC, NEW DRUG APPLICATION, IND # 119,361 CENTANAFADINE STAT-4.7 FINAL

CENTANAFADINE 6 OF 24


STAT-4.7

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, OC (Efficacy Sample)

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > FFolded F 126 131 1.38 0.0680

CENTANAFADINE 7 OF 24


STAT-4.7

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, OC (Efficacy Sample)

The TTEST Procedure

| | Va | riable: CHG | (Change | from Baselin | e) | |
|---|---|---|---|---|---|---|
| TRTP | PN N | Mean | Std Dev | Std Err | Minimum | Maximum |
| 1<br>3<br>Diff | 122<br>130 | -10.0492<br>-6.4462<br>-3.6030 | 10.4580<br>9.1313<br>9.7959 | 0.9468<br>0.8009<br>1.2348 | -44.0000<br>-37.0000 | 13.0000<br>13.0000 |
| TRTPN | Method | Mean | 95% CL | Mean | Std Dev | 95% CL Std Dev |
| 1<br>3<br>Diff (1-2)<br>Diff (1-2) | Pooled<br>Satterthwaite | -10.0492<br>-6.4462<br>-3.6030<br>-3.6030 | -11.9237<br>-8.0307<br>-6.0349<br>-6.0459 | | 10.4580<br>9.1313<br>9.7959 | 9.2900 11.9645<br>8.1400 10.3996<br>9.0073 10.7369 |
| | Method | Variances | D | F t Value | Pr > t | |
| | Pooled<br>Satterthwaite | Equal<br>Unequal | 25<br>240.5 | | 0.0038<br>0.0040 | |

CENTANAFADINE 8 OF 24


STAT-4.7

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, OC (Efficacy Sample)

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > FFolded F 121 129 1.31 0.1299

CENTANAFADINE 9 OF 24


STAT-4.7

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, OC (Efficacy Sample)

------ Analysis Visit (N)=35 ------

The TTEST Procedure

| | Vā | ariable: CHG | (Change | from Baselin | e) | |
|---|---|---|---|---|---|---|
| TRTPN | N N | Mean | Std Dev | Std Err | Minimum | Maximum |
| 1<br>3<br>Diff | 115<br>125<br>(1-2) | -10.1391<br>-7.1840<br>-2.9551 | 10.5945<br>9.3657<br>9.9732 | 0.9879<br>0.8377<br>1.2887 | -51.0000<br>-37.0000 | 11.0000<br>12.0000 |
| TRTPN | Method | Mean | 95% CL | Mean | Std Dev | 95% CL Std Dev |
| 1<br>3<br>Diff (1-2)<br>Diff (1-2) | Pooled<br>Satterthwaite | -10.1391<br>-7.1840<br>-2.9551<br>-2.9551 | -12.0962<br>-8.8420<br>-5.4938<br>-5.5074 | -0.4165 | 10.5945<br>9.3657<br>9.9732 | 9.3797 12.1737<br>8.3310 10.6962<br>9.1521 10.9574 |
| | Method | Variance | s D | F t Value | Pr > t | |
| | Pooled<br>Satterthwaite | Equal<br>Unequal | 23<br>228.3 | | | |

CENTANAFADINE 10 OF 24


STAT-4.7

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, OC (Efficacy Sample)

------ Analysis Visit (N)=35 ------

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F Folded F 114 124 1.28 0.1789

CENTANAFADINE 11 OF 24


STAT-4.7

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, OC (Efficacy Sample)

The TTEST Procedure

| | | Variable: CHG | (Change | from Baselin | e) | |
|---|---|---|---|---|---|---|
| TRTP | N N | Mean | Std Dev | Std Err | Minimum | Maximum |
| 1 3 | 113<br>123 | -10.5841<br>-7.3008 | 10.5117<br>10.1658 | 0.9889<br>0.9166 | -40.0000<br>-39.0000 | 11.0000<br>12.0000 |
| Diff | (1-2) | -3.2833 | 10.3328 | 1.3464 | | |
| TRTPN | Method | Mean | 95% CL | Mean | Std Dev | 95% CL Std Dev |
| 1 3 | | -10.5841<br>-7.3008 | -12.5434<br>-9.1153 | -8.6248<br>-5.4863 | 10.5117<br>10.1658 | 9.2969 12.0944<br>9.0346 11.6234 |
| Diff (1-2) | Pooled | -3.2833 | -5.9359 | -0.6306 | 10.3328 | 9.4754 11.3621 |
| Diff (1-2) | Satterthwaite | -3.2833 | -5.9399 | -0.6266 | | |
| | Method | Variance | s D | F t Value | Pr > t | |
| | Pooled<br>Satterthwa | Equal<br>ite Unequal | 23<br>230.7 | | | |

CENTANAFADINE 12 OF 24


STAT-4.7

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, OC (Efficacy Sample)

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F Folded F 112 122 1.07 0.7162

CENTANAFADINE 13 OF 24


STAT-4.7

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, OC (Efficacy Sample)

------ Analysis Visit (N)=7 ------

The TTEST Procedure

| | | Va | riable: CHG | (Change | from Baseline | e) | | |
|---|---|---|---|---|---|---|---|---|
| T | RTPN | N | Mean | Std Dev | Std Err | Minimum | Maximum | |
| 2<br>3<br>D | | 139<br>139 | -5.4460<br>-3.5612<br>-1.8849 | 6.6389<br>6.6693<br>6.6541 | 0.5631<br>0.5657<br>0.7982 | -24.0000<br>-31.0000 | 9.0000<br>10.0000 | |
| TRTPN | Meth | nod | Mean | 95% CL | Mean | Std Dev | 95% CL St | d Dev |
| 2<br>3<br>Diff (1-2<br>Diff (1-2 | | ed<br>erthwaite | -5.4460<br>-3.5612<br>-1.8849<br>-1.8849 | -6.5595<br>-4.6797<br>-3.4562<br>-3.4562 | -2.4426<br>-0.3136 | 6.6389<br>6.6693<br>6.6541 | 5.9667 | 7.5264<br>7.5609<br>7.2597 |
| | 1 | Method | Variances | D! | F t Value | Pr > t | | |
| | | Pooled<br>Satterthwaite | Equal<br>Unequal | 27<br>275.9 | | | | |

CENTANAFADINE 14 OF 24


STAT-4.7

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, OC (Efficacy Sample)

------ Analysis Visit (N)=7 ------

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > FFolded F 138 138 1.01 0.9572

CENTANAFADINE 15 OF 24


STAT-4.7

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, OC (Efficacy Sample)

The TTEST Procedure

| | | | | Variable: CHG | (Change | from Baselin | ie) | | |
|---|---|---|---|---|---|---|---|---|---|
| | TRTPN | | N | Mean | Std Dev | Std Err | Minimum | Maximum | |
| | 2<br>3<br>Diff | (1-2) | 125<br>132 | -8.0880<br>-4.8561<br>-3.2319 | 8.3396<br>7.9070<br>8.1202 | 0.7459<br>0.6882<br>1.0134 | -35.0000<br>-38.0000 | 12.0000<br>8.0000 | |
| TRTPN | | Method | | Mean | 95% CL | Mean | Std Dev | 95% CL S | td Dev |
| 2<br>3<br>Diff (1<br>Diff (1 | | Pooled<br>Satterth | waite | -8.0880<br>-4.8561<br>-3.2319<br>-3.2319 | -9.5644<br>-6.2175<br>-5.2277<br>-5.2307 | -6.6116<br>-3.4946<br>-1.2362<br>-1.2332 | 8.3396<br>7.9070<br>8.1202 | 7.4182<br>7.0545<br>7.4725 | 9.5243<br>8.9958<br>8.8919 |
| | | Metho | d | Variances | D! | F t Value | Pr > t | | |
| | | Poole<br>Satte | d<br>rthwai | Equal<br>te Unequal | 252.0° | | | | |

CENTANAFADINE 16 OF 24


STAT-4.7

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, OC (Efficacy Sample)

------ Analysis Visit (N)=14 ------

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F Folded F 124 131 1.11 0.5473

CENTANAFADINE 17 OF 24


STAT-4.7

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, OC (Efficacy Sample)

The TTEST Procedure

| | Va | riable: CHG | (Change | from Baseline | e) | |
|---|---|---|---|---|---|---|
| TRTP | N N | Mean | Std Dev | Std Err | Minimum | Maximum |
| 2<br>3<br>Diff | 116<br>132 | -10.5690<br>-5.9924<br>-4.5765 | 9.5555<br>8.8925<br>9.2084 | 0.8872<br>0.7740<br>1.1719 | -34.0000<br>-40.0000 | 17.0000<br>11.0000 |
| TRTPN | Method | Mean | 95% CL | Mean | Std Dev | 95% CL Std Dev |
| 2<br>3<br>Diff (1-2)<br>Diff (1-2) | Pooled<br>Satterthwaite | -10.5690<br>-5.9924<br>-4.5765<br>-4.5765 | -12.3264<br>-7.5236<br>-6.8848<br>-6.8960 | -4.4613<br>-2.2683 | 9.5555<br>8.8925<br>9.2084 | 8.4641 10.9727<br>7.9337 10.1169<br>8.4616 10.1008 |
| | Method | Variances | D. | F t Value | Pr > t | |
| | Pooled<br>Satterthwaite | Equal<br>Unequal | 24<br>236.4 | | | |

CENTANAFADINE 18 OF 24


STAT-4.7

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, OC (Efficacy Sample)

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F Folded F 115 131 1.15 0.4242

CENTANAFADINE 19 OF 24


STAT-4.7

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, OC (Efficacy Sample)

------ Analysis Visit (N)=28 ------

The TTEST Procedure

| | Vá | ariable: CHG | (Change | from Baseline | e) | |
|---|---|---|---|---|---|---|
| TRTE | PN N | Mean | Std Dev | Std Err | Minimum | Maximum |
| 2<br>3<br>Diff | 114<br>130<br>E (1-2) | -10.4298<br>-6.4462<br>-3.9837 | 10.0344<br>9.1313<br>9.5636 | 0.9398<br>0.8009<br>1.2271 | -42.0000<br>-37.0000 | 7.0000<br>13.0000 |
| TRTPN | Method | Mean | 95% CL | Mean | Std Dev | 95% CL Std Dev |
| 2<br>3<br>Diff (1-2)<br>Diff (1-2) | Pooled<br>Satterthwaite | -10.4298<br>-6.4462<br>-3.9837<br>-3.9837 | -6.4009 | -8.5679<br>-4.8616<br>-1.5664<br>-1.5508 | 10.0344<br>9.1313<br>9.5636 | 8.8794 11.5377<br>8.1400 10.3996<br>8.7822 10.4989 |
| | Method | Variance | es D | F t Value | Pr > t | |
| | Pooled<br>Satterthwaite | Equal<br>E Unequal | 24<br>230.3 | | | |

CENTANAFADINE 20 OF 24


STAT-4.7

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, OC (Efficacy Sample)

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > FFolded F 113 129 1.21 0.2991

CENTANAFADINE 21 OF 24


STAT-4.7

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, OC (Efficacy Sample)

The TTEST Procedure

| Variable: CHG (Change from Baseline) | | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | TRTPN | | N | Mean | Std Dev | Std Err | Minimum | Maximum |
| | 2<br>3<br>Diff | (1-2) | 104<br>125 | -12.0577<br>-7.1840<br>-4.8737 | 10.7666<br>9.3657<br>10.0256 | 1.0557<br>0.8377<br>1.3306 | -40.0000<br>-37.0000 | 10.0000 |
| TRTPN | | Method | | Mean | 95% CL | Mean | Std Dev | 95% CL Std Dev |
| 2<br>3<br>Diff (1-<br>Diff (1- | , | Pooled<br>Satterth | waite | -12.0577<br>-7.1840<br>-4.8737<br>-4.8737 | -14.1515<br>-8.8420<br>-7.4957<br>-7.5308 | -9.9639<br>-5.5260<br>-2.2517<br>-2.2166 | 10.7666<br>9.3657<br>10.0256 | 9.4757 12.4678<br>8.3310 10.6962<br>9.1821 11.0411 |
| | | Metho | d | Variance | s Di | F t Value | Pr > t | |
| | | Poole<br>Satte | d<br>rthwai | Equal<br>te Unequal | 22°<br>205.7° | | | |

CENTANAFADINE 22 OF 24


STAT-4.7

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, OC (Efficacy Sample)

------ Analysis Visit (N)=35 -----

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F Folded F 103 124 1.32 0.1375

CENTANAFADINE 23 OF 24


STAT-4.7

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, OC (Efficacy Sample)

------ Analysis Visit (N)=42 ------

The TTEST Procedure

| | 7 | /ariable: CHG | (Change | from Baseline | e) | |
|---|---|---|---|---|---|---|
| TRTP | N N | Mean | Std Dev | Std Err | Minimum | Maximum |
| 2<br>3<br>Diff | 102<br>123<br>(1-2) | -11.5490<br>-7.3008<br>-4.2482 | 11.6293<br>10.1658<br>10.8531 | 1.1515<br>0.9166<br>1.4534 | -41.0000<br>-39.0000 | 11.0000<br>12.0000 |
| TRTPN | Method | Mean | 95% CL | Mean | Std Dev | 95% CL Std Dev |
| 2<br>3<br>Diff (1-2)<br>Diff (1-2) | Pooled<br>Satterthwaite | -11.5490<br>-7.3008<br>-4.2482<br>-4.2482 | -13.8332<br>-9.1153<br>-7.1124<br>-7.1502 | -5.4863<br>-1.3840 | 11.6293<br>10.1658<br>10.8531 | 10.2229 13.4878<br>9.0346 11.6234<br>9.9325 11.9632 |
| | Method | Variance | s D | F t Value | Pr > t | |
| | Pooled<br>Satterthwait | Equal<br>ce Unequal | 22<br>202.3 | | | |

CENTANAFADINE 24 OF 24


STAT-4.7

Unadjusted Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, OC (Efficacy Sample)

\_\_\_\_\_

The TTEST Procedure

Variable: CHG (Change from Baseline)

Equality of Variances

Method Num DF Den DF F Value Pr > F Folded F 101 122 1.31 0.1554


STAT-4.8

Non-Parametric Stratified by Center Analysis of Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, LOCF (Efficacy Sample)

The FREQ Procedure

Summary Statistics for TRTP by CHG Controlling for POOLCNTR

Cochran-Mantel-Haenszel Statistics (Based on Rank Scores)

| Statistic | Alternative Hypothesis | DF | Value | Prob |
|-----------|------------------------|----|--------|--------|
| 1 | Nonzero Correlation | 1 | 0.4550 | 0.5000 |
| 2 | Row Mean Scores Differ | 2 | 4.9054 | 0.0861 |

<sup>1</sup> WILCOXON TEST STRATIFIED BY (POOLED) CENTER.


STAT-4.8

Non-Parametric Stratified by Center Analysis of Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, LOCF (Efficacy Sample)

------ Analysis Visit (N)=14 ------

The FREQ Procedure

Summary Statistics for TRTP by CHG Controlling for POOLCNTR

Cochran-Mantel-Haenszel Statistics (Based on Rank Scores)

| Statistic | Alternative Hypothesis | DF | Value | Prob |
|-----------|------------------------|----|---------|--------|
| 1 | Nonzero Correlation | 1 | 6.1912 | 0.0128 |
| 2 | Row Mean Scores Differ | 2 | 14.3978 | 0.0007 |

<sup>1</sup> WILCOXON TEST STRATIFIED BY (POOLED) CENTER.


STAT-4.8

Non-Parametric Stratified by Center Analysis of Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, LOCF (Efficacy Sample)

The FREQ Procedure

Summary Statistics for TRTP by CHG Controlling for POOLCNTR

Cochran-Mantel-Haenszel Statistics (Based on Rank Scores)

| Statistic | Alternative Hypothesis | DF | Value | Prob |
|-----------|------------------------|----|---------|--------|
| 1 | Nonzero Correlation | 1 | 7.3934 | 0.0065 |
| 2 | Row Mean Scores Differ | 2 | 17.6867 | 0.0001 |

<sup>1</sup> WILCOXON TEST STRATIFIED BY (POOLED) CENTER.

STAT-4.8

Non-Parametric Stratified by Center Analysis of Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, LOCF (Efficacy Sample)

The FREQ Procedure

Summary Statistics for TRTP by CHG Controlling for POOLCNTR

Cochran-Mantel-Haenszel Statistics (Based on Rank Scores)

| Statistic | Alternative Hypothesis | DF | Value | Prob |
|-----------|------------------------|----|---------|--------|
| 1 | Nonzero Correlation | 1 | 6.0289 | 0.0141 |
| 2 | Row Mean Scores Differ | 2 | 14.5765 | 0.0007 |

<sup>1</sup> WILCOXON TEST STRATIFIED BY (POOLED) CENTER.


STAT-4.8

Non-Parametric Stratified by Center Analysis of Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, LOCF (Efficacy Sample)

------ Analysis Visit (N)=35 ------

The FREQ Procedure

Summary Statistics for TRTP by CHG Controlling for POOLCNTR

Cochran-Mantel-Haenszel Statistics (Based on Rank Scores)

| Statistic | Alternative Hypothesis | DF | Value | Prob |
|-----------|------------------------|----|---------|--------|
| 1 | Nonzero Correlation | 1 | 3.2902 | 0.0697 |
| 2 | Row Mean Scores Differ | 2 | 11.9563 | 0.0025 |

<sup>1</sup> WILCOXON TEST STRATIFIED BY (POOLED) CENTER.

CENTANAFADINE 6 OF 6


STAT-4.8

Non-Parametric Stratified by Center Analysis of Mean Change from Baseline to Double Blind Tretmnet Period by Study Day in AISRS Total Score, LOCF (Efficacy Sample)

------

------ Analysis Visit (N)=42 ------

The FREQ Procedure

Summary Statistics for TRTP by CHG Controlling for POOLCNTR

Cochran-Mantel-Haenszel Statistics (Based on Rank Scores)

| Statistic | Alternative Hypothesis | DF | Value | Prob |
|-----------|------------------------|----|---------|--------|
| 1 | Nonzero Correlation | 1 | 2.7238 | 0.0989 |
| 2 | Row Mean Scores Differ | 2 | 10.7158 | 0.0047 |

<sup>1</sup> WILCOXON TEST STRATIFIED BY (POOLED) CENTER.

CENTANAFADINE 1 OF 11


### STAT-4.9

Residual at Day 42 from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

The UNIVARIATE Procedure
Variable: RESID (Residual)
 AVISITN = 42
 AVISIT = DAY 42

#### Moments

| N | 338 | Sum Weights | 338 |
|-----------------|------------|------------------|------------|
| Mean | 0.21994106 | Sum Observations | 74.3400787 |
| Std Deviation | 10.206485 | Variance | 104.172337 |
| Skewness | -0.4662637 | Kurtosis | -0.2816581 |
| Uncorrected SS | 35122.428 | Corrected SS | 35106.0776 |
| Coeff Variation | 4640.5546 | Std Error Mean | 0.5551596 |

### Basic Statistical Measures

# Location Variability

| Mean | 0.219941 | Std Deviation | 10.20649 |
|--------|----------|---------------------|-----------|
| Median | 2.116541 | Variance | 104.17234 |
| Mode | 7.859023 | Range | 51.41794 |
| | | Interguartile Range | 14.95136 |

#### Tests for Location: Mu0=0

| Test | -Statistic- | p Value |
|---------------------|-------------|-------------------------------------|
| Student's t<br>Sign | t 0.396176 | Pr > t 0.6922<br>Pr >= M 0.0256 |
| Signed Rank | S 1936.5 | |

CENTANAFADINE 2 OF 11


STAT-4.9

Residual at Day 42 from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

The UNIVARIATE Procedure
Variable: RESID (Residual)
 AVISITN = 42
 AVISIT = DAY 42

Quantiles (Definition 5)

| Level | Quantile |
|------------|-----------|
| 100% Max | 21.91943 |
| 99% | 20.45404 |
| 95% | 14.85949 |
| 90% | 12.11174 |
| 75% Q3 | 7.82680 |
| 50% Median | 2.11654 |
| 25% Q1 | -7.12456 |
| 10% | -14.10923 |
| 5% | -18.33244 |
| 1% | -27.07807 |
| 0% Min | -29.49851 |

#### Extreme Observations

| Lowest | | Highes | t |
|----------------------|------------|--------------------|-------------|
| Value | Obs | Value | Obs |
| -29.4985<br>-27.6116 | 961<br>257 | 19.4617<br>20.4540 | 1608<br>298 |
| -27.3096 | 1412 | 20.7976 | 1491 |
| -27.0781 | 401 | 21.6142 | 973 |

CENTANAFADINE 3 OF 11


STAT-4.9

Residual at Day 42 from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

\_\_\_\_\_\_

The UNIVARIATE Procedure
Variable: RESID (Residual)

AVISITN = 42

AVISIT = DAY 42

#### Extreme Observations

| nest | High | Lowest | |
|------|---------|--------|----------|
| Obs | Value | Obs | Value |
| 1066 | 21.9194 | 1117 | -25.9557 |

CENTANAFADINE 4 OF 11


-28 5

#### STAT-4.9

Residual at Day 42 from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

The UNIVARIATE Procedure



SOURCE: MMRMDX1; TABLE: stat1k.lis; RUN: 31AUG2020 08:32; ANALYSIS DATASET CREATED: 16JUN2020 08:14 PROGRAM: /opt/sas/Data/DAP/EB1020/P40520100014/STAT/Program.dev/DOC\_STAT/stat1.sas OPDC, NEW DRUG APPLICATION, IND # 119,361 CENTANAFADINE STAT-4.9 FINAL

-29+\*

CENTANAFADINE 5 OF 11 PROTOCOL 405-201-00014

STAT-4.9

Residual at Day 42 from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

\_\_\_\_\_\_

The UNIVARIATE Procedure
Variable: RESID (Residual)
 AVISITN = 42
 AVISIT = DAY 42

CENTANAFADINE 6 OF 11


STAT-4.9

Residual at Day 42 from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

The UNIVARIATE Procedure

Variable: STUDENTRESID (Studentized Residual)

AVISITN = 42 AVISIT = DAY 42

#### Moments

| N | 338 | Sum Weights | 338 |
|-----------------|------------|------------------|------------|
| Mean | 0.02186339 | Sum Observations | 7.38982701 |
| Std Deviation | 1.00255899 | Variance | 1.00512453 |
| Skewness | -0.4654092 | Kurtosis | -0.2701205 |
| Uncorrected SS | 338.888534 | Corrected SS | 338.726967 |
| Coeff Variation | 4585.55983 | Std Error Mean | 0.05453202 |

### Basic Statistical Measures

# Location Variability

| Mean | 0.021863 | Std Deviation | 1.00256 |
|--------|----------|---------------------|---------|
| Median | 0.204955 | Variance | 1.00512 |
| Mode | 0.760366 | Range | 5.13076 |
| | | Interguartile Range | 1.45333 |

#### Tests for Location: Mu0=0

| Test | -Statisti | cp Val | .ue |
|-------------|-----------|----------------|--------|
| Student's t | t 0.4009 | 28 Pr > t | 0.6887 |
| Sign | M | 21 Pr >= M | 0.0256 |
| Signed Rank | S 1930 | .5 $Pr >= S $ | 0.2836 |

CENTANAFADINE 7 OF 11


STAT-4.9

Residual at Day 42 from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

The UNIVARIATE Procedure

Variable: STUDENTRESID (Studentized Residual)

AVISITN = 42 AVISIT = DAY 42

Quantiles (Definition 5)

| Level | Quantile |
|------------|-----------|
| 100% Max | 2.170595 |
| 99% | 1.980822 |
| 95% | 1.444907 |
| 90% | 1.182725 |
| 75% Q3 | 0.762961 |
| 50% Median | 0.204955 |
| 25% Q1 | -0.690365 |
| 10% | -1.369158 |
| 5% | -1.794783 |
| 1% | -2.635345 |
| 0% Min | -2.960170 |

#### Extreme Observations

| nest | High | Lowest | |
|-------------|--------------------|-------------|----------------------|
| Obs | Value | Obs | Value |
| 1608<br>298 | 1.88413<br>1.98082 | 961<br>1412 | -2.96017<br>-2.72302 |
| 1491 | 2.07185 | 257 | -2.68489 |
| 1066 | 2.14336 | 401 | -2.63534 |

CENTANAFADINE 8 OF 11


STAT-4.9

Residual at Day 42 from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

\_\_\_\_\_\_

The UNIVARIATE Procedure

Variable: STUDENTRESID (Studentized Residual)

AVISITN = 42 AVISIT = DAY 42

Extreme Observations

| est | High | est | Lov |
|-----|---------|------|----------|
| Obs | Value | Obs | Value |
| 973 | 2.17059 | 1117 | -2.54132 |

CENTANAFADINE 9 OF 11


STAT-4.9

Residual at Day 42 from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

\_\_\_\_\_\_



CENTANAFADINE 10 OF 11


STAT-4.9

Residual at Day 42 from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

The UNIVARIATE Procedure
Variable: STUDENTRESID (Studentized Residual)

AVISITN = 42 AVISIT = DAY 42

CENTANAFADINE 11 OF 11


STAT-4.9

Residual at Day 42 from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

......





CENTANAFADINE 1 OF 26 PROTOCOL 405-201-00014

STAT-4.10

Proc Mixed Output Using Heterogeneous Variance Structure for Treatment Groups (Efficacy Sample)

The Mixed Procedure

Model Information

Data Set WORK.INDATA
Dependent Variable CHG
Covariance Structure Unstructured
Subject Effect SUBJID
Group Effect TRTPN
Estimation Method REML
Residual Variance Method None

Fixed Effects SE Method Kenward-Roger
Degrees of Freedom Method Kenward-Roger

Class Level Information

Class Levels Values

AVISITN 6 7 14 21 28 35 42

TRTPN 3 1 2 3

POOLCNTR 39

CENTANAFADINE 2 OF 26 PROTOCOL 405-201-00014

STAT-4.10

Proc Mixed Output Using Heterogeneous Variance Structure for Treatment Groups (Efficacy Sample)

\_\_\_\_\_

The Mixed Procedure

Class Level Information

Class Levels Values

SUBJID 421



CENTANAFADINE

3 OF 26

STAT-4.10

Proc Mixed Output Using Heterogeneous Variance Structure for Treatment Groups (Efficacy Sample)

\_\_\_\_\_

The Mixed Procedure



CENTANAFADINE
4 OF 26

STAT-4.10

Proc Mixed Output Using Heterogeneous Variance Structure for Treatment Groups (Efficacy Sample)

The Mixed Procedure



CENTANAFADINE 5 OF 26 PROTOCOL 405-201-00014

STAT-4.10

Proc Mixed Output Using Heterogeneous Variance Structure for Treatment Groups (Efficacy Sample)

\_\_\_\_\_

The Mixed Procedure



CENTANAFADINE 6 OF 26 PROTOCOL 405-201-00014

STAT-4.10

Proc Mixed Output Using Heterogeneous Variance Structure for Treatment Groups (Efficacy Sample)

\_\_\_\_\_\_

The Mixed Procedure



CENTANAFADINE 7 OF 26 PROTOCOL 405-201-00014

# STAT-4.10

Proc Mixed Output Using Heterogeneous Variance Structure for Treatment Groups (Efficacy Sample)

\_\_\_\_\_

#### The Mixed Procedure



#### Dimensions

| Covariance | Parameters | 63 |
|------------|------------|-----|
| Columns in | X | 73 |
| Columns in | Z | 0 |
| Subjects | | 421 |
| Max Obs pe | r Subject | 6 |

### Number of Observations

| Number | of | Observations | Read | 2227 |
|--------|----|--------------|----------|------|
| Number | of | Observations | Used | 2227 |
| Number | of | Observations | Not Used | 0 |

CENTANAFADINE 8 OF 26 PROTOCOL 405-201-00014

# STAT-4.10

Proc Mixed Output Using Heterogeneous Variance Structure for Treatment Groups (Efficacy Sample)

\_\_\_\_\_\_

#### The Mixed Procedure

#### Iteration History

| Iteration | Evaluations | -2 Res Log Like | Criterion |
|-----------|-------------|-----------------|------------|
| 0 | 1 | 15800.38727426 | |
| 1 | 4 | 13478.73670114 | 0.00213540 |
| 2 | 1 | 13467.00275618 | 0.00024731 |
| 3 | 1 | 13465.70016597 | 0.00001037 |
| 4 | 1 | 13465.64921223 | 0.00000003 |
| 5 | 1 | 13465.64904810 | 0.00000000 |

Convergence criteria met.

| | Estimated | R Matrix for | SUBJID | |
|-----|-----------|--------------|---------|---------|
| Row | Col1 | Col2 | Col3 | Col4 |
| 1 | 36.9737 | 26.0068 | 31.4785 | 33.3871 |
| 2 | 26.0068 | 59.7634 | 55.9805 | 56.6731 |
| 3 | 31.4785 | 55.9805 | 78.9073 | 73.4766 |
| 4 | 33.3871 | 56.6731 | 73.4766 | 94.5512 |

CENTANAFADINE 9 OF 26 PROTOCOL 405-201-00014

STAT-4.10

Proc Mixed Output Using Heterogeneous Variance Structure for Treatment Groups (Efficacy Sample)

#### The Mixed Procedure

| | Esti | mated R Corr | elation Matr | ix for SUBJII | | |
|---|---|---|---|---|---|---|
| | Row | Col1 | Co12 | Col3 | Col4 | |
| | 1 2 | 1.0000<br>0.5533 | 0.5533<br>1.0000 | 0.5828<br>0.8152 | 0.5647<br>0.7539 | |
| | 3<br>4 | 0.5828<br>0.5647 | 0.8152<br>0.7539 | 1.0000<br>0.8507 | 0.8507<br>1.0000 | |
| | | Estimated | R Matrix for | SUBJID | | |
| Row | Col1 | Col2 | Co13 | Col4 | Col5 | Col6 |
| 1<br>2<br>3<br>4<br>5<br>6 | 48.7945<br>45.9963<br>44.9550<br>46.9027<br>44.0988<br>44.7419 | 45.9963<br>92.0313<br>77.3240<br>75.1467<br>71.7701<br>69.6304 | 44.9550<br>77.3240<br>93.5276<br>87.1175<br>77.8069<br>80.6325 | 46.9027<br>75.1467<br>87.1175<br>101.83<br>91.1218<br>92.2892 | 44.0988<br>71.7701<br>77.8069<br>91.1218<br>101.52<br>89.0164 | 44.7419<br>69.6304<br>80.6325<br>92.2892<br>89.0164<br>109.05 |
| | | Estimated | R Matrix for | SUBJID | | |
| Row | Col1 | Col2 | Co13 | Col4 | Col5 | Col6 |
| 1<br>2 | 45.3296<br>42.2715 | 42.2715<br>58.5296 | 36.0407<br>46.1505 | 39.1670<br>46.4824 | 40.8245<br>51.7087 | 39.9697<br>50.9898 |

CENTANAFADINE 10 OF 26 PROTOCOL 405-201-00014

STAT-4.10

Proc Mixed Output Using Heterogeneous Variance Structure for Treatment Groups (Efficacy Sample)

# The Mixed Procedure

#### Estimated R Matrix for SUBJID Col1 Row Col2 Col3 Col4 Col5 Col6 36.0407 46.1505 71.3771 62.2249 65.8373 69.3392 39.1670 46.4824 62.2249 75.8237 70.2194 74.6922 40.8245 51.7087 65.8373 70.2194 84.4321 83.9356 39.9697 50.9898 69.3392 74.6922 83.9356 97.8853

#### Covariance Parameter Estimates

| Cov Parm | Subject | Group | Estimate |
|----------|---------|---------|----------|
| UN(1,1) | SUBJID | TRTPN 1 | 48.7945 |
| UN(2,1) | SUBJID | TRTPN 1 | 45.9963 |
| UN(2,2) | SUBJID | TRTPN 1 | 92.0313 |
| UN(3,1) | SUBJID | TRTPN 1 | 44.9550 |
| UN(3,2) | SUBJID | TRTPN 1 | 77.3240 |
| UN(3,3) | SUBJID | TRTPN 1 | 93.5276 |
| UN(4,1) | SUBJID | TRTPN 1 | 46.9027 |
| UN(4,2) | SUBJID | TRTPN 1 | 75.1467 |
| UN(4,3) | SUBJID | TRTPN 1 | 87.1175 |
| UN(4,4) | SUBJID | TRTPN 1 | 101.83 |
| UN(5,1) | SUBJID | TRTPN 1 | 44.0988 |
| UN(5,2) | SUBJID | TRTPN 1 | 71.7701 |
| UN(5,3) | SUBJID | TRTPN 1 | 77.8069 |
| UN(5,4) | SUBJID | TRTPN 1 | 91.1218 |

CENTANAFADINE 11 OF 26 PROTOCOL 405-201-00014

STAT-4.10

Proc Mixed Output Using Heterogeneous Variance Structure for Treatment Groups (Efficacy Sample)

\_\_\_\_\_

The Mixed Procedure

#### Covariance Parameter Estimates

| Cov Parm | Subject | Group | Estimate |
|----------|---------|---------|----------|
| UN(5,5) | SUBJID | TRTPN 1 | 101.52 |
| UN(6,1) | SUBJID | TRTPN 1 | 44.7419 |
| UN(6,2) | SUBJID | TRTPN 1 | 69.6304 |
| UN(6,3) | SUBJID | TRTPN 1 | 80.6325 |
| UN(6,4) | SUBJID | TRTPN 1 | 92.2892 |
| UN(6,5) | SUBJID | TRTPN 1 | 89.0164 |
| UN(6,6) | SUBJID | TRTPN 1 | 109.05 |
| UN(1,1) | SUBJID | TRTPN 2 | 36.9737 |
| UN(2,1) | SUBJID | TRTPN 2 | 26.0068 |
| UN(2,2) | SUBJID | TRTPN 2 | 59.7634 |
| UN(3,1) | SUBJID | TRTPN 2 | 31.4785 |
| UN(3,2) | SUBJID | TRTPN 2 | 55.9805 |
| UN(3,3) | SUBJID | TRTPN 2 | 78.9073 |
| UN(4,1) | SUBJID | TRTPN 2 | 33.3871 |
| UN(4,2) | SUBJID | TRTPN 2 | 56.6731 |
| UN(4,3) | SUBJID | TRTPN 2 | 73.4766 |
| UN(4,4) | SUBJID | TRTPN 2 | 94.5512 |
| UN(5,1) | SUBJID | TRTPN 2 | 32.3181 |
| UN(5,2) | SUBJID | TRTPN 2 | 56.3760 |
| UN(5,3) | SUBJID | TRTPN 2 | 72.7477 |
| UN(5,4) | SUBJID | TRTPN 2 | 86.8002 |
| UN(5,5) | SUBJID | TRTPN 2 | 107.38 |
| UN(6,1) | SUBJID | TRTPN 2 | 30.4643 |
| UN(6,2) | SUBJID | TRTPN 2 | 56.8611 |

CENTANAFADINE 12 OF 26 PROTOCOL 405-201-00014

STAT-4.10

Proc Mixed Output Using Heterogeneous Variance Structure for Treatment Groups (Efficacy Sample)

\_\_\_\_\_

The Mixed Procedure

Covariance Parameter Estimates

| Cov Parm | Subject | Group | Estimate |
|----------|---------|---------|----------|
| UN(6,3) | SUBJID | TRTPN 2 | 70.9567 |
| UN(6,4) | SUBJID | TRTPN 2 | 85.9523 |
| UN(6,5) | SUBJID | TRTPN 2 | 101.05 |
| UN(6,6) | SUBJID | TRTPN 2 | 117.94 |
| UN(1,1) | SUBJID | TRTPN 3 | 45.3296 |
| UN(2,1) | SUBJID | TRTPN 3 | 42.2715 |
| UN(2,2) | SUBJID | TRTPN 3 | 58.5296 |
| UN(3,1) | SUBJID | TRTPN 3 | 36.0407 |
| UN(3,2) | SUBJID | TRTPN 3 | 46.1505 |
| UN(3,3) | SUBJID | TRTPN 3 | 71.3771 |
| UN(4,1) | SUBJID | TRTPN 3 | 39.1670 |
| UN(4,2) | SUBJID | TRTPN 3 | 46.4824 |
| UN(4,3) | SUBJID | TRTPN 3 | 62.2249 |
| UN(4,4) | SUBJID | TRTPN 3 | 75.8237 |
| UN(5,1) | SUBJID | TRTPN 3 | 40.8245 |
| UN(5,2) | SUBJID | TRTPN 3 | 51.7087 |
| UN(5,3) | SUBJID | TRTPN 3 | 65.8373 |
| UN(5,4) | SUBJID | TRTPN 3 | 70.2194 |
| UN(5,5) | SUBJID | TRTPN 3 | 84.4321 |
| UN(6,1) | SUBJID | TRTPN 3 | 39.9697 |
| UN(6,2) | SUBJID | TRTPN 3 | 50.9898 |
| UN(6,3) | SUBJID | TRTPN 3 | 69.3392 |
| UN(6,4) | SUBJID | TRTPN 3 | 74.6922 |
| UN(6,5) | SUBJID | TRTPN 3 | 83.9356 |

CENTANAFADINE 13 OF 26 PROTOCOL 405-201-00014

STAT-4.10

Proc Mixed Output Using Heterogeneous Variance Structure for Treatment Groups (Efficacy Sample)

The Mixed Procedure

Covariance Parameter Estimates

Cov Parm Subject Group Estimate
UN(6,6) SUBJID TRTPN 3 97.8853

Fit Statistics

-2 Res Log Likelihood 13465.6 AIC (Smaller is Better) 13591.6 AICC (Smaller is Better) 13595.5 BIC (Smaller is Better) 13846.3

Null Model Likelihood Ratio Test

DF Chi-Square Pr > ChiSq 62 2334.74 <.0001

CENTANAFADINE 14 OF 26 PROTOCOL 405-201-00014

 ${\tt STAT-4.10}\\ {\tt Proc\ Mixed\ Output\ Using\ Heterogeneous\ Variance\ Structure\ for\ Treatment\ Groups}\\ ({\tt Efficacy\ Sample})$ 

\_\_\_\_\_\_

Parameter Code=AISRSTOT ------

# The Mixed Procedure

#### Solution for Fixed Effects

| | Pooled<br>Center | Analysis<br>Visit | Planned<br>Treatment | | Standard | | | |
|---|---|---|---|---|---|---|---|---|
| Effect | Number | (N) | (N) | Estimate | Error | DF | t Value | Pr > t |
| Intercept | | | | 2.2570 | 4.8279 | 484 | 0.47 | 0.6404 |
| AVISITN | | 7 | | 0.1158 | 2.6468 | 338 | 0.04 | 0.9651 |
| AVISITN | | 14 | | -1.0804 | 2.4063 | 361 | -0.45 | 0.6537 |
| AVISITN | | 21 | | 1.3469 | 2.0492 | 336 | 0.66 | 0.5115 |
| AVISITN | | 28 | | -1.3671 | 1.7371 | 334 | -0.79 | 0.4318 |
| AVISITN | | 35 | | -1.2228 | 1.5148 | 307 | -0.81 | 0.4202 |
| AVISITN | | 42 | | 0 | | | | |
| TRTPN | | | 1 | -3.9849 | 1.2601 | 249 | -3.16 | 0.0018 |
| TRTPN | | | 2 | -4.4036 | 1.3262 | 243 | -3.32 | 0.0010 |
| TRTPN | | | 3 | 0 | | | | |
| AVISITN*TRTPN | | 7 | 1 | 2.0812 | 1.0252 | 214 | 2.03 | 0.0436 |
| AVISITN*TRTPN | | 7 | 2 | 2.5703 | 1.1536 | 220 | 2.23 | 0.0269 |
| AVISITN*TRTPN | | 7 | 3 | 0 | | | | |
| AVISITN*TRTPN | | 14 | 1 | 0.3743 | 0.9708 | 239 | 0.39 | 0.7002 |
| AVISITN*TRTPN | | 14 | 2 | 0.8059 | 1.0165 | 221 | 0.79 | 0.4288 |
| AVISITN*TRTPN | | 14 | 3 | 0 | | | | |
| AVISITN*TRTPN | | 21 | 1 | -0.03336 | 0.7740 | 225 | -0.04 | 0.9657 |
| AVISITN*TRTPN | | 21 | 2 | -0.05933 | 0.8789 | 200 | -0.07 | 0.9462 |
| AVISITN*TRTPN | | 21 | 3 | 0 | | | | |
| AVISITN*TRTPN | | 28 | 1 | 0.04623 | 0.6580 | 232 | 0.07 | 0.9440 |
| AVISITN*TRTPN | | 28 | 2 | -0.08429 | 0.7725 | 199 | -0.11 | 0.9132 |
| AVISITN*TRTPN | | 28 | 3 | 0 | | | | |

SOURCE: MMRMDX2; TABLE: stat11.lis; RUN: 31AUG2020 08:32; ANALYSIS DATASET CREATED: 16JUN2020 08:14
PROGRAM: /opt/sas/Data/DAP/EB1020/P40520100014/STAT/Program.dev/DOC\_STAT/stat1.sas
OPDC, NEW DRUG APPLICATION, IND # 119,361 CENTANAFADINE STAT-4.10 FINAL

Dooled Applyais Dlanned

CENTANAFADINE 15 OF 26 PROTOCOL 405-201-00014

STAT-4.10

Proc Mixed Output Using Heterogeneous Variance Structure for Treatment Groups (Efficacy Sample)

\_\_\_\_\_\_

#### The Mixed Procedure

#### Solution for Fixed Effects

| | Pooled<br>Center | Analysis<br>Visit | Planned<br>Treatment | | Standard | | | |
|---|---|---|---|---|---|---|---|---|
| Effect | Number | (N) | (N) | Estimate | Error | DF | t Value | Pr > t |
| AVISITN*TRTPN | | 35 | 1 | 0.2367 | 0.6395 | 189 | 0.37 | 0.7117 |
| AVISITN*TRTPN | | 35 | 2 | -0.9126 | 0.5964 | 187 | -1.53 | 0.1276 |
| AVISITN*TRTPN | | 35 | 3 | 0 | | | | |
| AVISITN*TRTPN | | 42 | 1 | 0 | | | | |
| AVISITN*TRTPN | | 42 | 2 | 0 | | | | |
| AVISITN*TRTPN | | 42 | 3 | 0 | | | | |
| POOLCNTR | | | | 0.8283 | 3.8363 | 321 | 0.22 | 0.8292 |
| POOLCNTR | | | | -6.1914 | 5.3240 | 366 | -1.16 | 0.2456 |
| POOLCNTR | | | | 1.0964 | 3.7183 | 309 | 0.29 | 0.7683 |
| POOLCNTR | | | | -1.6031 | 4.5459 | 325 | -0.35 | 0.7246 |
| POOLCNTR | | | | -4.5469 | 4.4902 | 349 | -1.01 | 0.3119 |
| POOLCNTR | | | | 0.4501 | 3.8364 | 321 | 0.12 | 0.9067 |
| POOLCNTR | | | | -0.1036 | 3.7924 | 316 | -0.03 | 0.9782 |
| POOLCNTR | | | | -3.2912 | 4.3656 | 360 | -0.75 | 0.4514 |
| POOLCNTR | | | | 1.9748 | 5.2591 | 363 | 0.38 | 0.7075 |
| POOLCNTR | | | | -4.1388 | 3.8918 | 320 | -1.06 | 0.2884 |
| POOLCNTR | | | | -3.1507 | 4.2517 | 350 | -0.74 | 0.4592 |
| POOLCNTR | | | | -10.6697 | 5.2445 | 363 | -2.03 | 0.0426 |
| POOLCNTR | | | | -4.3208 | 4.3847 | 332 | -0.99 | 0.3251 |
| POOLCNTR | | | | 2.8042 | 4.0999 | 331 | 0.68 | 0.4945 |
| POOLCNTR | | | | -2.4878 | 4.1211 | 333 | -0.60 | 0.5465 |
| POOLCNTR | | | | -3.2434 | 4.7088 | 355 | -0.69 | 0.4914 |

SOURCE: MMRMDX2; TABLE: stat11.lis; RUN: 31AUG2020 08:32; ANALYSIS DATASET CREATED: 16JUN2020 08:14
PROGRAM: /opt/sas/Data/DAP/EB1020/P40520100014/STAT/Program.dev/DOC\_STAT/stat1.sas
OPDC, NEW DRUG APPLICATION, IND # 119,361 CENTANAFADINE STAT-4.10 FINAL

Dooled Applyais Dlanned

CENTANAFADINE 16 OF 26 PROTOCOL 405-201-00014

STAT-4.10

Proc Mixed Output Using Heterogeneous Variance Structure for Treatment Groups (Efficacy Sample)

Parameter Code=AISRSTOT ------

#### The Mixed Procedure

#### Solution for Fixed Effects

| | Pooled<br>Center | Analysis<br>Visit | Planned<br>Treatment | | Standard | | | |
|---|---|---|---|---|---|---|---|---|
| Effect | Number | (N) | (N) | Estimate | Error | DF | t Value | Pr > t |
| | | ` ' | ` ' | | | | | |
| POOLCNTR | | | | -4.6400 | 4.2765 | 342 | -1.08 | 0.2787 |
| POOLCNTR | | | | 0.3984 | 4.8159 | 338 | 0.08 | 0.9341 |
| POOLCNTR | | | | -1.9005 | 4.8163 | 339 | -0.39 | 0.6934 |
| POOLCNTR | | | | -1.4595 | 3.9964 | 336 | -0.37 | 0.7152 |
| POOLCNTR | | | | -4.0268 | 4.1976 | 338 | -0.96 | 0.3381 |
| POOLCNTR | | | | 8.7760 | 4.9299 | 391 | 1.78 | 0.0758 |
| POOLCNTR | | | | 2.1905 | 3.9947 | 328 | 0.55 | 0.5838 |
| POOLCNTR | | | | -5.0765 | 4.0162 | 322 | -1.26 | 0.2071 |
| POOLCNTR | | | | -3.2253 | 4.1899 | 338 | -0.77 | 0.4420 |
| POOLCNTR | | | | 5.7015 | 4.3994 | 342 | 1.30 | 0.1959 |
| POOLCNTR | | | | -7.0249 | 4.4804 | 348 | -1.57 | 0.1178 |
| POOLCNTR | | | | -4.1895 | 4.2580 | 328 | -0.98 | 0.3259 |
| POOLCNTR | | | | 1.1537 | 3.7287 | 314 | 0.31 | 0.7572 |
| POOLCNTR | | | | 2.2150 | 3.7161 | 311 | 0.60 | 0.5516 |
| POOLCNTR | | | | -2.3843 | 4.6802 | 355 | -0.51 | 0.6108 |
| POOLCNTR | | | | 1.3772 | 4.6860 | 354 | 0.29 | 0.7690 |
| POOLCNTR | | | | -5.2391 | 3.9702 | 332 | -1.32 | 0.1879 |
| POOLCNTR | | | | -0.5364 | 4.4506 | 351 | -0.12 | 0.9041 |
| POOLCNTR | | | | -1.5627 | 3.8965 | 323 | -0.40 | 0.6886 |
| POOLCNTR | | | | -3.9649 | 5.2626 | 363 | -0.75 | 0.4517 |
| POOLCNTR | | | | -5.0626 | 4.5384 | 368 | -1.12 | 0.2654 |
| POOLCNTR | | | | -4.3025 | 4.4648 | 310 | -0.96 | 0.3360 |

SOURCE: MMRMDX2; TABLE: stat11.lis; RUN: 31AUG2020 08:32; ANALYSIS DATASET CREATED: 16JUN2020 08:14
PROGRAM: /opt/sas/Data/DAP/EB1020/P40520100014/STAT/Program.dev/DOC\_STAT/stat1.sas
OPDC, NEW DRUG APPLICATION, IND # 119,361 CENTANAFADINE STAT-4.10 FINAL

Dooled Applyais Dlanned

CENTANAFADINE 17 OF 26 PROTOCOL 405-201-00014

# STAT-4.10

Proc Mixed Output Using Heterogeneous Variance Structure for Treatment Groups (Efficacy Sample)

\_\_\_\_\_

Parameter Code=AISRSTOT ------

# The Mixed Procedure

#### Solution for Fixed Effects

| | Pooled<br>Center | Analysıs<br>Visit | Planned<br>Treatment | | Standard | | | |
|---|---|---|---|---|---|---|---|---|
| Effect | Number | (N) | (N) | Estimate | Error | DF | t Value | Pr > t |
| POOLCNTR | | | | 0 | | | | |
| BASE*AVISITN | | 7 | | -0.1300 | 0.06016 | 371 | -2.16 | 0.0313 |
| BASE*AVISITN | | 14 | | -0.1294 | 0.07004 | 408 | -1.85 | 0.0655 |
| BASE*AVISITN | | 21 | | -0.2303 | 0.07607 | 431 | -3.03 | 0.0026 |
| BASE*AVISITN | | 28 | | -0.1649 | 0.08037 | 436 | -2.05 | 0.0408 |
| BASE*AVISITN | | 35 | | -0.1882 | 0.08325 | 439 | -2.26 | 0.0243 |
| BASE*AVISITN | | 42 | | -0.2273 | 0.08808 | 441 | -2.58 | 0.0102 |

### Type 3 Tests of Fixed Effects

| Effect | Num<br>DF | Den<br>DF | F Value | Pr > F |
|---------------|-----------|-----------|---------|--------|
| AVISITN | 5 | 347 | 1.35 | 0.2432 |
| TRTPN | 2 | 247 | 10.64 | <.0001 |
| AVISITN*TRTPN | 10 | 288 | 1.85 | 0.0523 |
| POOLCNTR | 38 | 361 | 2.24 | <.0001 |
| BASE*AVISITN | 6 | 372 | 2.28 | 0.0359 |

CENTANAFADINE 18 OF 26 PROTOCOL 405-201-00014

 ${\tt STAT-4.10}\\ {\tt Proc Mixed Output Using Heterogeneous Variance Structure for Treatment Groups}\\ ({\tt Efficacy Sample})$ 

\_\_\_\_\_

# The Mixed Procedure

#### Least Squares Means

| Effect | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
|---|---|---|---|---|---|---|---|---|---|---|
| AVISITN*TRTPN | 7 | 1 | -6.2343 | 0.6492 | 143 | -9.60 | <.0001 | 0.05 | -7.5175 | -4.9510 |
| AVISITN*TRTPN | 7 | 2 | -6.1638 | 0.5830 | 159 | -10.57 | <.0001 | 0.05 | -7.3153 | -5.0123 |
| AVISITN*TRTPN | 7 | 3 | -4.3306 | 0.6230 | 146 | -6.95 | <.0001 | 0.05 | -5.5618 | -3.0994 |
| AVISITN*TRTPN | 14 | 1 | -9.1119 | 0.8613 | 144 | -10.58 | <.0001 | 0.05 | -10.8143 | -7.4095 |
| AVISITN*TRTPN | 14 | 2 | -9.0991 | 0.7308 | 140 | -12.45 | <.0001 | 0.05 | -10.5441 | -7.6541 |
| AVISITN*TRTPN | 14 | 3 | -5.5013 | 0.6996 | 153 | -7.86 | <.0001 | 0.05 | -6.8835 | -4.1192 |
| AVISITN*TRTPN | 21 | 1 | -10.9137 | 0.8728 | 148 | -12.50 | <.0001 | 0.05 | -12.6385 | -9.1890 |
| AVISITN*TRTPN | 21 | 2 | -11.3585 | 0.8343 | 140 | -13.61 | <.0001 | 0.05 | -13.0079 | -9.7090 |
| AVISITN*TRTPN | 21 | 3 | -6.8955 | 0.7677 | 143 | -8.98 | <.0001 | 0.05 | -8.4130 | -5.3780 |
| AVISITN*TRTPN | 28 | 1 | -11.0717 | 0.9127 | 144 | -12.13 | <.0001 | 0.05 | -12.8758 | -9.2676 |
| AVISITN*TRTPN | 28 | 2 | -11.6209 | 0.9119 | 136 | -12.74 | <.0001 | 0.05 | -13.4243 | -9.8176 |
| AVISITN*TRTPN | 28 | 3 | -7.1331 | 0.7890 | 146 | -9.04 | <.0001 | 0.05 | -8.6924 | -5.5737 |
| AVISITN*TRTPN | 35 | 1 | -11.6202 | 0.9220 | 138 | -12.60 | <.0001 | 0.05 | -13.4433 | -9.7972 |
| AVISITN*TRTPN | 35 | 2 | -13.1883 | 0.9849 | 137 | -13.39 | <.0001 | 0.05 | -15.1358 | -11.2407 |
| AVISITN*TRTPN | 35 | 3 | -7.8720 | 0.8310 | 144 | -9.47 | <.0001 | 0.05 | -9.5146 | -6.2295 |
| AVISITN*TRTPN | 42 | 1 | -12.1124 | 0.9593 | 140 | -12.63 | <.0001 | 0.05 | -14.0089 | -10.2158 |
| AVISITN*TRTPN | 42 | 2 | -12.5311 | 1.0402 | 135 | -12.05 | <.0001 | 0.05 | -14.5884 | -10.4738 |
| AVISITN*TRTPN | 42 | 3 | -8.1275 | 0.8928 | 142 | -9.10 | <.0001 | 0.05 | -9.8925 | -6.3625 |

CENTANAFADINE 19 OF 26


STAT-4.10

Proc Mixed Output Using Heterogeneous Variance Structure for Treatment Groups (Efficacy Sample)

------ Parameter Code=AISRSTOT ------

# The Mixed Procedure

## Differences of Least Squares Means

| | Analysis<br>Visit | Planned<br>Treatment | Analysis<br>Visit | Planned<br>Treatment | | Standard | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Effect | (N) | (N) | (N) | (N) | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| AVISITN*TRTPN | 7 | 1 | 7 | 2 | -0.07041 | 0.7962 | 240 | -0.09 | 0.9296 | 0.05 | -1.6389 | 1.4980 |
| AVISITN*TRTPN | 7 | 1 | 7 | 3 | -1.9037 | 0.8264 | 248 | -2.30 | 0.0221 | 0.05 | -3.5313 | -0.2761 |
| AVISITN*TRTPN | 7 | 1 | 14 | 1 | 2.8777 | 0.6083 | 130 | 4.73 | <.0001 | 0.05 | 1.6742 | 4.0812 |
| AVISITN*TRTPN | 7 | 1 | 14 | 2 | 2.8648 | 0.9105 | 235 | 3.15 | 0.0019 | 0.05 | 1.0711 | 4.6586 |
| AVISITN*TRTPN | 7 | 1 | 14 | 3 | -0.7329 | 0.8853 | 251 | -0.83 | 0.4086 | 0.05 | -2.4765 | 1.0107 |
| AVISITN*TRTPN | 7 | 1 | 21 | 1 | 4.6795 | 0.6357 | 125 | 7.36 | <.0001 | 0.05 | 3.4213 | 5.9376 |
| AVISITN*TRTPN | 7 | 1 | 21 | 2 | 5.1242 | 0.9953 | 223 | 5.15 | <.0001 | 0.05 | 3.1629 | 7.0855 |
| AVISITN*TRTPN | 7 | 1 | 21 | 3 | 0.6613 | 0.9401 | 234 | 0.70 | 0.4825 | 0.05 | -1.1909 | 2.5134 |
| AVISITN*TRTPN | 7 | 1 | 28 | 1 | 4.8374 | 0.6689 | 107 | 7.23 | <.0001 | 0.05 | 3.5114 | 6.1635 |
| AVISITN*TRTPN | 7 | 1 | 28 | 2 | 5.3867 | 1.0612 | 209 | 5.08 | <.0001 | 0.05 | 3.2946 | 7.4788 |
| AVISITN*TRTPN | 7 | 1 | 28 | 3 | 0.8988 | 0.9577 | 232 | 0.94 | 0.3489 | 0.05 | -0.9880 | 2.7856 |
| AVISITN*TRTPN | 7 | 1 | 35 | 1 | 5.3860 | 0.7106 | 103 | 7.58 | <.0001 | 0.05 | 3.9767 | 6.7953 |
| AVISITN*TRTPN | 7 | 1 | 35 | 2 | 6.9540 | 1.1245 | 205 | 6.18 | <.0001 | 0.05 | 4.7370 | 9.1711 |
| AVISITN*TRTPN | 7 | 1 | 35 | 3 | 1.6378 | 0.9925 | 229 | 1.65 | 0.1003 | 0.05 | -0.3178 | 3.5934 |
| AVISITN*TRTPN | 7 | 1 | 42 | 1 | 5.8781 | 0.7520 | 100 | 7.82 | <.0001 | 0.05 | 4.3862 | 7.3700 |
| AVISITN*TRTPN | 7 | 1 | 42 | 2 | 6.2968 | 1.1733 | 197 | 5.37 | <.0001 | 0.05 | 3.9829 | 8.6107 |
| AVISITN*TRTPN | 7 | 1 | 42 | 3 | 1.8932 | 1.0448 | 220 | 1.81 | 0.0713 | 0.05 | -0.1659 | 3.9523 |
| AVISITN*TRTPN | 7 | 2 | 7 | 3 | -1.8333 | 0.7769 | 236 | -2.36 | 0.0191 | 0.05 | -3.3638 | -0.3028 |
| AVISITN*TRTPN | 7 | 2 | 14 | 1 | 2.9481 | 0.9769 | 217 | 3.02 | 0.0029 | 0.05 | 1.0226 | 4.8736 |
| AVISITN*TRTPN | 7 | 2 | 14 | 2 | 2.9352 | 0.5957 | 124 | 4.93 | <.0001 | 0.05 | 1.7563 | 4.1142 |
| AVISITN*TRTPN | 7 | 2 | 14 | 3 | -0.6625 | 0.8392 | 237 | -0.79 | 0.4306 | 0.05 | -2.3157 | 0.9907 |
| AVISITN*TRTPN | 7 | 2 | 21 | 1 | 4.7499 | 0.9872 | 222 | 4.81 | <.0001 | 0.05 | 2.8045 | 6.6953 |

CENTANAFADINE 20 OF 26 PROTOCOL 405-201-00014

STAT-4.10

Proc Mixed Output Using Heterogeneous Variance Structure for Treatment Groups (Efficacy Sample)

Parameter Code=AISRSTOT ------

#### The Mixed Procedure

#### Differences of Least Squares Means

| Analysis | Planned | Analysis | Planned | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| (N) | (N) | (N) | (N) | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| 7 | 2 | 21 | 2 | 5.1946 | 0.6623 | 127 | 7.84 | <.0001 | 0.05 | 3.8840 | 6.5052 |
| 7 | 2 | 21 | 3 | 0.7317 | 0.8968 | 222 | 0.82 | 0.4154 | 0.05 | -1.0357 | 2.4990 |
| 7 | 2 | 28 | 1 | 4.9078 | 1.0227 | 212 | 4.80 | <.0001 | 0.05 | 2.8918 | 6.9238 |
| 7 | 2 | 28 | 2 | 5.4571 | 0.7394 | 123 | 7.38 | <.0001 | 0.05 | 3.9936 | 6.9207 |
| 7 | 2 | 28 | 3 | 0.9692 | 0.9152 | 226 | 1.06 | 0.2907 | 0.05 | -0.8343 | 2.7727 |
| 7 | 2 | 35 | 1 | 5.4564 | 1.0312 | 202 | 5.29 | <.0001 | 0.05 | 3.4231 | 7.4897 |
| 7 | 2 | 35 | 2 | 7.0244 | 0.8369 | 117 | 8.39 | <.0001 | 0.05 | 5.3670 | 8.6819 |
| 7 | 2 | 35 | 3 | 1.7082 | 0.9516 | 218 | 1.80 | 0.0740 | 0.05 | -0.1674 | 3.5838 |
| 7 | 2 | 42 | 1 | 5.9485 | 1.0645 | 201 | 5.59 | <.0001 | 0.05 | 3.8495 | 8.0475 |
| 7 | 2 | 42 | 2 | 6.3673 | 0.9160 | 116 | 6.95 | <.0001 | 0.05 | 4.5531 | 8.1814 |
| 7 | 2 | 42 | 3 | 1.9637 | 1.0060 | 208 | 1.95 | 0.0523 | 0.05 | -0.01970 | 3.9470 |
| 7 | 3 | 14 | 1 | 4.7814 | 1.0016 | 225 | 4.77 | <.0001 | 0.05 | 2.8076 | 6.7551 |
| 7 | 3 | 14 | 2 | 4.7685 | 0.8936 | 227 | 5.34 | <.0001 | 0.05 | 3.0077 | 6.5293 |
| 7 | 3 | 14 | 3 | 1.1708 | 0.3843 | 131 | 3.05 | 0.0028 | 0.05 | 0.4106 | 1.9310 |
| 7 | 3 | 21 | 1 | 6.5832 | 1.0115 | 226 | 6.51 | <.0001 | 0.05 | 4.5899 | 8.5764 |
| 7 | 3 | 21 | 2 | 7.0279 | 0.9799 | 219 | 7.17 | <.0001 | 0.05 | 5.0966 | 8.9592 |
| 7 | 3 | 21 | 3 | 2.5650 | 0.5796 | 122 | 4.43 | <.0001 | 0.05 | 1.4176 | 3.7124 |
| 7 | 3 | 28 | 1 | 6.7411 | 1.0463 | 218 | 6.44 | <.0001 | 0.05 | 4.6790 | 8.8032 |
| 7 | 3 | 28 | 2 | 7.2904 | 1.0468 | 207 | 6.96 | <.0001 | 0.05 | 5.2266 | 9.3542 |
| 7 | 3 | 28 | 3 | 2.8025 | 0.5700 | 132 | 4.92 | <.0001 | 0.05 | 1.6749 | 3.9301 |
| 7 | 3 | 35 | 1 | 7.2897 | 1.0544 | 212 | 6.91 | <.0001 | 0.05 | 5.2111 | 9.3682 |
| 7 | 3 | 35 | 2 | 8.8577 | 1.1109 | 201 | 7.97 | <.0001 | 0.05 | 6.6671 | 11.0483 |
| | Analysis Visit (N) 7 7 7 7 7 7 7 7 7 7 7 7 7 7 7 7 7 7 | Visit Treatment (N) (N) 7 2 7 | Visit (N) (N) (N) 7 | Visit (N) Treatment (N) Visit (N) Treatment (N) 7 2 21 2 7 2 21 3 7 2 28 1 7 2 28 2 7 2 28 3 7 2 35 1 7 2 35 2 7 2 35 3 7 2 42 1 7 2 42 2 7 2 42 3 7 3 14 1 7 3 14 3 7 3 21 2 7 3 21 2 7 3 28 1 7 3 28 2 7 3 28 3 7 3 28 3 7 3 28 3 | Visit (N) Treatment (N) Visit (N) Treatment (N) Estimate 7 2 21 2 5.1946 7 2 21 3 0.7317 7 2 28 1 4.9078 7 2 28 2 5.4571 7 2 28 3 0.9692 7 2 28 3 0.9692 7 2 35 1 5.4564 7 2 35 2 7.0244 7 2 35 3 1.7082 7 2 42 1 5.9485 7 2 42 1 5.9485 7 2 42 2 6.3673 7 2 42 3 1.9637 7 3 14 1 4.7685 7 3 14 3 1.1708 7 3 21 2 <td>Visit Treatment (N) Visit (N) Treatment (N) Standard Error 7 2 21 2 5.1946 0.6623 7 2 21 3 0.7317 0.8968 7 2 28 1 4.9078 1.0227 7 2 28 2 5.4571 0.7394 7 2 28 3 0.9692 0.9152 7 2 28 3 0.9692 0.9152 7 2 35 1 5.4564 1.0312 7 2 35 2 7.0244 0.8369 7 2 35 3 1.7082 0.9516 7 2 42 1 5.9485 1.0645 7 2 42 2 6.3673 0.9160 7 2 42 3 1.9637 1.0060 7 3 14 1 4.7814 1.0016</td> <td>Visit (N) Treatment (N) Visit (N) Treatment (N) Standard (N) Error (N) DF 7 2 21 2 5.1946 0.6623 127 7 2 21 3 0.7317 0.8968 222 7 2 28 1 4.9078 1.0227 212 7 2 28 2 5.4571 0.7394 123 7 2 28 3 0.9692 0.9152 226 7 2 35 1 5.4564 1.0312 202 7 2 35 2 7.0244 0.8369 117 7 2 35 3 1.7082 0.9516 218 7 2 42 1 5.9485 1.0645 201 7 2 42 2 6.3673 0.9160 116 7 2 42 3 1.9637 1.0060 208</td> <td>Visit Treatment (N) Visit (N) Treatment (N) Standard (N) Error DF t Value 7 2 21 2 5.1946 0.6623 127 7.84 7 2 21 3 0.7317 0.8968 222 0.82 7 2 28 1 4.9078 1.0227 212 4.80 7 2 28 2 5.4571 0.7394 123 7.38 7 2 28 3 0.9692 0.9152 226 1.06 7 2 35 1 5.4564 1.0312 202 5.29 7 2 35 2 7.0244 0.8369 117 8.39 7 2 35 3 1.7082 0.9516 218 1.80 7 2 42 1 5.9485 1.0645 201 5.59 7 2 42 2 6.3673 0.9160<td>Visit (N) Treatment (N) Visit (N) Treatment (N) Standard (N) Estimate Error DF t Value Pr &gt; t 7 2 21 2 5.1946 0.6623 127 7.84 &lt;.0001</td> 7 2 21 3 0.7317 0.8968 222 0.82 0.4154 7 2 28 1 4.9078 1.0227 212 4.80 &lt;.0001</td> 7 2 28 2 5.4571 0.7394 123 7.38 <.0001 | Visit Treatment (N) Visit (N) Treatment (N) Standard Error 7 2 21 2 5.1946 0.6623 7 2 21 3 0.7317 0.8968 7 2 28 1 4.9078 1.0227 7 2 28 2 5.4571 0.7394 7 2 28 3 0.9692 0.9152 7 2 28 3 0.9692 0.9152 7 2 35 1 5.4564 1.0312 7 2 35 2 7.0244 0.8369 7 2 35 3 1.7082 0.9516 7 2 42 1 5.9485 1.0645 7 2 42 2 6.3673 0.9160 7 2 42 3 1.9637 1.0060 7 3 14 1 4.7814 1.0016 | Visit (N) Treatment (N) Visit (N) Treatment (N) Standard (N) Error (N) DF 7 2 21 2 5.1946 0.6623 127 7 2 21 3 0.7317 0.8968 222 7 2 28 1 4.9078 1.0227 212 7 2 28 2 5.4571 0.7394 123 7 2 28 3 0.9692 0.9152 226 7 2 35 1 5.4564 1.0312 202 7 2 35 2 7.0244 0.8369 117 7 2 35 3 1.7082 0.9516 218 7 2 42 1 5.9485 1.0645 201 7 2 42 2 6.3673 0.9160 116 7 2 42 3 1.9637 1.0060 208 | Visit Treatment (N) Visit (N) Treatment (N) Standard (N) Error DF t Value 7 2 21 2 5.1946 0.6623 127 7.84 7 2 21 3 0.7317 0.8968 222 0.82 7 2 28 1 4.9078 1.0227 212 4.80 7 2 28 2 5.4571 0.7394 123 7.38 7 2 28 3 0.9692 0.9152 226 1.06 7 2 35 1 5.4564 1.0312 202 5.29 7 2 35 2 7.0244 0.8369 117 8.39 7 2 35 3 1.7082 0.9516 218 1.80 7 2 42 1 5.9485 1.0645 201 5.59 7 2 42 2 6.3673 0.9160 <td>Visit (N) Treatment (N) Visit (N) Treatment (N) Standard (N) Estimate Error DF t Value Pr &gt; t 7 2 21 2 5.1946 0.6623 127 7.84 &lt;.0001</td> 7 2 21 3 0.7317 0.8968 222 0.82 0.4154 7 2 28 1 4.9078 1.0227 212 4.80 <.0001 | Visit (N) Treatment (N) Visit (N) Treatment (N) Standard (N) Estimate Error DF t Value Pr > t 7 2 21 2 5.1946 0.6623 127 7.84 <.0001 | Visit (N) Treatment (N) Visit (N) Treatment (N) Standard (N) Error DF t Value Pr > t Alpha 7 2 21 2 5.1946 0.6623 127 7.84 <.0001 | Visit (N) Treatment (N) Visit (N) Treatment (N) Standard Error DF t Value Pr > t Alpha Lower 7 2 21 2 5.1946 0.6623 127 7.84 <.0001 |

CENTANAFADINE 21 OF 26 PROTOCOL 405-201-00014

 ${\tt STAT-4.10}\\ {\tt Proc\ Mixed\ Output\ Using\ Heterogeneous\ Variance\ Structure\ for\ Treatment\ Groups}\\ ({\tt Efficacy\ Sample})$ 

Parameter Code=AISRSTOT ------

# The Mixed Procedure

#### Differences of Least Squares Means

| Analysis | Planned | Analysis | Planned | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| (N) | (N) | (N) | (N) | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| 7 | 3 | 35 | 3 | 3.5415 | 0.6078 | 121 | 5.83 | <.0001 | 0.05 | 2.3383 | 4.7447 |
| 7 | 3 | 42 | 1 | 7.7818 | 1.0871 | 208 | 7.16 | <.0001 | 0.05 | 5.6387 | 9.9249 |
| 7 | 3 | 42 | 2 | 8.2005 | 1.1603 | 193 | 7.07 | <.0001 | 0.05 | 5.9120 | 10.4891 |
| 7 | 3 | 42 | 3 | 3.7969 | 0.6986 | 121 | 5.44 | <.0001 | 0.05 | 2.4139 | 5.1800 |
| 14 | 1 | 14 | 2 | -0.01284 | 1.0728 | 241 | -0.01 | 0.9905 | 0.05 | -2.1262 | 2.1005 |
| 14 | 1 | 14 | 3 | -3.6106 | 1.0505 | 244 | -3.44 | 0.0007 | 0.05 | -5.6798 | -1.5414 |
| 14 | 1 | 21 | 1 | 1.8018 | 0.4983 | 124 | 3.62 | 0.0004 | 0.05 | 0.8156 | 2.7880 |
| 14 | 1 | 21 | 2 | 2.2465 | 1.1457 | 246 | 1.96 | 0.0510 | 0.05 | -0.01000 | 4.5031 |
| 14 | 1 | 21 | 3 | -2.2164 | 1.0971 | 248 | -2.02 | 0.0444 | 0.05 | -4.3773 | -0.05549 |
| 14 | 1 | 28 | 1 | 1.9598 | 0.5937 | 126 | 3.30 | 0.0013 | 0.05 | 0.7848 | 3.1347 |
| 14 | 1 | 28 | 2 | 2.5090 | 1.2033 | 242 | 2.09 | 0.0381 | 0.05 | 0.1387 | 4.8793 |
| 14 | 1 | 28 | 3 | -1.9789 | 1.1122 | 246 | -1.78 | 0.0764 | 0.05 | -4.1696 | 0.2119 |
| 14 | 1 | 35 | 1 | 2.5083 | 0.6469 | 124 | 3.88 | 0.0002 | 0.05 | 1.2279 | 3.7887 |
| 14 | 1 | 35 | 2 | 4.0764 | 1.2595 | 241 | 3.24 | 0.0014 | 0.05 | 1.5953 | 6.5574 |
| 14 | 1 | 35 | 3 | -1.2399 | 1.1423 | 252 | -1.09 | 0.2788 | 0.05 | -3.4897 | 1.0099 |
| 14 | 1 | 42 | 1 | 3.0004 | 0.7209 | 123 | 4.16 | <.0001 | 0.05 | 1.5735 | 4.4274 |
| 14 | 1 | 42 | 2 | 3.4192 | 1.3033 | 235 | 2.62 | 0.0093 | 0.05 | 0.8516 | 5.9868 |
| 14 | 1 | 42 | 3 | -0.9844 | 1.1881 | 252 | -0.83 | 0.4081 | 0.05 | -3.3243 | 1.3554 |
| 14 | 2 | 14 | 3 | -3.5977 | 0.9490 | 240 | -3.79 | 0.0002 | 0.05 | -5.4672 | -1.7283 |
| 14 | 2 | 21 | 1 | 1.8147 | 1.0821 | 244 | 1.68 | 0.0948 | 0.05 | -0.3168 | 3.9461 |
| 14 | 2 | 21 | 2 | 2.2594 | 0.4852 | 117 | 4.66 | <.0001 | 0.05 | 1.2985 | 3.2202 |
| 14 | 2 | 21 | 3 | -2.2036 | 1.0001 | 237 | -2.20 | 0.0285 | 0.05 | -4.1737 | -0.2334 |
| | Visit<br>(N) 7 7 7 14 14 14 14 14 14 14 1 | Visit (N) (N) 7 3 7 3 7 3 7 3 14 1 14 1 14 1 14 1 14 1 14 1 14 1 14 | Visit (N) (N) (N) 7 3 355 7 3 42 7 3 42 7 3 42 14 1 14 14 1 14 14 1 21 14 1 21 14 1 22 14 1 28 14 1 28 14 1 35 14 1 35 14 1 35 14 1 35 14 1 42 | Visit Treatment Visit Treatment (N) (N) (N) (N) 7 3 35 3 7 3 42 1 7 3 42 2 7 3 42 3 14 1 14 2 14 1 14 3 14 1 21 2 14 1 21 3 14 1 28 1 14 1 28 2 14 1 28 2 14 1 35 1 14 1 35 2 14 1 35 2 14 1 42 1 14 1 42 1 14 1 42 2 14 1 42 3 14 1 42 | Visit Treatment (N) Visit (N) Treatment (N) Estimate 7 3 35 3 3.5415 7 3 42 1 7.7818 7 3 42 2 8.2005 7 3 42 3 3.7969 14 1 14 2 -0.01284 14 1 14 3 -3.6106 14 1 21 1 1.8018 14 1 21 2 2.2465 14 1 21 3 -2.2164 14 1 21 3 -2.2164 14 1 28 1 1.9598 14 1 28 2 2.5090 14 1 28 2 2.5083 14 1 35 1 2.5083 14 1 35 2 4.0764 14 1 35 | Visit (N) Treatment (N) Visit (N) Treatment (N) Standard Error 7 3 35 3 3.5415 0.6078 7 3 42 1 7.7818 1.0871 7 3 42 2 8.2005 1.1603 7 3 42 3 3.7969 0.6986 14 1 14 2 -0.01284 1.0728 14 1 14 3 -3.6106 1.0505 14 1 14 3 -3.6106 1.0505 14 1 21 1 1.8018 0.4983 14 1 21 2 2.2465 1.1457 14 1 21 3 -2.2164 1.0971 14 1 21 3 -2.2164 1.0971 14 1 28 2 2.5090 1.2033 14 1 28 2 2.5090 1.2033 | Visit (N) Treatment (N) Visit (N) Treatment (N) Standard (N) Error (N) DF 7 3 35 3 3.5415 0.6078 121 7 3 42 1 7.7818 1.0871 208 7 3 42 2 8.2005 1.1603 193 7 3 42 3 3.7969 0.6986 121 14 1 14 2 -0.01284 1.0728 241 14 1 14 3 -3.6106 1.0505 244 14 1 21 1 1.8018 0.4983 124 14 1 21 2 2.2465 1.1457 246 14 1 21 3 -2.2164 1.0971 248 14 1 28 1 1.9598 0.5937 126 14 1 28 2 2.5090 1.2033 242 <t< td=""><td>Visit (N) Treatment (N) Visit (N) Treatment (N) Standard (N) Error (N) DF t Value 7 3 35 3 3.5415 0.6078 121 5.83 7 3 42 1 7.7818 1.0871 208 7.16 7 3 42 2 8.2005 1.1603 193 7.07 7 3 42 3 3.7969 0.6986 121 5.44 14 1 14 2 -0.01284 1.0728 241 -0.01 14 1 14 3 -3.6106 1.0505 244 -3.44 14 1 21 1 1.8018 0.4983 124 3.62 14 1 21 2 2.2465 1.1457 246 1.96 14 1 21 3 -2.2164 1.0971 248 -2.02 14 1 28 1 1.9598 0.5937</td><td>Visit (N) Treatment (N) Visit (N) Treatment (N) Standard (N) Error DF t Value Pr &gt; t 7 3 35 3 3.5415 0.6078 121 5.83 &lt;.0001</td> 7 3 42 1 7.7818 1.0871 208 7.16 &lt;.0001</t<> | Visit (N) Treatment (N) Visit (N) Treatment (N) Standard (N) Error (N) DF t Value 7 3 35 3 3.5415 0.6078 121 5.83 7 3 42 1 7.7818 1.0871 208 7.16 7 3 42 2 8.2005 1.1603 193 7.07 7 3 42 3 3.7969 0.6986 121 5.44 14 1 14 2 -0.01284 1.0728 241 -0.01 14 1 14 3 -3.6106 1.0505 244 -3.44 14 1 21 1 1.8018 0.4983 124 3.62 14 1 21 2 2.2465 1.1457 246 1.96 14 1 21 3 -2.2164 1.0971 248 -2.02 14 1 28 1 1.9598 0.5937 | Visit (N) Treatment (N) Visit (N) Treatment (N) Standard (N) Error DF t Value Pr > t 7 3 35 3 3.5415 0.6078 121 5.83 <.0001 | Visit (N) Treatment (N) Visit (N) Treatment (N) Standard Error DF t Value Pr > t Alpha 7 3 35 3 3.5415 0.6078 121 5.83 <.0001 | Visit |

CENTANAFADINE 22 OF 26 PROTOCOL 405-201-00014

 ${\tt STAT-4.10}\\ {\tt Proc\ Mixed\ Output\ Using\ Heterogeneous\ Variance\ Structure\ for\ Treatment\ Groups}\\ ({\tt Efficacy\ Sample})$ 

Parameter Code=AISRSTOT ------

#### The Mixed Procedure

#### Differences of Least Squares Means

| | Analysis<br>Visit | Planned<br>Treatment | Analysis<br>Visit | Planned<br>Treatment | | Standard | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Effect | (N) | (N) | (N) | (N) | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| AVISITN*TRTPN | 14 | 2 | 28 | 1 | 1.9726 | 1.1146 | 237 | 1.77 | 0.0780 | 0.05 | -0.2231 | 4.1683 |
| AVISITN*TRTPN | 14 | 2 | 28 | 2 | 2.5219 | 0.6012 | 117 | 4.19 | <.0001 | 0.05 | 1.3313 | 3.7125 |
| AVISITN*TRTPN | 14 | 2 | 28 | 3 | -1.9660 | 1.0166 | 246 | -1.93 | 0.0543 | 0.05 | -3.9684 | 0.03631 |
| AVISITN*TRTPN | 14 | 2 | 35 | 1 | 2.5211 | 1.1224 | 230 | 2.25 | 0.0256 | 0.05 | 0.3096 | 4.7327 |
| AVISITN*TRTPN | 14 | 2 | 35 | 2 | 4.0892 | 0.7094 | 112 | 5.76 | <.0001 | 0.05 | 2.6836 | 5.4949 |
| AVISITN*TRTPN | 14 | 2 | 35 | 3 | -1.2270 | 1.0495 | 241 | -1.17 | 0.2435 | 0.05 | -3.2945 | 0.8404 |
| AVISITN*TRTPN | 14 | 2 | 42 | 1 | 3.0133 | 1.1531 | 228 | 2.61 | 0.0096 | 0.05 | 0.7411 | 5.2855 |
| AVISITN*TRTPN | 14 | 2 | 42 | 2 | 3.4320 | 0.7779 | 110 | 4.41 | <.0001 | 0.05 | 1.8903 | 4.9737 |
| AVISITN*TRTPN | 14 | 2 | 42 | 3 | -0.9716 | 1.0991 | 236 | -0.88 | 0.3776 | 0.05 | -3.1369 | 1.1937 |
| AVISITN*TRTPN | 14 | 3 | 21 | 1 | 5.4124 | 1.0600 | 245 | 5.11 | <.0001 | 0.05 | 3.3245 | 7.5003 |
| AVISITN*TRTPN | 14 | 3 | 21 | 2 | 5.8571 | 1.0305 | 236 | 5.68 | <.0001 | 0.05 | 3.8269 | 7.8873 |
| AVISITN*TRTPN | 14 | 3 | 21 | 3 | 1.3942 | 0.5352 | 124 | 2.61 | 0.0103 | 0.05 | 0.3349 | 2.4535 |
| AVISITN*TRTPN | 14 | 3 | 28 | 1 | 5.5703 | 1.0932 | 237 | 5.10 | <.0001 | 0.05 | 3.4167 | 7.7240 |
| AVISITN*TRTPN | 14 | 3 | 28 | 2 | 6.1196 | 1.0943 | 225 | 5.59 | <.0001 | 0.05 | 3.9632 | 8.2760 |
| AVISITN*TRTPN | 14 | 3 | 28 | 3 | 1.6317 | 0.5625 | 130 | 2.90 | 0.0044 | 0.05 | 0.5189 | 2.7446 |
| AVISITN*TRTPN | 14 | 3 | 35 | 1 | 6.1189 | 1.1010 | 230 | 5.56 | <.0001 | 0.05 | 3.9495 | 8.2882 |
| AVISITN*TRTPN | 14 | 3 | 35 | 2 | 7.6869 | 1.1558 | 218 | 6.65 | <.0001 | 0.05 | 5.4090 | 9.9649 |
| AVISITN*TRTPN | 14 | 3 | 35 | 3 | 2.3707 | 0.5550 | 119 | 4.27 | <.0001 | 0.05 | 1.2717 | 3.4697 |
| AVISITN*TRTPN | 14 | 3 | 42 | 1 | 6.6110 | 1.1323 | 226 | 5.84 | <.0001 | 0.05 | 4.3799 | 8.8421 |
| AVISITN*TRTPN | 14 | 3 | 42 | 2 | 7.0298 | 1.2033 | 210 | 5.84 | <.0001 | 0.05 | 4.6576 | 9.4019 |
| AVISITN*TRTPN | 14 | 3 | 42 | 3 | 2.6262 | 0.6518 | 120 | 4.03 | <.0001 | 0.05 | 1.3357 | 3.9166 |
| AVISITN*TRTPN | 21 | 1 | 21 | 2 | 0.4447 | 1.1553 | 250 | 0.38 | 0.7006 | 0.05 | -1.8307 | 2.7201 |
CENTANAFADINE 23 OF 26 PROTOCOL 405-201-00014

 ${\tt STAT-4.10}\\ {\tt Proc\ Mixed\ Output\ Using\ Heterogeneous\ Variance\ Structure\ for\ Treatment\ Groups}\\ ({\tt Efficacy\ Sample})$ 

-----

Parameter Code=AISRSTOT ------

### The Mixed Procedure

### Differences of Least Squares Means

| | Analysis | Planned | Analysis | Planned | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Visit | Treatment | Visit | Treatment | | Standard | | | | | | |
| Effect | (N) | (N) | (N) | (N) | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| AVISITN*TRTPN | 21 | 1 | 21 | 3 | -4.0182 | 1.1060 | 249 | -3.63 | 0.0003 | 0.05 | -6.1964 | -1.8400 |
| AVISITN*TRTPN | 21 | 1 | 28 | 1 | 0.1579 | 0.4168 | 121 | 0.38 | 0.7054 | 0.05 | -0.6672 | 0.9831 |
| AVISITN*TRTPN | 21 | 1 | 28 | 2 | 0.7072 | 1.2123 | 246 | 0.58 | 0.5602 | 0.05 | -1.6806 | 3.0950 |
| AVISITN*TRTPN | 21 | 1 | 28 | 3 | -3.7807 | 1.1210 | 249 | -3.37 | 0.0009 | 0.05 | -5.9886 | -1.5728 |
| AVISITN*TRTPN | 21 | 1 | 35 | 1 | 0.7065 | 0.5769 | 114 | 1.22 | 0.2232 | 0.05 | -0.4362 | 1.8492 |
| AVISITN*TRTPN | 21 | 1 | 35 | 2 | 2.2745 | 1.2680 | 245 | 1.79 | 0.0741 | 0.05 | -0.2230 | 4.7721 |
| AVISITN*TRTPN | 21 | 1 | 35 | 3 | -3.0417 | 1.1509 | 253 | -2.64 | 0.0087 | 0.05 | -5.3083 | -0.7751 |
| AVISITN*TRTPN | 21 | 1 | 42 | 1 | 1.1986 | 0.5977 | 115 | 2.01 | 0.0473 | 0.05 | 0.01472 | 2.3825 |
| AVISITN*TRTPN | 21 | 1 | 42 | 2 | 1.6174 | 1.3116 | 239 | 1.23 | 0.2187 | 0.05 | -0.9664 | 4.2011 |
| AVISITN*TRTPN | 21 | 1 | 42 | 3 | -2.7862 | 1.1963 | 253 | -2.33 | 0.0206 | 0.05 | -5.1422 | -0.4303 |
| AVISITN*TRTPN | 21 | 2 | 21 | 3 | -4.4629 | 1.0784 | 244 | -4.14 | <.0001 | 0.05 | -6.5872 | -2.3387 |
| AVISITN*TRTPN | 21 | 2 | 28 | 1 | -0.2868 | 1.1855 | 247 | -0.24 | 0.8091 | 0.05 | -2.6218 | 2.0482 |
| AVISITN*TRTPN | 21 | 2 | 28 | 2 | 0.2625 | 0.4862 | 114 | 0.54 | 0.5903 | 0.05 | -0.7006 | 1.2256 |
| AVISITN*TRTPN | 21 | 2 | 28 | 3 | -4.2254 | 1.0936 | 251 | -3.86 | 0.0001 | 0.05 | -6.3792 | -2.0716 |
| AVISITN*TRTPN | 21 | 2 | 35 | 1 | 0.2618 | 1.1929 | 242 | 0.22 | 0.8265 | 0.05 | -2.0880 | 2.6115 |
| AVISITN*TRTPN | 21 | 2 | 35 | 2 | 1.8298 | 0.6210 | 112 | 2.95 | 0.0039 | 0.05 | 0.5995 | 3.0602 |
| AVISITN*TRTPN | 21 | 2 | 35 | 3 | -3.4864 | 1.1242 | 250 | -3.10 | 0.0021 | 0.05 | -5.7006 | -1.2723 |
| AVISITN*TRTPN | 21 | 2 | 42 | 1 | 0.7539 | 1.2219 | 242 | 0.62 | 0.5378 | 0.05 | -1.6529 | 3.1607 |
| AVISITN*TRTPN | 21 | 2 | 42 | 2 | 1.1726 | 0.7252 | 110 | 1.62 | 0.1087 | 0.05 | -0.2645 | 2.6098 |
| AVISITN*TRTPN | 21 | 2 | 42 | 3 | -3.2310 | 1.1706 | 250 | -2.76 | 0.0062 | 0.05 | -5.5365 | -0.9254 |
| AVISITN*TRTPN | 21 | 3 | 28 | 1 | 4.1762 | 1.1379 | 246 | 3.67 | 0.0003 | 0.05 | 1.9348 | 6.4175 |
| AVISITN*TRTPN | 21 | 3 | 28 | 2 | 4.7254 | 1.1393 | 234 | 4.15 | <.0001 | 0.05 | 2.4808 | 6.9701 |

CENTANAFADINE 24 OF 26


# STAT-4.10 Proc Mixed Output Using Heterogeneous Variance Structure for Treatment Groups (Efficacy Sample)

\_\_\_\_\_\_

## The Mixed Procedure

### Differences of Least Squares Means

| | Analysis<br>Visit | Planned<br>Treatment | Analysis<br>Visit | Planned<br>Treatment | | Standard | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Effect | (N) | (N) | (N) | (N) | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| AVISITN*TRTPN | 21 | 3 | 28 | 3 | 0.2375 | 0.4197 | 124 | 0.57 | 0.5725 | 0.05 | -0.5932 | 1.0683 |
| AVISITN*TRTPN | 21 | 3 | 35 | 1 | 4.7247 | 1.1454 | 239 | 4.12 | <.0001 | 0.05 | 2.4683 | 6.9811 |
| AVISITN*TRTPN | 21 | 3 | 35 | 2 | 6.2928 | 1.1985 | 231 | 5.25 | <.0001 | 0.05 | 3.9314 | 8.6541 |
| AVISITN*TRTPN | 21 | 3 | 35 | 3 | 0.9765 | 0.4363 | 125 | 2.24 | 0.0270 | 0.05 | 0.1131 | 1.8399 |
| AVISITN*TRTPN | 21 | 3 | 42 | 1 | 5.2168 | 1.1755 | 237 | 4.44 | <.0001 | 0.05 | 2.9011 | 7.5326 |
| AVISITN*TRTPN | 21 | 3 | 42 | 2 | 5.6356 | 1.2444 | 223 | 4.53 | <.0001 | 0.05 | 3.1832 | 8.0880 |
| AVISITN*TRTPN | 21 | 3 | 42 | 3 | 1.2320 | 0.4938 | 124 | 2.49 | 0.0139 | 0.05 | 0.2546 | 2.2093 |
| AVISITN*TRTPN | 28 | 1 | 28 | 2 | 0.5493 | 1.2420 | 246 | 0.44 | 0.6587 | 0.05 | -1.8971 | 2.9956 |
| AVISITN*TRTPN | 28 | 1 | 28 | 3 | -3.9386 | 1.1523 | 245 | -3.42 | 0.0007 | 0.05 | -6.2082 | -1.6690 |
| AVISITN*TRTPN | 28 | 1 | 35 | 1 | 0.5486 | 0.4314 | 115 | 1.27 | 0.2061 | 0.05 | -0.3059 | 1.4030 |
| AVISITN*TRTPN | 28 | 1 | 35 | 2 | 2.1166 | 1.2961 | 246 | 1.63 | 0.1037 | 0.05 | -0.4363 | 4.6695 |
| AVISITN*TRTPN | 28 | 1 | 35 | 3 | -3.1996 | 1.1814 | 251 | -2.71 | 0.0072 | 0.05 | -5.5264 | -0.8728 |
| AVISITN*TRTPN | 28 | 1 | 42 | 1 | 1.0407 | 0.4870 | 114 | 2.14 | 0.0347 | 0.05 | 0.07594 | 2.0054 |
| AVISITN*TRTPN | 28 | 1 | 42 | 2 | 1.4594 | 1.3388 | 242 | 1.09 | 0.2768 | 0.05 | -1.1778 | 4.0967 |
| AVISITN*TRTPN | 28 | 1 | 42 | 3 | -2.9442 | 1.2257 | 253 | -2.40 | 0.0170 | 0.05 | -5.3581 | -0.5303 |
| AVISITN*TRTPN | 28 | 2 | 28 | 3 | -4.4879 | 1.1541 | 240 | -3.89 | 0.0001 | 0.05 | -6.7614 | -2.2144 |
| AVISITN*TRTPN | 28 | 2 | 35 | 1 | -0.00071 | 1.2487 | 244 | -0.00 | 0.9995 | 0.05 | -2.4604 | 2.4590 |
| AVISITN*TRTPN | 28 | 2 | 35 | 2 | 1.5673 | 0.5233 | 106 | 3.00 | 0.0034 | 0.05 | 0.5299 | 2.6047 |
| AVISITN*TRTPN | 28 | 2 | 35 | 3 | -3.7489 | 1.1831 | 243 | -3.17 | 0.0017 | 0.05 | -6.0794 | -1.4184 |
| AVISITN*TRTPN | 28 | 2 | 42 | 1 | 0.4914 | 1.2765 | 245 | 0.38 | 0.7006 | 0.05 | -2.0229 | 3.0057 |
| AVISITN*TRTPN | 28 | 2 | 42 | 2 | 0.9101 | 0.6303 | 107 | 1.44 | 0.1516 | 0.05 | -0.3393 | 2.1596 |
| AVISITN*TRTPN | 28 | 2 | 42 | 3 | -3.4934 | 1.2273 | 247 | -2.85 | 0.0048 | 0.05 | -5.9108 | -1.0761 |

CENTANAFADINE 25 OF 26 PROTOCOL 405-201-00014

 ${\tt STAT-4.10}\\ {\tt Proc\ Mixed\ Output\ Using\ Heterogeneous\ Variance\ Structure\ for\ Treatment\ Groups}\\ ({\tt Efficacy\ Sample})$ 

Parameter Code=AISRSTOT ------

### The Mixed Procedure

### Differences of Least Squares Means

| | Analysis | Planned | Analysis | Planned | | G1 1 1 | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Visit | Treatment | Visit | Treatment | | Standard | | | | | _ | |
| Effect | (N) | (N) | (N) | (N) | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| AVISITN*TRTPN | 28 | 3 | 35 | 1 | 4.4872 | 1.1598 | 240 | 3.87 | 0.0001 | 0.05 | 2.2026 | 6.7718 |
| AVISITN TRITN AVISITN*TRTPN | 28 | 3 | 35 | 2 | 6.0552 | 1.2125 | 237 | 4.99 | <.0001 | 0.05 | 3.6666 | 8.4439 |
| | | 3 | | 2 | | | | | | | | |
| AVISITN*TRTPN | 28 | 3 | 35 | 3 | 0.7390 | 0.3985 | 123 | 1.85 | 0.0661 | 0.05 | -0.04985 | 1.5278 |
| AVISITN*TRTPN | 28 | 3 | 42 | 1 | 4.9793 | 1.1895 | 239 | 4.19 | <.0001 | 0.05 | 2.6361 | 7.3225 |
| AVISITN*TRTPN | 28 | 3 | 42 | 2 | 5.3980 | 1.2579 | 229 | 4.29 | <.0001 | 0.05 | 2.9194 | 7.8766 |
| AVISITN*TRTPN | 28 | 3 | 42 | 3 | 0.9944 | 0.4443 | 125 | 2.24 | 0.0270 | 0.05 | 0.1151 | 1.8738 |
| AVISITN*TRTPN | 35 | 1 | 35 | 2 | 1.5681 | 1.3037 | 244 | 1.20 | 0.2302 | 0.05 | -1.0000 | 4.1361 |
| AVISITN*TRTPN | 35 | 1 | 35 | 3 | -3.7482 | 1.1884 | 246 | -3.15 | 0.0018 | 0.05 | -6.0888 | -1.4075 |
| AVISITN*TRTPN | 35 | 1 | 42 | 1 | 0.4921 | 0.5403 | 111 | 0.91 | 0.3644 | 0.05 | -0.5785 | 1.5628 |
| AVISITN*TRTPN | 35 | 1 | 42 | 2 | 0.9109 | 1.3458 | 239 | 0.68 | 0.4992 | 0.05 | -1.7403 | 3.5620 |
| AVISITN*TRTPN | 35 | 1 | 42 | 3 | -3.4927 | 1.2325 | 249 | -2.83 | 0.0050 | 0.05 | -5.9203 | -1.0652 |
| AVISITN*TRTPN | 35 | 2 | 35 | 3 | -5.3162 | 1.2406 | 241 | -4.29 | <.0001 | 0.05 | -7.7601 | -2.8724 |
| AVISITN*TRTPN | 35 | 2 | 42 | 1 | -1.0759 | 1.3301 | 247 | -0.81 | 0.4193 | 0.05 | -3.6956 | 1.5438 |
| AVISITN*TRTPN | 35 | 2 | 42 | 2 | -0.6572 | 0.4852 | 99.7 | -1.35 | 0.1786 | 0.05 | -1.6198 | 0.3054 |
| AVISITN*TRTPN | 35 | 2 | 42 | 3 | -5.0608 | 1.2827 | 247 | -3.95 | 0.0001 | 0.05 | -7.5871 | -2.5344 |
| AVISITN*TRTPN | 35 | 3 | 42 | 1 | 4.2403 | 1.2175 | 244 | 3.48 | 0.0006 | 0.05 | 1.8421 | 6.6385 |
| AVISITN*TRTPN | 35 | 3 | 42 | 2 | 4.6591 | 1.2849 | 235 | 3.63 | 0.0004 | 0.05 | 2.1277 | 7.1905 |
| AVISITN*TRTPN | 35 | 3 | 42 | 3 | 0.2555 | 0.3442 | 121 | 0.74 | 0.4594 | 0.05 | -0.4260 | 0.9369 |
| AVISITN*TRTPN | 42 | 1 | 42 | 2 | 0.4187 | 1.3727 | 245 | 0.31 | 0.7606 | 0.05 | -2.2850 | 3.1225 |
| AVISITN*TRTPN | 42 | 1 | 42 | 3 | -3.9849 | 1.2601 | 249 | -3.16 | 0.0018 | 0.05 | -6.4667 | -1.5030 |
| AVISITN*TRTPN | 42 | 2 | 42 | 3 | -4.4036 | 1.3262 | 243 | -3.32 | 0.0010 | 0.05 | -7.0159 | -1.7913 |

CENTANAFADINE 26 OF 26 PROTOCOL 405-201-00014

# STAT-4.10 Proc Mixed Output Using Heterogeneous Variance Structure for Treatment Groups (Efficacy Sample)

Parameter Code=AISRSTOT ------

The Mixed Procedure

Tests of Effect Slices

| | Analysis | | | | |
|---------------|----------|-----|-----|---------|--------|
| | Visit | Num | Den | | |
| Effect | (N) | DF | DF | F Value | Pr > F |
| AVISITN*TRTPN | 7 | 2 | 243 | 3.60 | 0.0289 |
| AVISITN*TRTPN | 14 | 2 | 246 | 9.18 | 0.0001 |
| AVISITN*TRTPN | 21 | 2 | 248 | 10.57 | <.0001 |
| AVISITN*TRTPN | 28 | 2 | 246 | 9.47 | 0.0001 |
| AVISITN*TRTPN | 35 | 2 | 246 | 10.24 | <.0001 |
| AVISITN*TRTPN | 42 | 2 | 247 | 7.30 | 0.0008 |

CENTANAFADINE 1 OF 14 PROTOCOL 405-201-00014

STAT-5.1

Proc Mixed Output for Change from Baseline in CGI-S Scale, MMRM (UN)

(Efficacy Sample)

The Mixed Procedure

Model Information

WORK.INDATA Data Set Dependent Variable CHG Dependent Variable Covariance Structure Unstructured Subject Effect SUBJID Estimation Method REML

Residual Variance Method Fixed Effects SE Method Kenward-Roger Degrees of Freedom Method Kenward-Roger

> Class Level Information Values

6 AVISITN 3 TRTPN

Levels

POOLCNTR 39

Class



CENTANAFADINE

2 OF 14

STAT-5.1
Proc Mixed Output for Change from Baseline in CGI-S Scale, MMRM (UN)
(Efficacy Sample)

\_\_\_\_\_

------ Parameter Code=CGIO201 ------

The Mixed Procedure

Class Level Information

Class Levels Values

SUBJID 421



CENTANAFADINE

3 OF 14

STAT-5.1
Proc Mixed Output for Change from Baseline in CGI-S Scale, MMRM (UN)
(Efficacy Sample)

\_\_\_\_\_

The Mixed Procedure



CENTANAFADINE 4 OF 14 PROTOCOL 405-201-00014

STAT-5.1
Proc Mixed Output for Change from Baseline in CGI-S Scale, MMRM (UN)
(Efficacy Sample)

\_\_\_\_\_

The Mixed Procedure



CENTANAFADINE 5 OF 14 PROTOCOL 405-201-00014

STAT-5.1
Proc Mixed Output for Change from Baseline in CGI-S Scale, MMRM (UN)
(Efficacy Sample)

\_\_\_\_\_\_

The Mixed Procedure




STAT-5.1

Proc Mixed Output for Change from Baseline in CGI-S Scale, MMRM (UN)
(Efficacy Sample)

The Mixed Procedure




STAT-5.1
Proc Mixed Output for Change from Baseline in CGI-S Scale, MMRM (UN)
(Efficacy Sample)

\_\_\_\_\_

The Mixed Procedure



CENTANAFADINE 8 OF 14 PROTOCOL 405-201-00014

### STAT-5.1

| Proc Mixed | Output | for | Change | from | Baseline | in | CGI-S | Scale, | MMRM | (UN) |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | (Ef: | ficacy | z Sample) | | | | | |

-----

The Mixed Procedure

#### Dimensions

| Covariance | Parameters | 21 |
|-------------|------------|-----|
| Columns in | X | 73 |
| Columns in | Z | 0 |
| Subjects | | 421 |
| Max Obs per | Subject | 6 |

### Number of Observations

| Number | of | Observations | Read | 2220 |
|--------|----|--------------|----------|------|
| Number | of | Observations | Used | 2220 |
| Number | of | Observations | Not Used | 0 |

### Iteration History

| Criterion | -2 Res Log Like | Evaluations | Iteration |
|------------|-----------------|-------------|-----------|
| | 5534.17561525 | 1 | 0 |
| 0.00358545 | 3687.88676445 | 2 | 1 |
| 0.00001709 | 3687.36668372 | 1 | 2 |
| 0.00000000 | 3687.36429296 | 1 | 3 |


STAT-5.1

Proc Mixed Output for Change from Baseline in CGI-S Scale, MMRM (UN) (Efficacy Sample)

------ Parameter Code=CGIO201 ------

The Mixed Procedure

Convergence criteria met.

Covariance Parameter Estimates

| Cov Parm | Subject | Estimate |
|----------|---------|----------|
| UN(1,1) | SUBJID | 0.3911 |
| UN(2,1) | SUBJID | 0.2991 |
| UN(2,2) | SUBJID | 0.6117 |
| UN(3,1) | SUBJID | 0.3110 |
| UN(3,2) | SUBJID | 0.5237 |
| UN(3,3) | SUBJID | 0.7431 |
| UN(4,1) | SUBJID | 0.2804 |
| UN(4,2) | SUBJID | 0.5001 |
| UN(4,3) | SUBJID | 0.5893 |
| UN(4,4) | SUBJID | 0.7650 |
| UN(5,1) | SUBJID | 0.3206 |
| UN(5,2) | SUBJID | 0.5243 |
| UN(5,3) | SUBJID | 0.6146 |
| UN(5,4) | SUBJID | 0.6923 |
| UN(5,5) | SUBJID | 0.9120 |
| UN(6,1) | SUBJID | 0.2947 |
| UN(6,2) | SUBJID | 0.5097 |
| UN(6,3) | SUBJID | 0.5999 |

CENTANAFADINE 10 OF 14 PROTOCOL 405-201-00014

### STAT-5.1

Proc Mixed Output for Change from Baseline in CGI-S Scale, MMRM (UN) (Efficacy Sample)

The Mixed Procedure

#### Covariance Parameter Estimates

| Cov Parm | Subject | Estimate |
|----------|---------|----------|
| UN(6,4) | SUBJID | 0.7026 |
| UN(6,5) | SUBJID | 0.8049 |
| UN(6,6) | SUBJID | 0.9541 |

### Fit Statistics

| -2 Res Log Likelihood | 3687.4 |
|--------------------------|--------|
| AIC (Smaller is Better) | 3729.4 |
| AICC (Smaller is Better) | 3729.8 |
| BIC (Smaller is Better) | 3814.3 |

### Null Model Likelihood Ratio Test

| DF | Chi-Square | Pr > ChiSc |
|----|------------|------------|
| 20 | 1046 01 | < 0.001 |


# STAT-5.1 Proc Mixed Output for Change from Baseline in CGI-S Scale, MMRM (UN) (Efficacy Sample)

The Mixed Procedure

## Type 3 Tests of Fixed Effects

| | Num | Den | | |
|---------------|-----|-----|---------|---------|
| Effect | DF | DF | F Value | Pr > F |
| AVISITN | 5 | 352 | 0.16 | 0.9771 |
| TRTPN | 2 | 377 | 4.07 | 0.0179 |
| AVISITN*TRTPN | 10 | 522 | 1.44 | 0.1591 |
| POOLCNTR | 38 | 379 | 1.62 | 0.0135 |
| BASE*AVISITN | 6 | 378 | 6.13 | < .0001 |

## Estimates

| | | Standard | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Label | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| DAY7 1 vs 3 | -0.05184 | 0.07546 | 381 | -0.69 | 0.4925 | 0.05 | -0.2002 | 0.09652 |
| DAY7 2 vs 3 | -0.03062 | 0.07587 | 379 | -0.40 | 0.6868 | 0.05 | -0.1798 | 0.1186 |
| DAY14 1 vs 3 | -0.1951 | 0.09505 | 376 | -2.05 | 0.0408 | 0.05 | -0.3820 | -0.00824 |
| DAY14 2 vs 3 | -0.1611 | 0.09681 | 384 | -1.66 | 0.0968 | 0.05 | -0.3515 | 0.02920 |
| DAY21 1 vs 3 | -0.2313 | 0.1053 | 367 | -2.20 | 0.0286 | 0.05 | -0.4383 | -0.02432 |
| DAY21 2 vs 3 | -0.2400 | 0.1076 | 376 | -2.23 | 0.0262 | 0.05 | -0.4515 | -0.02852 |
| DAY28 1 vs 3 | -0.2650 | 0.1076 | 364 | -2.46 | 0.0142 | 0.05 | -0.4766 | -0.05345 |
| DAY28 2 vs 3 | -0.2665 | 0.1099 | 371 | -2.42 | 0.0158 | 0.05 | -0.4827 | -0.05034 |


# STAT-5.1 Proc Mixed Output for Change from Baseline in CGI-S Scale, MMRM (UN) (Efficacy Sample)

### The Mixed Procedure

#### Estimates

| Label | | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
|---|---|---|---|---|---|---|---|---|---|
| DAY35 | 1 vs 3 | -0.2626 | 0.1183 | 364 | -2.22 | 0.0271 | 0.05 | -0.4952 | -0.02991 |
| DAY35 | 2 vs 3 | -0.3555 | 0.1212 | 373 | -2.93 | 0.0036 | 0.05 | -0.5938 | -0.1173 |
| DAY42 | 1 vs 3 | -0.3287 | 0.1219 | 365 | -2.70 | 0.0073 | 0.05 | -0.5684 | -0.08902 |
| DAY42 | 2 vs 3 | -0.2820 | 0.1249 | 372 | -2.26 | 0.0245 | 0.05 | -0.5276 | -0.03644 |

### Least Squares Means

| Effect | Analysis<br>Visit<br>(N) | Planned<br>Treatment<br>(N) | Estimate | Standard<br>Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
|---|---|---|---|---|---|---|---|---|---|---|
| AVISITN*TRTPN | 7 | 1 | -0.4635 | 0.05831 | 389 | -7.95 | <.0001 | 0.05 | -0.5781 | -0.3488 |
| AVISITN*TRTPN | 7 | 2 | -0.4422 | 0.05866 | 386 | -7.54 | <.0001 | 0.05 | -0.5576 | -0.3269 |
| AVISITN*TRTPN | 7 | 3 | -0.4116 | 0.05774 | 385 | -7.13 | <.0001 | 0.05 | -0.5251 | -0.2981 |
| AVISITN*TRTPN | 14 | 1 | -0.7240 | 0.07107 | 405 | -10.19 | <.0001 | 0.05 | -0.8637 | -0.5843 |
| AVISITN*TRTPN | 14 | 2 | -0.6900 | 0.07311 | 420 | -9.44 | <.0001 | 0.05 | -0.8337 | -0.5463 |
| AVISITN*TRTPN | 14 | 3 | -0.5289 | 0.07093 | 407 | -7.46 | <.0001 | 0.05 | -0.6683 | -0.3894 |
| AVISITN*TRTPN | 21 | 1 | -0.8550 | 0.07830 | 405 | -10.92 | <.0001 | 0.05 | -1.0089 | -0.7010 |
| AVISITN*TRTPN | 21 | 2 | -0.8637 | 0.08093 | 419 | -10.67 | <.0001 | 0.05 | -1.0227 | -0.7046 |


# STAT-5.1 Proc Mixed Output for Change from Baseline in CGI-S Scale, MMRM (UN) (Efficacy Sample)

\_\_\_\_\_

The Mixed Procedure

Least Squares Means

| | Analysis<br>Visit | Planned<br>Treatment | | Standard | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Effect | (N) | (N) | Estimate | Error | DF | t Value | Pr > t | Alpha | Lower | Upper |
| AVISITN*TRTPN | 21 | 3 | -0.6236 | 0.07749 | 396 | -8.05 | <.0001 | 0.05 | -0.7760 | -0.4713 |
| AVISITN*TRTPN | 28 | 1 | -0.9048 | 0.08001 | 403 | -11.31 | <.0001 | 0.05 | -1.0621 | -0.7475 |
| AVISITN*TRTPN | 28 | 2 | -0.9063 | 0.08273 | 413 | -10.96 | <.0001 | 0.05 | -1.0689 | -0.7437 |
| AVISITN*TRTPN | 28 | 3 | -0.6398 | 0.07895 | 392 | -8.10 | <.0001 | 0.05 | -0.7950 | -0.4846 |
| AVISITN*TRTPN | 35 | 1 | -0.9406 | 0.08760 | 403 | -10.74 | <.0001 | 0.05 | -1.1128 | -0.7684 |
| AVISITN*TRTPN | 35 | 2 | -1.0336 | 0.09091 | 418 | -11.37 | <.0001 | 0.05 | -1.2123 | -0.8549 |
| AVISITN*TRTPN | 35 | 3 | -0.6781 | 0.08597 | 389 | -7.89 | <.0001 | 0.05 | -0.8471 | -0.5090 |
| AVISITN*TRTPN | 42 | 1 | -1.0402 | 0.09021 | 406 | -11.53 | <.0001 | 0.05 | -1.2176 | -0.8629 |
| AVISITN*TRTPN | 42 | 2 | -0.9935 | 0.09365 | 415 | -10.61 | <.0001 | 0.05 | -1.1776 | -0.8095 |
| AVISITN*TRTPN | 42 | 3 | -0.7115 | 0.08826 | 388 | -8.06 | <.0001 | 0.05 | -0.8851 | -0.5380 |


## STAT-5.1

Proc Mixed Output for Change from Baseline in CGI-S Scale, MMRM (UN) (Efficacy Sample)

\_\_\_\_\_

The Mixed Procedure

Tests of Effect Slices

| | Analysis | | | | |
|---------------|----------|-----|-----|---------|--------|
| | Visit | Num | Den | | |
| Effect | (N) | DF | DF | F Value | Pr > F |
| AVISITN*TRTPN | 7 | 2 | 380 | 0.24 | 0.7878 |
| AVISITN*TRTPN | 14 | 2 | 381 | 2.39 | 0.0931 |
| AVISITN*TRTPN | 21 | 2 | 374 | 3.30 | 0.0379 |
| AVISITN*TRTPN | 28 | 2 | 370 | 4.03 | 0.0186 |
| AVISITN*TRTPN | 35 | 2 | 372 | 4.73 | 0.0094 |
| AVISITN*TRTPN | 42 | 2 | 372 | 4.24 | 0.0150 |


-----

 $$\tt STAT-5.2$$  Proc GLM Output for Change from Baseline to Day 42 in CGI-S Scale, LOCF (Efficacy Sample)

\_\_\_\_\_

The GLM Procedure

Class Level Information

Class Levels Values
TRTPN 3 1 2 3

POOLCNTR 39

Number of Observations Read 421 Number of Observations Used 421

CENTANAFADINE 2 OF 6


 $$\tt STAT-5.2$$  Proc GLM Output for Change from Baseline to Day 42 in CGI-S Scale, LOCF (Efficacy Sample)

The GLM Procedure

Dependent Variable: CHG Change from Baseline

| Source | | DF | Sum<br>Squar | | Mean Sq | uare F | Value | Pr > F |
|---|---|---|---|---|---|---|---|---|
| Model | | 41 | 75.26697 | 25 | 1.835 | 7798 | 1.97 | 0.0006 |
| Error | | 379 | 352.90879 | 94 | 0.931 | 1578 | | |
| Corrected Total | | 420 | 428.17577 | 20 | | | | |
| | R-Square | Coef | f Var | Root | MSE | CHG Mean | | |
| | 0.175785 | -118 | .7866 | 0.964 | 965 | -0.812352 | | |
| Source | | DF | Type III | SS | Mean Sq | uare F | Value | Pr > F |
| TRTPN<br>POOLCNTR<br>BASE | | 2<br>38<br>1 | 6.970645<br>46.936465<br>17.187534 | 90 | 3.4853<br>1.2351<br>17.1875 | 7016 | 3.74<br>1.33<br>18.46 | 0.0246<br>0.0997<br><.0001 |


 $$\tt STAT-5.2$$  Proc GLM Output for Change from Baseline to Day 42 in CGI-S Scale, LOCF (Efficacy Sample)

### The GLM Procedure

| Level of | | СНО | ; | BASE | |
|----------|-----|-------------|------------|------------|------------|
| TRTPN | N | Mean | Std Dev | Mean | Std Dev |
| 1 | 140 | -0.92142857 | 1.10634441 | 4.55714286 | 0.56608498 |
| 2 | 140 | -0.89285714 | 0.97225118 | 4.65714286 | 0.54668956 |
| 3 | 141 | -0.62411348 | 0.92225660 | 4.52482270 | 0.55525490 |


STAT-5.2

Proc GLM Output for Change from Baseline to Day 42 in CGI-S Scale, LOCF (Efficacy Sample)

The GLM Procedure Least Squares Means

| | | Standard | | LSMEAN |
|-------|-------------|------------|---------|--------|
| TRTPN | CHG LSMEAN | Error | Pr > t | Number |
| 1 | -0.99635472 | 0.08963644 | <.0001 | 1 |
| 2 | -0.93139660 | 0.09048002 | <.0001 | 2 |
| 3 | -0.69523223 | 0.08917989 | <.0001 | 3 |

Least Squares Means for effect TRTPN
Pr > |t| for H0: LSMean(i)=LSMean(j)

### Dependent Variable: CHG

| i/j | 1 | 2 | 3 |
|---|---|---|---|
| 1<br>2<br>3 | 0.5780<br>0.0096 | 0.5780 | 0.0096<br>0.0437 |
| TRTPN | CHG LSMEAN | 95% Confidenc | ce Limits |
| 1 | -0.996355<br>-0.931397 | -1.172602<br>-1.109302 | -0.820108<br>-0.753491 |


STAT-5.2

Proc GLM Output for Change from Baseline to Day 42 in CGI-S Scale, LOCF (Efficacy Sample)

The GLM Procedure Least Squares Means

TRTPN CHG LSMEAN 95% Confidence Limits

3 -0.695232 -0.870582 -0.519883

Least Squares Means for Effect TRTPN

Difference
Between 95% Confidence Limits for
i j Means LSMean(i)-LSMean(j)

1 2 -0.064958 -0.294343 0.164427
1 3 -0.301122 -0.528624 -0.073621
2 3 -0.236164 -0.465593 -0.006735

NOTE: To ensure overall protection level, only probabilities associated with pre-planned comparisons should be used.


 $$\tt STAT-5.2$$  Proc GLM Output for Change from Baseline to Day 42 in CGI-S Scale, LOCF

(Efficacy Sample)

The GLM Procedure

Dependent Variable: CHG Change from Baseline

| Parameter | Estimate | Standard<br>Error | t Value | Pr > t |
|-----------|-------------|-------------------|---------|---------|
| 1 vs 3 | -0.30112249 | 0.11570382 | -2.60 | 0.0096 |
| 2 vs 3 | -0.23616436 | 0.11668402 | -2.02 | 0.0437 |

| CENTANAFADINE | 1 OF 6 |
|------------------------|--------|

STAT-5.3

Proc GLM Output for Change from Baseline to Day 42 in CGI-S Scale, OC (Efficacy Sample)

------ Parameter Code=CGI0201 Analysis Visit (N)=42 ------

The GLM Procedure

Class Level Information

Class Levels Values
TRTPN 3 1 2 3

Number of Observations Read 421 Number of Observations Used 421

CENTANAFADINE 2 OF 6


 $$\tt STAT-5.3$$  Proc GLM Output for Change from Baseline to Day 42 in CGI-S Scale, OC (Efficacy Sample)

The GLM Procedure

Dependent Variable: CHG Change from Baseline

| Source | | DF | Sum<br>Squai | | Mean | Square | F Value | Pr > F |
|---|---|---|---|---|---|---|---|---|
| Model | | 3 | 28.33050 | )66 | 9.4 | 435022 | 9.85 | <.0001 |
| Error | | 417 | 399.84526 | 553 | 0.9 | 588615 | | |
| Corrected Total | | 420 | 428.1757 | 720 | | | | |
| | R-Square | Coef | f Var | Root | MSE | CHG Me | an | |
| | 0.066166 | -120 | .5408 | 0.979 | 215 | -0.8123 | 52 | |
| Source | | DF | Type III | SS | Mean | Square | F Value | Pr > F |
| TRTPN | | 2 | 6.176562 | | | 828118 | 3.22 | 0.0409 |
| BASE | | 1 | 20.761320 | )28 | 20.76 | 132028 | 21.65 | <.0001 |


 $$\tt STAT-5.3$$  Proc GLM Output for Change from Baseline to Day 42 in CGI-S Scale, OC (Efficacy Sample)

......

### The GLM Procedure

| Level of | | СНО | ; | BAS | E |
|----------|-----|-------------|------------|------------|------------|
| TRTPN | N | Mean | Std Dev | Mean | Std Dev |
| 1 | 140 | -0.92142857 | 1.10634441 | 4.55714286 | 0.56608498 |
| 2 | 140 | -0.89285714 | 0.97225118 | 4.65714286 | 0.54668956 |
| 3 | 141 | -0.62411348 | 0.92225660 | 4.52482270 | 0.55525490 |


## STAT-5.3

Proc GLM Output for Change from Baseline to Day 42 in CGI-S Scale, OC (Efficacy Sample)

------

### The GLM Procedure Least Squares Means

| | | Standard | | LSMEAN |
|-------|-------------|------------|---------|--------|
| TRTPN | CHG LSMEAN | Error | Pr > t | Number |
| 1 | -0.93041807 | 0.08278130 | <.0001 | 1 |
| 2 | -0.86176789 | 0.08302801 | <.0001 | 2 |
| 3 | -0.64605649 | 0.08259948 | <.0001 | 3 |

Least Squares Means for effect TRTPN Pr > |t| for H0: LSMean(i)=LSMean(j)

### Dependent Variable: CHG

| i/j | 1 | 2 | 3 |
|---|---|---|---|
| 1<br>2<br>3 | 0.5589<br>0.0154 | 0.5589 | 0.0154<br>0.0668 |
| TRTPN | CHG LSMEAN | 95% Confidence | e Limits |
| 1 2 | -0.930418<br>-0.861768 | -1.093139<br>-1.024973 | -0.767697<br>-0.698562 |


STAT-5.3

Proc GLM Output for Change from Baseline to Day 42 in CGI-S Scale, OC (Efficacy Sample)

......

The GLM Procedure Least Squares Means

TRTPN CHG LSMEAN 95% Confidence Limits

3 -0.646056 -0.808420 -0.483693

Least Squares Means for Effect TRTPN

Difference
Between 95% Confidence Limits for
i j Means LSMean(i)-LSMean(j)

1 2 -0.068650 -0.299331 0.162031
1 3 -0.284362 -0.514078 -0.054646
2 3 -0.215711 -0.446452 0.015030

NOTE: To ensure overall protection level, only probabilities associated with pre-planned comparisons should be used.


STAT-5.3

Proc GLM Output for Change from Baseline to Day 42 in CGI-S Scale, OC (Efficacy Sample)

The GLM Procedure

Dependent Variable: CHG Change from Baseline

| Parameter | Estimate | Estimate Error t | | |
|-----------|-------------|------------------|-------|--------|
| 1 vs 3 | -0.28436158 | 0.11686401 | -2.43 | 0.0154 |
| 2 vs 3 | -0.21571140 | 0.11738543 | -1.84 | 0.0668 |

CENTANAFADINE 1 OF 1 PROTOCOL 405-201-00014

STAT-6.1.1

Shapiro-Wilk Test for Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

| | | | | GOODNESS OF FIT | |
|---|---|---|---|---|---|
| | | TEST | GOODNESS OF FIT | TEST | |
| PROTOCOL | Day | VARIABLE | TEST | STATISTICS | Pvalue |
| 40520100014 | DAY 7 | RESID | Shapiro-Wilk | 0.9618 | <0.0001 |
| | | STUDENTRESID | Shapiro-Wilk | 0.9619 | <0.0001 |
| | DAY 14 | RESID | Shapiro-Wilk | 0.9742 | <0.0001 |
| | | STUDENTRESID | Shapiro-Wilk | 0.9729 | <0.0001 |
| | DAY 21 | RESID | Shapiro-Wilk | 0.9755 | <0.0001 |
| | | STUDENTRESID | Shapiro-Wilk | 0.9754 | <0.0001 |
| | DAY 28 | RESID | Shapiro-Wilk | 0.9780 | <0.0001 |
| | | STUDENTRESID | Shapiro-Wilk | 0.9785 | <0.0001 |
| | DAY 35 | RESID | Shapiro-Wilk | 0.9772 | <0.0001 |
| | | STUDENTRESID | Shapiro-Wilk | 0.9776 | <0.0001 |
| | DAY 42 | RESID | Shapiro-Wilk | 0.9767 | <0.0001 |
| | | STUDENTRESID | Shapiro-Wilk | 0.9772 | <0.0001 |

------

FILE: normality\_ba.lis, RUN: 31AUG2020 08:32

| OF 48 |
|-------|
|-------|


STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

The UNIVARIATE Procedure Variable: RESID (Residual)

#### Moments

| N | 415 | Sum Weights | 415 |
|-----------------|------------|------------------|------------|
| Mean | 0.00590733 | Sum Observations | 2.45154156 |
| Std Deviation | 6.29621838 | Variance | 39.6423659 |
| Skewness | -0.7622497 | Kurtosis | 1.20879183 |
| Uncorrected SS | 16411.9539 | Corrected SS | 16411.9395 |
| Coeff Variation | 106583.167 | Std Error Mean | 0.3090692 |

### Basic Statistical Measures

### Location Variability

| Mean | 0.005907 | Std Deviation | 6.29622 |
|--------|----------|---------------------|----------|
| Median | 0.890327 | Variance | 39.64237 |
| Mode | 2.147650 | Range | 41.51301 |
| | | Interguartile Range | 6.74509 |

-----

FILE: normalitybc.lis, RUN: 31AUG2020 08:32

| CENTANAFADINE | 2 OF 4 |
|---------------|--------|
|---------------|--------|


STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

The UNIVARIATE Procedure Variable: RESID (Residual)

Tests for Location: Mu0=0

| Test | -S | tatistic- | p Valı | ue |
|-------------|----|-----------|----------|--------|
| Student's t | t | 0.019113 | Pr > t | 0.9848 |
| Sign | M | 31.5 | Pr >= M | 0.0023 |
| Signed Rank | S | 4203 | Pr >= S | 0.0856 |

### Tests for Normality

| Test | Sta | tistic | р | p Value |
|--------------------|------|----------|---------|------------|
| Shapiro-Wilk | W | 0.961785 | Pr < W | <0.0001 |
| Kolmogorov-Smirnov | D | 0.084284 | Pr > D | <0.0100 |
| Cramer-von Mises | W-Sq | 0.900816 | Pr > W- | Sq <0.0050 |
| Anderson-Darling | A-Sq | 5.031644 | Pr > A- | Sq <0.0050 |

-----

FILE: normalitybc.lis, RUN: 31AUG2020 08:32

| CENTANAFADINE | 3 OF 48 |
|------------------------|---------|

STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

\_\_\_\_\_\_

The UNIVARIATE Procedure Variable: RESID (Residual)

Quantiles (Definition 5)

| Level | Quantile |
|------------|-------------------------|
| 100% Max | 17.902786 |
| 99% | 11.786668 |
| 95% | 8.673196 |
| 90% | 6.633776 |
| 75% Q3 | 3.932496 |
| 50% Median | 0.890327 |
| 25% O1 | -2.812590 |
| 10% | -8.383850<br>-12.326090 |
| 1% | -17.376429 |
| 0% Min | -23.610226 |

\_\_\_\_\_

FILE: normalitybc.lis, RUN: 31AUG2020 08:32

CENTANAFADINE 4 OF 48 PROTOCOL 405-201-00014

STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

-----

------ Analysis Visit (N)=7 ------

The UNIVARIATE Procedure Variable: RESID (Residual)

Extreme Observations

| 20,000 | | | | nighted c | |
|----------|--------------|-----|---------|--------------|-----|
| Value | USUBJID | Obs | Value | USUBJID | Obs |
| -23.6102 | 40520100014- | 253 | 11.7867 | 40520100014- | 24 |
| -23.5381 | 40520100014- | 267 | 12.5707 | 40520100014- | 44 |
| -20.6914 | 40520100014- | 395 | 14.6909 | 40520100014- | 36 |
| -18.3791 | 40520100014- | 48 | 15.9070 | 40520100014- | 281 |
| -17.3764 | 40520100014- | 381 | 17.9028 | 40520100014- | 186 |

------

FILE: normalitybc.lis, RUN: 31AUG2020 08:32

CENTANAFADINE 5 OF 48


STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

......

The UNIVARIATE Procedure

Variable: STUDENTRESID (Studentized Residual)

Moments

| N | 415 | Sum Weights | 415 |
|-----------------|------------|------------------|------------|
| Mean | 0.00076876 | Sum Observations | 0.31903492 |
| Std Deviation | 1.01663979 | Variance | 1.03355646 |
| Skewness | -0.7470648 | Kurtosis | 1.26177724 |
| Uncorrected SS | 427.892621 | Corrected SS | 427.892376 |
| Coeff Variation | 132244.305 | Std Error Mean | 0.04990488 |

Basic Statistical Measures

Location Variability

| Mean | 0.000769 | Std Deviation | 1.01664 |
|--------|----------|---------------------|---------|
| Median | 0.138127 | Variance | 1.03356 |
| Mode | 0.330816 | Range | 6.97281 |
| | | Interguartile Range | 1.04756 |

------

FILE: normalitybc.lis, RUN: 31AUG2020 08:32
| 6 OF | 48 | 5 |
|------|----|---|
|------|----|---|

STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

The UNIVARIATE Procedure

Variable: STUDENTRESID (Studentized Residual)

Tests for Location: Mu0=0

| Test | -St | tatistic- | p Valı | 1e |
|-------------|-----|-----------|----------|--------|
| Student's t | t | 0.015404 | Pr > t | 0.9877 |
| Sign | M | 31.5 | Pr >= M | 0.0023 |
| Signed Rank | S | 4190 | Pr >= S | 0.0866 |

#### Tests for Normality

| Test | Sta | tistic | p V | alue |
|--------------------|------|----------|----------|-----------|
| Shapiro-Wilk | W | 0.961929 | Pr < W | <0.0001 |
| Kolmogorov-Smirnov | D | 0.086473 | Pr > D | <0.0100 |
| Cramer-von Mises | W-Sq | 0.912147 | Pr > W-S | q <0.0050 |
| Anderson-Darling | A-Sq | 5.104489 | Pr > A-S | q <0.0050 |

\_\_\_\_\_\_

FILE: normalitybc.lis, RUN: 31AUG2020 08:32

| CENTANAFADINE 7 OF 48 |
|-----------------------|

STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

The UNIVARIATE Procedure

Variable: STUDENTRESID (Studentized Residual)

Quantiles (Definition 5)

| Level | Quantile |
|------------|-----------|
| 100% Max | 3.049245 |
| 99% | 1.938606 |
| 95% | 1.444558 |
| 90% | 1.079590 |
| 75% Q3 | 0.613816 |
| 50% Median | 0.138127 |
| 25% Q1 | -0.433740 |
| 10% | -1.322380 |
| 5% | -2.093381 |
| 1% | -2.777724 |
| 0% Min | -3.923569 |

\_\_\_\_\_\_

FILE: normalitybc.lis, RUN: 31AUG2020 08:32

CENTANAFADINE

8 OF 48

STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

\_\_\_\_\_\_

------ Analysis Visit (N)=7 ------

The UNIVARIATE Procedure
Variable: STUDENTRESID (Studentized Residual)

Extreme Observations

| | Lowest | | | | Highest |
|----------|--------------|-----|---------|--------------|---------|
| Value | USUBJID | Obs | Value | USUBJID | Obs |
| -3.92357 | 40520100014- | 267 | 1.93861 | 40520100014- | 328 |
| -3.74529 | 40520100014- | 253 | 2.19553 | 40520100014- | 24 |
| -3.23957 | 40520100014- | 395 | 2.26410 | 40520100014- | 36 |
| -2.83208 | 40520100014- | 48 | 2.64914 | 40520100014- | 281 |
| -2.77772 | 40520100014- | 414 | 3.04925 | 40520100014- | 186 |

------

FILE: normalitybc.lis, RUN: 31AUG2020 08:32

CENTANAFADINE 9 OF 48


STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

The UNIVARIATE Procedure Variable: RESID (Residual)

#### Moments

| N | 389 | Sum Weights | 389 |
|-----------------|------------|------------------|------------|
| Mean | -0.0478972 | Sum Observations | -18.632024 |
| Std Deviation | 8.10987026 | Variance | 65.7699957 |
| Skewness | -0.6462853 | Kurtosis | 0.96373179 |
| Uncorrected SS | 25519.6508 | Corrected SS | 25518.7583 |
| Coeff Variation | -16931.814 | Std Error Mean | 0.41118674 |

## Basic Statistical Measures

Location Variability

| Mean | -0.04790 | Std Deviation | 8.10987 |
|--------|----------|---------------------|----------|
| Median | 1.17581 | Variance | 65.77000 |
| Mode | 5.07029 | Range | 55.06309 |
| | | Interquartile Range | 10.14964 |

------

FILE: normalitybc.lis, RUN: 31AUG2020 08:32

| CENTANAFADINE 10 | OF | 4 | 8 |
|------------------|----|---|---|
|------------------|----|---|---|

STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

The UNIVARIATE Procedure Variable: RESID (Residual)

Tests for Location: Mu0=0

| Student's t t $-0.11649$ Pr > t 0.9073<br>Sign M 25.5 Pr >= M 0.0111 | Test | -St | atistic- | p Valı | ıe |
|---|---|---|---|---|---|
| Signed Rank S 2399.5 Pr >= S 0.2801 | | | | 1 - 1 | |

## Tests for Normality

| Test | Sta | tistic | p Va | lue |
|--------------------|------|----------|-----------|-----------|
| Shapiro-Wilk | W | 0.974232 | Pr < W | <0.0001 |
| Kolmogorov-Smirnov | D | 0.075075 | Pr > D | <0.0100 |
| Cramer-von Mises | W-Sq | 0.543451 | Pr > W-Sc | 4 <0.0050 |
| Anderson-Darling | A-Sq | 2.960271 | Pr > A-Sc | 4 <0.0050 |

\_\_\_\_\_\_

FILE: normalitybc.lis, RUN: 31AUG2020 08:32

| CENTANAFADINE | 11 OF 48 |
|---------------|----------|

PROTOCOL 405-201-00014 STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

\_\_\_\_\_\_

The UNIVARIATE Procedure Variable: RESID (Residual)

Quantiles (Definition 5)

| Level | Quantile |
|------------|-----------|
| 100% Max | 22.23178 |
| 99% | 16.59354 |
| 95% | 11.12111 |
| 90% | 9.36192 |
| 75% Q3 | 5.23846 |
| 50% Median | 1.17581 |
| 25% Q1 | -4.91118 |
| 10% | -10.67147 |
| 5% | -15.17154 |
| 1% | -23.34365 |
| 0% Min | -32.83131 |

\_\_\_\_\_

FILE: normalitybc.lis, RUN: 31AUG2020 08:32

CENTANAFADINE 12 OF 48 PROTOCOL 405-201-00014

STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

-----

The UNIVARIATE Procedure Variable: RESID (Residual)

Extreme Observations

| Dwesc | | | | 11 | ignest |
|----------|-------------|-----|---------|--------------|--------|
| Value | USUBJID | Obs | Value | USUBJID | Obs |
| -32.8313 | 40520100014 | 437 | 16.5927 | 40520100014- | 451 |
| -29.4798 | 40520100014 | 665 | 16.5935 | 40520100014- | 459 |
| -25.1439 | 40520100014 | 796 | 17.5325 | 40520100014- | 470 |
| -23.3436 | 40520100014 | 651 | 17.8254 | 40520100014- | 589 |
| -22.7128 | 40520100014 | 482 | 22.2318 | 40520100014- | 678 |

------

FILE: normalitybc.lis, RUN: 31AUG2020 08:32

CENTANAFADINE 13 OF 48


STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

The UNIVARIATE Procedure

Variable: STUDENTRESID (Studentized Residual)

Moments

| N | 389 | Sum Weights | 389 |
|-----------------|------------|------------------|------------|
| Mean | -0.0058977 | Sum Observations | -2.2942086 |
| Std Deviation | 1.00702053 | Variance | 1.01409034 |
| Skewness | -0.6687682 | Kurtosis | 1.22213191 |
| Uncorrected SS | 393.480582 | Corrected SS | 393.467052 |
| Coeff Variation | -17074.776 | Std Error Mean | 0.05105797 |

Basic Statistical Measures

Location Variability

| Mean | -0.00590 | Std Deviation | 1.00702 |
|--------|----------|---------------------|---------|
| Median | 0.14300 | Variance | 1.01409 |
| Mode | 0.61175 | Range | 7.23960 |
| | | Interguartile Range | 1.23899 |

-----

FILE: normalitybc.lis, RUN: 31AUG2020 08:32

| CENTANAFADINE 14 O | OF | 1 4 | 48 |
|--------------------|----|-----|----|
|--------------------|----|-----|----|

STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

The UNIVARIATE Procedure

Variable: STUDENTRESID (Studentized Residual)

Tests for Location: Mu0=0

| Test | -Stat | istic- | | p Value | e |
|-------------|-------|--------|----|---------|--------|
| Student's t | t -0 | .11551 | Pr | > t | 0.9081 |
| Sign | M | 25.5 | Pr | >= M | 0.0111 |
| Signed Rank | S | 2371.5 | Pr | >= S | 0.2858 |

## Tests for Normality

| Test | Sta | tistic | p | Value |
|--------------------|------|----------|--------|-------------|
| Shapiro-Wilk | W | 0.972919 | Pr < W | <0.0001 |
| Kolmogorov-Smirnov | D | 0.075857 | Pr > D | <0.0100 |
| Cramer-von Mises | W-Sq | 0.550481 | Pr > W | -Sq <0.0050 |
| Anderson-Darling | A-Sq | 2.96986 | Pr > A | -Sq <0.0050 |

\_\_\_\_\_

FILE: normalitybc.lis, RUN: 31AUG2020 08:32

| CENTANAFADINE | 15 OF 48 |
|---------------|----------|
|---------------|----------|

STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

# The UNIVARIATE Procedure

Variable: STUDENTRESID (Studentized Residual)

Quantiles (Definition 5)

| Level | Quantile |
|------------|-----------|
| 100% Max | 2.814987 |
| 99% | 2.126709 |
| 95% | 1.349592 |
| 90% | 1.156538 |
| 75% Q3 | 0.635037 |
| 50% Median | 0.142997 |
| 25% Q1 | -0.603950 |
| 10% | -1.376566 |
| 5% | -1.830571 |
| 1% | -2.869759 |
| 0% Min | -4.424614 |

\_\_\_\_\_\_

FILE: normalitybc.lis, RUN: 31AUG2020 08:32

CENTANAFADINE 16 OF 48


STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

------

------ Analysis Visit (N)=14 ------

The UNIVARIATE Procedure

Variable: STUDENTRESID (Studentized Residual)

## Extreme Observations

| Lowest | | | | | | |
|--------|----------|--------------|-----|---------|--------------|-----|
| | Value | USUBJID | Obs | Value | USUBJID | Obs |
| | -4.42461 | 40520100014- | 437 | 2.00259 | 40520100014- | 459 |
| | -3.72916 | 40520100014- | 665 | 2.12671 | 40520100014- | 470 |
| | -3.07149 | 40520100014- | 796 | 2.13944 | 40520100014- | 558 |
| | -2.86976 | 40520100014- | 482 | 2.28195 | 40520100014- | 589 |
| | -2.86776 | 40520100014- | 651 | 2.81499 | 40520100014- | 678 |

------

FILE: normalitybc.lis, RUN: 31AUG2020 08:32

CENTANAFADINE 17 OF 48


STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

The UNIVARIATE Procedure Variable: RESID (Residual)

#### Moments

| N | 375 | Sum Weights | 375 |
|-----------------|------------|------------------|------------|
| Mean | 0.04424235 | Sum Observations | 16.5908809 |
| Std Deviation | 8.77628273 | Variance | 77.0231386 |
| Skewness | -0.5795826 | Kurtosis | 0.26916873 |
| Uncorrected SS | 28807.3879 | Corrected SS | 28806.6538 |
| Coeff Variation | 19836.8372 | Std Error Mean | 0.45320529 |

## Basic Statistical Measures

## Location Variability

| Mean | 0.04424 | Std Deviation | 8.77628 |
|--------|----------|---------------------|----------|
| Median | 0.97708 | Variance | 77.02314 |
| Mode | -4.26252 | Range | 53.44257 |
| | | Interguartile Range | 12.23517 |

Note: The mode displayed is the smallest of 3 modes with a count of 2.

\_\_\_\_\_\_

FILE: normalitybc.lis, RUN: 31AUG2020 08:32

| 48 |
|----|

STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

The UNIVARIATE Procedure Variable: RESID (Residual)

Tests for Location: Mu0=0

| Test | -Sta | tistic- | p V | alue |
|-------------|------|---------|----------|--------|
| Student's t | t 0 | .097621 | Pr > t | 0.9223 |
| Sign | M | 14.5 | Pr >= M | 0.1481 |
| Signed Rank | S | 2381 | Pr >= S | 0.2575 |

## Tests for Normality

| Test | Sta | tistic | р | Value |
|--------------------|------|----------|---------|-------------|
| Shapiro-Wilk | W | 0.975477 | Pr < W | <0.0001 |
| Kolmogorov-Smirnov | D | 0.067214 | Pr > D | <0.0100 |
| Cramer-von Mises | W-Sq | 0.379476 | Pr > W- | -Sq <0.0050 |
| Anderson-Darling | A-Sq | 2.479975 | Pr > A- | -Sq <0.0050 |

\_\_\_\_\_

FILE: normalitybc.lis, RUN: 31AUG2020 08:32

| CENTANAFADINE | 19 OF 48 |
|---------------|----------|
|---------------|----------|

STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

The UNIVARIATE Procedure Variable: RESID (Residual)

Quantiles (Definition 5)

| Level | Quantile |
|------------|------------|
| 100% Max | 23.818333 |
| 95% | 12.320121 |
| 90% | 10.028486 |
| 75% Q3 | 6.741001 |
| 50% Median | 0.977085 |
| 25% Q1 | -5.494165 |
| 10% | -11.975058 |
| 5% | -16.506856 |
| 1% | -25.986745 |
| 0% Min | -29.624234 |

\_\_\_\_\_

FILE: normalitybc.lis, RUN: 31AUG2020 08:32

CENTANAFADINE 20 OF 48


STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

-----

------ Analysis Visit (N)=21 ------

The UNIVARIATE Procedure Variable: RESID (Residual)

Extreme Observations

| Howest | | | | nighest | |
|----------|--------------|------|---------|--------------|------|
| Value | USUBJID | Obs | Value | USUBJID | Obs |
| -29.6242 | 40520100014- | 1043 | 14.0883 | 40520100014- | 1081 |
| -26.7808 | 40520100014- | 966 | 15.3032 | 40520100014- | 921 |
| -26.7543 | 40520100014- | 825 | 17.2591 | 40520100014- | 1076 |
| -25.9867 | 40520100014- | 848 | 20.5261 | 40520100014- | 1056 |
| -23.7829 | 40520100014- | 832 | 23.8183 | 40520100014- | 856 |

------

FILE: normalitybc.lis, RUN: 31AUG2020 08:32

CENTANAFADINE 21 OF 48


STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

The UNIVARIATE Procedure

Variable: STUDENTRESID (Studentized Residual)

Moments

| N | 375 | Sum Weights | 375 |
|-----------------|------------|------------------|------------|
| Mean | 0.00487939 | Sum Observations | 1.82977148 |
| Std Deviation | 1.00562938 | Variance | 1.01129045 |
| Skewness | -0.5952846 | Kurtosis | 0.35653957 |
| Uncorrected SS | 378.231556 | Corrected SS | 378.222628 |
| Coeff Variation | 20609.7331 | Std Error Mean | 0.05193048 |

Basic Statistical Measures

Location Variability

| Mean | 0.00488 | Std Deviation | 1.00563 |
|--------|----------|---------------------|---------|
| Median | 0.11437 | Variance | 1.01129 |
| Mode | -0.47879 | Range | 6.14534 |
| | | Interquartile Range | 1.39912 |

Note: The mode displayed is the smallest of 3 modes with a count of 2.

FILE: normalitybc.lis, RUN: 31AUG2020 08:32

| OF 48 |
|-------|
|-------|

STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

The UNIVARIATE Procedure

Variable: STUDENTRESID (Studentized Residual)

Tests for Location: Mu0=0

| Test | -St | tatistic- | p Val | ue |
|-------------|-----|-----------|----------|--------|
| Student's t | t | 0.09396 | Pr > t | 0.9252 |
| Sign | M | 14.5 | Pr >= M | 0.1481 |
| Signed Rank | S | 2414 | Pr >= S | 0.2510 |

## Tests for Normality

| Test | Sta | tistic | | -p Val | ue |
|--------------------|------|----------|------|--------|---------|
| Shapiro-Wilk | M | 0.97535 | Pr < | W | <0.0001 |
| Kolmogorov-Smirnov | D | 0.067951 | Pr > | D | <0.0100 |
| Cramer-von Mises | W-Sq | 0.375553 | Pr > | W-Sq | <0.0050 |
| Anderson-Darling | A-Sq | 2.435138 | Pr > | A-Sq | <0.0050 |

\_\_\_\_\_\_

FILE: normalitybc.lis, RUN: 31AUG2020 08:32

| CENTANAFADINE | 23 OF 48 |
|---------------|----------|
|---------------|----------|

STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

\_\_\_\_\_

# The UNIVARIATE Procedure

Variable: STUDENTRESID (Studentized Residual)

Quantiles (Definition 5)

| Level | Quantile |
|------------|-----------|
| 100% Max | 2.685261 |
| 99% | 1.737520 |
| 95% | 1.409697 |
| 90% | 1.150881 |
| 75% Q3 | 0.773889 |
| 50% Median | 0.114367 |
| 25% Q1 | -0.625233 |
| 10% | -1.363214 |
| 5% | -1.907909 |
| 1% | -2.928031 |
| 0% Min | -3.460083 |

\_\_\_\_\_

FILE: normalitybc.lis, RUN: 31AUG2020 08:32

CENTANAFADINE 24 OF 48 PROTOCOL 405-201-00014

STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

\_\_\_\_\_

------ Analysis Visit (N)=21 -----

The UNIVARIATE Procedure
Variable: STUDENTRESID (Studentized Residual)

Extreme Observations

| | | -Lowest | | | Highest |
|----------|--------------|---------|---------|--------------|---------|
| Value | USUBJID | Obs | Value | USUBJID | Obs |
| -3.46008 | 40520100014- | 1043 | 1.72616 | 40520100014- | 914 |
| -3.30052 | 40520100014- | 825 | 1.73752 | 40520100014- | 921 |
| -3.15665 | 40520100014- | 966 | 1.93699 | 40520100014- | 1076 |
| -2.92803 | 40520100014- | 848 | 2.39535 | 40520100014- | 1056 |
| -2.67885 | 40520100014- | 868 | 2.68526 | 40520100014- | 856 |

\_\_\_\_\_

FILE: normalitybc.lis, RUN: 31AUG2020 08:32

CENTANAFADINE 25 OF 48


STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

......

The UNIVARIATE Procedure Variable: RESID (Residual)

#### Moments

| N | 366 | Sum Weights | 366 |
|-----------------|------------|------------------|------------|
| Mean | 0.10619435 | Sum Observations | 38.8671306 |
| Std Deviation | 9.24929929 | Variance | 85.5495374 |
| Skewness | -0.504134 | Kurtosis | -0.0661248 |
| Uncorrected SS | 31229.7086 | Corrected SS | 31225.5812 |
| Coeff Variation | 8709.78509 | Std Error Mean | 0.48346862 |

## Basic Statistical Measures

Location Variability

| Mean | 0.106194 | Std Deviation | 9.24930 |
|--------|----------|---------------------|----------|
| Median | 1.270199 | Variance | 85.54954 |
| Mode | 6.917760 | Range | 50.29097 |
| | | Interguartile Range | 12.74462 |

\_\_\_\_\_\_

FILE: normalitybc.lis, RUN: 31AUG2020 08:32

| CENTANAFADINE 26 OF | F 48 |
|---------------------|------|
|---------------------|------|

STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

The UNIVARIATE Procedure Variable: RESID (Residual)

Tests for Location: Mu0=0

| Test | -Stat | istic- | p Val | ue |
|-------------|-------|--------|----------|--------|
| Student's t | t 0. | 219651 | Pr > t | 0.8263 |
| Sign | M | 24 | Pr >= M | 0.0139 |
| Signed Rank | S | 2320.5 | Pr >= S | 0.2525 |

#### Tests for Normality

| Test | Sta | tistic | p Val | lue |
|--------------------|------|----------|-----------|---------|
| Shapiro-Wilk | M | 0.977981 | Pr < W | <0.0001 |
| Kolmogorov-Smirnov | D | 0.069596 | Pr > D | <0.0100 |
| Cramer-von Mises | W-Sq | 0.475034 | Pr > W-Sq | <0.0050 |
| Anderson-Darling | A-Sq | 2.720452 | Pr > A-Sq | <0.0050 |

\_\_\_\_\_

FILE: normalitybc.lis, RUN: 31AUG2020 08:32

| CENTANAFADINE | 27 OF 48 |
|---------------|----------|
|---------------|----------|

STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

The UNIVARIATE Procedure Variable: RESID (Residual)

Quantiles (Definition 5)

| Level | Quantile |
|---|---|
| 100% Max<br>99%<br>95%<br>90%<br>75% Q3<br>50% Median | 23.67290<br>17.88792<br>13.05207<br>10.51949<br>7.10617<br>1.27020 |
| 25% Q1<br>10%<br>5% | -5.63845<br>-12.94030<br>-16.83098<br>-24.63841 |
| 0% Min | -26.61808 |

\_\_\_\_\_\_

FILE: normalitybc.lis, RUN: 31AUG2020 08:32

CENTANAFADINE 28 OF 48


STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

------

------ Analysis Visit (N)=28 -----

The UNIVARIATE Procedure Variable: RESID (Residual)

Extreme Observations

| Iowesc | | | | nighesc | |
|----------|--------------|------|---------|--------------|------|
| Value | USUBJID | Obs | Value | USUBJID | Obs |
| -26.6181 | 40520100014- | 1408 | 17.6443 | 40520100014- | 1440 |
| -26.2893 | 40520100014- | 1199 | 17.8879 | 40520100014- | 1350 |
| -24.9814 | 40520100014- | 1242 | 18.4836 | 40520100014- | 1213 |
| -24.6384 | 40520100014- | 1245 | 20.7367 | 40520100014- | 1421 |
| -24.6213 | 40520100014- | 1334 | 23.6729 | 40520100014- | 1336 |

------

FILE: normalitybc.lis, RUN: 31AUG2020 08:32

CENTANAFADINE 29 OF 48


STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

......

The UNIVARIATE Procedure

Variable: STUDENTRESID (Studentized Residual)

Moments

| N | 366 | Sum Weights | 366 |
|-----------------|------------|------------------|------------|
| Mean | 0.010984 | Sum Observations | 4.02014573 |
| Std Deviation | 1.00683954 | Variance | 1.01372586 |
| Skewness | -0.5138819 | Kurtosis | 0.01054228 |
| Uncorrected SS | 370.054095 | Corrected SS | 370.009937 |
| Coeff Variation | 9166.41575 | Std Error Mean | 0.05262835 |

Basic Statistical Measures

Location Variability

| Mean | 0.010984 | Std Deviation | 1.00684 |
|--------|----------|---------------------|---------|
| Median | 0.140686 | Variance | 1.01373 |
| Mode | 0.737348 | Range | 5.69482 |
| | | Interguartile Range | 1.37277 |

-----

FILE: normalitybc.lis, RUN: 31AUG2020 08:32

| ٥F | ' 4 | 18 | i | |
|----|-----|-----|----|------|
| ٥F | 7 | ? 4 | 48 | 7 48 |

STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

The UNIVARIATE Procedure

Variable: STUDENTRESID (Studentized Residual)

Tests for Location: Mu0=0

| Test | -S | tatistic- | p Valu | ıe |
|-------------|----|-----------|----------|--------|
| Student's t | t | 0.208709 | Pr > t | 0.8348 |
| Sign | M | 24 | Pr >= M | 0.0139 |
| Signed Rank | S | 2326.5 | Pr >= S | 0.2513 |

## Tests for Normality

| Test | Sta | tistic | р | Value |
|--------------------|------|----------|---------|------------|
| Shapiro-Wilk | W | 0.978466 | Pr < W | <0.0001 |
| Kolmogorov-Smirnov | D | 0.069808 | Pr > D | <0.0100 |
| Cramer-von Mises | W-Sq | 0.472312 | Pr > W- | Sq <0.0050 |
| Anderson-Darling | A-Sq | 2.687998 | Pr > A- | Sq <0.0050 |

\_\_\_\_\_\_

FILE: normalitybc.lis, RUN: 31AUG2020 08:32

| CENTANAFADINE | 31 OF 48 |
|---------------|----------|
|---------------|----------|

STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

\_\_\_\_\_

------ Analysis Visit (N)=28 ------

## The UNIVARIATE Procedure

Variable: STUDENTRESID (Studentized Residual)

Quantiles (Definition 5)

| Level | Quantile |
|---------------|------------------------|
| 100% Max | 2.640998 |
| 95% | 1.401831 |
| 90%<br>75% O3 | 1.157699 |
| 50% Median | 0.140686 |
| 25% Q1<br>10% | -0.609115<br>-1.386098 |
| 5% | -1.825071 |
| 1%<br>0% Min | -2.744377<br>-3.053825 |

\_\_\_\_\_\_

FILE: normalitybc.lis, RUN: 31AUG2020 08:32

CENTANAFADINE 32 OF 48 PROTOCOL 405-201-00014

STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

------

------ Analysis Visit (N)=28 ------

The UNIVARIATE Procedure
Variable: STUDENTRESID (Studentized Residual)

Extreme Observations

| Lowest | | | | | Highest |
|----------|--------------|------|---------|--------------|---------|
| Value | USUBJID | Obs | Value | USUBJID | Obs |
| -3.05383 | 40520100014- | 1199 | 1.88200 | 40520100014- | 1440 |
| -2.94301 | 40520100014- | 1408 | 1.97041 | 40520100014- | 1213 |
| -2.77174 | 40520100014- | 1242 | 2.02350 | 40520100014- | 1350 |
| -2.74438 | 40520100014- | 1334 | 2.29077 | 40520100014- | 1421 |
| -2.64333 | 40520100014- | 1245 | 2.64100 | 40520100014- | 1336 |

------

FILE: normalitybc.lis, RUN: 31AUG2020 08:32

CENTANAFADINE 33 OF 48


STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

The UNIVARIATE Procedure Variable: RESID (Residual)

#### Moments

| N | 344 | Sum Weights | 344 |
|-----------------|------------|------------------|------------|
| Mean | 0.22073119 | Sum Observations | 75.9315287 |
| Std Deviation | 9.61866843 | Variance | 92.5187824 |
| Skewness | -0.4952975 | Kurtosis | -0.1237985 |
| Uncorrected SS | 31750.7028 | Corrected SS | 31733.9424 |
| Coeff Variation | 4357.63905 | Std Error Mean | 0.51860385 |

## Basic Statistical Measures

Location Variability

| Mean | 0.220731 | Std Deviation | 9.61867 |
|--------|----------|---------------------|----------|
| Median | 1.701746 | Variance | 92.51878 |
| Mode | 7.432365 | Range | 54.67437 |
| | | Interguartile Range | 14.33341 |

-----

FILE: normalitybc.lis, RUN: 31AUG2020 08:32

CENTANAFADINE 34 OF 48


STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

The UNIVARIATE Procedure Variable: RESID (Residual)

Tests for Location: Mu0=0

| Test | -S | tatistic- | p Val | ue |
|-------------|----|-----------|----------|--------|
| Student's t | t | 0.425626 | Pr > t | 0.6706 |
| Sign | M | 16 | Pr >= M | 0.0945 |
| Signed Rank | S | 2217 | Pr >= S | 0.2302 |

## Tests for Normality

| Test | Sta | tistic | p Va | lue |
|--------------------|------|----------|-----------|---------|
| Shapiro-Wilk | W | 0.977242 | Pr < W | <0.0001 |
| Kolmogorov-Smirnov | D | 0.067652 | Pr > D | <0.0100 |
| Cramer-von Mises | W-Sq | 0.438875 | Pr > W-Sq | <0.0050 |
| Anderson-Darling | A-Sq | 2.629038 | Pr > A-Sq | <0.0050 |

\_\_\_\_\_\_

FILE: normalitybc.lis, RUN: 31AUG2020 08:32

| CENTANAFADINE | 35 OF 48 |
|---------------|----------|
|---------------|----------|

STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

------ Analysis Visit (N)=35 ------

The UNIVARIATE Procedure Variable: RESID (Residual)

Quantiles (Definition 5)

| Level | Quantile |
|------------|-----------|
| 100% Max | 22.53512 |
| 99% | 18.03788 |
| 95% | 13.41618 |
| 90% | 11.23166 |
| 75% Q3 | 7.76020 |
| 50% Median | 1.70175 |
| 25% Q1 | -6.57321 |
| 10% | -13.76659 |
| 5% | -16.80512 |
| 1% | -23.07843 |
| 0% Min | -32.13925 |

\_\_\_\_\_

FILE: normalitybc.lis, RUN: 31AUG2020 08:32

CENTANAFADINE 36 OF 48


STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

------

------ Analysis Visit (N)=35 -----

The UNIVARIATE Procedure Variable: RESID (Residual)

Extreme Observations

| Value | USUBJID | Obs | Value | USUBJID | Obs |
|----------|--------------|------|---------|--------------|------|
| -32.1393 | 40520100014- | 1562 | 17.1124 | 40520100014- | 1590 |
| -28.7832 | 40520100014- | 1691 | 18.0379 | 40520100014- | 1575 |
| -24.7266 | 40520100014- | 1606 | 21.5556 | 40520100014- | 1707 |
| -23.0784 | 40520100014- | 1569 | 22.1875 | 40520100014- | 1693 |
| -21.5722 | 40520100014- | 1663 | 22.5351 | 40520100014- | 1775 |

------

FILE: normalitybc.lis, RUN: 31AUG2020 08:32

CENTANAFADINE 37 OF 48


STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

......

The UNIVARIATE Procedure

Variable: STUDENTRESID (Studentized Residual)

Moments

| N | 344 | Sum Weights | 344 |
|-----------------|------------|------------------|------------|
| Mean | 0.02322776 | Sum Observations | 7.99034796 |
| Std Deviation | 1.00148516 | Variance | 1.00297252 |
| Skewness | -0.5068561 | Kurtosis | -0.0234398 |
| Uncorrected SS | 344.205173 | Corrected SS | 344.019575 |
| Coeff Variation | 4311.58814 | Std Error Mean | 0.05399646 |

Basic Statistical Measures

Location Variability

| Mean | 0.023228 | Std Deviation | 1.00149 |
|--------|----------|---------------------|---------|
| Median | 0.176296 | Variance | 1.00297 |
| Mode | 0.759057 | Range | 5.93096 |
| | | Interguartile Range | 1.49444 |

-----

FILE: normalitybc.lis, RUN: 31AUG2020 08:32

| 38 01 | 48 |
|-------|----|
|-------|----|

STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

The UNIVARIATE Procedure

Variable: STUDENTRESID (Studentized Residual)

Tests for Location: Mu0=0

| Test | -St | atistic- | p Val | ue |
|-------------|-----|----------|----------|--------|
| Student's t | t | 0.430172 | Pr > t | 0.6673 |
| Sign | M | 16 | Pr >= M | 0.0945 |
| Signed Rank | S | 2252 | Pr >= S | 0.2230 |

## Tests for Normality

| Test | Sta | tistic | p V | alue |
|--------------------|------|----------|----------|-----------|
| Shapiro-Wilk | W | 0.977591 | Pr < W | <0.0001 |
| Kolmogorov-Smirnov | D | 0.069272 | Pr > D | <0.0100 |
| Cramer-von Mises | W-Sq | 0.428574 | Pr > W-S | q <0.0050 |
| Anderson-Darling | A-Sq | 2.550366 | Pr > A-S | q <0.0050 |

-----

FILE: normalitybc.lis, RUN: 31AUG2020 08:32

| CENTANAFADINE | 39 OF 48 |
|---------------|----------|
|---------------|----------|

STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

\_\_\_\_\_\_

# The UNIVARIATE Procedure

Variable: STUDENTRESID (Studentized Residual)

Quantiles (Definition 5)

| Level | Quantile |
|---|---|
| 100% Max<br>99%<br>95%<br>90%<br>75% Q3<br>50% Median<br>25% Q1<br>10% | 2.378000<br>1.842423<br>1.414009<br>1.195080<br>0.813832<br>0.176296<br>-0.680604<br>-1.427671<br>-1.744891 |
| 1% | -2.358551 |
| 0% Min | -3.552963 |

\_\_\_\_\_\_

FILE: normalitybc.lis, RUN: 31AUG2020 08:32

CENTANAFADINE 40 OF 48


STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

------

------ Analysis Visit (N)=35 ------

The UNIVARIATE Procedure

Variable: STUDENTRESID (Studentized Residual)

Extreme Observations

| | | Lowest | | | Highest |
|----------|--------------|--------|---------|--------------|---------|
| Value | USUBJID | Obs | Value | USUBJID | Obs |
| -3.55296 | 40520100014- | 1562 | 1.74930 | 40520100014- | 1590 |
| -3.06229 | 40520100014- | 1691 | 1.84242 | 40520100014- | 1575 |
| -2.54111 | 40520100014- | 1606 | 2.22747 | 40520100014- | 1707 |
| -2.35855 | 40520100014- | 1569 | 2.36251 | 40520100014- | 1693 |
| -2.26636 | 40520100014- | 1663 | 2.37800 | 40520100014- | 1775 |

------

FILE: normalitybc.lis, RUN: 31AUG2020 08:32

CENTANAFADINE 41 OF 48


STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

......

The UNIVARIATE Procedure Variable: RESID (Residual)

#### Moments

| N | 338 | Sum Weights | 338 |
|-----------------|------------|------------------|------------|
| Mean | 0.21994106 | Sum Observations | 74.3400787 |
| Std Deviation | 10.206485 | Variance | 104.172337 |
| Skewness | -0.4662637 | Kurtosis | -0.2816581 |
| Uncorrected SS | 35122.428 | Corrected SS | 35106.0776 |
| Coeff Variation | 4640.5546 | Std Error Mean | 0.5551596 |

## Basic Statistical Measures

## Location Variability

| Mean | 0.219941 | Std Deviation | 10.20649 |
|--------|----------|---------------------|-----------|
| Median | 2.116541 | Variance | 104.17234 |
| Mode | 7.859023 | Range | 51.41794 |
| | | Interguartile Range | 14.95136 |

------

FILE: normalitybc.lis, RUN: 31AUG2020 08:32

| CENTANAFADINE | 42 OF 48 |
|---------------|----------|
|---------------|----------|

STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

The UNIVARIATE Procedure Variable: RESID (Residual)

Tests for Location: Mu0=0

| Test | -S | tatistic- | p Valı | ıe |
|---|---|---|---|---|
| Student's t<br>Sign<br>Signed Rank | t<br>M<br>S | 0.396176<br>21<br>1936.5 | Pr > t <br>Pr >= M <br>Pr >= S | 0.6922<br>0.0256<br>0.2821 |

## Tests for Normality

| Test | Statistic | | p Value | |
|--------------------|-----------|----------|----------|------------|
| Shapiro-Wilk | W | 0.976668 | Pr < W | <0.0001 |
| Kolmogorov-Smirnov | D | 0.076295 | Pr > D | <0.0100 |
| Cramer-von Mises | W-Sq | 0.500683 | Pr > W-9 | Sq <0.0050 |
| Anderson-Darling | A-Sq | 2.723085 | Pr > A-3 | Sq <0.0050 |

\_\_\_\_\_

FILE: normalitybc.lis, RUN: 31AUG2020 08:32

| CENTANAFADINE | 43 OF 48 |
|---------------|----------|
|---------------|----------|

STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

\_\_\_\_\_

The UNIVARIATE Procedure Variable: RESID (Residual)

Quantiles (Definition 5)

| Level | Quantile |
|--------------------------------|-------------------------------------|
| 100% Max<br>99%<br>95%<br>90% | 21.91943<br>20.45404<br>14.85949 |
| 75% Q3<br>50% Median<br>25% O1 | 7.82680<br>2.11654<br>-7.12456 |
| 10%<br>5%<br>1% | -14.10923<br>-18.33244<br>-27.07807 |
| 0% Min | -29.49851 |

\_\_\_\_\_\_

FILE: normalitybc.lis, RUN: 31AUG2020 08:32

CENTANAFADINE 44 OF 48


STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

------

------ Analysis Visit (N)=42 -----

The UNIVARIATE Procedure Variable: RESID (Residual)

Extreme Observations

| Lowest | | | nignest | | | |
|--------|----------|--------------|---------|---------|--------------|------|
| | Value | USUBJID | Obs | Value | USUBJID | Obs |
| | -29.4985 | 40520100014- | 2031 | 19.4617 | 40520100014- | 2128 |
| | -27.6116 | 40520100014- | 1928 | 20.4540 | 40520100014- | 1934 |
| | -27.3096 | 40520100014- | 2099 | 20.7976 | 40520100014- | 2111 |
| | -27.0781 | 40520100014- | 1950 | 21.6142 | 40520100014- | 2033 |
| | -25.9557 | 40520100014- | 2054 | 21.9194 | 40520100014- | 2046 |

\_\_\_\_\_\_

FILE: normalitybc.lis, RUN: 31AUG2020 08:32

| CENTANAFADINE | 45 OF 48 |
|---------------|----------|
|---------------|----------|

STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

# The UNIVARIATE Procedure

Variable: STUDENTRESID (Studentized Residual)

#### Moments

| N | 338 | Sum Weights | 338 |
|-----------------|------------|------------------|------------|
| Mean | 0.02186339 | Sum Observations | 7.38982701 |
| Std Deviation | 1.00255899 | Variance | 1.00512453 |
| Skewness | -0.4654092 | Kurtosis | -0.2701205 |
| Uncorrected SS | 338.888534 | Corrected SS | 338.726967 |
| Coeff Variation | 4585.55983 | Std Error Mean | 0.05453202 |

## Basic Statistical Measures

| Location | Variability |
|----------|-------------|
|----------|-------------|

| Mean | 0.021863 | Std Deviation | 1.00256 |
|--------|----------|---------------------|---------|
| Median | 0.204955 | Variance | 1.00512 |
| Mode | 0.760366 | Range | 5.13076 |
| | | Interguartile Range | 1.45333 |

------

FILE: normalitybc.lis, RUN: 31AUG2020 08:32

| CENTANAFADINE | 46 OF | 48 |
|---------------|-------|----|
|---------------|-------|----|

STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

The UNIVARIATE Procedure

Variable: STUDENTRESID (Studentized Residual)

Tests for Location: Mu0=0

| Test | -Sta | tistic- | p Valı | ıe |
|-------------|------|---------|----------|--------|
| Student's t | t C | .400928 | Pr > t | 0.6887 |
| Sign | M | 21 | Pr >= M | 0.0256 |
| Signed Rank | S | 1930.5 | Pr >= S | 0.2836 |

## Tests for Normality

| Test | Sta | tistic | p Val | ue |
|--------------------|------|----------|-----------|---------|
| Shapiro-Wilk | M | 0.977218 | Pr < W | <0.0001 |
| Kolmogorov-Smirnov | D | 0.075766 | Pr > D | <0.0100 |
| Cramer-von Mises | W-Sq | 0.494181 | Pr > W-Sq | <0.0050 |
| Anderson-Darling | A-Sq | 2.68251 | Pr > A-Sq | <0.0050 |

\_\_\_\_\_

FILE: normalitybc.lis, RUN: 31AUG2020 08:32

| CENTANAFADINE | 47 OF 48 |
|---------------|----------|
|---------------|----------|

STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

\_\_\_\_\_

# The UNIVARIATE Procedure

Variable: STUDENTRESID (Studentized Residual)

Quantiles (Definition 5)

| Level | Quantile |
|---|---|
| 100% Max<br>99%<br>95%<br>90%<br>75% Q3 | 2.170595<br>1.980822<br>1.444907<br>1.182725<br>0.762961<br>0.204955 |
| 25% Q1<br>10%<br>5% | -0.690365<br>-1.369158<br>-1.794783<br>-2.635345 |
| 0% Min | -2.960170 |

\_\_\_\_\_\_

FILE: normalitybc.lis, RUN: 31AUG2020 08:32

CENTANAFADINE 48 OF 48


STAT-6.1.2

Residual by Week from Proc Mixed for Change from Baseline in AISRS Total Score, Primary Efficacy Analysis Model (Efficacy Sample)

------

------ Analysis Visit (N)=42 -----

The UNIVARIATE Procedure

Variable: STUDENTRESID (Studentized Residual)

Extreme Observations

| Value USUBJID Obs Value USUBJID -2.96017 40520100014 2031 1.88413 40520100014- -2.72302 40520100014 2099 1.98082 40520100014- -2.68489 40520100014 1928 2.07185 40520100014- | mignese |
|---|---|
| -2.72302 40520100014 2099 1.98082 40520100014- | Obs |
| | 2128 |
| -2.68489 40520100014 1928 2.07185 40520100014- | 1934 |
| | 2111 |
| -2.63534 40520100014 1950 2.14336 40520100014- | 2046 |
| -2.54132 40520100014 2054 2.17059 40520100014- | 2033 |

------

FILE: normalitybc.lis, RUN: 31AUG2020 08:32



# This page is a manifestation of an electronically captured signature

# **SIGNATURE PAGE**

Document Name: P40520100014\_DOC\_STAT

Document Number: 1000088241

**Document Version: 3.0** 

| Signed by | Meaning of Signature | Server Date<br>(dd-MMM-<br>yyyy hh:min) -<br>UTC timezone |
|---|---|---|
| | Safety Approval | 22-Sep-2020<br>14:15:24 |
| | Biostatistics Approval | 22-Sep-2020<br>00:48:53 |
| | Clinical Programming<br>Approval | 22-Sep-2020<br>16:17:04 |
| | Clinical Approval | 23-Sep-2020<br>00:10:52 |